## Janssen Research & Development \*

#### **Clinical Protocol**

A Phase 2 Randomized, Open-label, Parallel-group, Multicenter Study to Assess Intrahepatic and Peripheral Changes of Immunologic and Virologic Markers in Response to Combination Regimens Containing JNJ-73763989 and Nucleos(t)ide Analog With or Without JNJ-56136379 in Patients With Chronic Hepatitis B Virus Infection

## The INSIGHT Study

# Protocol 73763989HPB2003; Phase 2 AMENDMENT 6

#### JNJ-73763989 and JNJ-56136379

\*Janssen Research & Development is a global organization that operates through different legal entities in various countries. Therefore, the legal entity acting as the sponsor for Janssen Research & Development studies may vary, such as, but not limited to Janssen Biotech, Inc.; Janssen Products, LP; Janssen Biologics, BV; Janssen-Cilag International NV; Janssen, Inc; Janssen Pharmaceutica NV; Janssen Sciences Ireland UC; Janssen Biopharma Inc.; or Janssen Research & Development, LLC. The term "sponsor" is used throughout the protocol to represent these various legal entities; the sponsor is identified on the Contact Information page that accompanies the protocol.

United States (US) sites of this study will be conducted under US Food & Drug Administration Investigational New Drug (IND) regulations (21 CFR Part 312).

**EudraCT NUMBER: 2019-004475-39** 

**Status:** Approved

**Date:** 25 November 2021

**Prepared by:** Janssen Research & Development, a division of Janssen Pharmaceutica NV

**EDMS number:** EDMS-ERI-200320376, 16.0

**GCP Compliance:** This study will be conducted in compliance with Good Clinical Practice, and applicable regulatory requirements.

#### **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

## PROTOCOL AMENDMENT SUMMARY OF CHANGES TABLE

| DOCUMENT HISTORY | |
|-------------------|------------------|
| Document | Date |
| Amendment 6 | This document |
| Amendment 5 | 01 October 2021 |
| Amendment 4 | 30 July 2021 |
| Amendment 3 | 14 August 2020 |
| Amendment 2 | 07 May 2020 |
| Amendment 1 | 10 April 2020 |
| Original Protocol | 12 February 2020 |

## **Amendment 6 (This document)**

**Overall Rationale for the Amendment:** The primary reason for this amendment is to update the criteria for post-treatment monitoring and for nucleos(t)ide analog (NA) re-treatment for participants who discontinued NA treatment at Week 48.

With Amendment 5, changes were introduced to the criteria for post-treatment monitoring and NA retreatment for patients who discontinued NA treatment. These changes were triggered by a case of hepatitis B reactivation with subacute hepatic failure (initially reported as severe clinical ALT flare) following NA treatment cessation as per protocol in the REEF-2 (73763989PAHPB2002) study which led to listing of the patient for high urgency liver transplantation. The patient received a donor liver at Week 14 post-stopping NA and has since then showed an uneventful post-operative recovery.

To further protect the safety of study participants, the current amendment includes additional changes to the criteria for post-treatment monitoring and for NA re-treatment for participants who discontinued NA treatment.

These changes are based on additional follow-up information from participants in the REEF-2 study who stopped all treatment including NA per protocol and is incorporating recommendations from Health Authorities and the independent data monitoring committee.

| <b>Description of Change</b> | Brief Rationale | Section Number and Name |
|---|---|---|
| Update of criteria for post- | In further off-treatment analysis of | 1.1 Synopsis |
| treatment monitoring and for | REEF-2 with all participants | 1.3.2 Schedule of Activities - Follow-up |
| NA re-treatment | having reached at least 12 weeks of | Phase |
| | follow-up post stopping NA, some | 2.3.3 Benefit-risk Assessment for Study |
| | participants show a pattern of fast | Participation |
| | increase of HBV DNA followed by | 4.2 Scientific Rationale for Study Design |
| | significant elevations of ALT that | 6.6.2 NA Re-treatment Criteria |
| | improved after re-starting of NA | 10.12 Appendix 12: NA Re-treatment and |
| | treatment. Based on these | Monitoring After Stopping of NA |
| | observations it was decided to | |
| | implement more conservative rules | |
| | for post-treatment monitoring and | |
| | re-treatment criteria for all | |
| | participants who met NA treatment | |
| | completion criteria and stopped NA | |
| | treatment. | |
| Minor errors were corrected | Correction and clarification. | Throughout the protocol |
| and minor clarifications | | |
| were made. | | |

# **TABLE OF CONTENTS**

| PROTOCOL AMENDMENT SUMMARY OF CHANGES TABLE | <mark>2</mark> |
|---|---|
| TABLE OF CONTENTS | 3 |
| LIST OF IN-TEXT TABLES AND FIGURES | 6 |
| 1. PROTOCOL SUMMARY | 7 |
| 1.1. Synopsis | |
| 1.2. Schema | |
| 1.3. Schedule of Activities | |
| 1.3.1. Schedule of Activities - Screening and Study Intervention Phase | |
| 1.3.2. Schedule of Activities - Follow-up Phase | |
| 1.3.3. Schedule of Activities – Optional PegIFN-α2a Treatment | |
| 2. INTRODUCTION | |
| 2.1. Study Rationale | |
| 2.2. Background | |
| 2.2.1. Nonclinical Studies | |
| 2.2.1.1. JNJ-3989 and JNJ-6379 | 41 |
| 2.2.1.2. Combination of JNJ-3989 or JNJ-6379 with Entecavir, Tenofovir Disoproxil, or Tenofovir Alafenamide | 46 |
| 2.2.1.3. Combination of JNJ-3989 with PegIFN-α2a | |
| 2.2.1.4. Combination of JNJ-6379 with PegIFN-α2a | |
| 2.2.2. Clinical Studies | |
| 2.2.2.1. JNJ-3989 and JNJ-6379 | |
| 2.2.2.2. Combination of JNJ-3989 and JNJ-6379 with Entecavir, Tenofovir Disoproxil, or Tenofovir Alafenamide | |
| 2.2.2.3. Combination of JNJ-3989 and JNJ-6379 with PegIFN-α2a | 54 |
| 2.3. Benefit-Risk Assessment | |
| 2.3.1. Benefits for Study Participation | |
| 2.3.1.1. Known Benefits | |
| 2.3.1.2. Potential Benefits | |
| 2.3.2. Risks for Study Participation | |
| 2.3.2.1. Known Risks | |
| 2.3.2.2. Potential Risks | |
| 2.3.2.2.1. Potential Risks for JNJ-3989 | |
| 2.3.2.2.2. Potential Risks for JNJ-6379 | 59 |
| 2.3.2.2.3. Potential Risks for Tenofovir Disoproxil and PegIFN-α2a | 61 |
| 2.3.2.3. Risks Due to Study Procedures | 61 |
| 2.3.2.3.1. Potential Risks and Inconvenience Associated with the Liver Biopsy Procedures | 61 |
| 2.3.2.3.2. Potential Risks and Inconvenience Associated with the Optional Leukapheresis Procedure | 62 |
| 2.3.3. Benefit-risk Assessment for Study Participation | |
| 3. OBJECTIVES AND ENDPOINTS | 64 |
| 4. STUDY DESIGN | |
| 4.1. Overall Design | |
| <ul><li>4.2. Scientific Rationale for Study Design</li></ul> | |
| 4.2.1. Study-Specific Ethical Design Considerations | |
| 4.3.1. JNJ-3989 | |
| 4.3.2. JNJ-6379 | |
| 4.4. End of Study Definition | |
| 5. STUDY POPULATION | 76 |

| 5.1. | Inclusion Criteria | |
|---|---|---|
| 5.2. | Exclusion Criteria | |
| 5.3. | Lifestyle Considerations | |
| 5.4. | Screen Failures | 84 |
| 6. S | TUDY INTERVENTION | 85 |
| 6.1. | Study Intervention(s) Administered | 85 |
| 6.2. | Preparation/Handling/Storage/Accountability | |
| 6.3. | Measures to Minimize Bias: Randomization and Blinding | |
| 6.4. | Study Intervention Compliance | |
| 6.5. | Concomitant Therapy | |
| 6.6. | Dose Modification | |
| 6.6.1. | Study Intervention Completion at Week 48 | ๋อง |
| 6.6.2. | | |
| 6.7. | NA Re-treatment Criteria and Monitoring after Stopping of NA Study Intervention After the End of the Study | |
| 0.7. | Study Intervention After the End of the Study | . 90 |
| | ISCONTINUATION OF INVESTIGATIONAL INTERVENTION AND PARTICIPANT | |
| | ISCONTINUATION/WITHDRAWAL | |
| 7.1. | Discontinuation of Study Intervention | |
| 7.2. | Participant Discontinuation/Withdrawal From the Study | |
| 7.2.1. | Withdrawal From the Use of Research Samples | |
| 7.3. | Lost to Follow-up | 99 |
| 8. S | TUDY ASSESSMENTS AND PROCEDURES | 99 |
| 8.1. | Liver Biopsy and Fine Needle Aspiration Biopsy | |
| 8.2. | Blood Efficacy Assessments | |
| 8.2.1. | Sequencing | |
| 8.3. | Blood Immune Assessments | |
| 8.3.1. | Peripheral Blood Mononuclear Cell Immune Analyses | |
| 8.3.2. | Leukapheresis (Optional With Separate Consent) | |
| 8.4. | Safety Assessments | |
| 8.4.1. | Physical Examinations | |
| 8.4.2. | Vital Signs | |
| 8.4.3. | Electrocardiograms | |
| 8.4.4. | Clinical Safety Laboratory Assessments | |
| 8.5. | Adverse Events and Serious Adverse Events | |
| 8.5.1. | Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event | 100 |
| 0.5.1. | InformationInformation | 107 |
| 8.5.2. | Method of Detecting Adverse Events and Serious Adverse Events | |
| 8.5.3. | Follow-up of Adverse Events and Serious Adverse Events | 100<br>100 |
| 8.5.4. | Regulatory Reporting Requirements for Serious Adverse Events | |
| 8.5.5.<br>8.5.6. | PregnancyAdverse Events of Special Interest | 100<br>100 |
| 8.5.6.1 | , | |
| 8.5.6.2 | | |
| 8.5.6.3 | · | |
| 8.5.6.4 | · | |
| 8.5.6.5 | | |
| 8.5.7. | Other Toxicities | |
| 8.5.7.1 | | |
| 8.5.7.2 | , | |
| 8.6. | Treatment of Overdose | |
| 8.7. | Pharmacokinetics | |
| 8.7.1. | Evaluations | |
| 8.7.2. | Analytical Procedures | 1 14<br>1 1 4 |
| 8.7.3. | Pharmacokinetic Parameters and Evaluations | |
| 8.8. | Pharmacokinetics/Pharmacodynamics | |
| 8.9. | Host Genetics | ı 14 |

| 8.10.<br>8.11. | Host Biomarkers | |
|---|---|---|
| 9. S | TATISTICAL CONSIDERATIONS | 115 |
| 9.1. | Statistical Hypotheses | |
| 9.2. | Sample Size Determination | |
| 9.3. | Populations for Analyses. | |
| 9.4. | Statistical Analyses | |
| 9.4.1. | Analysis of Efficacy and Antiviral Activity | |
| 9.4.1.1. | · | |
| 9.4.1.2. | | |
| 9.4.1.3. | Analysis of Exploratory Endpoints | 118 |
| 9.4.2. | Safety Analyses | |
| 9.4.3. | Other Analyses | |
| 9.5. | Interim Analysis | |
| 9.6. | Independent Flare Expert Panel | 122 |
| 10. S | UPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 122 |
| 10.1. | Appendix 1: Abbreviations and Definitions of Terms | |
| 10.2. | Appendix 2: Clinical Laboratory Tests | |
| 10.3. | Appendix 3: Regulatory, Ethical, and Study Oversight Considerations | 128 |
| REGUL | ATORY AND ETHICAL CONSIDERATIONS | 128 |
| FINANG | CIAL DISCLOSURE | 131 |
| | MED CONSENT PROCESS | |
| DATA F | PROTECTION | 132 |
| | TERM RETENTION OF SAMPLES FOR ADDITIONAL FUTURE RESEARCH | |
| COMM | ITTEES STRUCTURE | 133 |
| | CATION POLICY/DISSEMINATION OF CLINICAL STUDY DATA | |
| | QUALITY ASSURANCE | |
| | REPORT FORM COMPLETION | |
| | CE DOCUMENTS | |
| | ORING | |
| | E AUDITSRD RETENTION | |
| | AND SITE START AND CLOSURE | |
| 10.4. | Appendix 4: Adverse Events: Definitions and Procedures for Recording, Evaluating, | 130 |
| 10.4. | Follow-up, and Reporting | 140 |
| ADVER | RSE EVENT DEFINITIONS AND CLASSIFICATIONS | 140 |
| | BUTION DEFINITIONS | |
| SEVER | RITY CRITERIA | 141 |
| SPECIA | AL REPORTING SITUATIONS | 141 |
| | EDURES | |
| | ACTING SPONSOR REGARDING SAFETY | |
| | JCT QUALITY COMPLAINT HANDLING | |
| 10.5. | Appendix 5: Rash Management | 144 |
| 10.6. | Appendix 6: Intervention-emergent ALT/AST Elevations | |
| 10.7. | Appendix 7: Cardiovascular Safety Abnormalities | |
| 10.8. | Appendix 8: Contraceptive and Barrier Guidance and Collection of Pregnancy Information | |
| 10.9. | Appendix 9: DAIDS Table | |
| 10.10. | Appendix 10: Protocol Amendment History | |
| 10.11. | Appendix 11: Covid Appendix | 103<br>107 |
| 10.12. | Appendix 12. NA Re-freatment and Monitoring After Stopping of NA | 107 |
| 11. R | EFERENCES | 188 |
| INVES | TIGATOR AGREEMENT | 191 |

# **LIST OF IN-TEXT TABLES AND FIGURES**

# **TABLES**

| Table 1: | Various Stages of HBV Infection – Terminology and Characteristics (EASL 2017) <sup>5</sup> | |
|---|---|---|
| Table 2: | Animal/Human Exposure Ratios at NOAEL for JNJ-3989 | 42 |
| Table 3: | Animal/Human Ratios at the NOAEL in Rat and Dog (Human Exposure at 250 mg | |
| | JNJ-6379 Once Daily for 28 Days [Study 56136379HPB1001]) | 44 |
| Table 4: | Disallowed Medication | 92 |
| Table 5: | PegIFN-α2a Hematological Dose Modification Guidelines | 93 |
| Table 6: | Management of Rash Events by Severity Grade | 144 |
| FIGURES | <b>;</b> | |
| Figure 1: | Schematic Overview of the Study – Prior to Protocol Amendment 5 | 23 |
| Figure 2: | Schematic Overview of the Study – As of Protocol Amendment 5 | 24 |

## 1. PROTOCOL SUMMARY

# 1.1. Synopsis

A Phase 2 Randomized, Open-label, Parallel-group, Multicenter Study to Assess Intrahepatic and Peripheral Changes of Immunologic and Virologic Markers in Response to Combination Regimens Containing JNJ-73763989 and Nucleos(t)ide Analog With or Without JNJ-56136379 in Patients With Chronic Hepatitis B Virus Infection.

JNJ-73763989 (JNJ-3989) is a liver-targeted antiviral therapeutic for subcutaneous (SC) injection designed to treat chronic hepatitis B virus (HBV) infection via a ribonucleic acid interference (RNAi) mechanism. Engagement of the cellular RNAi machinery by JNJ-3989 results in specific cleavage of HBV ribonucleic acid (RNA) transcripts, thereby reducing the levels of HBV proteins and the pre-genomic RNA (pgRNA), the precursor of viral relaxed circular deoxyribonucleic acid (DNA). The RNAi triggers in JNJ-3989, JNJ-73763976 (JNJ-3976) and JNJ-73763924 (JNJ-3924), are designed to target all HBV RNA transcripts derived from covalently closed circular DNA (cccDNA), as well as transcripts derived from integrated viral DNA. The latter has been suggested to be a significant source of hepatitis B surface antigen (HBsAg) in hepatitis B e antigen (HBeAg) negative patients or patients on long term treatment with nucleos(t)ide analogs (NAs), the current standard of care.<sup>35</sup>

JNJ-56136379 (JNJ-6379) is an orally administered capsid assembly modulator (CAM) that is being developed for the treatment of chronic HBV infection. JNJ-6379 binds to hepatitis B core protein (HBc) and interferes with the viral capsid assembly process, thereby preventing the polymerase-bound pgRNA encapsidation. This results in the formation of HBV capsids, devoid of HBV DNA or RNA (non-functional capsids), and ultimately in the inhibition of HBV replication. In addition, JNJ-6379 also acts at an early stage of the viral life cycle by inhibiting the de-novo formation of cccDNA potentially by interfering with the capsid disassembly process. JNJ-6379 was initially part of the study intervention for participants but has been removed as study intervention with the implementation of an urgent safety measure, as described in Protocol Amendment 5.

Prior to Protocol Amendment 5: The term "study intervention" throughout the protocol, refers to JNJ-3989, JNJ-6379, NA, and optional PegIFN- $\alpha 2a^a$ .

As of Protocol Amendment 5: The term "study intervention" throughout the protocol, refers to JNJ-3989, NA, and optional PegIFN  $\alpha 2a$ .

#### **OBJECTIVES AND ENDPOINTS**

The study will be conducted in 3 phases for all participants: a screening phase (4 weeks), an open-label study intervention phase (48 weeks), and a follow-up phase (48 weeks). Note that the follow-up period will be extended for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation.

The following objectives and endpoints will be assessed overall and by study panel:

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess changes in intrahepatic HBsAg between baseline and on-treatment liver | |

<sup>&</sup>lt;sup>a</sup> Note: Optional PegIFN α2a was introduced as 'study intervention' as of Protocol Amendment 4.

| | Objectives | | Endpoints |
|---|---|---|---|
| | biopsy in response to JNJ-3989-based combination treatment | | |
| Sec | condary | | |
| • | To assess changes in intrahepatic immune response between baseline and on-treatment liver biopsy | • | Changes between baseline and on-treatment liver biopsy in intrahepatic immune response (eg, CD45+ T-cells, CD4+ T-cells, CD8+ T-cells, Natural Killer cells, and dendritic cells) in terms of proportion of cells, cell types, and spatial redistribution |
| • | To assess changes in intrahepatic viral nucleic acids and proteins between baseline and on-treatment liver biopsy | • | Changes from baseline in intrahepatic viral parameters (such as cccDNA, pgRNA, intrahepatic RNA, or HBsAg in terms of copy number, or number of positive cells) |
| | | • | Changes from baseline in intrahepatic cccDNA levels and transcriptional activity (pgRNA/cccDNA ratio) |
| • | To evaluate the efficacy of the study intervention as measured in blood | • | The proportion of participants during the study intervention and follow-up phases with: |
| | | | HBsAg seroclearance at Week 72 (ie, 24 weeks after completion of all study interventions at Week 48) without restarting NA treatment. |
| | | | (Sustained) Reduction, suppression, and/or seroclearance considering single and multiple markers (such as HBsAg, HBeAg, HBV DNA and ALT) |
| | | | HBsAg and HBeAg seroconversion |
| | | | Flares (virologic, biochemical, and clinical) |
| | | • | Time to first HBsAg seroclearance |
| • | To evaluate the frequency of virologic breakthrough during study intervention | • | Proportion of participants with virologic breakthrough |
| • | To assess HBV-specific T-cell responses | • | Changes from baseline in HBV-specific peripheral blood T-cell responses during the study intervention and follow-up phases |
| • | To evaluate the safety and tolerability of the study intervention | • | Proportion of participants with (S)AEs and abnormalities in clinical laboratory tests (including hematology, blood biochemistry, blood coagulation, urinalysis, urine chemistry, and renal biomarkers), 12-lead ECGs, vital signs, and physical examinations throughout the study |
| • | To evaluate the plasma PK of JNJ-3989 (ie, JNJ-3976 and JNJ-3924) and | • | Plasma PK parameters of JNJ-3976, JNJ-3924, and optionally of JNJ-6379, NA and PegIFN-α2a, as applicable |

| Objectives | Endpoints |
|---|---|
| optionally of JNJ-6379, NA and PegIFN- $\alpha$ 2a, as applicable | |
| Exploratory | |
| To explore the relationship of intrahepatic<br>markers with blood markers (immune and<br>viral) | Association between levels and changes in intrahepatic and blood markers |
| To explore the association of baseline characteristics and intrahepatic and/or blood (immune and viral) biomarkers at baseline and on/off-treatment with selected on/off-treatment efficacy variables | Association of baseline characteristics and baseline and on/off-treatment viral blood markers (such as baseline NA treatment duration, age, and baseline and on/off-treatment HBsAg levels) with selected off-treatment efficacy variables |
| | Association of intrahepatic and blood biomarkers<br>(such as cccDNA levels, T-cell frequency) with<br>selected on/off-treatment efficacy variables |
| To explore intrahepatic immune and viral<br>changes at Week 72 and/or during off-<br>treatment flares (only for participants with<br>Week 72 biopsy available) | • Changes from baseline and on-treatment liver biopsy in intrahepatic immune and viral markers at Week 72 and/or during off-treatment flares (only for participants with Week 72 biopsy available) |
| To explore changes in the severity of liver disease | Changes in fibrosis (according to Fibroscan liver stiffness measurements) at the end of study intervention (EOSI) and end of follow-up versus screening/baseline* |
| To explore the efficacy in terms of changes<br>in HBV RNA and hepatitis B core-related<br>antigen (HBcrAg) levels. | Changes from baseline in HBV RNA and HBcrAg levels during study intervention and follow-up phases. |
| • To explore the relationship between plasma PK parameters (JNJ-3989 [ie, JNJ-3976 and JNJ-3924] and/or JNJ-6379 and/or NA and/or PegIFN-α2a) and selected pharmacodynamic (PD) parameters of efficacy and/or safety, as applicable | • Relationship between various plasma PK parameters (JNJ-3976 and JNJ-3924, and/or JNJ-6379, and/or NA, and/or PegIFN-α2a) and selected efficacy and/or safety endpoints, as applicable |
| To explore the HBV genome sequence | The emergence of intervention-associated<br>mutations during the study intervention and<br>follow-up phases |
| | To assess the impact of baseline HBV genome<br>polymorphisms on selected on/off-treatment<br>efficacy variables |

<sup>\*</sup> Only applicable to participants who are enrolled at a site with an on-site Fibroscan device.

# **Hypothesis**

As this is an exploratory study, no hypothesis will be tested.

#### **OVERALL DESIGN**

As of Protocol Amendment 5, this study is a Phase 2 single-arm, open-label, multicenter, study to assess intrahepatic and peripheral changes of immunologic and virologic markers in response to a combination regimen containing JNJ-3989 and NA in chronic HBV-infected participants.

With the implementation of an urgent safety measure, as described in Protocol Amendment 5, JNJ-6379 has been removed as study intervention and the study will continue as a single-arm study. Participants randomized to Arm 1 had to stop JNJ-6379 treatment immediately but continue JNJ-3989 + NA treatment.

In addition, participants who provide separate consent may receive optional treatment with PegIFN- $\alpha$ 2a starting after the Week 40 biopsy (or after the optional leukapheresis if applicable) but before the Week 48 visit. The duration (either 12 or 24 weeks) will be at the investigator's discretion.

A target of 24 chronic HBV-infected male and female participants, 18-65 years (inclusive) of age will be enrolled in 2 panels, approximately 12 participants in each panel. Panel 1 will consist of participants who are HBeAg positive and not currently treated and Panel 2 will consist of participants who are HBeAg negative and virologically suppressed by entecavir (ETV), tenofovir disoproxil, or tenofovir alafenamide (TAF) treatment.

The study will be conducted in 3 phases for all participants: a screening phase (4 weeks), an open-label study intervention phase (48 weeks), and a follow-up phase (48 weeks). If necessary, eg, for operational reasons, the screening phase may be extended up to a maximum of 6 weeks on a case-by-case basis and in agreement with the sponsor. The duration of individual participation will be up to 102 weeks. Note that the follow-up period will be extended for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation. For those participants, the duration of individual participation may be extended up to 126 weeks.

Prior to Protocol Amendment 5, participants were randomized in a 1:1 ratio within each panel to receive one of the following interventions (ie, treatments) for 48 weeks:

• Intervention arm 1, combination regimen JNJ-3989+JNJ-6379+NA (target of 12 participants):

200 mg JNJ-3989 (SC injection once every 4 weeks [Q4W], with the last injection at Week 44), AND

250 mg JNJ-6379 (tablets once daily [qd]), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

• Intervention arm 2, combination regimen JNJ-3989+NA (target of 12 participants):

200 mg JNJ-3989 (SC injection O4W, with the last injection at Week 44), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

As of Protocol Amendment 5:

• Participants who were randomized to study intervention with JNJ-6379 prior to Protocol Amendment 5, had to stop JNJ-6379 treatment immediately but will still receive the following interventions (ie, treatments) for 48 weeks:

200 mg JNJ-3989 (SC injection Q4W, with the last injection at Week 44), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

• New participants will enroll without randomization within each panel to receive the combination regimen JNJ-3989 + NA as study intervention for 48 weeks:

200 mg JNJ-3989 (SC injection Q4W, with the last injection at Week 44), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

For participants who consented to receive optional PegIFN- $\alpha$ 2a, the PegIFN- $\alpha$ 2a treatment will be completed after 12 or 24 weeks at the investigator's discretion.

All participants will complete treatment with JNJ-3989 after a fixed duration of 48 weeks. If the NA treatment completion criteria (see "Study Intervention Completion at Week 48") are met based on clinical laboratory tests performed at Week 44, treatment with NA will also be completed at Week 48. In participants not meeting these criteria, NA treatment will continue during the follow-up phase. Participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who have not met NA treatment completion criteria at Week 48 may have NA treatment completion criteria assessed at the end of treatment with PegIFN- $\alpha$ 2a and stop NA if criteria are met.

All participants will have sparse PK sampling on Day 1 and at Weeks 4, 12, and 24 (and at early withdrawal). All participants who consent to participate in the intensive PK substudy (optional) will undergo intensive PK sampling at Week 4.

All participants will be monitored closely during the follow-up phase and, if applicable, should restart NA treatment in accordance with the NA re-treatment criteria mentioned below.

Prior to Protocol Amendment 5, randomization within each panel was stratified by Fibroscan score (<7 kPa vs ≥7 kPa). Randomization and stratification are not applicable anymore per Protocol Amendment 5.

A participant will be considered to have completed the study if he or she has completed the assessments at Follow-up Week 48. The follow-up phase will be extended by 24 weeks (ie, up to Follow-up Week 72) for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA + PegIFN- $\alpha$ 2a.

An Independent Flare Expert Panel (IFLEP) will be appointed for this study.

### **Study Intervention Completion at Week 48**

Participants will complete treatment with JNJ-3989 after a fixed duration of 48 weeks. If all of the below criteria are met based on clinical laboratory tests performed at Week 44, treatment with NA will also be completed at the next scheduled visit (ie, Week 48):

- The participant has ALT <3x upper limit of normal (ULN), AND
- The participant has HBV DNA < lower limit of quantification (LLOQ), AND
- The participant is HBeAg negative, AND
- The participant has HBsAg <10 International Units Per Milliliter (IU/mL).

**Note:** In case of ALT elevation  $\ge 3x$  ULN at Week 44 the investigator must consider different potential causes of increased ALT to ensure appropriate work up and management as needed. If the ALT elevation is unrelated to HBV activity and/or <3x ULN by Week 48, NA completion may be considered at the discretion of the investigator and in consultation with the sponsor.

Participants who do not meet the above criteria at Week 48 should continue NA treatment during the 48-week follow-up phase. Participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who have not met NA treatment completion criteria at Week 48 may have NA treatment completion criteria assessed at the end of treatment with PegIFN- $\alpha$ 2a and stop NA if criteria are met. The follow-up phase will be extended up by 24 weeks (ie, up to Follow-up Week 72) for participants who are receiving optional

treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA + PegIFN- $\alpha$ 2a.

## NA Re-treatment Criteria and Monitoring After Stopping of NA

Participants who meet the NA treatment completion criteria (as described above) will be monitored closely during the follow-up phase.

After stopping NA treatment, participants should be monitored as follows:

- Regular monitoring visits will be every 4 weeks during the follow-up phase in accordance with the schedule of activities.
- A post-treatment HBV DNA value of >20,000 IU/mL should trigger re-testing of ALT/AST, HBV DNA, and total and direct bilirubin within a maximum of 7 days from receipt of the data and further repeats as necessary (ie, weekly until HBV DNA returns to <20,000 IU/mL).
- A post-treatment HBV DNA value of >2,000 IU/mL (but <20,000 IU/mL) should trigger a re-test within 14 days from receipt of the data and further repeats as necessary (ie, every other week until HBV DNA returns to <2,000 IU/mL).
- A post-treatment ALT value of >5x ULN should trigger re-testing of ALT, AST, ALP, total and direct bilirubin, international normalized ratio (INR), albumin, and HBV DNA on a weekly basis until ALT and AST levels have returned to <5x ULN.

After stopping NA treatment, participants should re-start NA treatment:

- Immediately with signs of decreasing liver function based on laboratory findings (eg, INR, direct bilirubin) or clinical assessment (eg, ascites, hepatic encephalopathy).
- Immediately with an HBV DNA value of >100,000 IU/mL (irrespective of confirmation and/or ALT increase).
- With confirmed post-treatment HBeAg seroreversion (HBeAg positive after it was negative at NA completion)
- With confirmed\* post-treatment increases in HBV DNA >2,000 IU/mL and ALT >5x ULN
- With confirmed\* post-treatment increases in HBV DNA >20,000 IU/mL.
- \* At least 4 weeks apart frequency of visits as described above

*Note:* Additional re-testing and/or earlier restarting of NA treatment is at the investigator's discretion, even if the above cut-offs are not yet met.

To avoid delays in decision making, sites are encouraged to run local re-testing in parallel with central retesting in the situations described above that require more frequent re-testing. Local test results are to be recorded in the CRF and/or source documents, including information on the HBV DNA assay used. In addition, to avoid delays in NA re-treatment, it should be considered to dispense NA to participants who potentially met the NA re-treatment criteria (eg, pending confirmation) and who will not be available to come to the study site immediately at the time the confirmatory test results will become available. This should ensure that the participant can immediately restart NA treatment if indicated, upon direct confirmation by the investigator.

In case NA treatment is re-started, participants will be followed until the end of the study or until clinical stabilization, whichever comes later.

NA re-treatment criteria during follow-up are presented graphically in Section 10.12, Appendix 12: NA Re-treatment During Follow-up.

# NUMBER OF PARTICIPANTS

A target of 24 chronic HBV-infected adult male and female participants will be randomized or enrolled.

# **Description of Interventions**

Status: Approved, Date: 25 November 2021

| Intervention name | JNJ-3989 | JNJ-6379**** | PegIFN-α2a | Entecavir (ETV)<br>monohydrate | Tenofovir<br>disoproxil | Tenofovir<br>alafenamide (TAF)* |
|---|---|---|---|---|---|---|
| Туре | Drug | Drug | Drug | Drug | Drug | Drug |
| Dosage | Solution for | Tablets | Solution for | Film-coated tablets | Film-coated tablets | Film-coated tablets |
| formulation | injection | | injection | | | |
| Unit dose | 200 mg/vial | 25 and 100 mg | 180 μg/0.5 mL | 0.5 mg | 245 mg | 25 mg |
| strength(s) | | | | | | |
| Dosage level | 200 mg once every | 250 mg once daily | 180 μg once weekly | Nucleoside-naïve patients: | 245 mg qd | 25 mg qd |
| | 4 weeks (Q4W) | (qd) | (QW)** | 0.5 mg qd | | |
| | | | | <u>Lamivudine-refractory</u> | | |
| | | | | patients: | | |
| | | | | 1 mg* qd (but should<br>preferably be treated with<br>tenofovir disoproxil or<br>TAF instead) | | |
| | | | | Other indications: | | |
| | | | | 1 mg* qd (must be agreed upon by the sponsor) | | |
| Route of administration | Subcutaneous injection preferably in the abdomen | Oral | Subcutaneous<br>injection (in the<br>thigh or abdomen) | Oral | Oral | Oral |
| Use | Investigational | Investigational | Investigational | Background intervention | Background | Background |
| | intervention | intervention | intervention | | intervention | intervention |
| Sourcing | Provided centrally | Provided centrally | Provided centrally | Provided centrally by the | Provided centrally | Provided centrally |
| | by the sponsor | by the sponsor | by the sponsor*** | sponsor | by the sponsor | by the sponsor |
| Packaging and | Each unit will be | Each unit will be | Commercial | Commercial supplies will | Commercial supplies | Commercial supplies |
| Labeling | labeled with unique | labeled with unique | supplies will be | be sourced. Each unit will | will be sourced. | will be sourced. |
| | medication ID | medication ID | sourced. Each unit | be labeled with unique | Each unit will be | Each unit will be |
| | number | number | will be labeled with | medication ID number | labeled with unique | labeled with unique |
| | | | unique medication | | medication ID | medication ID |
| | | | ID number*** | | number | number |
| | | In child-resistant | In child-resistant | In child-resistant | In child-resistant | In child-resistant |
| | | packaging | packaging*** | packaging | packaging | packaging |
| | | Labels will c | contain information to m | neet the applicable regulatory | requirements. | |

 $CONFIDENTIAL-FOIA\ Exemptions\ Apply\ in\ U.S.$ 

| Intervention name | JNJ-3989 | JNJ-6379**** | PegIFN-α2a | Entecavir (ETV)<br>monohydrate | Tenofovir<br>disoproxil | Tenofovir<br>alafenamide (TAF)* |
|---|---|---|---|---|---|---|
| Food/Fasting | Regardless of food | Regardless of food | Per the prescribing | Per prescribing | Per prescribing | Per prescribing |
| instructions | intake | intake | information | information | information | information |

Q4W: once every 4 weeks; qd: once daily; QW: once weekly

In countries where TAF is available, it will be one of the NA treatment options.

For PegIFN α2a, dose adjustment may be applicable for participants who develop laboratory abnormalities during PegIFN α2a treatment.

May vary based on local regulations.

Participants enrolled before Protocol Amendment 5 was in effect, may have received JNJ 6379 as part of their study intervention. As of Protocol Amendment 5: study intervention includes JNJ 3989, NA and optionally PegIFN α2a.

#### LIVER BIOPSY AND FINE NEEDLE ASPIRATION BIOPSY

Percutaneous core liver biopsies and fine needle aspiration biopsies (FNABs) will be performed at Week -1 and Week 40. If participants agree to undergo an additional optional liver biopsy, FNAB and/or core liver biopsy samples may be taken at the selected location at Follow-up Week 24 or at the time points clinically indicated.

Following local standard practice the biopsy location will be identified with ultrasound (which will also be used to rule out contraindicating conditions for a biopsy) and after application of local anesthesia the FNAB samples and core liver biopsy samples will be collected.

The liver biopsy procedure should be preceded and followed by standard medical monitoring according to local medical practice. This may include an overnight stay at the investigator's discretion. The use of low-dose aspirin is allowed with exception of 7 days prior to biopsies (see Section 6.5).

The liver tissue will be used to assess HBsAg. Changes from baseline in the proportion of HBsAg positive hepatocytes under therapy will be assessed.

In addition, the liver tissue may also be used to assess other HBV markers in the liver such as, but not limited to, total intracellular HBV RNA and DNA, HBeAg, and HBc. Changes in the quantity and potentially changes in the spatial distribution of these markers (including HBsAg) under therapy may be assessed. Viral genome (RNA or DNA) or transcript sequencing/analyses as well as assessment of HBV integrants in the host genome may be performed.

Intrahepatic immune status at baseline and response to treatment will be assessed. Both innate and adaptive immune compartment will be characterized, by measuring the relative number of specific cells and the expression of functional markers in each cell population using various single cell approaches, such as single cells transcriptomics in FNABs and Immunofluorescence staining, and transcriptomics and proteomics profiling in core needle biopsies. Depending on the latest platform developments (spatial transcriptomics, *in situ* sequencing approaches, etc.), methods for immune cells characterization might be adjusted.

Hepatitis B virus-specific T-cells, although very rare in FNABs, may be characterized and counted by multimers binding assays, staining and sorting for positive cells. Downstream profiling of collected HBV-specific T-cells may be performed by T-cell receptor sequencing and RNA sequencing.

Infiltrating immune cells will be used for the evaluation of innate and adaptive immune responses, which can be compared to responses in peripheral blood mononuclear cell (PBMCs).

Hepatitis B virus cccDNA levels may be assessed using quantitative polymerase chain reaction (qPCR) methods on a single cell level using laser capture microdissection or bulk analyses. The exact protocol of cccDNA measurement will be determined based on the latest method available considering the performance characteristics and the validation status of the assay. Southern Blot-based methods or novel methods for cccDNA detection (eg, fluorescent in situ hybridization [FiSH]) might be used depending on the availability of sample and established methodology. Quantification of intracellular pre-genomic HBV RNA can be used to determine transcriptional activity of HBV cccDNA by assessing the ratio of pgRNA levels over cccDNA levels.

Immune and virologic markers in the liver and/or changes thereof on-treatment will be used to assess association with blood markers and/or treatment response and outcome.

Remaining samples may be used for determination of liver JNJ-3989 (ie, JNJ-3976 and JNJ-3924) and/or JNJ-6379 concentrations and/or research on viral and host biomarkers and immune markers at the viral and/or host RNA/DNA, protein, and cell level.

#### **BLOOD EFFICACY ASSESSMENTS**

Qualitative and quantitative HBsAg and HBeAg, and quantitative HBcrAg as well as antibodies against HBsAg and HBeAg will be determined using validated serologic assays in a central laboratory. Samples for the determination of HBsAg and HBeAg will be processed in real-time. Samples for the determination of HBcrAg can be analyzed in batch and at the sponsor's discretion.

Hepatitis B virus DNA and HBV RNA will be quantified at central laboratories using validated assays for the quantification of HBV DNA and HBV RNA. Samples for the determination of HBV DNA will be processed in real-time. Samples for the determination of HBV RNA can be analyzed in batch and at the sponsor's discretion.

Hepatitis B virus DNA, HBsAg, HBeAg, anti-HBs, and anti-HBe antibody testing results will be provided to the investigator and the sponsor from screening until the end of follow-up.

In participants enrolled at a site with an on-site Fibroscan device, Fibroscan assessments will be performed to determine changes in fibrosis levels.

Samples may be used by the sponsor for additional exploratory assessments analyzing the serologic and virologic characteristics of HBV infection and efficacy or safety of the study intervention.

Viral genome sequence analysis will be performed to identify pre-existing baseline polymorphisms and to evaluate emergence of mutations associated with JNJ-3989, and/or JNJ-6379, and/or NA treatment.

#### **BLOOD IMMUNE ASSESSMENTS**

#### Peripheral Blood Mononuclear Cell Immune Analyses

Samples for PBMC immune analyses will be collected during the study intervention and follow-up phases and will be analyzed centrally for HBV-specific responses by enzyme-linked immunospot (ELISpot) and/or intracellular cytokine staining (ICS) after stimulation with HBV-specific antigens. ELISpot detects T-cells that secrete gamma interferon (IFN- $\gamma$ ) in response to a specific antigenic stimulation, whereas ICS determines the frequency of CD4+ and CD8+ T-cells secreting cytokines such as IFN- $\gamma$ , interleukin (IL)-2 and tumor necrosis factor (TNF)- $\alpha$  in response to a specific antigenic stimulation. Hepatitis B virus-specific T-cells may be characterized in PBMCs by binding assays (multimer staining) combined with downstream TCR and transcriptome profiling.

Additional experiments may be performed to further phenotypically and functionally characterize PBMCs using proliferation or cytotoxic assays or other methods such as cytometry by time of flight to evaluate innate and adaptive immune responses. Leftover samples may be used at the sponsor's discretion for additional exploratory research related to HBV infection or study intervention (safety/efficacy).

Additional PBMC samples may be taken in case of ALT flares, upon discussion with the sponsor, which may require an unscheduled visit.

## **Leukapheresis (Optional With Separate Consent)**

Leukapheresis allows to selectively collect higher quantities of PBMCs from participants without withdrawing large volumes of blood.

Leukapheresis will only be performed for participants who consent separately to this component of the study. Participants may withdraw such consent at any time without affecting their participation in other aspects of the study.

Leukapheresis may be done at least 1 week (and up to 3 weeks) after the liver biopsies (see Schedule of Activities). Prior to the procedure, the participant's wellbeing will be checked and leukapheresis will only

be offered if there is no clinical reason against it. If a participant has had a recent febrile illness, the leukapheresis should be postponed until body temperature is normal for at least 72 hours.

The leukapheresis procedure should mainly follow local standard procedures. Additional guidelines will be provided via a separate manual in order to standardize this process across sites.

One leukapheresis session is expected to last between 1.5 - 5 hours.

During the procedure, the participant will receive intravenous saline infusions and citrate-based anticoagulant. Use of heparin for anticoagulation is not allowed. A specialized leukapheresis trained research nurse or physician will be in attendance and in charge of the participant's immediate medical care to monitor the leukapheresis.

After completion of the leukapheresis procedure, participants will stay at the site for at least 30 minutes to monitor for any relevant safety events. Additional safety procedures may be performed at the discretion of the site staff. Participants are advised to refrain from exercise and strenuous activities for 3 day after the leukapheresis visit.

### **SAFETY EVALUATIONS**

Safety and tolerability will be assessed throughout the study from the time that the informed consent form is signed until completion of the last study-related activity, which may include contact for follow-up of safety. The evaluations of safety and tolerability will include monitoring of (S)AEs, physical examinations (including body weight), vital signs measurements, triplicate 12-lead ECGs, and clinical laboratory tests (including hematology, blood biochemistry, blood coagulation, urinalysis, urine chemistry, and renal biomarkers). Any clinically relevant changes occurring during the study must be recorded in the AE section of the case report form.

Specific toxicity management plans in line with the known pharmacological profile of the study intervention (and the drug classes) evaluated in this study are implemented.

#### PHARMACOKINETIC EVALUATIONS

Venous blood samples will be collected for measurement of plasma concentrations of JNJ-3989 (ie, JNJ-3976 and JNJ-3924), NA (ETV, TAF, or tenofovir) and PegIFN- $\alpha$ 2a, as applicable, at time points specified in the Schedule of Activities. Bioanalysis of NA and PegIFN- $\alpha$ 2a is optional at the discretion of the sponsor. Bioanalysis of JNJ-6379 may also be done on samples collected from participants who received JNJ-6379 up to Protocol Amendment 4.

All participants will have sparse PK sampling on Day 1 and at Weeks 4, 12, and 24 (and at early withdrawal). All participants who consent to participate in the intensive PK substudy (optional) will undergo intensive PK sampling at Week 4. If necessary (eg, for operational reasons), this visit may be scheduled at Week 8, 12, or 16.

Plasma concentration-time data for JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a will be analyzed via noncompartmental methods for all participants who underwent intensive PK sampling. The main PK parameter will be area under the plasma concentration-time curve over 24 hours (AUC<sub>24h</sub>),  $C_{max}$ ,  $t_{max}$ , plasma trough concentration ( $C_{0h}$ ), plasma concentration at the end of the dosing interval ( $\tau$ ) ( $C_{\tau}$ ), and minimum plasma concentration ( $C_{min}$ ). Additional exposure parameters may be calculated if applicable.

Data from this study may be combined with data from a selection of Phase 1 and 2 studies via population PK modelling. Individual estimates of PK parameters may be generated from the population PK analysis for potential use in exposure-response analysis.

#### PHARMACOKINETIC/PHARMACODYNAMIC EVALUATIONS

Relationships of individual PK parameters for JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a, with selected liver and blood biomarkers, and/or with selected safety endpoints may be evaluated.

### **HOST GENETICS**

A pharmacogenomic blood sample will be collected (preferably at baseline) to allow for the identification of genetic factors that may influence the efficacy, safety, or PK of the study intervention, to identify genetic factors associated with HBV infection, or to develop assays for the study intervention or HBV infection.

A blood sample will be taken for human leukocyte antigen (HLA) typing. In addition, host DNA blood samples to allow for epigenetic analyses will be collected.

#### HOST BIOMARKERS

The study includes collection of blood samples for exploratory analysis of host blood biomarkers at the host RNA, protein, and cell level.

Samples can only be used for research related to study intervention or HBV infection or may be used to develop tests/assays related to study intervention or HBV infection.

Blood samples will be taken that can be used to explore immunogenicity of JNJ-3989. The emergence of antibodies to JNJ-3989 (antidrug antibodies) might be analyzed using assays such as an enzyme-linked immunosorbent assay.

#### STATISTICAL METHODS

The primary analysis will be performed at the time when all participants have completed Week 48 or discontinued earlier. The final analysis will be performed when all participants have completed the last study visit (Follow-up Week 48) or discontinued earlier.

Given the exploratory nature of the study and the limited sample size per intervention arm per panel, no statistical testing will be performed. All data will be summarized descriptively including 90% confidence intervals as appropriate.

# **Statistical Hypotheses**

As this is an exploratory study, no hypothesis will be tested.

#### **Sample Size Determination**

This study aims to enroll 18 to 24 participants in total across Panels 1 and 2, ie, 8 to 12 participants per study panel. Due to the exploratory nature of the study, the sample size was determined based on clinical and feasibility considerations related to the liver biopsy procedures performed multiple times during the study, rather than a formal statistical calculation.

#### **Analyses of Efficacy and Antiviral Activity**

To evaluate the efficacy and antiviral activity in blood and liver, the primary analysis set will be the intent-to-treat (ITT) population.

All efficacy summaries will be presented with descriptive statistics, overall and by study panel.

If the endpoint is continuous, the descriptive statistics will include the number of participants, mean, standard deviation (SD), median, range, and interquartile range. If the endpoint is binary or categorical, the frequency distribution with the number and percentage of participants in each category will be calculated.

Graphic displays will also be used to summarize the data and to visualize trends by study panel.

Where applicable, additional specifics for analyses of primary, secondary, and exploratory endpoints are detailed below.

Analysis of the Primary Endpoint

The primary endpoint is the change between baseline and on-treatment liver biopsy (Week 40) in terms of the proportion of HBsAg-positive hepatocytes. The primary endpoint will be summarized descriptively and modelled with an appropriate statistical model accounting for the number of hepatocytes sampled in each liver biopsy. The change from baseline will be summarized for the overall study population and within each panel, together with the between-panel difference in the change.

Analysis of Secondary Endpoints

## Changes in Intrahepatic Immune Response

Variation in proportion of major cell populations, such as but not limited to CD4+ T-cells, CD8+ T-cells, CD45+ T-cells, Natural Killer cells, and dendritic cells, defined by single cell transcriptomics (in FNABs) and immunofluorescence staining (in core needle biopsies), will be assessed at Week 40 and compared to baseline, overall and by study panel.

The functional characterization of major cell populations will be assessed by transcriptomics and/or proteomics for major cell populations of interest at Week 40 and compared to baseline similarly.

### Changes in Intrahepatic Viral Nucleic Acids and Proteins

Changes from baseline in cccDNA level and/or transcriptional activity will be assessed using the general considerations outlined above.

Furthermore, the difference in the level of infected hepatocytes at baseline will be assessed by comparing cccDNA level and/or transcriptional activity.

Analyses of other viral markers will be performed descriptively. Statistical analyses will depend on the assay technology applied and the scope of the analyses.

Analysis of Exploratory Endpoints

The association between intrahepatic markers and blood (immune and viral) markers will be explored both at baseline and on-treatment by study panel using graphical displays and relevant correlation coefficients.

Impact of baseline characteristics on selected efficacy variables and their association with intrahepatic and blood markers will also be evaluated using similar methods.

Identification of markers (either intrahepatic or blood) that could potentially be associated with selected efficacy variables (such as decrease in blood HBsAg levels, intrahepatic cccDNA levels or any other relevant variables) will be conducted. Impact of treatment on different blood and hepatic markers will also be evaluated.

#### **Safety Analyses**

The Safety Population will be used for all safety analyses and includes all participants who received at least one dose of study intervention.

Safety will be evaluated by means of descriptive summaries of AEs including AEs of special interest to any of the study interventions, clinical laboratory tests, ECGs, vital signs, and physical examinations. The safety

analysis will be done by study phase. Results will be presented in tabular format and/or graphically over time, as appropriate.

# Other Analyses

### Pharmacokinetic Analyses

Descriptive statistics (number of participants, mean, SD, coefficient of variation, geometric mean, median, minimum, and maximum) will be calculated for the plasma concentrations of JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a, as applicable, and for the derived plasma PK parameters (noncompartmental analysis).

Special attention will be paid to the plasma concentrations and PK parameters of those participants who discontinued the study for an AE, or who experienced an AE ≥grade 3 or an SAE.

For each participant with intensive PK sampling, plasma concentration-time data of JNJ-3976, JNJ-3924, and/or JNJ-6379, and/or NA and/or PegIFN- $\alpha$ 2a will be graphically presented. Similarly, graphs of the mean plasma concentration-time profiles and overlay graphs with combined individual plasma concentration time profiles will be produced. Pharmacokinetic parameters will be subjected to an exploratory graphical analysis, including various transformations, to get a general overview.

Population PK analysis of plasma concentration-time data JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN-α2a may be performed using nonlinear mixed-effects modeling. Data may be combined with those from Phase 1 and/or 2 studies to support a relevant structural model. Available baseline characteristics (eg, demographics, laboratory variables, genotypes) may be included in the model as necessary. Details will be given in a population PK analysis plan and results of the population PK analysis, if applied, will be presented in a separate report.

Individual estimates of PK parameters may be generated from the population PK analysis for potential use in exposure-response analysis.

#### Pharmacokinetic/Pharmacodynamic Analyses

Relationships of PK parameters for JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a with selected efficacy and with selected safety endpoints may be evaluated and graphically displayed.

Modeling of key PD parameters (eg, HBsAg, HBV DNA) may be performed using population PK/PD. If PK/PD modeling of key efficacy endpoints is performed, treatment effect and possible covariates such as disease progression may be investigated. Other biomarkers may be explored at the sponsor's discretion.

#### Resistance Analysis

The results of HBV viral sequencing will be evaluated by the sponsor virologist. Relevant changes in amino acid and/or nucleic acid variations (eg., substitutions) in the HBV genome will be tabulated and described.

Additional exploratory characterization of the HBV viral sequence and phenotype may be performed and reported separately.

# Pharmacogenomic Analyses

The statistical approach for analyzing the exploratory host DNA research may depend on the objective of the analyses (efficacy, safety, and PK) and possibly relevant genes at the time of analysis. Analyses will be conducted at the sponsor's discretion, will always be under the sponsor's supervision, and results will be presented either in the clinical study report or a separate report.

## Host Exploratory Biomarker Analyses

Statistical approaches to explore associations between treatment response/clinical outcome and blood and liver biomarkers vary and depend on the different data types of the applied technology platforms, as well as on the extent of observed differences between participants. Analyses will be conducted at the sponsor's discretion, will always be under the sponsor's supervision, and results will be presented either in the clinical study report or a separate report.

#### **Interim Analysis**

Two interim analyses (IAs) may be performed: when all participants have completed Week 20 in the intervention phase (or discontinued earlier) and when they have completed Week 72 in the follow-up phase (ie, Follow-up Week 24) (or discontinued earlier). These IAs will be performed by the sponsor to support interactions with health authorities, as well as to support internal decisions about additional studies and/or investigation of other combination regimens.

Both primary and interim analyses will be based on all data available at the predefined cut-off time points and may include data at later time points for those participants who have reached subsequent visits.

## **Independent Flare Expert Panel**

An IFLEP will be appointed for this study. The IFLEP is composed of 3 independent medical experts with experience and expertise in hepatitis B and its treatment. The IFLEP will monitor ALT flares and will make recommendations regarding flare management based on an analysis of aggregate data.

In order to allow for an unbiased assessment, members of the IFLEP will not serve as study investigators.

Further details on the IFLEP process will be included in the IFLEP charter.

## 1.2. Schema

Figure 1: Schematic Overview of the Study – Prior to Protocol Amendment 5



ETV: entecavir; N: number of participants; LB: (planned) liver biopsy; NA=nucleos(t)ide analog; Q4W: once every 4 weeks; qd: once daily; TAF: tenofovir alafenamide; TD: tenofovir disoproxil; QW: once weekly

<sup>\*</sup> Participants who provide separate consent may receive optional treatment with PegIFN- $\alpha$ 2a starting after the Week 40 biopsy (or after the optional leukapheresis visit if applicable) for a duration of either 12 or 24 weeks at the investigator's discretion.

<sup>\*\*</sup> Treatment with JNJ-3989 (and JNJ-6379 if applicable) will be stopped at Week 48. Optional treatment with PegIFN-α2a will be stopped after 12 or 24 weeks (at the investigator's discretion). NA treatment may be stopped at Week 48 (or later for participants on PegIFN-α2a treatment) if NA treatment completion criteria are met.



Schematic Overview of the Study - As of Protocol Amendment 5 Figure 2:

ETV: entecavir; N: number of participants; LB: (planned) liver biopsy; NA=nucleos(t)ide analog; Q4W: once every 4 weeks; qd: once daily; TAF: tenofovir alafenamide; TD: tenofovir disoproxil; QW: once weekly

- \* Participants who provide separate consent may receive optional treatment with PegIFN-α2a starting after the Week 40 biopsy (or after the optional leukapheresis visit if applicable) for a duration of either 12 or 24 weeks at the investigator's discretion.
- \*\* Treatment with JNJ-3989 will be stopped at Week 48. Optional treatment with PegIFN-α2a will be stopped after 12 or 24 weeks (at the investigator's discretion). NA treatment may be stopped at Week 48 (or later for participants on PegIFN-α2a treatment) if NA treatment completion criteria are met.
- \*\*\* The follow-up phase will be extended for participants who are receiving optional treatment with PegIFN-α2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation.

Note: Former Arm 1 participants will now be joining Arm 2, both in terms of treatment assignment as well as how they will be statistically analyzed.

# 1.3. Schedule of Activities

Status: Approved, Date: 25 November 2021

# 1.3.1. Schedule of Activities - Screening and Study Intervention Phase

For additional visits and assessments in case of optional PegIFN- $\alpha$ 2a treatment, refer to Section 1.3.3.

| Phase | Scr | eening | | | | | | | 10 | Open-la | abel Stu | dy Inte | rventio | n <mark>a</mark> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | W 1 | | | | | | | | | | | | | | +/ W40 | j | | |
| Visit Day (D)/Week (W) | W 4<br>to 0 <sup>b</sup> | Biopsy | D1° | W2 | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | Pre<br>biopsy<br>Visit | Biopsy | Post<br>biopsy<br>Visit | W44 | W48/<br>WD <sup>d</sup> |
| Study Day (Window) | 28<br>to 1 | 7<br>to 1 | 1 | 15<br>(+/ 3d) | 29<br>(+/ 3d) | 57<br>(+/ 3d) | 85<br>(+/ 3d) | 113<br>(+/ 3d) | 141<br>(+/ 3d) | 169<br>(+/ 3d) | 197<br>(+/ 3d) | 225<br>(+/ 3d) | 253<br>(+/ 3d) | 281<br>(+/ 3d) | <7d Prior<br>to Biopsy | A CONTRACTOR | ≥1w ≤3w<br>After<br>Biopsy | 309<br>(+/ 3d) | 337<br>(+/ 3d) |
| Screening/Administrative | | | | | | | | | | | | | | | | | | 8 | |
| ICFe | X | | | | | | | | | | | | X X | X X | | | | | |
| ICF for optional liver biopsyf | (X) | | | | | | | | | | 3 | | 3 10<br>3 50 | 53 33<br>55 22 | | | | | |
| Inclusion/exclusion criteriag | X | X | | | | | | | | | | | S S | 2 3 | | | | | |
| Prestudy therapy (including prior anti HBV therapy) | X | | | | | | | | | | | | | | | | | | |
| Medical/surgical history and demographicsh | X | | | | | | | | | | | | | 33 33 | | | | | |
| Preplanned surgery/procedure(s) | X | | | | | | | | | | | | | | * | | | | |
| Fibroscan <sup>i,j</sup> | X | | | | | | | | | | | | | | | | | | (X) |
| Ultrasound | Xk | | | | | | | | ii<br>D | $X^1$ | 8 | | | | | | | | XI |
| Study Intervention | | | | | | | | | | | | | | | | | | | |
| Enrollment without randomizationpp | | | X | | | | | | | | | | | | | | | | |
| Administer JNJ 3989 | | | X | | X | X | X | X | X | X | X | X | X | X | | | | X | |
| Intake of NA <sup>n,</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Intake of JNJ 6379 <sup>n,o</sup> (stopped per Amendment 5) | | | X | | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Dispense NA (for at home use) <sup>n</sup> | | | X | | X | X | X | X | X | X | X | X | X | X | C. | | | X | (X)p |
| Dispense JNJ 6379 (stopped per<br>Amendment 5) n.o | | | X | | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Study intervention accountability | | | | | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Safety Assessments | | | | | | | | | | | | | | | | | | | |
| Complete physical examination <sup>q</sup> | X | | | | | | | | | X | | | | | | | | | X |
| Body weight and Symptom directed physical examination | | X | X | X | X | X | X | X | X | 2 | X | X | X | X | | | | X | |
| Vital signs <sup>r</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Phase | Scr | eening | | | | | | | 10 | Open-la | abel Stu | dy Inte | rventio | nª | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | W 1 | | | | | | | | | | | | | | +/ W40 | | | |
| Visit Day (D)/Week (W) | W 4<br>to 0 <sup>b</sup> | Biopsy | D1° | W2 | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | Pre<br>biopsy<br>Visit | Biopsy | Post<br>biopsy<br>Visit | W44 | W48/<br>WD <sup>d</sup> |
| Study Day (Window) | 28<br>to 1 | 7<br>to 1 | 1 | 15<br>(+/ 3d) | 29<br>(+/ 3d) | 57<br>(+/ 3d) | 85<br>(+/ 3d) | 113<br>(+/ 3d) | 141<br>(+/ 3d) | 169<br>(+/ 3d) | 197<br>(+/ 3d) | 225<br>(+/ 3d) | 253<br>(+/ 3d) | 281<br>(+/ 3d) | <7d Prior<br>to Biopsy | | ≥1w ≤3w<br>After<br>Biopsy | 309<br>(+/ 3d) | 337<br>(+/ 3d) |
| Triplicate 12 lead ECG <sup>s</sup> | X | | X | X | X | | X | | | X | Ĵ | ì | X | 08 80 | | | ~ | | X |
| Injection site reactions for JNJ 3989 | | | | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Clinical Laboratory Tests | | | | | | | | | | | | | | | | | | | |
| Hematology | X | | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>m</sup> | | | X | X |
| Blood chemistry (including liver function tests) <sup>t,u,v</sup> | X | | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Blood coagulation | X | | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>m</sup> | | | X | X |
| Urinalysis <sup>w</sup> | X | | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Urine chemistry <sup>x</sup> | X | | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Renal biomarkers <sup>y</sup> | | | X | | | | X | | | X | | | X | | | | | | X |
| Serum IgM anti HBc antibody test | X | | | | | | | | | | | | 3 3 | 2, 3 | | | | | |
| Testing for hepatitis A, B, C, D, and E virus,<br>HIV 1 and 2 | X | | | | | | | | | | | | | | | | | | |
| FSH test (postmenopausal women only) <sup>z</sup> | X | | | | | | | | 2 | | × | × | | | | | | | |
| AFP <sup>v</sup> | X | | | | | | | | | X | | | .15 | | | | | | X |
| Hemoglobin A1c | X | | | | | | | | | | | | | | | | | | |
| Serum pregnancy test (women of<br>childbearing potential only) | X | | | | | | | | | | | | | | | | | | |
| Urine pregnancy test (women of childbearing potential only) | | | X | | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| HBV genotype <sup>aa</sup> | | | X | | | | | | | | | | . X | | | | | | 14. |
| Liver Biopsy | | | | | | | | | | | | | | | | | | | |
| FNAB sample | | X <sup>m</sup> | | | | | | | | | | | 10 80 | 33 80 | | X <sup>m</sup> | | 3 | |
| Percutaneous core liver biopsy sample | | X <sup>m</sup> | | | | | | | 2 | | | | 8 | S8 83 | | X <sup>m</sup> | | | |
| Platelet aggregation test (local laboratory) | | | | | | | | | | | | | | | X <sup>m</sup> | | | | |
| Efficacy Assessments | | | | | | | | | | | | | | | | | | | |
| HBV Virology | | | | | | | | | | | | | | | | | | | |
| Blood sampling for HBV DNA | X | | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| Blood sampling for HBV RNAbb | X | | X | X | X | X | X | X | X | X | | X | | X | | | | X | X |

| Phase | Scr | eening | | | | | | | li) | Open-la | abel Stu | dy Inte | rventio | nª | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | W 1 | | | | | | | | | | | | | | +/ W40 | | | |
| Visit Day (D)/Week (W) | W 4<br>to 0 <sup>b</sup> | Biopsy | D1° | W2 | W4 | W8 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | Pre<br>biopsy<br>Visit | Biopsy | Post<br>biopsy<br>Visit | W44 | W48/<br>WD <sup>d</sup> |
| Study Day (Window) | 28<br>to 1 | 7<br>to 1 | 1 | 15<br>(+/ 3d) | 29<br>(+/ 3d) | 57<br>(+/ 3d) | 85<br>(+/ 3d) | 113<br>(+/ 3d) | 141<br>(+/ 3d) | 169<br>(+/ 3d) | 197<br>(+/ 3d) | 225<br>(+/ 3d) | 253<br>(+/ 3d) | | <7d Prior<br>to Biopsy | 281<br>(+/ 4w) | ≥1w ≤3w<br>After<br>Biopsy | 309<br>(+/ 3d) | 337<br>(+/ 3d) |
| Sampling for viral genome<br>sequencing <sup>cc</sup> | X | | X | | | | X | | | X | | X | .0 20 | X | | | | | X |
| HBV Serology | | | | | | | | | | | | | | | | | | | |
| Blood sampling for: | | | | | | | | | <i>3</i> | 2 | 3 | | | 10 (0)<br>10 (0) | | | | | |
| Anti HBs and anti HBe | X | | X | | | | | | | X | ~ | | 16 16 | 200 900 | | | | ec. | X |
| HBsAg (qualitative) | X | | | | | | | | | | | | | | | | | | X |
| HBeAg (qualitative) <sup>dd</sup> | X | | | | | | | | | X | | | | | | | | X | X |
| HBsAg (quantitative) | X | | X | X | X | X | X | X | X | X | X | X | X | X | | | | X | X |
| HBeAg (quantitative)ee | | | X | | (X) | (X) | (X) | | | (X) | | | | | | | | | (X) |
| HBcrAgbb | X | | X | | X | | X | | | X | | X | | X | | | | X | X |
| Exploratory serologyff | X | | X | X | X | X | X | X | X | X | 8 | X | | X | | | | X | X |
| Clinical Pharmacology<br>Assessments | | | | | | | | | | | | | | | * | | | | |
| Blood sampling for sparse PK of JNJ 3989, and NAgg | | | Xhh | | Xhh | | Xhh | | | Xhh | | | | | | | | | Xii |
| Blood sampling for intensive PK of JNJ 3989, and NA (PK substudy) <sup>ij</sup> | | | | | X | | | | | | | | | | | | | | |
| Exploratory Host Biomarkers | | | | | | | | | | | | | | | | | | | |
| Whole blood RNA gene expression | | | X | X | | | X | , | | X | | | | X | | | | | X |
| Whole blood single cell profiling | | X | X | X | X | X | X | | | X | | X | | X | | X | | | X |
| Host serum proteins (eg, cytokines) | | | X | | X | X | X | | | X | | X | | X | | | | | X |
| Antidrug antibodies (to JNJ 3989) | | | X | | | | | | | X | | | | | | | | | X |
| Immune Monitoring | | | | | | | | | | | | | | | | | | | |
| Leukapheresis (optional)kk | į, | | (X) | | | | | | | | 2 | | 2 10 | | | | (X) | | |
| Immune cells (PBMCs) <sup>II</sup> | | X | | | | | | | | X | | | | X | | | | | |
| Pharmacogenomics (Host DNA) | | | | | | | | | | | | | | | | | | | |
| HLA typing | | | X | | | | | | | | | | | | | | | | |
| Exploratory host genotyping <sup>mm</sup> | | | X | | | | | | | | | | 100 | | | | | | |
| Epigenetic research | | | X | - 1 | | | | | 2 | X | | | 5 10<br>5 5 | X | | | | ž. | X |
| Ongoing Participant Review | | | | | | | | | | | | | | | | | | 8 | |
| Concomitant therapy <sup>nn</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events <sup>nn,oo</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

ALP: alkaline phosphatase; ALT: alanine aminotransferase; AST: aspartate aminotransferase; CKD-EPI: Chronic Kidney Disease Epidemiology Collaboration; CRF: case report form; CT: computed tomography; D/d: day; DBP: diastolic blood pressure; DNA: deoxyribonucleic acid; ECG: electrocardiogram; eGFR: estimated glomerular filtration rate; FSH: follicle-stimulating hormone; HBc: hepatitis B core protein; HBe(Ag): hepatitis B e (antigen); HBcrAg: hepatitis B core-related antigen; HBs(Ag): hepatitis B surface (antigen); HBV: hepatitis B virus; HCC hepatocellular carcinoma; HIV-1 (-2): human immunodeficiency virus type 1 (type 2); HLA: human leukocyte antigen; ICF: informed consent form; IgM: immunoglobulin M; MRI: magnetic resonance imaging; NA: nucleos(t)ide analog; PBMC: peripheral blood mononuclear cell; PK: pharmacokinetic; RNA: ribonucleic acid; SBP: systolic blood pressure; ULN: upper limit of normal; W/w: week; WD: withdrawal.

- a. All study visits are to be scheduled relative to the baseline (Day 1) visit date.
- b. If necessary (eg, for operational reasons), the screening phase may be extended up to a maximum of 6 weeks in agreement with the sponsor.
- c. Day 1 samples are to be collected before the first dose of study intervention.
- d. End of study intervention. If NA treatment completion criteria are not met at Week 48 (see Section 6.6.1), participants will continue NA treatment during the follow-up phase. Participants who discontinue study intervention early will have an early WD visit and will enter follow-up (see the Schedule of Activities Follow-up Phase) unless they withdraw consent. Participants who withdraw consent will be offered an optional safety follow-up visit to occur on the day of consent withdrawal. For the optional safety follow-up visit, assessments are at the investigator's discretion and could be similar to the early WD visit.
- e. The ICF must be signed before the first study-related activity.

- f. If participants agree to undergo an optional liver biopsy, they must sign a separate ICF at screening or at any time prior to the optional liver biopsy (which may take place at Follow-up Week 24, or at any time during the study when clinically indicated). Refusal to give consent for these optional liver biopsy samples does not exclude a participant from participation in the study.
- g. Minimum criteria for the availability of documentation supporting the eligibility criteria will be described in Section 10.3, Appendix 3, Regulatory, Ethical and Study Oversight Considerations. Clinical status will be checked at screening and again before the first liver biopsies at Week -1 and before the first dose of study intervention. If a participant's clinical status changes (including any available laboratory results or receipt of additional medical records) after the start of screening but before the first liver biopsies at Week -1 or before the first dose of study intervention is given such that he or she no longer meets all eligibility criteria, then the participant should be excluded from participation in the study. Retesting to assess eligibility will be allowed once, using an unscheduled visit during the screening period.
- h. Medical history also includes mode of HBV transmission, stage of liver fibrosis, and alcohol consumption. Historical HBV DNA data and available data on previous HBV genotype assessments will be recorded in the CRF. Historical HBsAg, HBeAg, and ALT data, if available, will be recorded in the source document.
- i. Liver disease staging assessments will be performed based on Fibroscan obtained within 6 months prior to screening or at the time of screening.
- j. Only applicable to participants who are enrolled at a site with an on-site Fibroscan device.
- k. Participants must have absence of signs of cirrhosis or portal hypertension (absence of nodules, smooth liver contour, normal portal vein, spleen size <12 cm), absence of signs of HCC or clinically relevant renal abnormalities on an abdominal ultrasound performed within 6 months prior to screening or at the time of screening. In case of suspicious findings on conventional ultrasound the participant may still be eligible if HCC or clinically relevant renal abnormalities have been ruled out by a more specific imaging procedure (contrast enhanced ultrasound, CT or MRI). Additional ultrasound assessments may be performed when clinically indicated.
- 1. A liver ultrasound is recommended approximately every 24 weeks for HCC screening.
- m. Following local standard practice the biopsy location will be identified with ultrasound (which will also be used to rule out contraindicating conditions for a biopsy) and after application of local anesthesia the FNAB samples and core liver biopsy samples will be collected. Prior to any on-treatment biopsy, a recent (≤ 1 week) coagulation and hematology panel, and a platelet aggregation test are required (pre-biopsy visit). Prior to the off-treatment biopsies, blood coagulation and platelets will be assessed at a local laboratory according to local practice. On-treatment (pre)biopsy can either occur during a regularly scheduled visit or an unscheduled visit.
- n. In between study visits, participants will take oral study intervention at home. Participants will be requested to bring their study intervention with them to each study visit. At study visits, the study intervention should be taken on site.

- o. Participants enrolled before Protocol Amendment 5 was in effect, may have received JNJ-6379 as part of their study intervention. Dispensation of JNJ-6379 stopped immediately with the removal of JNJ-6379 as study intervention through an urgent safety measure. Participants have to return JNJ-6379 tablets to the site at the next scheduled visit.
- p. NA will be dispensed at Week 48 for intake during the follow-up phase in case the participant cannot stop NA treatment at Week 48.
- q. Complete physical examination, including height (only at screening), body weight, skin examination, and other body systems (see Section 8.4.1).
- r. Vital signs include supine SBP, DBP, pulse rate, and body temperature.
- s. All ECGs will be read centrally; ECGs should be completed before any tests, procedures or other consultation for that visit.
- t. Biochemistry samples must be taken after fasting for at least 10 hours for measurement of phosphate, calcium, creatinine, and lipids. Participants should bring their oral study intervention with them to each visit and have that day's intake at the site with breakfast.
- u. Creatinine clearance (eGFR calculated by the CKD-EPI formula) will be assessed.
- v. Intervention-emergent ALT/AST elevations (ie, ALT and/or AST ≥3x ULN and ≥3x nadir [ie, lowest value during study participation]), should trigger an assessment of confounding factors (alcohol intake, change in concomitant medication, and comorbidities) and a confirmatory visit, to be scheduled preferably within 7 days of the receipt of the initial ALT/AST results, to repeat laboratory testing of AFP, ALT, AST, ALP, bilirubin (total and direct), INR, albumin, and HBV DNA until ALT and AST levels have returned to <5x ULN and HBV DNA is <20,000 IU/mL. Additional tests should be considered based on clinical judgement. For more details and further management guidance refer to Section 8.5.6.2 and Section 10.6.
- w. Urinalysis by dipstick: specific gravity, pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase, and microscopic analysis if needed. The dipstick reading should be done as soon as possible and in accordance with the manufacturer's recommendation. In case of a positive dipstick result, a urine sample will be set aside for additional examination of the positive parameter (eg, quantification as applicable).
- x. Urine chemistry sample (quantitative measurement): creatinine, sodium, phosphate, glucose, protein, and albumin.
- y. Urine sample for selected renal biomarkers including retinol binding protein and beta-2-microglobulin.
- z. For postmenopausal women only: an FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a woman is not of childbearing potential.
- aa. HBV genotype will be determined at baseline using standard genotyping assay if HBV DNA levels are sufficiently high. For participants with low HBV DNA levels, available historical data on previous HBV genotype assessment will be collected in the CRF. Exploratory genotyping assays might be performed.
- bb. HBcrAg and HBV RNA samples may be batched and only selected samples may be tested at the sponsor's request. Samples can be used for assessment of other serologic/virologic markers of HBV.
- cc. Samples may be sequenced based on the sponsor virologist's request, considering the HBV DNA levels.
- dd. Participants must first complete HBeAg testing and have results reviewed by the investigator to confirm if they qualify for study participation.
- ee. Quantitative HBeAg assessment will only be performed in participants who are defined HBeAg positive at screening or who become HBeAg positive post-baseline based on a qualitative HBeAg assay.
- ff. Exploratory serology samples may be analyzed at the sponsor's discretion. Samples may be used to assess virologic or serologic markers of HBV.
- gg. All participants will have sparse PK sampling for JNJ-3976, JNJ-3924, and NA (ETV, TAF, or tenofovir). Bioanalysis of NA and/or PegIFN-α2a is optional at the discretion of the sponsor. Bioanalysis of JNJ-6379 may also be done on samples collected from participants who received JNJ-6379 up to Protocol Amendment 4 For all samples, the date and time of the preceding intake of oral study intervention (NA), the date and time of the previous JNJ-3989 administration, and the date and time of PK sampling should be recorded. Sparse PK sampling is not required if the participant is part of the intensive PK subgroup and has an extensive PK sampling at the same visit.
- hh. One sample at any time between 2 and 8 hours after JNJ-3989 dosing. Before leaving the study site, the participant's wellbeing should be confirmed.
- ii. Only in case of early withdrawal.

- jj. All participants who consent to participate in the intensive PK subgroup (optional) will undergo intensive PK sampling at Week 4. If necessary (eg, for operational reasons), this visit may be scheduled at Week 8, 12, or 16. The study intervention should be taken on site and time of dosing should be recorded. Pharmacokinetic samples will be taken predose and 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8,\* 10,\* and 24 hours postdose (\*the 8 and 10 hours postdose samples are optional). All efforts will be made to obtain the PK samples at the exact nominal time relative to dosing. However, samples obtained within 20% of the nominal time from dosing (eg, +/- 12 minutes of a 60-minute time point) will not be captured as a protocol deviation if the exact time of the sample collection is noted on the source document and CRF.
- kk. Leukapheresis is optional and will only be performed for participants who provided separate consent for this procedure. Refusal to give consent for leukapheresis does not exclude a participant from participation in the study. The leukapheresis procedure will be performed at least 1 week (and up to 3 weeks) after the liver biopsies; this can either occur during a regularly scheduled visit or an unscheduled visit. Prior to the procedure, the participant's wellbeing will be checked and leukapheresis will only be offered if there is no clinical reason against it. If a participant has had a recent febrile illness, the leukapheresis should be postponed until body temperature is normal for at least 72 hours. One leukapheresis session is expected to last between 1.5 5 hours. During the procedure, the participant will receive intravenous saline infusions and citrate-based anticoagulant. Use of heparin for anticoagulation is not allowed. After completion of the leukapheresis procedure, participants will stay at the site for at least 30 minutes to monitor for any relevant safety events. Participants are advised to refrain from exercise and strenuous activities for 3 days after the leukapheresis visit.
- 11. Additional PBMC samples may be taken in case of ALT flares, upon discussion with the sponsor, and may require an unscheduled visit.
- mm. The pharmacogenomic (DNA) sample should preferably be collected at baseline.
- nn. Adverse events and concomitant medications will be monitored from the time a signed and dated ICF is obtained until completion of the participant's last study-related procedure.
- oo. Includes close monitoring for neuropsychiatric adverse events during the optional PegIFN-α2a treatment period. Participants who develop a neuropsychiatric adverse event during optional PegIFN-α2a treatment, will be monitored closely until the neuropsychiatric adverse event resolves, with frequent (at least weekly) follow-up phone calls.
- pp. As of Protocol Amendment 5, new participants will enroll without randomization within each panel to receive the combination regimen JNJ-3989 + NA as study intervention for 48 weeks.

# 1.3.2. Schedule of Activities - Follow-up Phase

After study intervention completion (or early discontinuation), all participants will enter the 48-week follow-up phase (unless they withdraw consent). Participants who could not stop NA treatment or restarted NA treatment during the follow-up period, provided that their HBV DNA and ALT values have stabilized. will have less frequent visits (every 12 weeks).

For additional visits and assessments in case of optional PegIFN- $\alpha$ 2a treatment, refer to Section 1.3.3.

| Phase | | | | | | | | F | ollow-up | a,b | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 8 | | - | | * | | | +/ FU | W24d | | | | 3 3 | | | |
| Follow up (FU) Week (W) | FU<br>W2 | FU<br>W4 | FU<br>W8 | FU<br>W12 | FU<br>W16 | FU<br>W20 | FU<br>W24 | Optional<br>Biopsy | Post<br>biopsy<br>Visit | FU<br>W28 | FU<br>W32 | FU<br>W36 | FU<br>W40 | FU<br>W44 | FU<br>W48<br>EOS <sup>aa</sup> | Extended<br>FU to<br>maximum<br>FU W72 <sup>y</sup> |
| FU Study Day (Window) | 15<br>(+/<br>4d) | 29<br>(+/<br>4d) | 57<br>(+/<br>4d) | 85<br>(+/<br>4d) | 113<br>(+/<br>4d) | 141<br>(+/<br>4d) | 169<br>(+/<br>4d) | 169<br>(+/ 4w) | ≥1w<br>≤3w<br>After<br>Biopsy | 197<br>(+/<br>4d) | 225<br>(+/ 4d) | 253<br>(+/<br>4d) | 281<br>(+/<br>4d) | 309<br>(+/ 4d) | 337<br>(+/ 4d) | maximum<br>505 (+/<br>4d) |
| Visits in case all treatments including NA stopped | X | X | X | X | X | X | X | | | X | X | X | X | X | X | X |
| Visits in case NA is not stopped | X | X | (X) <sup>c</sup> | X | (X) <sup>c</sup> | (X) <sup>c</sup> | X | | | (X) <sup>c</sup> | (X) <sup>c</sup> | X | (X) <sup>c</sup> | (X) <sup>c</sup> | X | X |
| Study Intervention Administration | | | | | | | | | | | | | | | | |
| Administer/Dispense NA, as applicable <sup>e</sup> | (X) | (X) | (X) | (X) | (X) | (X) | (X) | | | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| NA accountability, as applicable | (X) | (X) | (X) | (X) | (X) | (X) | (X) | | * | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| Assess NA re treatment criteria, as applicable | (X) | (X) | (X) | (X) | (X) | (X) | (X) | | | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| Safety Assessments | | | | | | | | | | | | | | | | |
| Body weight and Symptom directed physical examination (if applicable) | X | X | X | X | X | X | X | | | X | X | X | X | X | X | X |
| Vital signsf | X | X | X | X | X | | X | | | X | X | X | X | X | X | X |
| Triplicate 12 lead ECGg | | X | Tes. | | 100 | | | | | | | | | | | |
| Liver ultrasoundh | | | 10 | | | | X | | | | | | | | X | |
| Clinical Laboratory Tests | | | | | | | | | | | | | | | | |
| Hematology | X | X | X | X | X | | X | | | X | | X | | X | X | X |
| Blood chemistry (including liver function tests) <sup>j,k,1</sup> | X | X | X <sup>m</sup> | X | X <sup>m</sup> | X <sup>m</sup> | X | | | X <sup>m</sup> | X <sup>m</sup> | X | X <sup>m</sup> | X <sup>m</sup> | X | X <sup>m</sup> |
| Blood coagulation | X | X | | X | | | X | | | | | X | | X | X | |
| Urinalysis <sup>n</sup> | | Xp | (X) | (X) | (X) | (X) | (X) | | | (X) | (X) | (X) | (X) | (X) | X | (X) |
| Urine chemistry <sup>o</sup> | | Xp | (X) | (X) | (X) | (X) | (X) | | | 0.8 100 | (X) | (X) | | (X) | X | |

| Phase | | | | | | | | F | ollow-ur | ) <sup>a,b</sup> | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | , | N. | | | 1 | | +/ FU | | | | | I | | | |
| Follow up (FU) Week (W) | FU<br>W2 | FU<br>W4 | FU<br>W8 | FU<br>W12 | FU<br>W16 | FU<br>W20 | FU<br>W24 | Optional<br>Biopsy | Post<br>biopsy<br>Visit | FU<br>W28 | FU<br>W32 | FU<br>W36 | FU<br>W40 | FU<br>W44 | FU<br>W48<br>EOS <sup>aa</sup> | Extended<br>FU to<br>maximum<br>FU W72 <sup>y</sup> |
| FU Study Day (Window) | 15<br>(+/<br>4d) | 29<br>(+/<br>4d) | 57<br>(+/<br>4d) | 85<br>(+/<br>4d) | 113<br>(+/<br>4d) | 141<br>(+/<br>4d) | 169<br>(+/<br>4d) | 169<br>(+/ 4w) | ≥1w<br>≤3w<br>After<br>Biopsy | 197<br>(+/<br>4d) | 225<br>(+/ 4d) | 253<br>(+/<br>4d) | 281<br>(+/<br>4d) | 309<br>(+/ 4d) | 337<br>(+/ 4d) | maximum<br>505 (+/<br>4d) |
| Visits in case all treatments including NA stopped | X | X | X | X | X | X | X | | | X | X | X | X | X | X | X |
| Visits in case NA is not stopped | X | X | (X)° | X | (X)° | (X) <sup>c</sup> | X | | | (X) <sup>c</sup> | (X) <sup>c</sup> | X | (X) <sup>c</sup> | (X) <sup>c</sup> | X | X |
| Urine pregnancy test (women of childbearing potential only) | | X | X | X | X | X | Χq | | | Хq | Xq | Xq | Χq | Χq | X | Xq |
| Liver Biopsy | | | | | | | | | | | | | | | | |
| FNAB sample | | | 18 | | 58 S | | | (X)i | | | | | | | | |
| Percutaneous core liver biopsy sample | | | | | | | | (X)i | | | | | | | | |
| Efficacy Assessments | | | | | | | | | | | | | | | | |
| Fibroscan <sup>r</sup> | | | | | | | (X) | | | | | | | | (X) | |
| HBV Virology | | | | | | | | | | | | | | | 10 50 | |
| Blood sample collection for HBV DNA <sup>z</sup> and HBV RNA <sup>s</sup> | X | X | X | Х | X | X | X | | | X | X | X | X | X | X | X |
| Sampling for viral genome sequencing <sup>t</sup> | | X | | X | | X | | | | | X | | X | | X | |
| HBV Serology | | | | | | | | | | | | | | | | |
| Blood sample collection for: | | | | | | | | | | | | | | | | |
| Anti HBs and anti HBe | | X | | X | | | X | | | | | X | | | X | |
| HBsAg (qualitative) | | | | | | | X | The state of the s | | | | | | | X | |
| HBeAg (qualitative) | | | 24 | X | | | X | | | | | | 1 | | X | |
| HBsAg (quantitative) | X | X | X | X | X | X | X | * | | X | X | X | X | X | X | X |
| HBeAg (quantitative) | X | X | X | X | X | X | X | | | X | X | X | X | X | X | X |
| HBcrAg <sup>s</sup> | | X | 2 | X | 2 | | X | | | | | X | | | X | |
| Exploratory serology <sup>u</sup> | X | X | X | X | X | X | X | | | | | X | | | X | |
| Exploratory Host Biomarkers | | | | | | | | | | | | | | | | |
| Whole blood RNA gene expression | | X | | | | | X | | | | | | | | X | |
| Whole blood single cell profiling | | X | X | X | X | İ | X | X | | | | X | | | X | |
| Host serum proteins (eg, cytokines) | | X | X | X | X | | X | | | | | X | | | X | |
| Antidrug antibodies (to JNJ 3989) | | | | | | | X | | | | | | | | X | |
| Immune Monitoring | | | | | | | | | | | | | | | | |
| Leukapheresis (optional) <sup>v</sup> | | | 1 | | | | | | (X) | | | | | | | |

| Phase | | 95 | | | | | | F | ollow-up | a,b | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | +/ FU | W24d | | | | | | | |
| Follow up (FU) Week (W) | FU<br>W2 | FU<br>W4 | FU<br>W8 | FU<br>W12 | FU<br>W16 | FU<br>W20 | FU<br>W24 | Optional<br>Biopsy | Post<br>biopsy<br>Visit | FU<br>W28 | FU<br>W32 | FU<br>W36 | FU<br>W40 | FU<br>W44 | FU<br>W48<br>EOS <sup>aa</sup> | Extended<br>FU to<br>maximum<br>FU W72 <sup>y</sup> |
| FU Study Day (Window) | 15<br>(+/<br>4d) | 29<br>(+/<br>4d) | 57<br>(+/<br>4d) | 85<br>(+/<br>4d) | 113<br>(+/<br>4d) | 141<br>(+/<br>4d) | 169<br>(+/<br>4d) | 169<br>(+/ 4w) | ≥1w<br>≤3w<br>After<br>Biopsy | 197<br>(+/<br>4d) | 225<br>(+/ 4d) | 253<br>(+/<br>4d) | 281<br>(+/<br>4d) | 309<br>(+/ 4d) | 337<br>(+/ 4d) | maximum<br>505 (+/<br>4d) |
| Visits in case all treatments including NA stopped | X | X | X | X | X | X | X | | | X | X | X | X | X | X | X |
| Visits in case NA is not stopped | X | X | (X) <sup>c</sup> | X | (X)° | (X)° | X | | | (X) <sup>c</sup> | (X) <sup>c</sup> | X | (X) <sup>c</sup> | (X)° | X | X |
| Immune cells (PBMCs)w | X | | | X | | | X | | | | | | | | | |
| Pharmacogenomics (Host DNA) | | | | | | | | | | | | | | | | |
| Epigenetic research | X | | | X | | | X | | | | | | | | X | |
| Ongoing Participant Review | | | | | | | | | | | | | | | | |
| Concomitant therapy <sup>x</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events <sup>x</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

ALP: alkaline phosphatase; ALT: alanine aminotransferase; AST: aspartate aminotransferase; d: days; DBP: diastolic blood pressure; DNA: deoxyribonucleic acid; ECG: electrocardiogram; eGFR: estimated glomerular filtration rate; EOS: end of study; FU: follow-up; HBcrAg: hepatitis B core-related antigen; HBe(Ag): hepatitis B e (antigen); HBs(Ag): hepatitis B surface (antigen); HBV: hepatitis B virus; HCC: hepatocellular carcinoma; ICF: informed consent form; NA: nucleos(t)ide analog; PBMC: peripheral blood mononuclear cells; RNA: ribonucleic acid; SBP: systolic blood pressure; ULN: upper limit of normal; W: Week.

- a. All follow-up study visits are to be scheduled relative to the last dose of JNJ-3989. An unscheduled visit can be performed upon the investigator's discretion, in case of HBV DNA elevations, ALT elevations, other signs of worsening of liver disease, or for any other reason during follow-up.
- b. Participants who withdraw consent during follow-up will be offered an optional safety follow-up visit.
- c. Visit is optional for participants who continue NA treatment and for participants who have restarted NA treatment during the follow-up period, provided that their HBV DNA and ALT values are stable.
- d. An optional liver biopsy (core liver biopsy and/or FNAB) may be performed at Follow-up Week 24 or at any time during the study if the participant provided consent.
- e. No JNJ-3989 will be administered or dispensed during follow-up. Administration/Dispensation of NA is only applicable for participants who could not stop NA treatment at Week 48 (Section 6.6.1), or for those who met the NA re-treatment criteria (Section 6.6.2). In between study visits, participants will take NA treatment at home. Participants will be requested to bring their NA treatment with them to each study visit. At study visits, the NA treatment should be taken on site.
- f. Vital signs include supine SBP, DBP, pulse rate, and body temperature.
- g. All ECGs will be read centrally; ECGs should be completed before any tests, procedures or other consultation for that visit.
- A liver ultrasound is recommended approximately every 24 weeks for HCC screening.
- i. Following local standard practice the biopsy location will be identified with ultrasound (which will also be used to rule out contraindicating conditions for a biopsy) and after application of local anesthesia the FNAB samples and core liver biopsy samples will be collected. Prior to the biopsy, blood coagulation and platelets will be assessed at a local laboratory according to local practice. The (post)biopsy visit can either occur during a regularly scheduled visit or an unscheduled visit.

- j. Biochemistry samples must be taken after fasting for at least 10 hours for measurement of phosphate, calcium, creatinine, and lipids.
- k. Creatinine clearance (eGFR calculated by the CKD-EPI formula) will be assessed.
- 1. ALT/AST elevations (ie, ALT and/or AST ≥3x ULN and ≥3x nadir [ie, lowest value during study participation]), should trigger an assessment of confounding factors (alcohol intake, change in concomitant medication, and comorbidities) and a confirmatory visit, to be scheduled preferably within 7 days of the receipt of the initial ALT/AST results, to repeat laboratory testing of AFP, ALT, AST, ALP, bilirubin (total and direct), INR, albumin, and HBV DNA until ALT and AST levels have returned to <5x ULN and HBV DNA is <20,000 IU/mL. Additional tests should be considered based on clinical judgement. For more details and further management guidance refer to Section 8.5.6.2 and Section 10.6.
- m. Liver function tests only.

- n. Urinalysis by dipstick: specific gravity, pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase, and microscopic analysis if needed. The dipstick reading should be done as soon as possible and in accordance with the manufacturer's recommendation. In case of a positive dipstick result, a urine sample will be set aside for additional examination of the positive parameter at the central laboratory (eg, quantification as applicable).
- o. Urine chemistry sample (quantitative measurement): creatinine, sodium, phosphate, glucose, protein, and albumin.
- p. A urinalysis and urine chemistry sample will be taken at Follow-up Week 4. In case of abnormalities, the tests should be repeated at the following visits.
- q. Urine pregnancy tests for at-home use will be provided to the participants as necessary to ensure urine pregnancy tests are performed at least every 4 weeks. Results will be reported at the next visit. If positive, the participant should contact the site immediately.
- r. Only applicable to participants who are enrolled at a site with an on-site Fibroscan device.
- s. HBcrAg and HBV RNA samples may be batched and only selected samples may be tested at the sponsor's request. Samples can be used for assessment of other serologic/virologic markers of HBV.
- t. Samples may be sequenced based on the sponsor virologist's request, considering the HBV DNA levels. A sample for viral genome sequencing will be taken at an unscheduled visit for confirmation of virologic relapse.
- u. Exploratory serology samples may be analyzed at the sponsor's discretion. Samples may be used to assess virologic or serologic markers of HBV.
- v. Leukapheresis is optional and will only be performed for participants who provided separate consent for this procedure. Refusal to give consent for these optional procedures does not exclude a participant from participation in the study. The leukapheresis procedure will be performed at least 1 week (and up to 3 weeks) after the liver biopsy; this can either occur during a regularly scheduled visit or an unscheduled visit. If no liver biopsy is being performed during follow-up, leukapheresis should take place around the FU W24 time point. Prior to the procedure, the participant's wellbeing will be checked and leukapheresis will only be offered if there is no clinical reason against it. If a participant has had a recent febrile illness, the leukapheresis should be postponed until body temperature is normal for at least 72 hours. One leukapheresis session is expected to last between 1.5 5 hours. During the procedure, the participant will receive intravenous saline infusions and citrate-based anticoagulant. Use of heparin for anticoagulation is not allowed. After completion of the leukapheresis procedure, participants will stay at the site for at least 30 minutes to monitor for any relevant safety events. Participants are advised to refrain from exercise and strenuous activities for 3 days after the leukapheresis visit.
- w. Additional PBMC samples may be taken in case of ALT flare, upon discussion with the sponsor, and may require an unscheduled visit.
- x. Adverse events and concomitant medications will be monitored from the time a signed and dated ICF is obtained until completion of the participant's last study-related procedure.
- y. With implementation of Protocol Amendment 5, the follow-up phase of 48 weeks will be extended for participants who are receiving optional treatment with PegIFN-α2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN-α2a to ensure all study participants will be followed for at least one year after NA treatment cessation. Visits will be scheduled at least every 4 weeks and assessments will be similar to assessments performed at the FU W28 visit. At the respective EOS visit for these participants, assessments as described in the FU W48 EOS visit will be performed.
- z. NA treatment should be re-started in accordance with the NA re-treatment criteria (refer to Section 6.6.2 and Section 10.12 Appendix 12 for guidance after stopping NA treatment.)

aa. The investigator should consider to re start NA treatment per local standard of care at the EOS visit (Follow up Week 48 up to maximum Follow up Week 72) for participants who met the NA treatment completion criteria at the end of treatment with PegIFN α2a during the follow up phase, who did not re start NA treatment during the follow up phase, and who did not achieve and maintain HBsAg seroclearance. NA will not be provided by the sponsor after the final study visit.

# 1.3.3. Schedule of Activities – Optional PegIFN-α2a Treatment

Participants who provide separate consent, may receive treatment with optional PegIFN- $\alpha$ 2a starting after the Week 40 biopsy (or after the optional leukapheresis if applicable) but before the Week 48 visit. The duration (either 12 or 24 weeks) will be at the investigator's discretion.

In addition to the main schedules of activities (refer to Sections 1.3.1 and 1.3.2), the following visits and assessments will be performed for participants receiving PegIFN- $\alpha$ 2a.

| Phase | | O | ptional Pe | egIFN α2 | a treatment | Comments |
|---|---|---|---|---|---|---|
| Additional visits | Before | Start | +2 wks | +4 wks | End<br>(+12 or 24 wks) | |
| Study Day (relative to start of PegIFN α2a treatment) | | 1 | 15 | 29 | 85 or 169 | |
| ICF for PegIFN α2a treatment | X | | | | | Participants must sign a separate ICF prior to the start of PegIFN 02a treatment. Refusal to give consent for this optional treatment does not exclude a participant from participation in the study. |
| Exclusion criteria for PegIFN α2a treatment | X | 20 | 2 13 | | | To be checked prior to the start of PegIFN α2a treatment (refer to Section 5.2). |
| Administer PegIFN α2a for 12 or 24 weeks | | | | (Weekly) | | All PegIFN a2a administrations (on study visits and in between study visits) should preferably be done in the evening by self injection. If desired, participants can also choose to have the weekly administration of PegIFN a2a performed on site irrespective of the time of day. |
| Dispense PegIFN α2a | | (E | Every 4 we | eeks) | | Participants will receive PegIFN α2a supply for self administration at home in between study visits. |
| Study intervention accountability | | | X | X | X | |
| Body weight and Symptom directed physical examination | | X | X | X | X | |
| Ophthalmic examination | X | | (As | applicab | le) | Periodic ophthalmologic examinations during PegIFN 0.2a treatment are at the investigator's discretion. Any patient who develops ocular symptoms should receive a prompt and complete eye examination. |
| Injection site reactions for PegIFN α2a | | - | (A | t every vi | sit) | |
| Hematology | | | X | X | | |
| Blood chemistry (including liver function tests) | | | | X | | |
| Blood sampling for HBV DNA | | X | | | X | |
| Blood sampling for HBsAg (quantitative) | | X | | | X | |
| Blood sampling for HBeAg (quantitative) | | X | × | | X | |
| Blood sampling for sparse PK of PegIFN α2a <sup>a</sup> | | | | X | X | For all samples, the date and time of the previous PegIFN $\alpha 2a$ administration, and the date and time of PK sampling should be recorded. Optional PegIFN $\alpha 2a$ should preferably be administered in the evening prior to the sparse PK visit, or alternatively in the morning of the visit on site. |
| Antidrug antibodies to PegIFN α2a | | | | | X | |

 $CONFIDENTIAL-FOIA\ Exemptions\ Apply\ in\ U.S.$
| Phase | | O | ptional Pe | gIFN α2 | a treatment | Comments |
|---|---|---|---|---|---|---|
| Additional visits | Start | +2 wks | +4 wks | End<br>(+12 or 24 wks) | | |
| Study Day (relative to start of PegIFN α2a treatment) | | 1 | 15 | 29 | 85 or 169 | |
| ECG | | 100 | | | X | |
| TSH and T4 | X | | 10 | | X | |
| AFP | | | | | X | |
| Concomitant therapy | | X | X | X | X | |
| Adverse events <sup>b</sup> | | X | X | X | X | |

AFP: alpha-fetoprotein; DNA: deoxyribonucleic acid; ECG: electrocardiogram; HBeAg: hepatitis B e antigen; HBsAg: hepatitis B surface antigen; HBV: hepatitis B virus; ICF: informed consent form; PegIFN-α2a: pegylated interferon alpha-2a; PK: pharmacokinetic; T4: thyroid-stimulating hormone; TSH: thyroxine; wks: week

- a. Bioanalysis of PegIFN-α2a is optional at the discretion of the sponsor.
- b. Includes close monitoring for neuropsychiatric adverse events during the optional PegIFN-α2a treatment period. Participants who develop a neuropsychiatric adverse event during optional PegIFN-α2a treatment, will be monitored closely until the neuropsychiatric adverse event resolves, with frequent (at least weekly) follow-up phone calls.

*Note:* Visits should preferably coincide with a regularly scheduled visit (as per the main schedules of activities in Sections 1.3.1 and 1.3.2). In case assessments coincide with the main schedule of activities, they only need to be performed once.

*Note:* Unscheduled visits for additional assessments are at the investigator's discretion as per local standard practice and following the prescribing information of PegIFN- $\alpha$ 2a.

#### 2. INTRODUCTION

## **Chronic Hepatitis B Infection**

Hepatitis B virus (HBV) is a small deoxyribonucleic acid (DNA) virus that specifically infects the human liver. It consists of a nucleocapsid in which the viral DNA is packed with hepatitis B core protein (HBc) and a membraneous envelope containing hepatitis B surface antigen (HBsAg). The acute phase of the infection (less than 6 months) is either followed by an immune controlled state (spontaneous cure from the infection) or progresses to chronic hepatitis B (more than 6 months). Chronic HBV infection may lead to serious illnesses such as liver cirrhosis and decompensation, and hepatocellular carcinoma (HCC), often with fatal outcome.<sup>33</sup>

The worldwide estimated prevalence of chronic HBV infection is 4.9% with about 292 million people affected.<sup>28</sup> Despite the availability of an efficacious prophylactic vaccine, yearly rates of new infections remain high. Approximately 680,000 people per year worldwide die from cirrhosis and HCC due to chronic HBV infection.<sup>31</sup>

The natural course of chronic HBV infection is the consequence of a complex interaction between the virus and the host which in the chronic setting might evolve over a duration of decades. This is associated with different disease phases or stages. The European Association for the Study of the Liver (EASL) guidelines differentiate between chronic infection and chronic hepatitis (Table 1).

| Table 1: Various Stages of HBV Infection – Terminology and Characteristics (EAS |
|---|
|---|

| | НВ | eAg positive | НВе | eAg negative |
|---|---|---|---|---|
| | Chronic infection | Chronic hepatitis | Chronic infection | Chronic hepatitis |
| HBsAg | High | High/intermediate | Low | Intermediate |
| HBeAg | Positive | Positive | Negative | Negative |
| HBV DNA | >10 <sup>7</sup> IU/mL | 10 <sup>4</sup> -10 <sup>7</sup> IU/mL | <2,000 IU/mL°° | >2,000 IU/mL |
| ALT | Normal | Elevated | Normal | Elevated* |
| Liver disease | None/minimal | Moderate/severe | None | Moderate/severe |
| Old | Immune tolerant | Immune reactive HBeAg | Inactive carrier | HBeAg negative chronic |
| terminology | | positive | | hepatitis |

ALT: alanine aminotransferase; DNA: deoxyribonucleic acid; EASL: European Association for the Study of the Liver; HBeAg: hepatitis B e antigen; HBsAg: hepatitis B surface antigen; HBV: hepatitis B virus; IU/mL: International Units Per Milliliter

Note that different definitions and naming of HBV disease phases may be used across different countries/regions.

According to the EASL treatment guidelines, the primary treatment goal for patients with chronic HBV infection is to improve survival and quality of life by preventing progression of liver disease, particularly to cirrhosis, liver failure, and HCC.

Irrespective of the hepatitis B e antigen (HBeAg) status, antiviral therapy is recommended for all patients with signs of active chronic hepatitis. <sup>2,5,30,33</sup> Approved therapies for chronic HBV infection are pegylated interferon alpha (PEG-IFN-α) and nucleos(t)ide analog (NA) inhibitors (ie, NA)

<sup>\*</sup> Persistently or intermittently. °°HBV deoxyribonucleic acid (DNA) levels can be between 2,000 and 20,000 IU/mL in some patients without signs of chronic hepatitis.

treatment) of the HBV polymerase/reverse transcriptase, the enzyme synthesizing HBV DNA from pre-genomic ribonucleic acid (pgRNA).

Oral treatment with NAs is effective at suppressing viral DNA formation and lowering virus concentration in the blood to levels below the lower limit of quantification (LLOQ) of the HBV DNA assays commonly used. This is associated with normalization of liver enzymes and reduced or halted progression of liver disease to cirrhosis and/or decompensation and even with regression of cirrhotic transformation. 4,18,22,25,36 While the risk of HCC development is reduced as well, it is not eliminated. 18,22,25

Hepatitis B surface antigen seroclearance 24 weeks after end of treatment is currently considered to be associated with the most thorough suppression of HBV replication and has been termed "functional cure". Unfortunately, with currently available NA treatment strategies the rate of HBsAg seroclearance remains very low (around 3%) even under long-term treatment.

Pegylated IFN is associated with a slightly higher rate of HBsAg seroclearance compared to NAs and is recommended for a fixed treatment duration of 48 weeks, but is administered subcutaneously (SC) and is associated with higher toxicity than NAs.<sup>27</sup>

With the low rate of functional cure with current treatments, and persistently high global prevalence of HBV-associated mortality, 5,33 there is a medical need for more effective finite treatment options that lead to sustained seroclearance of HBsAg and HBV DNA off treatment ("functional cure"). In order to achieve an effective finite treatment, combination of therapies with different mechanisms of action, as is standard of care for other chronic viral infections like hepatitis C virus (HCV) and human immunodeficiency virus (HIV), is deemed required.

A challenge for the clinical development of novel HBV agents is that while blood markers are used to assess their efficacy and immune response induced by these agents, their target organ is the liver. Although some of the efficacy blood markers are very well established from a clinical perspective, questions remain on how good these markers correlate with intrahepatic events, such as HBV covalently closed circular DNA (cccDNA) level and transcriptional activity. In addition, the immune response measured in the periphery is known to insufficiently reflect the situation in the liver. For example, the frequency of HBV-specific T-cells as well as liver resident immune cells cannot be adequately assessed by measuring immune response in the periphery. Multiple studies have shown the value of full needle core biopsies as well as fine needle aspirates to assess intrahepatic virologic and immunologic events of HBV. A wide range of methods are currently available, such as polymerase chain reaction (PCR) based methods, single cell analyses and high multiplex fluorescence-based methods.

JNJ-73763989 (JNJ-3989) is a liver-targeted antiviral therapeutic for SC injection designed to treat chronic HBV infection via a ribonucleic acid interference (RNAi) mechanism. JNJ-3989 consists of two RNAi triggers, one targeting the HBsAg open reading frame (JNJ-73763976 [JNJ-3976]), and one targeting the HBV X protein open reading frame (JNJ-73763924 [JNJ-3924]). Hence, engagement of the cellular RNAi machinery by JNJ-3989 results in specific cleavage of HBV ribonucleic acid (RNA) transcripts, thereby reducing the levels of HBV proteins and the pgRNA,

the precursor of viral relaxed circular DNA. The RNAi triggers in JNJ-3989 injection are designed to target all HBV RNA transcripts derived from cccDNA, as well as transcripts derived from integrated viral DNA. The latter has been suggested to be a significant source of HBsAg in HBeAg negative patients or patients on long term treatment with NAs, the current standard of care. <sup>35</sup>

JNJ-56136379 (JNJ-6379) is an orally administered capsid assembly modulator (CAM) that is being developed for the treatment of chronic HBV infection. JNJ-6379 binds to HBc and interferes with the viral capsid assembly process, thereby preventing the polymerase-bound pgRNA encapsidation. This results in the formation of HBV capsids, devoid of HBV DNA or RNA (nonfunctional capsids), and ultimately in the inhibition of HBV replication. In addition, JNJ-6379 also acts at an early stage of the viral life cycle by inhibiting the de-novo formation of cccDNA potentially by interfering with the capsid disassembly process. JNJ-6379 was initially part of the study intervention but has been removed as study intervention with the implementation of an urgent safety measure, as described in Protocol Amendment 5.

Prior to Protocol Amendment 5, the term "study intervention" throughout the protocol, refers to JNJ-3989, JNJ-6379, NA, and optional PegIFN- $\alpha 2a^a$ .

As of Protocol Amendment 5, the term "study intervention" throughout the protocol, refers to JNJ-3989, NA, and optional PegIFN- $\alpha$ 2a.

The term "sponsor" used throughout this document refers to the entities listed in the Contact Information page(s), which will be provided as a separate document.

The term "participant" throughout the protocol refers to the common term "subject".

## 2.1. Study Rationale

This liver biopsy study is primarily performed to assess changes in intrahepatic viral and host immune markers in response to JNJ-3989-based combination treatment. This analysis can be used to characterize mode of action (MoA) of the treatment. Furthermore, this study aims to explore association of hepatic and peripheral viral and/or host markers with selected efficacy variables, identify subpopulations that show a defined response, and identify cellular and molecular determinants of response. Hepatic and peripheral viral and immune markers and their correlations will be assessed. In addition, changes in liver histology may be assessed. The totality of results may be used to inform on the optimal use of therapeutics in current or future combinations. This study aims to assess intrahepatic events in the context of a full (48-week) treatment regimen as used in 2 ongoing Phase 2b studies in a similar HBV population to facilitate comparison of the results across studies.

The efficacy and safety of finite treatment duration will be assessed with a fixed 48-week treatment duration for JNJ-3989, in combination with NA treatment. Participants meeting pre-defined response criteria (outlined in Section 6.6.1) will also complete NA treatment after 48 weeks. The

<sup>&</sup>lt;sup>a</sup> Note: Optional PegIFN α2a was introduced as 'study intervention' as of Protocol Amendment 4.

participants may also receive optional treatment with PegIFN- $\alpha$ 2a for either 12 or 24 weeks at the investigator's discretion, to investigate whether addition of PegIFN- $\alpha$ 2a towards the end of the existing treatment regimen further decreases HBsAg.

## 2.2. Background

For the most comprehensive nonclinical and clinical information regarding JNJ-3989 and JNJ-6379, refer to the latest version of the Investigator's Brochure (IB) and addenda. <sup>14</sup> <sup>16,39</sup>

**Note:** JNJ-6379 was initially part of the study intervention but has been removed as study intervention with the implementation of an urgent safety measure, as described in Protocol Amendment 5. For completeness, background information on JNJ-6379 is still included in this section.

#### 2.2.1. Nonclinical Studies

#### 2.2.1.1. JNJ-3989 and JNJ-6379

Nonclinical assessments to support clinical development have been performed for the single agents JNJ-3989 and JNJ-6379, and also for their combination (up to 3 months studies).

#### JNJ-3989

Little potential for off-target inhibition of human gene expression in participants is expected, based on in silico human genome database screening.

The nonclinical safety profile of JNJ-3989 has been evaluated through a series of in vitro and in vivo studies. Repeat-dose SC toxicity studies of 2 weeks up to 24 or 37 weeks were conducted in rat and monkey, respectively. In the 2-week studies, JNJ-3989 was administered once weekly via SC injection at profile to commonly the profile profile profile month, followed by once monthly thereafter at the common monthly the common mont

In the 2-week and the 24-week studies in rat, JNJ-3989-related target organs were the liver, the kidney, and the injection site. The mandibular and mesenteric lymph nodes were identified as target organ in the 24-week study only. In the liver, hepatocyte alteration and hepatocyte mitosis, accompanied by an increase in hepatocellular vacuoles, oval cell hyperplasia, Kupffer cell vacuolation and/or increased liver weights were observed. The hepatocyte findings correlated to increased alkaline phosphatase (ALP) activity levels seen in the 24-week study. Kidney findings were characterized by cytoplasmic alteration of the cortical tubule epithelium. At the injection site, mononuclear cell or vacuolated macrophage infiltrates, epidermal exudate, hemorrhages and/or interstitial granules were observed. Macrophage vacuolation was observed in the sinus spaces of the mandibular and mesenteric lymph nodes.

Liver findings persisted throughout the recovery period. Partial recovery was observed in the kidney. No findings were present anymore at the injection sites and the lymph nodes at the end of the recovery period.

All these changes likely represented the distribution, accumulation, and clearance of JNJ-3989 and were considered not to be adverse due to the nature of the findings and the low severity. These are commonly described findings for N-acetylgalactosamine-conjugated RNAi.<sup>17</sup> The no observed adverse effect level (NOAEL) was therefore considered to be the highest dose tested, ie, commonly in the 24-week study.

In the 2-week study in monkey, apart from a minimally increased ALP activity which was considered not adverse, no JNJ-3989-related effects were observed. In the 37-week study, JNJ-3989-related target organs were the liver, mandibular and/or mesenteric lymph nodes, and the SC injection site. Findings included Kupffer cell basophilia/hypertrophy in the liver, vacuolated macrophages in the lymph nodes, and macrophage infiltrates in the injection site. Partial reversibility was observed for these findings. This likely represented the distribution, accumulation, and clearance of JNJ-3989 and was considered not to be adverse due to the low severity and/or nature of the findings. These are commonly described findings for N-acetylgalactosamine-conjugated RNAi. A non-adverse minimally increased ALP activity was observed at observed at observed at observed at observed at observed to be the highest dose tested, ie, or mg/kg in the 37-week study.

In the embryofetal development (EFD) studies, JNJ-3989 was not teratogenic in rats and rabbits.

The fertility study showed no effects on parental and reproductive parameters in male and female rats given JNJ-3989 up to a dose of CCI mg/kg/week.

JNJ-3989 was shown to be non-genotoxic when tested in the bacterial reverse mutation assay, and in vitro and in vivo micronucleus test.

Results of the non-Good Laboratory Practice (GLP) in vitro studies demonstrated there is no potential for induction of the innate immune system (cytokine and complement activation), mitochondrial toxicity/cytotoxicity, or platelet aggregation associated with JNJ-3989 exposure at concentrations up to CCI µg/mL.

The animal-to-human exposure ratios were calculated using rat and monkey exposures at NOAEL from the 24-week and 37-week studies, respectively, and human exposures after a single SC injection of 200 mg JNJ-3989 in human volunteers (Study AROHBV1001) (Table 2).

Table 2: Animal/Human Exposure Ratios at NOAEL for JNJ-3989

| | | | | | Ratio Total Concentration | |
|---|---|---|---|---|---|---|
| | Sex | NOAEL<br>(mg/kg) | C <sub>max</sub><br>(ng/mL) | AUC <sup>b</sup><br>(ng.h/mL) | C <sub>max</sub><br>A/H Ratio | AUC <sup>b</sup><br>A/H Ratio |
| JNJ-3976 | | | | | | |
| Human expo | sure <sup>a</sup> | | 1,315 | 20,136 | - | - |
| 24-week | M | CCI | 41,100 | 437,000 | 31.3 | 21.7 |
| rat <sup>c</sup> | F | | 43,100 | 270,000 | 32.8 | 13.4 |
| 37-week | M | | 73,200 | 1,230,000 | 55.7 | 61.1 |
| monkeyd | F | | 65,800 | 988,000 | 50.0 | 49.1 |

| | | | | | <b>Ratio Total Concentration</b> | |
|---|---|---|---|---|---|---|
| | Sex | NOAEL<br>(mg/kg) | C <sub>max</sub><br>(ng/mL) | AUC <sup>b</sup><br>(ng.h/mL) | C <sub>max</sub> A/H Ratio | AUC <sup>b</sup><br>A/H Ratio |
| JNJ-3924 | | | | | | |
| Human expo | sure <sup>a</sup> | | 363 | 4,605 | | |
| 24-week | M | CCI | 25,200 | 271,000 | 69.4 | 58.8 |
| rat <sup>c</sup> | F | | 26,200 | 163,000 | 72.2 | 35.4 |
| 37-week | M | | 21,600 | 383,000 | 59.5 | 83.2 |
| monkey <sup>d</sup> | F | | 23,000 | 392,000 | 63.4 | 85.1 |

Table 2: Animal/Human Exposure Ratios at NOAEL for JNJ-3989

AUC: area under the plasma concentration time curve;  $AUC_{0-24h}$ : area under the plasma concentration time curve from administration to 24 h;  $AUC_{0-last}$ : area under the plasma concentration time curve from administration to last quantifiable sampling point; A/H: animal/human ratio;  $C_{max}$ : maximum plasma concentration; F: female; M: male; M: male; M: male; M: male; M: pharmacokinetics; M: subcutaneous

- <sup>a</sup> Single dose of 200 mg JNJ 3989 in healthy volunteers via SC injection (Study AROHBV1001; based on recent clean dataset with data cut off 29 October 2019. Clinical PK update will be included in next revision of the IB).
- b AUC<sub>0-last</sub> for human exposure; AUC<sub>0-24h</sub> for animal exposures
- <sup>c</sup> Once weekly dosing for 4 weeks, followed by once monthly dosing, up to a total of 24 weeks
- d Once weekly dosing for 5 weeks followed by once monthly dosing, up to a total of 37 weeks

## JNJ-6379

Following 6 months of treatment in rats, the kidney and female reproductive tract (irregular estrous cycle) were identified as target organs. However, after further assessment of the kidney findings and their clinical relevance, it is deemed unlikely that the retrograde nephropathy seen in 1 out of 20 male rats following 6 months of dosing with JNJ-6379 at 100 mg eq./kg/day are relevant for the clinical studies. The retrograde nephropathy was partially recovered after a 9-week recovery period. In the 6-month rat study, female rats (at 200 mg eq./kg/day) showed an irregular estrous cycle, from which they recovered at the end of the 9-week treatment-free period. These irregular estrous cycles were also apparent in the female fertility studies (main and mechanistic). These changes were related to lowered hormone levels (luteinizing hormone, progesterone, estradiol). JNJ-6379, however, did not affect female fertility. The fetal loss seen during the early stages of pregnancy was considered to result from low hormone levels. In the dog study, no changes were observed in the reproductive tract at higher exposures in dogs.

In the 9-month dog study, the target organs identified were the adrenal glands and bone marrow. The adrenal glands did not show degenerative changes or loss of function and were therefore considered as non-adverse target organs. One female dog out of 4 dosed at 25 mg eq./kg/day (the highest dose) was sacrificed on Day 61, after showing poor health condition. A JNJ-6379 plasma level of 42,000 ng/mL was observed for this animal on Day 61, at approximately 24 hours after last dosing. Pronounced clinical pathologic changes, including pancytopenia, were noted. Marked increase in plasma cell-like cells was seen in the bone marrow during histopathologic examination, resulting in a marked reduction of hematopoietic tissue and extramedullary hematopoiesis in liver and spleen. The cause of the deteriorating condition was likely related to changes in the bone marrow. A second dog in the same dose group with pancytopenia recovered after a drug holiday and was re-exposed uneventfully.

In the EFD studies, JNJ-6379 was not teratogenic in rats and rabbits.

JNJ-6379 was not genotoxic in the in vitro micronucleus and Ames tests, and in the in vivo micronucleus tests in rats.

Animal/human ratios at the NOAEL in rat and dog for human exposure at 250 mg JNJ-6379 once daily (qd) for 28 days are displayed in Table 3.

Table 3: Animal/Human Ratios at the NOAEL in Rat and Dog (Human Exposure at 250 mg JNJ-6379 Once Daily for 28 Days [Study 56136379HPB1001])

| | | | | | | Ratio Ratio Total Concentration Concentration Concentration Bindin | | entration<br>ected for<br>a Protein |
|---|---|---|---|---|---|---|---|---|
| | Sex | NOAEL<br>(mg eq./kg/day) | C <sub>max</sub> (ng/mL) | AUC <sub>0-24h</sub><br>(ng.h/mL) | C <sub>max</sub> A/H Ratio | AUC <sub>0-24h</sub><br>A/H<br>Ratio | C <sub>max</sub><br>A/H<br>Ratio | AUC <sub>0-24h</sub><br>A/H<br>Ratio |
| Human exposure <sup>a</sup> | 2411 | | 13,798 | 267,180 | - | - | 110110 | 1100110 |
| - | M | CCI | 7,540 | 93,100 | 0.6 | 0.3 | 0.9 | 0.6 |
| 6M rat | M | | $13,600^{d}$ | 180,000 <sup>d</sup> | 1.0 | 0.7 | 1.7 | 1.1 |
| | F | | 19,900 | 233,000 | 1.4 | 0.9 | 2.4 | 1.5 |
| 9M dog | M | | 30,000 | 606,000 | 2.2 | 2.3 | 3.3 | 3.4 |
| | F | | 22,500 | 383,000 | 1.6 | 1.4 | 2.5 | 2.2 |

AUC: area under the plasma concentration time curve; AUC<sub>0-24h</sub>: area under the plasma concentration time curve from administration to 24 h; A/H: animal/human ratio; C<sub>max</sub>: maximum plasma concentration; F: female; M: male; NOAEL: no observed adverse effect level; qd: once daily.

## Combination of JNJ-3989 and JNJ-6379

A 1-month repeat-dose combination toxicity study of JNJ-6379 and JNJ-3989 was conducted in male and female Sprague-Dawley rats. JNJ-6379 (in PEG400 + 10% PVP-VA) was administered daily via oral gavage at colomy/kg, alone or in combination with JNJ-3989 (in phosphate-buffered saline) which was administered weekly via SC injections a colomy/kg. In addition, colomy/kg JNJ-3989 (SC, weekly) was dosed as well in a monotherapy group. Control animals received both vehicles via the respective routes.

The data showed that weekly SC injections with JNJ-3989 a CCI mg/kg in combination with daily administration of JNJ-6379 at CCI mg/kg (oral) for one month were well tolerated with no clinical signs or treatment-related mortality. Changes in clinical pathology and histopathology were mostly similar to the findings for the monotherapy groups dosed with JNJ-6379 at CCI mg/kg (oral) alone or with JNJ-3989 at CCI mg/kg (SC) alone. The only synergistic changes included a slight decrease in body weight (gain) at CCI mg/kg, in food consumption at CCI mg/kg, and a further decrease in lymphoid cellularity in the thymus of females at CCI mg/kg. These alterations were minor and non-adverse in nature. Based on these results, the NOAEL was

<sup>&</sup>lt;sup>a</sup> 250 mg JNJ 6379 qd for 28 days (Study 56136379HPB1001).

Ratio of the total C<sub>max</sub> or AUC corrected for species difference in plasma unbound fraction. Calculation: [animal C<sub>max</sub> or AUC<sub>0-24h</sub> x human free fraction].

A dose of mg eq./kg/day in male rats is considered to be above the NOAEL due to kidney findings in male rats, which are likely elevant for human.

The plasma C<sub>max</sub> of 13,600 ng/mL and AUC<sub>0-24h</sub> of 180,000 ng.h/mL in male rats at 100 mg eq./kg/day corresponds to an unbound C<sub>max</sub> of 1,754 ng/mL and AUC<sub>0-24h</sub> of 23,220 ng.h/mL (fraction unbound rat plasma 12.9%). This unbound plasma exposure will be achieved in humans at a total plasma C<sub>max</sub> of 22,784 ng/ml and AUC<sub>0-24h</sub> of 301,558 ng.h/mL (fraction unbound in human plasma 7.7%).

considered to be CC mg/kg. Maximum plasma concentration ( $C_{max}$ ) and AUC<sub>0 24h</sub> values for JNJ-6379 in males were 13,200 ng/mL and 181,000 ng·h/mL, and for females 15,500 ng/mL and 206,000 ng·h/mL, respectively, after 1 month of treatment. The mean  $C_{max}$  and AUC<sub>0 24h</sub> values for analyte JNJ-3924 in males were 20,900 ng/mL and 160,000 ng·h/mL, and for females 21,300 ng/mL and 125,000 ng·h/mL, respectively. For analyte JNJ-3976, the mean  $C_{max}$  and AUC<sub>0 24h</sub> values in males were 35,200 ng/mL and 258,000 ng·h/mL, and for females 35,300 ng/mL and 201,000 ng·h/mL, respectively.

A 3-month combination toxicity study of JNJ-3989 and JNJ-6379 is ongoing, preliminary data is available. In this study, JNJ-3989 was initially administered weekly (ie, a total of 6 doses) and monthly thereafter, via SC injections at dose levels o and monthly thereafter, via SC injections at dose levels o and monthly data is combination with JNJ-6379, and at 180 mg/kg for the monotherapy group. JNJ-6379 was administered daily via oral gavage at a dose level of mg/kg in the monotherapy and combination groups. Control animals received both vehicles via the respective routes.

No test article-related mortalities were noted among animals dosed with JNJ-6379 alone, JNJ-3989 alone, or with JNJ-6379 + JNJ-3989 at mg/kg. One male receiving JNJ-3989 alone at mg/kg died on Day 45, after a rapid change in its clinical condition. The death of this animal was considered to reflect an acute stress response without a relationship to the test article. One accidental death due to a possible gavage error was noted among the toxicokinetic animals in the mg/kg combination group. No bone marrow abnormalities were seen in these 2 animals.

One male rat dosed at company mg/kg JNJ-6379/JNJ-3989 was euthanized on Day 24 after showing severe clinical signs in the morning (decreased activity, erected fur, pallor, and cold to touch). No clinical signs were noted for this animal until Day 23, and body weight and weight gain were unaffected during the first 3 weeks of the study. The cause of moribundity was considered to be a markedly decreased hematopoietic cellularity of the bone marrow with pancytopenia, including markedly reduced platelet counts and consequent hemorrhages and blood loss. A relation to the treatment with JNJ-6379 and/or JNJ-3989 cannot be excluded.

Clinical pathology analysis in this rat revealed a marked decrease in white blood cells (WBCs) (neutrophil, lymphocyte, and monocyte counts), marked decreases in red blood cell (RBC) mass parameters (hemoglobin, hematocrit, and RBC count) including reticulocyte count, and platelet count. There was a mildly increased fibrinogen concentration and mildly prolonged prothrombin time. Other clinical pathology findings were observed for this animal, but they are not related to the bad condition and euthanasia.

At necropsy, the rat showed dark red discoloration/dark red foci in a wide variety of organs and tissues, and dark red material in the abdominal cavity adhered to the spleen (freshly clotted blood). This correlated to minimal to marked hemorrhages in multiple tissues, including brain.

At microscopic examination, the bone marrow of this animal showed markedly decreased cellularity of hematopoietic tissue. Based on the morphology of the remaining hematopoietic tissue and the absence of necrosis, this bone marrow finding was considered not acute but rather subacute or subchronic in nature. In absence of pre-values or earlier time points for hematology, it was not

possible to define the onset of the initiating event. Minimal to marked acute hemorrhages were noted in a wide range of tissues. Some other microscopic findings unrelated to the event were identified.

Altogether, the decreased cellularity of hematopoietic tissue in the bone marrow and the hematology/coagulation data indicate that reduced hematopoiesis resulted in decreases in WBC, reticulocyte, and platelet counts. The hemorrhages were interpreted to be the result of a deficit in primary hemostasis, consistent with the markedly reduced platelet counts. None of the remaining animals of this study showed decreased cellularity of the bone marrow.

In addition to the changes described above, decreased platelet counts were seen in females at and column mg/kg JNJ-6379/JNJ-3989. However, the decrease in platelet counts for these groups was mild, similar across animals within the groups and to those seen in a previous 1-month combination toxicity study with JNJ-6379/JNJ-3989, and not accompanied by other cytopenia nor bone marrow abnormalities. The decrease in platelet counts for these groups are likely caused by a different mechanism than for the male rat that was euthanized on Day 24, as described above.

No relevant changes on urinary biomarkers were detected in male and female rats given JN-6379 at CCI mg/kg/day (clusterin, albumin, ß2-microglobulin, Kidney Injury Molecule-1 [KIM-1], Neutrophil Gelatinase Associated Lipocalin [NGAL] and cystatin-C).

Based on the observation of pancytopenia in 1 rat and a mild platelet decrease in the combination groups in the 3-month combination toxicity study, the sponsor is implementing additional monitoring of significant on-treatment hematologic changes in clinical studies with dosing longer than 4 weeks (see Section 8.5.6.5). However, no significant abnormalities of hematologic parameters have been observed in clinical studies to date.

For further information, refer to the IBs and addenda. 14 16,39

# 2.2.1.2. Combination of JNJ-3989 or JNJ-6379 with Entecavir, Tenofovir Disoproxil, or Tenofovir Alafenamide

There is no common target organ between JNJ-6379 or JNJ-3989 and entecavir (ETV).<sup>23</sup> The single common toxicity target organ between JNJ-6379, JNJ-3989, and tenofovir disoproxil or tenofovir alafenamide (TAF) is the kidney.

In the chronic rat studies with JNJ-3989, slight alteration of the renal tubular epithelium was characterized by basophilic stippling and/or microvacuolation of the cytoplasm of renal tubules in the outer cortex in rats. These findings were not considered toxicologically meaningful since they were related to compound accumulation, there was no evidence of cellular damage (degeneration/necrosis) and there were no correlated clinical pathology indicators of changes in renal function. These kidney findings have been observed in both the 2-week and 6-month studies and did not worsen over time. No kidney findings were observed in monkeys.

In the chronic rat study (6 months) with JNJ-6379, retrograde nephropathy, secondary to papillary or pelvic calculi/precipitates, was noted in male rats but not in dogs or female rats. This finding is

mainly due to precipitation or calculi formation in distal parts of the kidney/lower urinary tract and is of limited relevance to man, due to differences in urinary composition and functional anatomy between (male) rats and humans. In general, compounds or metabolites of low solubility and high renal clearance may cause concretions in the kidneys/ urinary tract, especially at high doses, as the urine concentrates in the distal nephron and supersaturation of the compound can occur. Urinary pH, proteins and osmolality can also influence the formation of urinary concretions. Male rat urine normally has a high concentration of protein and high osmolality. In addition, rats may be predisposed to retrograde nephropathy because they are known to experience spontaneous urine reflux during micturition or urinary bladder contraction, and this reflux phenomenon can be increased or exacerbated by treatment induced obstructions. The retrograde nephropathy in male rats correlated with increased urea and creatinine in plasma and with urinary changes (red/brown discolored urine, increased volume, decreased pH, presence of blood and white and RBCs in sediment).<sup>3,32</sup> No kidney findings were observed in dogs.

Although both compounds (JNJ-3989 and JNJ-6379) showed histological kidney findings in the rat, the primary anatomical location, mechanism and severity are different. For JNJ-3989 the renal findings are without anticipated clinical or clinicopathological consequences and located in the proximal part of the nephron (outer cortex) and intracellular (not in the tubular lumen). For JNJ-6379, the main findings are restricted to male rats and initiate in distal parts of the kidney (renal pelvis/ papilla) and/or in the lumen of the lower urinary tract with secondary more proximal changes due to reflux.

For tenofovir disoproxil, renal tubular epithelial karyomegaly was observed in rats, dogs, and monkeys.<sup>24</sup> In dogs, the species most sensitive to tenofovir disoproxil-related effects on the kidney, additional microscopic alterations following chronic administration of tenofovir disoproxil (10 mg/kg/day for 42 weeks) included individual tubular cell necrosis, tubular dilatation, tubular degeneration/regeneration, pigment accumulation, and interstitial nephritis. This was associated with biochemical changes such as slight elevation in serum creatinine, glucosuria, proteinuria, and increased urine volume. The incidence and severity of nephrotoxicity was dose-related. Effects were reversible following cessation of treatment. In Rhesus monkeys, biochemical and/or histopathologic evidence of nephrotoxicity was observed at high doses. In rats, slight elevations in serum creatinine were observed without any histopathology correlation.

For TAF, minimal renal cortical tubular karyomegaly and/or basophilia was seen in rats and dogs. In addition, minimal renal cortical tubular degeneration/regeneration were reported in dogs. No renal findings were reported in monkeys.<sup>6</sup>

Based on the available toxicology data, there are no specific concerns about additive or synergistic toxicities in the kidney when JNJ-6379 or JNJ-3989 are combined with ETV, tenofovir disoproxil or TAF.

## 2.2.1.3. Combination of JNJ-3989 with PeglFN-α2a

A 3-month combination toxicity study of JNJ-3989 and PegIFN-α2a (Pegasys®) was conducted in male and female Cynomolgus monkeys (Study TOX14273). JNJ-3989 was administered at or mg/kg (SC, monthly) in combination with PegIFN-α2a at 0.015 mg/kg (SC, twice weekly). In addition, mg/kg JNJ-3989 (SC, monthly) or PegIFN-α2a (0.015 mg/kg; SC, twice weekly) were dosed in monotherapy groups. The study was conducted in monkeys as the toxicity profile of both PegIFN-α2a and JNJ-3989 were known in monkeys (rat studies were not performed with PegIFN-α2a).

There were no test item-related mortalities. JNJ-3989 (alone or combined with PegIFN- $\alpha$ 2a) was well tolerated and did not induce effects on clinical signs, body weight, food consumption, ophthalmoscopic examination, electrocardiology evaluation, coagulation, clinical chemistry or urinallysis parameters, as well as organ weight and macroscopic examination.

Transient local reactions (edema and erythema) were observed at the administration site a and/or commg/kg JNJ-3989. These reactions were also observed with PegIFN-α2a alone and incidentally in control females (erythema only). They were not correlated with microscopic findings.

Administration of JNJ-3989 alone or combined with PegIFN- $\alpha$ 2a elicited minimal to mild, transient (on Day 30 only), non-dose-related increases in neutrophils and total WBCs. Similar findings were observed in the group administered 0.015 mg/kg PegIFN- $\alpha$ 2a alone.

The combination of JNJ-3989 with PegIFN- $\alpha$ 2a did not induce any further effects on biomarkers (interferon gamma inducible protein 10 and interferon alpha) than the increases observed with PegIFN- $\alpha$ 2a treatment alone on Day 1.

JNJ-3989-related microscopic findings were observed in the lymph nodes (minimal to mild vacuolation of macrophages) at  $\geq$ 60 mg/kg and in the liver (minimal hypertrophy of Kupffer cells) at CCI mg/kg in single agent and combination groups. The microscopic changes were comparable between the animals administered with JNJ-3989 alone or combined with PegIFN- $\alpha$ 2a indicating an absence of synergistic effect.

Systemic exposure to JNJ-3924 and JNJ-3976 in plasma was similar after single and repeated dosing following administration of JNJ-73763989 alone or combined with reference item PegIFN- $\alpha$ 2a.

In conclusion, the intermittent SC administration of JNJ-3989 up to  $\Box$  mg/kg given alone or combined with PegIFN- $\alpha$ 2a for 3 months was well tolerated in Cynomolgus monkeys at up to  $\Box$  mg/kg. Treatment only induced transient local reactions at the injection site, transient hematological changes and microscopic findings in liver and lymph nodes, all considered as non-adverse. In addition, the administration of PegIFN- $\alpha$ 2a in combination with test item did not amplify any toxicological effect. Based on these results, there were no additive or synergistic effects on the toxicity profile and no drug-drug interactions when JNJ-3989 is combined with PegIFN- $\alpha$ 2a.

For further information, refer to the latest version of the IB and IB addendum for JNJ-3989<sup>15,16</sup>.

## 2.2.1.4. Combination of JNJ-6379 with PeglFN-α2a

As there is no appropriate species for studying the combination of JNJ-6379 with PegIFN- $\alpha$ 2a, an in vitro study on human bone marrow derived erythroid and myeloid progenitors using colony forming assays was done. JNJ-6379 (5-100  $\mu$ M) and PegIFN- $\alpha$ 2a (Pegasys<sup>®</sup>, 0.00005-0.1  $\mu$ M) were tested in combination in order to evaluate their potential additive or synergistic effects (study TOX14629).

The IC<sub>50</sub> values of the combination treatment were markedly lower compared to JNJ-6379 alone for all tested concentrations but similar to the values with PegIFN- $\alpha$ 2a alone. When the higher concentrations of PegIFN- $\alpha$ 2a were tested in combination with JNJ-6379, the reduction in colonies was mainly due to the strong toxicity of PegIFN- $\alpha$ 2a at these concentrations.

Comparing the predicted (adding the percent of reduction of JNJ-6379 and PegIFN- $\alpha$ 2a alone) and the actual percent reduction in colonies relative to the solvent control, it became clear that there were only minimal differences, pointing more to an additive effect and not a synergistic effect when JNJ-6379 and PegIFN- $\alpha$ 2a were combined.

#### 2.2.2. Clinical Studies

#### 2.2.2.1. JNJ-3989 and JNJ-6379

#### JNJ-3989

Clinical data on pharmacokinetics (PK), efficacy, and safety of JNJ-3989 are available from the ongoing Phase 1/2a AROHBV1001 study with a data cut-off date of 29 October 2019. All dosing with JNJ-3989 has been completed and ongoing participants are in the follow-up. Twenty adult healthy participants have received single SC injections of JNJ-3989 (35, 100, 200, 300, and 400 mg) and 84 adult chronic HBV-infected participants have received multiple doses of JNJ-3989 (25, 50, 100, 200, 300, and 400 mg), administered as 3 SC injections separated by either 7-day, 14-day, or 28-day intervals. All participants either continued or started ETV or tenofovir disoproxil on Day 1.

JNJ-3989 was generally safe and well tolerated with no deaths, serious adverse events (SAEs) considered at least possibly related to the study intervention, or adverse events (AEs) leading to study intervention discontinuation. All AEs were mild to moderate, with exception of 1 severe blood creatine phosphokinase increased in 1 chronic HBV-infected participant. All reported injection site reactions (ISRs) were mild. Adverse events and laboratory abnormalities were distributed across all dose levels and also occurred on placebo treatment, except for mild ISRs, which were only reported in participants on JNJ-3989 treatment. Most reported laboratory abnormalities were isolated incidents and resolved while on study intervention.

Antiviral-activity data were available for 56 chronic HBV-infected participants who received 3 SC injections of 25 to 400 mg JNJ-3989 every 4 weeks (Q4W).<sup>8,37</sup> In general, mean HBsAg declines reached nadir at Day 113 (ie, 8 weeks after last JNJ-3989). Mean HBsAg levels remained

suppressed (below baseline levels) at least until Day 392 (ie, 9 months after last dose) in a substantial proportion of patients.

#### JNJ-6379

At the time of protocol writing, 126 adult healthy and 41 chronic HBV-infected participants have been dosed with JNJ-6379 in 5 completed Phase 1 studies (56136379HPB1001, 56136379HPB1002, 56136379HPB1003, 56136379HPB1004, and 56136379HPB1005). In addition, data are available from 148 adult chronic HBV-infected participants in the ongoing Phase 2a study, 56136379HPB2001, also referred to as JADE.

#### Human Pharmacokinetics and Product Metabolism

Single Dose Studies in Healthy Participants

In Study 56136379HPB1001, single ascending doses (25, 50, 150, 300 and 600 mg) of JNJ-6379 (or placebo) were administered under fasting conditions to healthy participants. No major differences were observed in the shape of the mean JNJ-6379 plasma concentration-time curves for the different dose levels. Mean and individual PK profiles showed minimal lag-time. A single rather flat concentration peak was observed in the PK profiles of most participants. Plasma concentrations in the terminal phase declined generally in parallel for all dose levels. The C<sub>max</sub> and AUC from administration to 24 hours (AUC<sub>0.24h</sub>) increased proportionally with dose after single-dose administration of JNJ-6379 doses of 25 mg to 300 mg and less than dose proportionally at the dose of 600 mg. The AUC from administration to last quantifiable sampling point (AUC<sub>0 last</sub>) and the AUC to last sampling point from time zero extrapolated to infinity (AUC<sub>∞</sub>) increased proportionally between the JNJ-6379 25-mg and 600-mg dose levels. Mean values for terminal half-life (t<sub>1/2term</sub>) were comparable for the 25-mg to 300-mg dose levels, and averaged between 93.3 hours and 110.5 hours. For the 600-mg dose group, the average t<sub>1/2term</sub> was 141.3 hours. Mean values for the total apparent oral clearance (CL/F) were comparable for the 25-mg, 50-mg and 150-mg dose level, and appeared to decrease at higher dose levels. Mean values of the apparent volume of distribution were generally comparable for the different dose groups.

In Study 56136379HPB1002, study intervention exposure levels using a novel tablet formulation, containing hydroxypropylmethylcellulose E5 based spray-dried powder, were similar to exposure levels observed in study 56136379HPB1001 using the original formulation, both in fed conditions. The relative bioavailability of new 25-mg oral tablets of JNJ-6379 administered as a 150-mg dose under fasting and fed conditions, and of new 100-mg oral tablets of JNJ-6379 administered as a 300-mg dose under fasting conditions, was assessed in healthy adult participants. Assuming proportionality, based on the geometric mean ratios between the 3x 100-mg dose, fasting (test) and the 6x 25-mg dose, fasting (reference) of the dose-normalized PK parameters,  $C_{max}$  was 21.56% lower for the 100-mg tablet strength compared to the 25-mg tablet strength, and AUC<sub>0 last</sub> and AUC<sub>∞</sub> were similar. The median time to reach  $C_{max}$  ( $t_{max}$ ) was around 1.75 hours when 150 mg JNJ-6379 was dosed as 6x 25-mg oral tablets, and around 3.00 hours when 300 mg JNJ-6379 was dosed as 3x 100-mg oral tablets.

In Study 56136379HPB1005, the oral bioavailability of a single 300-mg dose of JNJ-6379 administered as a 100-mg tablet containing hydroxypropylmethylcellulose-acetate succinate based spray-dried powder (test tablet) was assessed. All 14 healthy adult participants received a 300-mg dose of JNJ-6379 under fasted conditions. Preliminary PK analysis was performed and mean  $C_{max}$  was 3,105 ng/mL, mean  $AUC_{0.72h}$  was 111,286 ng.h/mL and mean  $AUC_{\infty}$  was 280,926 ng.h/mL. The median  $t_{max}$  was around 3.00 hours. These preliminary PK parameter values are comparable to the PK parameters obtained after administration of JNJ-6379 formulated as hydroxypropylmethylcellulose E5 based spray-dried powder tablet.

## Multiple Dose Studies in Healthy Participants

In Session 7 of Study 56136379HPB1001, participants received 150 mg JNJ-6379 twice daily under fed conditions for the first 2 days of treatment, followed by 100 mg JNJ-6379 qd until Day 12. JNJ-6379 plasma concentrations accumulated during the study (accumulation ratio of approximately 6). The CL/F at steady-state and the  $t_{1/2\text{term}}$  were similar to values observed after single-dose administration, suggesting time-linear PK.

In Study 56136379HPB1004, participants received 250 mg of JNJ-6379 twice daily on Days 6 and 7 (fed conditions), followed by 170 mg qd on Day 8 to 25 in fed conditions (with exception of Day 21). On Day 21, a single dose of JNJ-6379 170 mg and a single dose of drospirenone/ethinylestradiol 3 mg/0.02 mg and a single dose of midazolam 2 mg were administered under fasted conditions. Mean JNJ-6379 C<sub>max</sub> and area under the plasma analyte concentration-time curve over the dose interval (AUC<sub>t</sub>) increased between Day 6 (first dose of JNJ-6379) and Day 20 as JNJ-6379 plasma concentrations accumulated due to the multiple-dose regimen administered in this study. Steady-state was reached before Day 20. Plasma concentration-time profiles of JNJ-6379 were similar those to observed Study 56136379HPB1001.

#### Multiple Dose Studies in chronic HBV-infected Participants

In Sessions 8, 9, 10, 11, and A of Study 56136379HPB1001, treatment-naïve chronic HBV-infected-infected participants were administered multiple-dose regimens (25, 75, 150, and 250 mg) of JNJ-6379 for 28 days. Pharmacokinetics of JNJ-6379 were not markedly different between healthy participants and chronic HBV-infected participants. Mean JNJ-6379 exposures in chronic HBV-infected participants could be predicted from data in healthy participants. The PK data show that exposure of JNJ-6379 in chronic HBV-infected participants is dose proportional and CL/F is constant over time.

#### Food Interaction

Although Study 56136379HPB1001 suggested slightly higher exposure of JNJ-6379 in fed conditions, data from Study 56136379HBP1002 with a higher number of participants showed that there is no food effect on JNJ-6379 exposure, and a preliminary PK analysis from Study 56136379HBP1005 suggests the same.

#### Drug-drug Interaction

Oral contraceptives: When administered simultaneously with 3 mg drospirenone/0.02 mg ethinylestradiol in Study 56136379HPB1004, JNJ-6379 increases the extent of exposure and decreases the CL/F of ethinylestradiol while the peak plasma concentration decreased. In contrast, JNJ-6379 has no clear effect on the extent of exposure and CL/F of drospirenone, a cytochrome P450 (CYP)3A4 sensitive progestin: peak plasma concentration decreased while no change in exposure and apparent clearance was observed. Consequently, oral contraceptives are still considered to be effective when administered simultaneously with JNJ-6379. However, as a precaution to avoid high exposure to ethinylestradiol, ethinylestradiol-containing contraceptives are only allowed if the ethinylestradiol content is ≤20 μg.

*Midazolam:* In Study 56136379HPB1004, coadministration of 170 mg JNJ-6379 qd with oral midazolam as a CYP3A4 probe substrate showed a reduction of 41.7% in  $C_{max}$  and 53.9% in AUC of midazolam, implying that JNJ-6379 may induce the metabolism of CYP3A4 sensitive substrates.

## Efficacy Studies

Antiviral activity data are available from Part II of Study 56136379HPB1001 (final analysis, 57 treatment-naïve participants treated with multiple-dose regimens of 25 to 250 mg JNJ-6379 qd for 28 days, unblinded). Available antiviral activity data for 4 weeks of treatment with JNJ-6379 in this study showed potent HBV DNA and RNA reductions but no changes in HBsAg, indicating that longer treatments are needed.

Interim efficacy data are available from the Phase 2a JADE study. Interim analysis (IA) 2 (cut-off date: 8 February 2019) includes Week 12 data from 64 chronic HBV-infected participants not treated at screening of whom 26 received 75 mg qd JNJ-6379 monotherapy (open-label) and 38 received 75 mg qd JNJ-6379 or placebo in addition to an NA (blinded). Interim analysis 2 also includes unblinded Week 24 data from 44 virologically suppressed chronic HBV-infected participants of whom 33 received 75 mg qd JNJ-6379 and 11 received placebo in addition to an NA. Interim analysis 3 (cut-off date: 7 March 2019) includes blinded Week 12 data from 40 virologically suppressed chronic HBV-infected participants who received 250 mg qd JNJ-6379 or placebo in addition to an NA.

The 12-week interim efficacy data in currently not treated participants on 75 mg JNJ-6379 monotherapy showed a mean reduction from baseline of HBV DNA of >3.5 log<sub>10</sub> International Units Per Milliliter (IU/mL) at Week 12. This decline was similar to the mean decline in participants treated with JNJ-6379 or placebo in combination with an NA (data still blinded).

The 24-week interim efficacy data in virologically suppressed participants on 75 mg JNJ-6379 showed that most participants had HBV DNA levels below the limit of quantification at baseline. At 24 weeks of treatment, 5 (23.8%) of 21 participants on JNJ-6379 experienced a mean reduction from baseline in HBV RNA of  $>2 \log_{10} IU/mL$  versus 1 (14.3%) of 7 participants on placebo. Hepatitis B virus RNA levels at Week 24 were undetectable for 21 (100.0%) of 21 participants on

JNJ-6379 and 4 (57.1%) of 7 participants on placebo. No relevant mean changes from baseline in HBsAg and HBeAg were noted so far.

In the monotherapy arm with 75 mg JNJ-6379, 5 of 28 participants (status after IA cut-off date) experienced a virologic breakthrough defined as confirmed on-treatment HBV DNA increase by >1 log<sub>10</sub> from nadir level or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had HBV DNA level below the LLOQ of the HBV DNA assay. All 5 participants with virologic breakthrough had an emerging core amino acid mutation T33N, which is known to confer reduced JNJ-6379 activity in vitro. All 5 participants discontinued JNJ-6379 and started NA treatment. An urgent safety measure was implemented to discontinue JNJ-6379 treatment in all participants in this arm and offer NA treatment. No cases of virologic breakthrough were observed in any of the arms combining JNJ-6379/placebo with NA treatment. A futility rule was implemented in the 250 mg JNJ-6379 monotherapy arm (if ≥1 participant in the 250 mg monotherapy arm experiences virologic breakthrough during the first 24 weeks of treatment, NA treatment will be added to JNJ-6379 treatment as soon as possible for all remaining participants).

In the monotherapy arm with 250 mg JNJ-6379, 1 participant experienced virologic breakthrough (status after IA cut-off date). The participant discontinued JNJ-6379 treatment and started NA treatment at the withdrawal visit, due to meeting non-response criteria. Nucleos(t)ide analog treatment will be added for all remaining participants in the JNJ-6379 250 mg monotherapy arm in accordance with the futility rule mentioned above.

## Safety Studies

Data from 5 completed Phase 1 studies (56136379HPB1001, 56136379HPB1002, 56136379HPB1003, 56136379HPB1004, and 56136379HPB1005) in healthy and chronic HBV-infected participants (N 126 and 41, respectively), indicate that orally administered JNJ-6379 as single doses up to 600 mg or as multiple doses (250 mg twice daily for 2 days followed by 170 mg qd for 18 days or 150 mg twice daily for 2 days followed by 100 mg qd for 10 days) in healthy participants and as multiple doses up to 250 mg for 28 days in chronic HBV-infected participants was safe and well tolerated. No SAEs considered at least possibly related to the study intervention were reported. Most AEs were mild and not considered treatment-related, with no dose-related trends.

Safety data are also available from IAs 2 and 3 conducted for the Phase 2a JADE study, which were mentioned above. There were no deaths, SAEs considered at least possibly related to the study intervention, or AEs leading to discontinuation. Most AEs were grade 1 or 2 in severity. The majority of reported AEs were considered unrelated to JNJ-6379 by the investigator. Grade 2 to 4 AEs considered at least possibly related to JNJ-6379 by the investigator were grade 2 asthenia (3 participants), grade 4 alanine aminotransferase (ALT) increased, grade 2 headache, grade 2 vertigo, grade 3 anemia (corrected to grade 2 by the investigator after the IA cut-off date), grade 2 hypertension, and grade 2 fatigue (all observed in 1 participant each).

Increased cholesterol is considered a laboratory abnormality of interest for JNJ-6379, based on safety review from nonclinical and clinical trials. Cholesterol increased was reported as an AE in

4 (4.1%) participants on JNJ-6379 for the pooled Phase 1 studies, in 1 (2.4%) participant on JNJ-6379 for the Phase 1 study 56136379HPB1005, and in none of the participants in the Phase 2a JADE study.

# Combination of JNJ-3989 and JNJ-6379

Clinical data of triple combination treatment of JNJ-3989, JNJ-6379, and NA are available from the ongoing Phase 1/2a AROHBV1001 study (Cohort 12). Twelve adult chronic HBV mono-infected participants have received 3 SC injections of JNJ-3989 (200 mg Q4W) in combination with oral JNJ-6379 (250 mg qd) and oral NA treatment (ETV or tenofovir disoproxil).

Up to the interim analysis (IA) cut-off date of 29 October 2019, no deaths, SAEs, or treatment-emergent adverse events (TEAEs) leading to study intervention discontinuation were reported. Two (16.7%) participants reported at least 1 TEAE during the treatment phase. The TEAEs (upper respiratory tract infection and hypertension) were of mild severity and considered not related to the study intervention by the investigator.

The triple combination treatment of JNJ-3989, JNJ-6379, and NA is currently being investigated in chronic HBV mono-infected participants in the ongoing Phase 2 clinical studies 73763989HPB2001 (REEF-1, 90 participants in triple combination Arm 1) and 73763989PAHPB2002 (REEF-2, 80 participants in triple combination Arm 1). Up to 48-week hematology data from the ongoing Phase 2 clinical study REEF-1 are available and overall around 5% of the participants experienced AEs or laboratory abnormalities related to hematology, the majority of mild to moderate severity. The hematologic abnormalities resolved on continued JNJ-3989+JNJ-6379+NA treatment. <sup>16</sup>

Since the initial protocol writing, interim results of the REEF-1 and REEF-2 studies had become available. In the primary REEF-1 analysis (Week 48, end of treatment) the mean reduction of HBsAg levels in the triple arm (JNJ-6379+JNJ-3989 100mg+NA) appeared to be less than in the dual arm (JNJ-3989 100mg+NA). More recent interim results of the REEF-2 study (Week 48, end of treatment) confirmed this observation when the effect of JNJ-6379+JNJ-3989 200mg+NA on mean HBsAg level reduction in REEF-2 study is compared to JNJ-3989 200mg+NA in the REEF-1 study. To match with the REEF-2 population, this cross-study comparison focused on the REEF-1 subpopulation of HBeAg negative, virologically suppressed participants with chronic hepatitis B. PK-PD modelling analyses accounting for variability in baseline characteristics further support this observation. Therefore, a negative effect of JNJ-6379 on the HBsAg lowering effect of JNJ-3989+NA is suspected.

# 2.2.2.2. Combination of JNJ-3989 and JNJ-6379 with Entecavir, Tenofovir Disoproxil, or Tenofovir Alafenamide

Entecavir monohydrate is an HBV NA reverse transcriptase inhibitor indicated for the treatment of chronic HBV infection in adults and children at least 2 years of age with evidence of active viral replication and either evidence of persistent elevations in serum aminotransferases (ALT or aspartate aminotransferase [AST]) or histologically active disease. The most common adverse reactions ( $\geq$ 3% of participants) are headache, fatigue, dizziness, and nausea.

There is no common target organ between JNJ-6379 or JNJ-3989 and ETV.<sup>23</sup>

Tenofovir disoproxil (available in several salt forms including tenofovir disoproxil fumarate and tenofovir disoproxil maleate) is a first-generation oral prodrug of the NA tenofovir that is indicated for the treatment of chronic HBV infection in adult and pediatric patients at least 12 years of age. In addition, tenofovir disoproxil in combination with other antiretrovirals is indicated for the treatment of HIV type 1 (HIV-1) infection in adult and pediatric patients at least 2 years of age. The most common adverse reactions (≥10% of participants) are abdominal pain, nausea, insomnia, pruritus, vomiting, dizziness, and pyrexia.

TAF is an ester prodrug of the NA tenofovir that is indicated for the treatment of chronic HBV-infected in adults and that is characterized by a better safety profile than tenofovir disoproxil. The most common adverse reaction ( $\geq 10\%$  of participants) is headache.

The single common toxicity target organ between JNJ-6379, JNJ-3989, and tenofovir disoproxil or TAF is the kidney (see Section 2.2.1.2).

Clinical data on dual combination treatment of JNJ-6379 and NA are available from the ongoing Phase 2a 56136379HPB2001 study (JADE).<sup>14</sup> In participants treated with tenofovir disoproxil, C<sub>trough</sub> concentrations of tenofovir at Week 12 were higher in participants receiving tenofovir disoproxil in combination with JNJ-6379 than in participants receiving tenofovir disoproxil as monotherapy (94.2 [30.0] and 115 [66.0] ng/mL for 75- and 250-mg JNJ-6379, respectively in combination with tenofovir disoproxil, vs 66.8 [37.0] ng/mL as tenofovir disoproxil monotherapy).

Clinical data of triple combination treatment of JNJ-3989, JNJ-6379, and NA are available from the ongoing Phase 1/2a AROHBV1001 study (see Section 2.2.2.1). Dosing JNJ-6379 or JNJ-3989 with NA for 12 weeks, did not show any clinically relevant changes in kidney parameters/glomerular function.

For further information regarding ETV, tenofovir disoproxil, and TAF, refer to the respective currently approved prescribing information.

## Overall Assessment of the Combination Therapy

Based on the points listed below, no clinically relevant drug-drug interactions (DDIs) and no specific concerns about additive or synergistic toxicities in the kidney are expected when JNJ-6379 or JNJ-3989 are combined with ETV, or tenofovir disoproxil, or TAF:

- Available toxicology data, described in Section 2.2.2.1
- In vitro drug transporters
- Metabolic interaction data
- Absence of relevant DDIs in the combination toxicity studies up to 3 months with JNJ-6379 and JNJ-3989
- Absence of synergistic or additive histology findings in the kidney observed in the combination toxicity studies up to 3 months with JNJ-6379 and JNJ-3989

- Available clinical data with JNJ-6379 (JADE study [56136379HPB2001]) up to 48 weeks treatment on the absence of changes in kidney parameters/glomerular function
- Available clinical data of triple combination treatment of JNJ-3989, JNJ-6379, and NA described in Section 2.2.2.1.

In addition, pancytopenia in 1 rat and a mild platelet decrease were seen in the combination groups in the 3-month combination toxicity study (preliminary data, Section 2.2.1). No significant abnormalities of hematologic parameters have been observed in clinical studies to date. The sponsor is implementing additional monitoring of significant on-treatment hematologic changes in clinical studies with dosing longer than 4 weeks (see Section 8.5.6.5). For further information, refer to the IBs and addenda. 14 16,39

## 2.2.2.3. Combination of JNJ-3989 and JNJ-6379 with PeglFN-α2a

PegIFN- $\alpha$ 2a is a covalent conjugate of recombinant alfa-2a interferon that is indicated for the treatment of chronic hepatitis B in adult and pediatric patients at least 3 years of age. In addition, PegIFN- $\alpha$ 2a in combination with other medicinal products is indicated for the treatment of chronic hepatitis C virus (HCV)-infection in adult and pediatric patients at least 5 years of age and not treated before. The most common adverse reactions ( $\geq$ 10% of participants) are anorexia, anxiety, headache, concentration impairment, dyspnea, cough, alopecia, dermatitis, pruritis, dry skin, myalgia, arthralgia, asthenia, pyrexia, and fatigue. For further information regarding PegIFN- $\alpha$ 2a, refer to the currently approved prescribing information.

Treatment with PegIFN-α2a has been associated with decreases in platelet count (common adverse reaction). In the ongoing Phase 1/2a AROHBV1001 study (see Section 2.2.2.1), no effect on platelet count has been observed in the triple combination treatment cohort 12 (JNJ-3989, JNJ-6379, and NA). Of the 84 adult chronic HBV-infected participants that received 3 subcutaneous injections of JNJ-3989, 6 participants developed grade 1 platelet reduction with no general trend towards a continuous decline. For JNJ-6379, no effect on platelet count has been observed in the ongoing Phase 2a study 56136379HPB2001 (JADE) for the 189 adult chronic HBV-infected participants that were dosed with JNJ-6379.

Based on preclinical data, a potential common toxicity target organ between JNJ-6379, JNJ-3989, and PegIFN- $\alpha$ 2a is the bone marrow (see Section 2.2.1.1). Bone marrow suppression is a known side effect of PegIFN- $\alpha$ 2a (rare).

No pharmacokinetic (PK) interaction is expected between JNJ-3989 and PegIFN- $\alpha$ 2a based on the known pharmacologic profile of JNJ-3989<sup>15,16,41</sup>.

At the time of protocol amendment 4 writing, no clinical data on the combination of JNJ-3989 and JNJ-6379 with PegIFN-α2a are available. Nonclinical studies to investigate the effect on platelet count decreases and on bone marrow in non-human primates (JNJ-3989) and bone marrow stem cells (JNJ-6379) were completed, and results are summarized in Section 2.2.1.1.

#### 2.3. Benefit-Risk Assessment

More detailed information about the known and expected benefits and risks of JNJ-3989 and JNJ-6379 may be found in the respective IBs and addenda. 14 16,39

For the benefit-risk evaluation of ETV, tenofovir disoproxil, TAF, and PegIFN- $\alpha$ 2a refer to the respective prescribing information.

JNJ-6379 was initially part of the study intervention but has been removed as study intervention with the implementation of an urgent safety measure, as described in Protocol Amendment 5. Emerging data from the REEF-1 and REEF-2 studies resulted in an unfavorable benefit-risk balance of JNJ-6379 in combination with JNJ-3989+NA, compared to JNJ-3989+NA alone. Therefore, the Sponsor decided to discontinue treatment with JNJ-6379 in all ongoing clinical studies effective immediately. Participants who were on treatment with JNJ-6379 were contacted and requested to stop taking JNJ-6379, while continuing treatment with NA, JNJ-3989 and PegIFN-α2a. For newly enrolled participants, JNJ-6379 was taken out of the treatment regimen. For completeness, the benefit-risk assessment for JNJ-6379 is still included in this section.

## 2.3.1. Benefits for Study Participation

#### 2.3.1.1. Known Benefits

The clinical benefit of JNJ-3989 and JNJ-6379 remains to be established.

#### 2.3.1.2. Potential Benefits

Results from clinical studies with JNJ-3989, JNJ-6379, NAs, and optional PegIFN-α2a may be useful for the development of a novel therapeutic approach for chronic HBV infection.

The combination of JNJ-6379 and JNJ-3989 on a background of NAs would target different stages of the viral life cycle. While NA treatment reduces HBV DNA to levels close to or below the LLOQ of the HBV DNA assay, HBV replication is not completely inhibited, resulting in replenishment of the cccDNA pool. The addition of JNJ-6379, which targets the HBV capsid assembly ("primary" MoA) and the de novo cccDNA formation ("secondary" MoA), is expected to block HBV replication more profoundly by inhibiting formation of HBV RNA and DNA containing particles, and to inhibit de novo cccDNA formation, ultimately leading to reduction in cccDNA levels/transcriptional activity and HBsAg seroclearance ("intensified viral suppression"). The addition of JNJ-3989 to an NA, or to JNJ-6379 in combination with an NA, is expected to intensify viral suppression (further) by downregulating levels of the HBV DNA precursor pgRNA. In addition, JNJ-3989 reduces levels of all viral proteins including HBsAg, which is known to interfere with the host immune responses. 7,20,34 By acting on both viral replication and by reducing barriers to the host immune-responses, higher functional cure rates may be achieved.

The addition of short-term PegIFN- $\alpha$ 2a (for 12 or 24 weeks) to the regimen at a time when HBsAg is already significantly reduced or eliminated, may lead to further improvement of the immune response (such as reactivation of NK-cells and further activation of endogenous HBV-specific T-cells) and ultimately could lead to immune control of HBV (ie, functional cure). In addition,

PegIFN- $\alpha$ 2a has shown to have direct antiviral effects on HBV which could also contribute to the efficacy of the regimen. By adding short-term PegIFN- $\alpha$ 2a to the regimen, higher efficacy may be achieved.

# 2.3.2. Risks for Study Participation

#### 2.3.2.1. Known Risks

No known risks associated with JNJ-3989 or JNJ-6379 have been identified from clinical observations so far in the Phase 1 and 2 studies. Injection site reactions were identified as adverse drug reactions for JNJ-3989.

The side effect profile of PegIFN- $\alpha$ 2a is well established and includes, but is not limited to, neuropsychiatric, autoimmune, ischemic, ophthalmologic, hematological, and infectious disorders. Exacerbations of hepatitis during hepatitis B therapy are common and characterized by transient and potentially severe increases in serum ALT. Marked increases in ALT were sometimes accompanied by bilirubin elevation and other liver test abnormalities. In many, but not all cases, these disorders resolve after stopping PegIFN- $\alpha$ 2a therapy. For a full list of known risks for PegIFN- $\alpha$ 2a, refer to the respective prescribing information.

#### 2.3.2.2. Potential Risks

All therapies have the potential to cause adverse experiences. In addition, the discontinuation of NA treatment bares a risk of hepatitis B flares.

Patients with positive HBV DNA and positive HBsAg can always experience increases in liver transaminases which may indicate immune activation and may result in the reduction of viral parameters such as HBV DNA and/or HBsAg. Whether this occurs at higher frequency during or after treatment with JNJ-6379 and JNJ-3989 is not known.

Please refer to Section 2.2 for details on the safety results in the studies conducted to date.

## **2.3.2.2.1.** Potential Risks for JNJ-3989

#### **ALT Elevations**

ALT elevations are considered an important potential risk for JNJ-3989. Two distinct patterns of ALT elevations have been observed in participants receiving JNJ-3989: a rapidly rising and resolving ALT elevation or a more sustained pattern of ALT elevation. The latter has been observed in HBV/HDV co-infected participants in study 73763989HPB2004 during double-blind treatment phase. A causal association of ALT elevations with JNJ-3989 has not been confirmed and the underlying mechanism for ALT elevations being more frequent in the context of HBV/HDV co-infection is not yet understood. <sup>16</sup>

## **Reproductive Risks and Pregnancy**

In the EFD studies, JNJ-3989 was not teratogenic in rats and rabbits. The fertility in male and female rats is not impacted with JNJ-3989 up to a dose of CCI mg/kg/week.

Based on the difference in metabolic pathways and in vitro data indicating absence of impact of JNJ-3989 on CYP enzymes and transporters, no clinically relevant interactions are anticipated between JNJ-3989 and oral contraceptives.

## **Potential Genotoxicity**

JNJ-3989 is considered to be devoid of genotoxic activity. Nonclinical carcinogenicity studies have not been conducted.

#### Other Potential Toxicity/Events of Special Interest

JNJ-3989 is considered non-cytotoxic, did not activate human platelet aggregation, did not activate the innate immune system to a significant degree in vitro, and did not activate complement in vitro.

Hematologic abnormalities are an event of special interest for JNJ-3989 and JNJ-6379 based on animal studies (refer to Section 2.3.2.2.2 for further information).

#### **Viral Resistance**

Treatment with JNJ-3989 may lead to viral resistance, but resistance to JNJ-3989 is not anticipated to impact treatment with other small interfering RNAs (siRNAs). Using these agents in combination, especially in combination with ETV or tenofovir is expected to minimize the risk of emerging resistant viral variants.

#### 2.3.2.2.2. Potential Risks for JNJ-6379

Since the initial protocol writing, interim results of the REEF-1 and REEF-2 studies had become available. The data suggested that JNJ-6379 has a negative impact on the HBsAg lowering effect of JNJ-3989+NA (see Section 2.2.2.1). In addition, there were new insights in the adverse renal profile of JNJ-6379 (see below). Taken together, it was concluded that JNJ-6379 had an unfavorable benefit-risk balance in combination with JNJ-3989+NA, compared to JNJ-3989+NA alone. Therefore, the Sponsor decided to discontinue treatment with JNJ-6379 in all ongoing clinical studies effective immediately. For completeness, the potential risks for JNJ-6379 are still described in this section.

#### **Reproductive Risks and Pregnancy**

In the fertility study in females, early embryonic development was affected: an increase in pre- and post-implantation loss, reduction in implantation and live fetuses at common eq./kg/day. The fetal loss seen during the early stages of pregnancy was considered the result of low hormone levels (decreased luteinizing hormone, progesterone, estradiol) induced by treatment with JNJ-6379.

In the EFD studies, JNJ-6379 was not teratogenic in rats and rabbits.

In the EFD study in rats, fetal weights at CCI mg eq./kg/day were lowered, and there was retarded ossification from CCI mg eq./kg/day onwards. The NOAEL for EFD was considered to be CCI mg eq./kg/day. At this dose, the AUC<sub>0 24h</sub> was 84,000 ng.h/mL and the  $C_{max}$  was 5,190 ng/mL.

In the EFD study in rabbits, the NOAEL for EFD was considered to be the highest dose tested, ie, occluding eq./kg/day. At this dose, the AUC<sub>0.24h</sub> was 99,200 ng.h/mL and the C<sub>max</sub> was 6,880 ng/mL.

## **Potential Genotoxicity**

JNJ-6379 was not genotoxic in the in vitro and in vivo tests.

JNJ-6379 did not affect male or female fertility. Carcinogenicity studies are not yet conducted.

## Other Potential Toxicity/Events of Special Interest

Based on nonclinical findings in rats and dogs and based on clinical findings, increased cholesterol was identified as a laboratory abnormality of interest.

Renal complications are considered an event of special interest for JNJ-6379. Immediate treatment-emergent decrease in mean eGFR, which was initially observed in the JADE study, has also been observed in both JNJ-6379 treatment arms in the ongoing REEF-1 study. The eGFRcr values remained reduced during treatment, with a fast rebound after end of treatment. The eGFR decrease (calculated from serum creatinine) may be an anomaly due to JNJ-6379 possibly interfering with tubular excretion of creatinine via inhibition of MATE-1 transporter.<sup>39</sup> This hypothesis was supported by the absence of a pattern of increased biomarkers of proximal tubulotoxicity (the beta-2microglobulin/creatinine and the retinol binding protein/creatinine ratios), suggesting that the eGFRcr reduction was due to transporter inhibition at the level of creatinine excretion from the proximal tubule rather than renal toxicity.

Emerging data from the REEF-2 study became available, confirming the transient pattern of eGFRcr declines but, in addition, showing an increase of the beta-2microglobulin/creatinine and the retinol binding protein/creatinine ratios in some participants when TDF was continued and combined with JNJ-6379+JNJ-3989. These new data are suggesting that JNJ-6379 in combination with TDF may contribute to renal tubulo-toxicity.

Hematologic abnormalities are considered an event of special interest for JNJ-3989 and JNJ-6369. Mild thrombocytopenia was observed in recently conducted non-clinical toxicology studies with the combination of JNJ-3989 and JNJ-6379. In addition, in a 3-month combination study with 80 rats, 1 rat developed pancytopenia related to bone marrow depletion after 23 days of dosing. Previously, in a 9-month dog study in 24 dogs treated with JNJ-6379 alone, pancytopenia which correlated with a marked increase in plasma cell-like cells in the bone marrow was observed in 1 dog after 60 days of dosing. Refer to Section 8.5.6.5. A minor additive effect was observed in vitro in human bone marrow derived erythroid and myeloid progenitors when combining JNJ-6379 and Peg-IFN- $\alpha$ 2a. <sup>14</sup>

#### **Viral Resistance**

Treatment with JNJ-6379 may lead to emergence of viral variants with reduced susceptibility or resistance to JNJ-6379. Based on nonclinical data, these variants remain susceptible to tenofovir and ETV but might affect treatment options with CAMs in the future. All 5 participants with virologic breakthrough in the JADE study who received 75 mg JNJ-6379 monotherapy, had an

emerging core amino acid mutation T33N, which is known to confer reduced JNJ-6379 activity in vitro (see Section 2.2.2.1 for the results of the IAs).

## **Drug-drug Interactions**

Based on results from DDI study 56136379HPB1004 investigating the potential effect of coadministration of JNJ-6379 with oral contraceptives, it is not anticipated that the efficacy of oral contraceptives will be impacted during coadministration with JNJ-6379 since the exposure of a progestin sensitive to CYP3A4 induction was not significantly affected by coadministration of JNJ-6379. In contrast, it is anticipated that coadministration with ethinylestradiol-containing contraceptives will result in an increased exposure to ethinylestradiol. Therefore, specific requirements on the use of ethinylestradiol-containing contraceptives are included in Section 6.5.

## 2.3.2.2.3. Potential Risks for Tenofovir Disoproxil and PeglFN-α2a

For the general potential risks of tenofovir disoproxil and PegIFN- $\alpha$ 2a refer to the respective prescribing information.

Risks specific for this study design are listed below:

- PegIFN-α2a might increase the immunogenicity of JNJ-3989.
- Combination of PegIFN-α2a with JNJ-3989 and JNJ-6379 might increase the risk of hematologic abnormalities and/or of bone marrow suppression.
- JNJ-6379 might increase tenofovir plasma concentrations.

# 2.3.2.3. Risks Due to Study Procedures

# 2.3.2.3.1. Potential Risks and Inconvenience Associated with the Liver Biopsy Procedures

Percutaneous core liver biopsies and fine needle aspiration biopsies (FNAB) will be performed during this study for research purposes.

The risks and complications related to these procedures will be described in the informed consent form (ICF) and may include:

- Pain and discomfort located at or near the puncture site and radiating upwards toward the right shoulder region, which may last for up to a few hours or rarely days after the procedure.
- Bleeding at the biopsy site.
- Infection and internal bleeding and/or puncture of other internal organs (gall bladder, lung, intestine or kidney) which can lead to serious complications (uncommon 1 in 1000 to 1 in 100) including the need for emergency surgery, blood transfusion, or removal of organs. Deaths directly related to liver biopsy occur rarely (approximately 1 in every 10,000 biopsies).

# 2.3.2.3.2. Potential Risks and Inconvenience Associated with the Optional Leukapheresis Procedure

Participants who provide separate consent may undergo leukapheresis. The risks and complications related to this procedure will be described in the ICF and may include:

- Frequent side effects (~5% of participants): chills, reactions to the citratebased anticoagulant (eg, prolonged bleeding for up to 20 minutes after the procedure), numbness or tingling of the lips, face, or on the fingertips, muscle cramps, abnormal heart rhythm, or metallic taste in the mouth
- Occasional side effects (<5% of participants): bruising or discomfort at the injection sites, pain/numbness in the arm (usually of short duration), tiredness the day following the procedure, weakness, nausea/vomiting, fainting due to decreased blood pressure, pink or red coloration of urine, hemolysis
- Rare side effects (≤1% of participants): superficial inflammation of the vein in the arm that is being used for the procedure which may result in pain, heat, and redness, pulmonary embolism, rapid breathing, chest pain, or cough

## 2.3.3. Benefit-risk Assessment for Study Participation

Based on the available data and proposed safety measures, the overall risk/benefit assessment for JNJ-3989 and JNJ-6379 clinical studies is deemed acceptable for the following reasons:

- At the time of protocol writing, JNJ-3989 was generally safe and well tolerated during the ongoing Phase 1/2a Study AROHBV1001 (see Section 2.2.2). All but one AE were mild or moderate in severity. All ISRs, identified as adverse drug reactions for JNJ-3989, were mild in intensity.
- No clinically significant safety concerns had been raised for JNJ-6379 at the time of initial protocol writing, based on the safety information from studies in healthy adult participants and adult participants with chronic HBV infection. Most observed AEs at that time were mild in severity and considered not related to JNJ-6379 by the investigator (see Section 2.2.2). At the time of Protocol Amendment 5 writing, it was concluded that JNJ-6379 has an unfavorable benefit-risk balance in combination with JNJ-3989+NA, compared to JNJ-3989+NA alone (see Section 2.3.2.2.2). Therefore, the Sponsor decided to discontinue treatment with JNJ-6379 in all ongoing clinical studies effective immediately, as a measure to minimize risk to participants of this and other studies.
- Events of Special Interest are significant AEs that are judged to be of special interest because of clinical importance, known class effects or based on nonclinical signals. Events of Special Interest that will be carefully monitored during the study include ISRs, ALT/AST elevations, renal complications, hematological abnormalities, and events related to cholesterol increase (Section 8.5.6 and Section 8.4.4). In addition, the following toxicities will also be carefully monitored: rash and acute systemic allergic reactions (Section 8.5.7).
- Continued careful assessment of the safety, efficacy, and PK during treatment is included in this study.
- To minimize potential risk and stress to participants, the following measures are in place:

Utilization of selection criteria which exclude participants who may potentially be at higher risk of an AE (see Section 5).

Utilization of withdrawal criteria (see Section 7). If a participant drops out due to withdrawal of consent, he/she retains the option to participate in the safety follow-up procedures.

Following local standard practice the biopsy location will be identified with ultrasound (which will also be used to rule out contraindicating conditions for a biopsy). At the off-treatment biopsy, blood coagulation and platelets will be assessed according to local practice. Prior to the on-treatment biopsy, a recent ( $\leq 1$  week) coagulation and hematology panel and a platelet aggregation test are required, to ensure normal count and function of platelets and normal coagulation parameters. Site selection will be based on their experience in the performance of core liver biopsies and FNABs.

Participants will be monitored closely during the optional leukapheresis. In case of serious complications, the leukapheresis procedure will be stopped immediately. Participants will stay on site for at least 30 minutes after leukapheresis to monitor for potential side effects. Additional safety-related assessments may be performed at the discretion of the investigator and may include additional laboratory tests after the procedure to measure hematologic parameters.

At regular time points throughout the study (see Schedule of Activities), blood samples for biochemistry, blood coagulation, and hematology and urine samples for urinalysis, urine chemistry, and renal biomarkers will be collected. Vital signs (systolic and diastolic blood pressure [SBP and DBP]), pulse rate, and body temperature), height (only at screening), body weight, and electrocardiograms (ECGs) will be recorded throughout the study. Physical examinations will be performed and AEs will be assessed (see Section 8.3, Safety Assessments). Events of Special Interest will be closely monitored (Section 8.5.6, Adverse Events of Special Interest).

Based on pre-clinical and clinical data available today, the combination of JNJ-3989, JNJ-6379, tenofovir disoproxil, and short-term PegIFN- $\alpha$ 2a is considered safe. Data from nonclinical combination toxicity studies showed a minimal additive effect on myeloid and erythroid cells in vitro when combining JNJ-6379 and PegIFN- $\alpha$ 2a (Section 2.2.1.4) and confirmed that combination of PegIFN- $\alpha$ 2a with JNJ-3989 did not induce any synergistic or additive effect in monkeys up to 3 months of treatment (Section 2.2.1.3). Review of 48-week hematology data from the ongoing Phase 2 clinical study REEF-1 (Section 2.2.2.1) did not identify any safety concerns.

The impact of PegIFN-α2a addition to JNJ-3989 on ALT elevations is not known in the context of HBV monoinfection. Strict rules for management of ALT elevation are in place (refer to Section 8.5.6.2, Intervention-emergent ALT/AST Elevations).

An Independent Flare Expert Panel (IFLEP) will be appointed to characterize and adjudicate each ALT flare (see Section 9.6).

After stopping treatment with NA, JNJ-3989, JNJ-6379 (if applicable), and PegIFN- $\alpha$ 2a (if applicable), participants will be monitored closely during the follow-up phase, with frequent follow-up visits and pre-defined NA re-treatment criteria in case of flares (Section 6.6.2).

The post-treatment monitoring and NA re-treatment criteria (Section 6.6.2) were further updated based on findings from a case of post-treatment HBV reactivation with subacute hepatic failure and assessment of additional REEF-2 study data.

JNJ-3989 will be administered using a proper SC technique to decrease the risk of ISRs. Injection site reactions will be managed as outlined in Section 8.5.6.1.

Any clinically significant abnormalities persisting at the end of the study/early discontinuation will be followed up by the investigator until resolution (return to baseline) or until stabilization (to be agreed upon with the sponsor).

## 3. OBJECTIVES AND ENDPOINTS

The following objectives and endpoints will be assessed overall and by study panel:

| | Objectives | | Endpoints |
|---|---|---|---|
| Pri | mary | | |
| • | To assess changes in intrahepatic HBsAg between baseline and on-treatment liver biopsy in response to JNJ-3989-based combination treatment | • | Changes in the proportion of HBsAg positive hepatocytes between baseline and on-treatment Week 40 |
| Sec | ondary | | |
| • | To assess changes in intrahepatic immune response between baseline and on-treatment liver biopsy | • | Changes between baseline and on-treatment liver biopsy in intrahepatic immune response (eg, CD45+ T-cells, CD4+ T-cells, CD8+ T-cells, Natural Killer cells, and dendritic cells) in terms of proportion of cells, cell types, and spatial redistribution |
| • | To assess changes in intrahepatic viral nucleic acids and proteins between baseline and on-treatment liver biopsy | • | Changes from baseline in intrahepatic viral parameters (such as cccDNA, pgRNA, intrahepatic RNA, or HBsAg in terms of copy number, or number of positive cells) |
| | | • | Changes from baseline in intrahepatic cccDNA levels and transcriptional activity (pgRNA/cccDNA ratio) |
| • | To evaluate the efficacy of the study intervention as measured in blood | • | The proportion of participants during the study intervention and follow-up phases with: |
| | | | HBsAg seroclearance at Week 72 (ie, 24 weeks after completion of all study interventions at Week 48) without restarting NA treatment. |
| | | | (Sustained) Reduction, suppression, and/or seroclearance considering single and multiple markers (such as HBsAg, HBeAg, HBV DNA and ALT) |
| | | | HBsAg and HBeAg seroconversion |
| | | | Flares (virologic, biochemical, and clinical) |

| | Objectives | | Endpoints |
|---|---|---|---|
| | | • | Time to first HBsAg seroclearance |
| • | To evaluate the frequency of virologic breakthrough during study intervention | • | Proportion of participants with virologic breakthrough |
| • | To assess HBV-specific T-cell responses | • | Changes from baseline in HBV-specific peripheral blood T-cell responses during the study intervention and follow-up phases |
| • | To evaluate the safety and tolerability of the study intervention | • | Proportion of participants with (S)AEs and abnormalities in clinical laboratory tests (including hematology, blood biochemistry, blood coagulation, urinalysis, urine chemistry, and renal biomarkers), 12-lead ECGs, vital signs, and physical examinations throughout the study |
| • | To evaluate the plasma PK of JNJ-3989 (ie, JNJ-3976 and JNJ-3924) and optionally of JNJ-6379, NA and/or PegIFN-α2a, as applicable | • | Plasma PK parameters of JNJ-3976, JNJ-3924, and optionally of JNJ-6379, NA and/or PegIFN-α2a, as applicable |
| Exp | loratory | 1 | |
| • | To explore the relationship of intrahepatic markers with blood markers (immune and viral) | • | Association between levels and changes in intrahepatic and blood markers |
| • | To explore the association of baseline characteristics and intrahepatic and/or blood (immune and viral) biomarkers at baseline and on/off-treatment with selected on/off-treatment efficacy variables | • | Association of baseline characteristics and baseline and on/off-treatment viral blood markers (such as baseline NA treatment duration, age, and baseline and on/off-treatment HBsAg levels) with selected off-treatment efficacy variables |
| | | • | Association of intrahepatic and blood biomarkers (such as cccDNA levels, T-cell frequency) with selected on/off-treatment efficacy variables |
| • | To explore intrahepatic immune and viral changes at Week 72 and/or during off-treatment flares (only for participants with Week 72 biopsy available) | • | Changes from baseline and on-treatment liver<br>biopsy in intrahepatic immune and viral markers<br>at Week 72 and/or during off-treatment flares<br>(only for participants with Week 72 biopsy<br>available) |
| • | To explore changes in the severity of liver disease | • | Changes in fibrosis (according to Fibroscan liver stiffness measurements) at the end of study intervention (EOSI) and end of follow-up versus screening/baseline* |
| • | To explore the efficacy in terms of changes in HBV RNA and hepatitis B core-related antigen (HBcrAg) levels. | • | Changes from baseline in HBV RNA and HBcrAg levels during study intervention and follow-up phases. |
| • | To explore the relationship between plasma PK parameters (JNJ-3989 [ie, JNJ-3976 and JNJ-3924] and/or JNJ-6379 and/or NA and/or PegIFN-α2a) and selected pharmacodynamic (PD) | • | Relationship between various plasma PK parameters (JNJ-3976 and JNJ-3924, and/or JNJ-6379, and/or NA, and/or PegIFN-α2a) and |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Objectives | Endpoints |
|---|---|
| parameters of efficacy and/or safety, as applicable | selected efficacy and/or safety endpoints, as applicable |
| To explore the HBV genome sequence | The emergence of intervention-associated<br>mutations during the study intervention and<br>follow-up phases |
| | To assess the impact of baseline HBV genome<br>polymorphisms on selected on/off-treatment<br>efficacy variables |

<sup>\*</sup> Only applicable to participants who are enrolled at a site with an on-site Fibroscan device.

Refer to Section 8 for evaluations related to endpoints.

#### **HYPOTHESIS**

As this is an exploratory study, no hypothesis will be tested.

#### 4. STUDY DESIGN

## 4.1. Overall Design

As of Protocol Amendment 5, the study is a Phase 2 single-arm, open-label, multicenter, study to assess intrahepatic and peripheral changes of immunologic and virologic markers in response to a combination regimen containing JNJ-3989 and NA in chronic HBV-infected participants.

With the implementation of an urgent safety measure, as described in Protocol Amendment 5, JNJ-6379 has been removed as study intervention and the study will continue as a single-arm study. Participants randomized to Arm 1 had to stop JNJ-6379 treatment immediately but continue JNJ-3989 + NA treatment.

In addition, participants who provide separate consent may receive optional treatment with PegIFN- $\alpha$ 2a starting after the Week 40 biopsy (or after the optional leukapheresis if applicable) but before the Week 48 visit. The duration (either 12 or 24 weeks) will be at the investigator's discretion.

A target of 24 chronic HBV-infected male and female participants, 18-65 years (inclusive) of age will be enrolled in 2 panels, approximately 12 participants in each panel. Panel 1 will consist of participants who are HBeAg positive and not currently treated and Panel 2 will consist of participants who are HBeAg negative and virologically suppressed by ETV, tenofovir disoproxil, or TAF treatment.

The study will be conducted in 3 phases for all participants: a screening phase (4 weeks), an open-label study intervention phase (48 weeks), and a follow-up phase (48 weeks). If necessary, eg, for operational reasons, the screening phase may be extended up to a maximum of 6 weeks on a case-by-case basis and in agreement with the sponsor. The duration of individual participation will be up to 102 weeks. Note that the follow-up period will be extended for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of

treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation. For those participants, the duration of individual participation may be extended up to 126 weeks.

Prior to Protocol Amendment 5, participants were randomized in a 1:1 ratio within each panel to receive one of the following interventions (ie, treatments) for 48 weeks:

• Intervention arm 1, combination regimen JNJ-3989+JNJ-6379+NA (target of 12 participants):

200 mg JNJ-3989 (SC injection Q4W, with the last injection at Week 44), AND

250 mg JNJ-6379 (tablets qd), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

• Intervention arm 2, combination regimen JNJ-3989+NA (target of 12 participants):

200 mg JNJ-3989 (SC injection Q4W, with the last injection at Week 44), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

#### As of Protocol Amendment 5:

• Participants who were randomized to study intervention with JNJ-6379 prior to Protocol Amendment 5, had to stop JNJ-6379 treatment immediately but will still receive the following interventions (ie, treatments) for 48 weeks:

200 mg JNJ-3989 (SC injection Q4W, with the last injection at Week 44), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

• New participants will enroll without randomization within each panel to receive the combination regimen JNJ-3989 + NA as study intervention for 48 weeks:

200 mg JNJ-3989 (SC injection Q4W, with the last injection at Week 44), AND

NA: ETV, tenofovir disoproxil, or TAF (tablets qd)

In addition, participants who provide separate consent may receive optional treatment with PegIFN- $\alpha$ 2a starting after the Week 40 biopsy (or after the optional leukapheresis if applicable). The duration (either 12 or 24 weeks) will be at the investigator's discretion. This will allow to investigate whether addition of PegIFN- $\alpha$ 2a for 12 or 24 weeks may increase the participant's chance to achieve HBsAg loss.

All participants will complete treatment with JNJ-3989 after a fixed duration of 48 weeks. If the NA treatment completion criteria (outlined in Section 6.6.1) are met based on clinical laboratory tests performed at Week 44, treatment with NA will also be completed at Week 48. In participants not meeting these criteria, NA treatment will continue during the follow-up phase. Participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who have not met NA treatment completion criteria at Week 48 may have NA treatment completion criteria assessed at the end of treatment with PegIFN- $\alpha$ 2a and stop NA if criteria are met.

All participants will be monitored closely during the follow-up phase and, if applicable, should restart NA treatment in accordance with the NA re-treatment criteria (see Section 6.6.2 for more details).

Prior to Protocol Amendment 5, randomization within each panel was stratified by Fibroscan score (<7 kPa vs  $\ge$ 7 kPa). Randomization and stratification are not applicable anymore per Protocol Amendment 5.Safety and tolerability, including (S)AEs, laboratory assessments, ECGs, vital signs, and physical examination, will be assessed throughout the study from the time of signing the ICF until completion of the last study-related activity (see Section 8.4 and Section 8.5).

At Week-1 and Week 40, FNAB samples and core liver biopsy samples will be taken. Additional optional FNAB and/or core liver biopsy samples may be taken (eg, at follow-up Week 24) from participants who provide separate consent (see Section 8.1).

Efficacy will be evaluated using different parameters including HBsAg and HBeAg (see Section 8.2).

Samples for HBV genome sequencing will be taken at the time points indicated in the Schedule of Activities (see Section 8.2.1). Sequencing of samples obtained may be triggered by the sponsor's virologist based on changes in HBV DNA levels observed in each individual participant and the limits of the sequencing assay.

Peripheral blood mononuclear cell (PBMC) samples for immune analyses will be collected at the time points indicated in the Schedule of Activities (see Section 8.3).

The study includes collection of blood samples for exploratory analysis of viral markers (see Section 8.1) and host blood biomarkers at the host RNA, protein, and cell level (see Section 8.10).

All participants will have sparse PK sampling on Day 1 and at Weeks 4, 12, and 24 (and at early withdrawal). All participants who consent to participate in the intensive PK substudy (optional) will undergo intensive PK sampling at Week 4.

A population PK analysis may be performed based on the available data for JNJ-6379, JNJ-3989, and optionally, NA and/or PegIFN- $\alpha$ 2a, potentially in combination with data from a selection of Phase 1 and/or 2 studies. PK parameters in participants undergoing intensive PK sampling will be calculated via noncompartmental methods.

Pharmacokinetic/pharmacodynamic relations may be explored (see Section 8.8).

Host DNA samples will be collected to allow for the identification of genetic factors (see Section 8.9). In addition, host DNA blood samples to allow for epigenetic analyses will be collected.

Human leukocyte antigen (HLA) typing will be performed as indicated in the Schedule of Activities.

In case of premature discontinuation of investigational intervention (before Week 48), follow-up assessments should be obtained until 48 weeks after EOSI unless the participant withdraws consent.

If a participant withdraws before completing the study intervention, the reason for withdrawal (if known) is to be documented in the case report form (CRF) and in the source document. Participants who withdraw consent will be offered an optional safety follow-up visit.

An IFLEP will be appointed for this study (see Section 9.6).

A diagram of the study design is provided in Section 1.2.

## 4.2. Scientific Rationale for Study Design

#### **Study Population**

Patients with chronic HBV infection will be eligible if (1) they are HBeAg positive and not currently being treated or (2) if they are HBeAg negative and virologically suppressed by NA treatment.

Patients with advanced liver fibrosis or liver cirrhosis are excluded, as the goal of the study is to assess the potential of a finite treatment to achieve functional cure, and discontinuation of treatment in patients with cirrhosis is not current practice due to concerns about poor tolerability of liver flares associated with increased viral replication. The safety of the combination regimens evaluated in this study will first be established in patients without liver cirrhosis prior to initiating studies in patients with more advanced liver disease.

### Study Design Change – Protocol Amendment 5

Based on emerging data from the REEF-1 (73763989HPB2001) and REEF-2 (73763989PAHPB2002) studies, the study design has been adapted in Protocol Amendment 5.

In summary, the data from the REEF-1 and REEF-2 studies suggested that JNJ-6379 has a negative impact on the HBsAg lowering effect of JNJ-3989+NA (see details in Section 2.2.2.1) and that JNJ-6379 in combination with TDF may further contribute to renal tubulo-toxicity (see details in Section 2.3.2.2.2). Together, this led to a conclusion of an unfavorable benefit-risk balance of JNJ-6379 in combination with JNJ-3989+NA, compared to JNJ-3989+NA alone. Therefore, the Sponsor decided to discontinue treatment with JNJ-6379 in all ongoing clinical studies effective immediately. Participants currently on treatment with JNJ-6379 were contacted and requested to stop taking JNJ-6379, while continuing treatment with NA, JNJ-3989, and PegIFN-α2a. For newly enrolled participants, JNJ-6379 was taken out of the treatment regimen.

Furthermore, the sponsor decided to make additional changes to the study design because of a severe clinical ALT flare that was reported following discontinuation of NA treatment in a participant who was randomized to the control arm (placebo + placebo + NA) in the REEF-2 study. Discontinuation of NA treatment was following the protocol-defined criteria and in line with recent EASL treatment guidelines<sup>5</sup>. Flares following NA discontinuation are not unexpected, but the

rapid evolution and clinical deterioration seen in this participant who had no history or evidence of liver cirrhosis was unforeseeable. Therefore, to protect the safety of participants, the protocol was amended: more frequent monitoring of participants who discontinued NA treatment during follow-up was included and the NA re-treatment criteria for all participants who discontinued NA treatment were revised.

In addition, the follow-up phase in this study has been extended to ensure that all participants have at least one year of follow-up after NA treatment cessation.

#### Randomization, Stratification Factors and Blinding

Note that randomization and stratification are not applicable anymore per Protocol Amendment 5. Prior to Protocol Amendment 5, randomization and stratification were performed as described below.

Within each of the two study panels (ie, HBeAg positive patients who are not currently being treated and HBeAg negative patients being virologically suppressed by NA treatment), randomization was used to minimize bias in the assignment of participants to intervention arms, to increase the likelihood that known and unknown participant attributes (eg, demographic and baseline characteristics) were evenly balanced across intervention groups, and to enhance the validity of statistical comparisons across intervention arms.

Randomization within each panel was stratified by Fibroscan score (<7 kPa vs  $\ge$ 7 kPa).

As this is an exploratory study, participants will be treated in an open-label fashion. In addition, most relevant assessments will be based on objective markers (biopsy and peripheral immunology) and are not subject to bias from the participants or observers.

### **Criteria for Completion of NA Treatment**

To explore the possibility of finite treatment, all participants who completed the 48-week study intervention will stop all study interventions including NAs at Week 48 if they meet NA treatment completion criteria (described in Section 6.6.1). The treatment completion criteria which take ALT, HBV DNA, HBeAg and HBsAg levels into consideration, have been selected to ensure that only participants with a chance of sustained off-treatment response are allowed to complete all study intervention. Across a range of studies, HBsAg levels below 100 IU/mL are consistently associated with favorable off treatment response. <sup>19,26</sup> The stringent HBsAg cutoff of 10 IU/mL for NA treatment completion was chosen to account for the direct effect of JNJ-3989 on HBsAg levels.

Participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who have not met NA treatment completion criteria at Week 48 may have NA treatment completion criteria assessed at the end of treatment with PegIFN- $\alpha$ 2a and stop NA if criteria are met.

After stopping all study interventions, participants will be monitored closely during the 48-week follow-up phase and should restart NA treatment in accordance with the NA re treatment criteria (see Section 6.6.2, for more details).

## Follow-up Procedures and Criteria for Re-initiation of NA Treatment

The follow-up period will be extended for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation.

To ensure safety of patients during the follow-up phase, an ALT flare management plan is in place, including a high visit frequency for patients after completion of NA treatment (at Week 48), and weekly visits for patients with ALT/AST  $\geq 3x$  upper limit of normal (ULN) and  $\geq 3x$  nadir until stabilization.

Increases in ALT and HBV DNA are frequently seen in patients after discontinuation of NA treatment. These ALT elevations can be reflecting an activation of the host cellular immune response and can as such lead to functional cure. Cases of fulminant HBV reactivation with fatal outcome were described after cessation of NA treatment, but the vast majority of such cases were described in patients with decompensated liver disease at the time of NA discontinuation. These patients are not eligible to participate in the study. Still, a vigilant follow-up of patients during this phase of the study is critical to ensure patient safety. Increases in ALT that are accompanied by signs of decreased liver function, or an HBV DNA value of >100,000 IU/mL (irrespective of confirmation and/or ALT increase), will trigger immediate re-initiation of NA treatment based on protocol-defined NA re-treatment criteria (see Section 6.6.2).

Re-initiation of NA treatment is also required in case of confirmed HBeAg seroconversion (HBeAg positive after it was negative at NA completion), in case of confirmed\* ALT increase (>5x ULN) in combination with increased HBV DNA replication (>2,000 IU/mL), and in case of confirmed\* increased HBV DNA replication at higher levels (>20,000 IU/mL).

### \* At least 4 weeks apart

A post-treatment HBV DNA value of >20,000 IU/mL should trigger re-testing of ALT/AST, HBV DNA, and total and direct bilirubin within a maximum of 7 days from receipt of the data and further repeats as necessary (ie, weekly until HBV DNA returns to <20,000 IU/mL). A post-treatment HBV DNA value of >2,000 IU/mL (but <20,000 IU/mL) should trigger a re-test within 14 days from receipt of the data and further repeats as necessary (ie, every other week until HBV DNA returns to <2,000 IU/mL). A post-treatment ALT value of >5x ULN should trigger re-testing of ALT, AST, ALP, total and direct bilirubin, INR, albumin, and HBV DNA on a weekly basis until ALT and AST levels have returned to <5x ULN. Additional re-testing and/or earlier restarting of NA treatment is at the investigator's discretion, even if the above cut-offs are not yet met.

To avoid delays in decision making, sites are encouraged to run local re-testing in parallel with central re-testing in the situations described above that require more frequent re-testing. Local test results are to be recorded in the CRF and/or source documents, including information on the HBV DNA assay used. In addition, to avoid delays in NA re-treatment, it should be considered to dispense NA to participants who potentially met the NA re-treatment criteria (eg, pending confirmation) and who will not be available to come to the study site immediately at the time the

confirmatory test results will become available. This should ensure that the participant can immediately restart NA treatment if indicated, upon direct confirmation by the investigator.

The decision to re-start NA treatment should take into consideration the dynamics of HBV DNA and/or ALT values and should be discussed with the sponsor. Refer to Section 6.6.2.

NA re-treatment criteria during follow-up are presented graphically in Section 10.12, Appendix 12: NA Re-treatment During Follow-up.

## **Liver Biopsy**

HBV is a hepatropic virus, with the liver being the site of its replication which requires a modulation of intrahepatic immune response to allow the establishment of a chronic persistent infection. Although some of the viral blood markers are well established from a clinical perspective, questions remain on the relationship of these markers with intrahepatic events, such as expression of viral proteins (eg, HBsAg), HBV pgRNA, DNA and cccDNA level and transcriptional activity in the liver, ie, the target organ of HBV infection. Similarly, while assessment of peripheral immune response can provide insights into the HBV related immune response, it is well accepted that a large proportion of the relevant immune responses are enriched and/or restricted to the liver environment. 10,11,29 For example, many HBV specific CD8+ T-cells have a tissue-resident phenotype and innate-like populations such as mucosal associated invariant T (MAIT) cells and Natural Killer cells are enriched with the latter having also a specialized liver-resident component. 11,29

Collecting liver biopsy samples will allow to perform critical assessments of intrahepatic virologic and immune events occurring in response to treatment with JNJ-3989, JNJ-6379 and NA, and to correlate the findings in the liver with treatment response and to viral and immune blood markers. In addition, these analyses are expected to improve the understanding of the molecular mechanisms of the treatment interventions and to provide important insight into the HBV pathology.

Both core liver biopsies and fine needle aspirates will be collected for high dimensional profiling of the liver tissue. The cryopreserved core biopsies will allow characterization of the infected hepatocytes compartment and phenotyping of the major immune cell populations (proportion of cells and spatial distribution). The liver tissue will be used to assess changes from baseline in the proportion of HBsAg positive hepatocytes under therapy. In addition, the liver tissue will also be used to assess other HBV markers in the liver such as, but not limited to, pgRNA, total intracellular HBV RNA and DNA, and HBc. Changes in the quantity and potentially changes in the spatial distribution of these markers (including HBsAg) under JNJ-3989 and JNJ-6379 (if applicable) containing therapy or NA treatment will be assessed. Viral genome (RNA or DNA) sequencing of the samples as well as assessment of HBV viral transcripts and HBV DNA integrants in the host genome may be performed. This will also allow to compare viral parameters assessed in the liver with viral parameters in the blood compartment.
From an immune perspective, both, the innate and adaptive intrahepatic immune compartment will be characterized. These analyses will include cells such as CD4+ T-cells, CD8+ T-cells, CD45+ cells, dendritic cells, and Natural Killer cells. Characterization of infiltrating immune cells will be used for the evaluation of innate and adaptive immune responses, which can be compared to responses in the PBMCs collected during the study.

Fine needle aspirates biopsies will be profiled by single cell transcriptomics approaches to better understand the innate and adaptive immune cells composition and functional status<sup>9</sup> (very few hepatocytes are expected to be collected with fine needle aspirates). Hepatitis B virus-specific T-cells will be one of the main targeted cell populations, detected and sorted by multimers binding assays. Downstream transcriptomic profiling of collected HBV specific T-cells may be performed by T-cell receptor sequencing and RNA sequencing. Similar multimer binding assays approaches might be applied to leukapheresis collected PBMCs, as HBV specific T-cells are present in very low frequency in patients with chronic HBV infection.<sup>9</sup>

Remaining samples may be used for determination of liver JNJ-3989 (ie, JNJ-3976 and JNJ-3924) and/or JNJ-6379 concentrations and/or research on viral and host biomarkers and immune markers at the viral and/or host RNA/DNA, protein, and cell level.

#### **Host DNA and Biomarker Collection**

It is recognized that genetic variation can be an important contributory factor to interindividual differences in intervention distribution and response and can also serve as a marker for disease susceptibility and prognosis. Pharmacogenomic research may help to explain interindividual variability in clinical outcomes and may help to identify population subgroups that respond differently to an intervention. The goal of the pharmacogenomic component is to collect DNA to allow the identification of genetic factors that may influence the efficacy, safety, or PK of JNJ-3989 and JNJ-6379, to identify genetic and epigenetic factors associated with HBV infection, or to develop assays for the study intervention or HBV infection.

Biomarker samples will be collected to evaluate the MoA of JNJ-3989 and JNJ-6379 (if applicable) in combination with NA, help to explain interindividual variability in clinical outcomes, or may help to identify population subgroups that respond differently to an intervention. The biomarker research can be used to address questions related to the safety, PK, and efficacy of the study intervention and HBV infection or to develop assays for the study intervention or HBV infection.

Host DNA (pharmacogenomic) and biomarker samples may be used to help address emerging issues and to enable the development of safer, more effective, and ultimately individualized therapies.

### 4.2.1. Study-Specific Ethical Design Considerations

Potential participants will be fully informed of the risks and requirements of the study and, during the study, participants will be given any new information that may affect their decision to continue participation. They will be told that their consent to participate in the study is voluntary and may be

withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only participants who are fully able to understand the risks, benefits, and potential AEs of the study, and provide their consent voluntarily will be enrolled.

Percutaneous core liver biopsies and FNABs will be performed during this study for research purposes. The risks and complications related to these procedures are described in Section 2.3.2.3. These risks and complications will be described in the ICF and will be clearly explained to potential participants prior to enrollment.

While all participants will receive the study intervention in combination with an approved therapy for HBV infection, some ethical consideration should be given to the fact that participants will not have access to potentially alternative or new effective therapies for the duration of the study (intervention and follow-up phase) since they may not begin any other approved or investigational therapies for treatment of HBV infection during this time. Participants with worsening HBV infection can discontinue the investigational intervention at any time, and the investigational intervention should be discontinued if a participant requires additional therapy for HBV infection.

The total blood volume to be collected is considered to be an acceptable amount of blood to be collected over this time period from the population in this study based upon the standard of the American Red Cross standard blood donation.<sup>1</sup>

#### 4.3. Justification for Dose

The proposed dose and treatment duration are selected to maximize the chance for patients to achieve functional cure and are supported by scientific understanding of available data. For both compounds, doses are selected that are currently being tested in ongoing Phase 2b studies REEF-1(73763989HPB2001) and REEF-2 (73763989PAHPB2002) (ie, 200 mg for JNJ-3989 and 250 mg for JNJ-6379).

**Note:** JNJ-6379 was initially part of the study intervention but has been removed as study intervention with the implementation of an urgent safety measure, as described in Protocol Amendment 5.

#### 4.3.1. JNJ-3989

Clinical data on PK, efficacy, and safety of JNJ-3989 are available from the ongoing Phase 1/2a AROHBV1001 study with a data cut-off date of 29 October 2019. All dosing with JNJ-3989 has been completed and ongoing participants are in the follow-up phase. Twenty adult healthy participants have received single SC injections of JNJ-3989 (35, 100, 200, 300, and 400 mg) and 84 adult chronic HBV-infected participants have received multiple doses of JNJ-3989 (25, 50, 100, 200, 300, and 400 mg), administered as 3 SC injections separated by either 7 day, 14-day, or 28-day intervals. All participants either continued or started on ETV or tenofovir disoproxil on Day 1.

JNJ-3989 was generally safe and well tolerated at all doses. No clinically relevant safety signal was identified.

Antiviral activity data were available for 56 chronic HBV-infected participants who received 3 SC injections of 25 to 400 mg JNJ-3989 Q4W. In general, mean HBsAg declines reached nadir at Day 113 (ie, 8 weeks after last JNJ-3989). Mean HBsAg levels remained suppressed (below baseline levels) at least until Day 392 (ie, 9 months after last dose) in a substantial proportion of patients.<sup>8,37</sup>

A dose of 200 mg JNJ-3989 Q4W is chosen based on the observed decline in HBsAg in study AROHBV1001 at this dose over 3 injections, and the lack of a substantial incremental efficacy response at higher doses.

The Phase 2b study REEF-1 is designed to establish the optimal dose of JNJ-3989. Based on data from the Phase 1/2a study AROHBV1001 with limited treatment duration, 200 mg was selected as the highest dose of JNJ-3989 tested in REEF-1. Until lower doses are proven equivalently effective in REEF-1, additional combination studies with JNJ-3989 and JNJ-6379 are conducted with 200 mg of JNJ-3989.

#### 4.3.2. JNJ-6379

**Note:** JNJ-6379 was initially part of the study intervention but has been removed as study intervention with the implementation of an urgent safety measure, as described in Protocol Amendment 5.

At the time of initial protocol writing, a dose of 250 mg JNJ-6379 qd was chosen for this study.

A dose of 250 mg of JNJ-6379 was being considered to ensure maximal viral inhibition via "primary" MoA (ie, interfering with the capsid assembly process). In addition, it ensured sufficient high exposures to engage the "secondary" MoA (ie, inhibition of de novo cccDNA formation). This dose selection was supported by translational PK/PD analyses and viral kinetic modeling. Analyses of the HBV DNA data from the 4-week 56136379HPB1001 study showed a profound but slightly less substantial reduction of plasma HBV DNA, as a measure of the "primary" MoA, in the 25 mg dose group compared to the 75 mg and higher dose groups, suggesting that for JNJ-6379 maximum effect (E<sub>max</sub>) in terms of HBV DNA inhibition via primary MoA was approached starting from a dose of 75 mg onwards. Since it was not possible to derive the engagement of the "secondary" MoA from the available short term data, the in vitro primary human hepatocyte 90% effective concentration values in the presence of serum proteins obtained for both MoAs were used to translate from the "primary" to the "secondary" MoA.

Participants were to be treated with JNJ-6379 for 48 weeks. Based on the MoA of JNJ-6379, it was expected that continued complete suppression of virus production and de novo cccDNA formation over many months was required to achieve reduction of the transcriptional active cccDNA pool, which was considered a prerequisite for HBsAg reduction and/or seroclearance.

Interim analysis data were at that time available from the ongoing Phase 2a JADE study in which the 250-mg dose was being tested for 48 weeks. Blinded Week 12 data from 40 virologically suppressed chronic HBV-infected participants who received 250 mg qd JNJ-6379 or placebo in addition to an NA showed that there were no deaths, grade 4 AEs, or AEs leading to discontinuation. Most AEs were mild or moderate in severity.

## 4.4. End of Study Definition

#### **End of Study Definition**

The end of study (EOS) is considered as the last visit (Follow-up Week 48 or early discontinuation) for the last participant in the study. With implementation of Protocol Amendment 5, the last visit for the last participant in the study may be up to Follow-up Week 72 (see Study Completion Definition below for rationale). The final data from the study site will be sent to the sponsor (or designee) after completion of the final participant visit at that study site, in the time frame specified in the Clinical Trial Agreement.

#### **Study Completion Definition**

A participant will be considered to have completed the study if he or she has completed the assessments at Follow-up Week 48. With implementation of Protocol Amendment 5, the follow-up phase of 48 weeks will be extended with a maximum of 24 weeks (ie, Follow-up Week 72) for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation.

#### 5. STUDY POPULATION

Screening for eligible participants will be performed within 4 weeks before administration of the study intervention. If necessary, eg, for operational reasons, the screening phase may be extended up to a maximum of 6 weeks on a case-by-case basis and in agreement with the sponsor.

The inclusion and exclusion criteria for enrolling participants in this study are described below. If there is a question about these criteria, the investigator must consult with the appropriate sponsor representative and resolve any issues before enrolling a participant in the study. Waivers are not allowed.

Retesting to assess eligibility will be allowed once, using an unscheduled visit during the screening period.

For a discussion of the statistical considerations of participant selection, refer to Section 9.2.

#### 5.1. Inclusion Criteria

Each potential participant must satisfy all of the following criteria to be enrolled in the study:

- 1. Adult participants  $\ge$ 18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place) to  $\le$ 65 years of age.
- 2. Participants must be medically stable on the basis of physical examination, medical history, vital signs, and triplicate 12-lead ECG performed at screening. Any abnormalities must be consistent with the underlying illness in the study population and this

determination must be recorded in the participant's source documents and initialed by the investigator.

- 3. Participants must have HBV infection documented by serum HBsAg positivity at screening. In addition, chronicity must be documented by any of the following at least 6 months prior to screening: serum HBsAg positivity, HBeAg positivity or HBV DNA positivity, ALT elevation above ULN without another cause than HBV infection, documented transmission event, liver biopsy with changes consistent with chronic HBV. If none of the above are available, the following ways of documenting chronicity are acceptable at the time of screening: absence of marker for acute infection such as immunoglobulin M (IgM) anti-HBs and anti-HBc antibodies, which can be tested at screening.
- 4. Participants who are not currently treated (defined as not having been on HBV treatment, including NAs and IFN products within 6 months prior to screening), including treatment-naïve participants (defined as never having received HBV treatment, including NAs and IFN products) should:
  - a. be HBeAg positive, AND
  - b. have serum HBV DNA at screening ≥20,000 IU /mL, AND
  - c. have ALT levels at screening <10x ULN, AND
  - d. have indication for NA treatment according to local standard practice.
- 5. Virologically suppressed participants should:
  - a. be HBeAg negative, AND
  - b. be on stable HBV treatment, defined as currently receiving NA treatment (ETV, tenofovir disoproxil, or TAF) for at least 6 months prior to screening and have been on the same NA treatment regimen (at the same dose) for at least 3 months at the time of screening, AND
  - c. have serum HBV DNA <60 IU/mL on 2 measurements at least 3 months apart (one of which is at screening), AND
  - d. have documented ALT values <2.0x ULN on 2 measurements at least 3 months apart (one of which is at screening).
- 6. Participants must have HBsAg > 100 IU/mL at screening.
- 7. Participants must have a body mass index (weight in kg divided by the square of height in meters) between 18.0 and 35.0 kg/m², extremes included.
- 8. Participants must have fibroscan liver stiffness measurement ≤9.0 kPa within 6 months prior to screening or at the time of screening.

*Note:* Other radiologic liver staging modalities (eg, acoustic radiation force impulse) might be used if standard practice at the site or if otherwise validated and agreed with the

sponsor. Results should be equivalent to Metavir F0-F2 with absence of signs of portal hypertension.

**Note:** Conventional imaging procedures (eg, conventional liver ultrasound, computed tomography [CT] or magnetic resonance imaging [MRI]) and serum marker panels are not allowed to rule out severe fibrosis or cirrhosis.

- 9. Female participants of childbearing potential must have a negative highly sensitive serum pregnancy test ( $\beta$ -human chorionic gonadotropin [ $\beta$ -hCG]) at screening and a negative urine pregnancy test on Day 1 before the first dose of study intervention.
- 10. Criterion modified per Amendment 5
  - 10.1 A woman must be (as defined in Section 10.8, Appendix 8, Contraceptive and Barrier Guidance and Collection of Pregnancy Information):
  - a. not of childbearing potential
  - b. of childbearing potential and practicing a highly effective, preferably user-independent method of contraception (failure rate of <1% per year when used consistently and correctly) for at least 30 days prior to screening and agrees to remain on a highly effective method while receiving study intervention and until 90 days after last dose of study intervention.

Examples of highly effective methods of contraception are located in Section 10.8, Appendix 8, Contraceptive and Barrier Guidance and Collection of Pregnancy Information.

**Note:** Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants in clinical studies.

Note (no longer applicable as of Protocol Amendment 5, because of the removal of JNJ-6379 as study intervention): Female participants of childbearing potential who are on a stable treatment regimen with hormonal contraceptives (ie, same dose and not starting or stopping hormonal contraceptive use for at least 30 days prior to screening) should continue the same dose regimen until 90 days after the last dose of study intervention. Ethinylestradiol-containing contraceptives are only allowed if the ethinylestradiol content is  $\leq 20~\mu g$ . Female participants stable on an ethinylestradiol-containing regimen with a dose  $\geq 20~\mu g$  who switch to an ethinylestradiol-containing regimen with a dose  $\leq 20~\mu g$ , should be on that new regimen for at least 1 week before the first dose of study intervention. For female participants of childbearing potential who will start a hormonal contraceptive treatment during the study, ethinylestradiol-containing contraceptives are not allowed.

11. Male participants must agree to wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study intervention period and until 90 days after last dose of study intervention.

- 12. Female participants must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study intervention period and until 90 days after last dose of study intervention.
- 13. Male participants must agree not to donate sperm for the purpose of reproduction during the study intervention phase and until 90 days after last dose of study intervention.
- 14. Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.
- 15. Participants must separately consent if he or she agrees to undergo optional study procedures (ie, leukapheresis, intensive PK, and/or optional biopsy). Refusal to give consent to one or all of these optional study procedures does not exclude from participation in the study.
- 16. In the investigator's opinion, the participant is able to understand and comply with protocol requirements, instructions, and study restrictions and is likely to complete the procedures as planned for this this study.

#### 5.2. Exclusion Criteria

Any potential participant who meets any of the following criteria will be excluded from participating in the study:

- 1. Criterion modified per Amendment 4
  - 1.1 Criterion modified per Amendment 5
  - 1.2 Participants with evidence of hepatitis A virus infection (hepatitis A antibody IgM), HCV infection (HCV antibody), hepatitis D virus (HDV) infection (HDV antibody), or hepatitis E virus (HEV) infection (HEV antibody IgM), or HIV-1 or HIV-2 infection (laboratory confirmed) at screening.

*Note:* Participants with a positive HCV antibody test can be enrolled if they have negative HCV RNA at screening and documented negative HCV RNA at least 6 months prior to screening.

*Note:* Participants with a positive HDV antibody test may be enrolled after discussion with the sponsor if an active HDV co-infection can be ruled out by documentation of negative HDV RNA.

*Note:* Participants with a positive IgM antibody test for HEV infection may be enrolled after discussion with the sponsor if an active HEV infection can be ruled out by documentation of negative anti-HEV IgG.<sup>a</sup>

\_

<sup>&</sup>lt;sup>a</sup> Negative HEV RNA may also be acceptable to rule out active HEV infection depending on local standard practices.

*Note:* Participants with a positive HIV-1 or HIV-2 antibody/antigen test at screening should have a confirmatory HIV RNA test, to rule out false positive results. They can be enrolled if they have a negative HIV RNA test at screening. Participants with evidence of HIV-1 or HIV-2 infection who are on antiretroviral treatment are excluded.

- 2. Participants with any of the following laboratory abnormalities within 12 months prior to screening or at the time of screening:
  - a. Total bilirubin >1.5x ULN<sup>a</sup>, OR
  - b. Direct bilirubin >1.2x ULN<sup>a</sup>, OR
  - c. Serum albumin <3.2 g/dL<sup>a</sup>,
- History or evidence of clinical signs/symptoms of hepatic decompensation including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices.
- 4. Participants with evidence of liver disease of non-HBV etiology. This includes but is not limited to hepatitis virus infections mentioned in exclusion criterion 1, drug- or alcohol related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, Gilbert's syndrome (mild cases are allowed, see exclusion criterion 2a), or any other non-HBV liver disease considered clinically significant by the investigator.
- 5. Participants with history or signs of cirrhosis or portal hypertension (nodules, no smooth liver contour, no normal portal vein, spleen size ≥12 cm), signs of HCC or clinically relevant renal abnormalities on an abdominal ultrasound performed within 6 months prior to screening or at the time of screening.

*Note:* In case of suspicious findings on conventional ultrasound the participant may still be eligible if HCC or clinically relevant renal abnormalities have been ruled out by a more specific imaging procedure (contrast enhanced ultrasound, CT or MRI).

- 6. Participants with one or more of the following laboratory abnormalities at screening as defined by the Division of Acquired Immunodeficiency Syndrome (DAIDS) Toxicity Grading Scale:
  - a. Estimated glomerular filtration rate (eGFR<sub>cr</sub>) ≥grade 3 (<60 mL/min/1.73m²), calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula;
  - b. Pancreatic lipase elevation ≥grade 3;
  - c. Pancreatic amylase elevation ≥grade 3
  - d. Hemoglobin  $\leq 10.9 \text{ g/dL (males)}, \leq 10.4 \text{ g/dL (females)};$

<sup>&</sup>lt;sup>a</sup> Unless explained by a clinical setting that is not hepatic decompensation.

- e. Platelet count ≤lower limit of normal (LLN);
- f. Alpha-fetoprotein (AFP) >100 ng/mL;
  - *Note:* Participants with AFP >ULN but ≤100 ng/mL may be eligible if HCC can be ruled out based on a sensitive imaging study (eg, contrast enhanced ultrasound, CT, or MRI) during screening.
- g. Any other laboratory abnormality considered to be clinically significant by the investigator.
- 7. Participants with presence of coagulopathy or bleeding disorder as indicated by:
  - a. International normalized ratio (INR)  $\geq$ 1.1 x ULN;
  - b. Partial thromboplastin time  $> 1.1 \times ULN$ ;
  - c. Any signs of prolonged bleeding (>10 minutes).
- 8. Participants with presence of hemoglobinopathy (including sickle cell disease, thalassemia).
- 9. Participants who had a liver biopsy performed prior to screening that led to complications and that in the opinion of the investigator would prohibit another liver biopsy.
- 10. Participants with history of amyloidosis.
- 11. Participant refusal to accept blood transfusions.
- 12. Participants with hemoglobin A1c >8% at screening.
- 13. Participants with a history of malignancy within 5 years prior to screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which are considered cured with minimal risk of recurrence).
- 14. Participants with abnormal sinus rhythm (heart rate <45 or >100 beats per minute [bpm]); QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 ms for males and >470 ms for females; QRS interval ≥120 ms; PR interval >220 ms; abnormal conduction; or any other clinically significant abnormalities on a 12-lead ECG at screening.
- 15. Participants with a history of or current cardiac arrhythmias (eg, extrasystole, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome) or history or other clinical evidence of significant or unstable cardiac disease (eg, angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia and/or coronary heart disease), moderate to severe valvular disease, or uncontrolled hypertension at screening.

- 16. Participants with any current or previous illness for which, in the opinion of the investigator and/or sponsor, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol specified assessments. This may include but is not limited to significant vascular, pulmonary (eg, chronic obstructive pulmonary disease), gastrointestinal (eg, significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine (eg, thyroid disease), neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances. Any condition possibly affecting drug absorption (eg, gastrectomy or other significant gastrointestinal tract surgery, such as gastroenterostomy, small bowel resection, or active enterostomy) will also lead to exclusion.
- 17. Participants who have received an organ transplant (except for skin, hair, or cornea transplants).
- 18. Participants with any history of or current clinically significant skin disease requiring regular or periodic treatment.
- 19. Participants with clinically relevant drug or alcohol abuse within 12 months before screening.
- 20. Participants with history of clinically relevant drug rash.
- 21. Participants who have taken any disallowed therapies as noted in Section 6.5 before the planned first dose of study intervention.
- 22. Participants having used any invasive investigational medical device within 3 months, or having received an investigational intervention or a biological product, immunoglobulin or other blood product not intended for the treatment of HBV within 6 months or 5 half-lives (whichever is longer), before the planned first dose of study intervention, or is currently enrolled in an interventional clinical study with an investigational product.
- 23. Female participants who are pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study intervention.
- 24. Male participants who plan to father a child while enrolled in this study or within 90 days after the last dose of study intervention.
- 25. Participants who had major surgery (eg, requiring general anesthesia), excluding diagnostic surgery, within 12 weeks before screening; or who have not fully recovered from surgery; or have surgery planned during the time of expected participation in the study.

- *Note:* Participants with planned surgical procedures to be conducted under local anesthesia may participate.
- 26. Participant is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.
- 27. Vulnerable participants (eg, incarcerated individuals, individuals under a legal protection measure).
- 28. Criterion modified per Amendment 5
  - 28.1 Participants with known allergies, hypersensitivity, or intolerance to JNJ-3989 or its excipients (refer to the IBs and addendum). 14 16
- 29. Participants with contraindications to the use of ETV, tenofovir disoproxil, or TAF per local prescribing information.
- 30. <u>For participants undergoing optional leukapheresis:</u> contraindications to the use of citrate-based anticoagulation per local prescribing information.

#### Additional exclusion criteria for optional PegIFN-a2a treatment:

31. Criterion added per Amendment 4

Criterion modified per Amendment 5

- 31.1 The following needs to be checked after the participant has signed the separate consent to receive the optional PegIFN- $\alpha$ 2a treatment.
- a. Patients with signs or symptoms compatible with autoimmune disorders.
- b. Participants with bone marrow suppression.
- c. Patients with hypoglycemia, hyperglycemia, and/or diabetes mellitus, who cannot be effectively controlled by medication.
- d. Participants with pre-existing ophthalmologic disorders.
- e. Participants with one or more of the following laboratory abnormalities:
  - ANC <1,500 cells/mm<sup>3</sup> (<1,000 cells/mm<sup>3</sup> for black or African American participants).
  - Serum creatinine >1.5xULN.
  - Inadequately controlled thyroid function (TSH and T4).
- f. Participants with a history of a severe psychiatric disorder, including severe depression, suicidal ideation and attempted suicide, or a current depression or other

psychiatric disorders that is not adequately controlled on a stable medication regimen.

**NOTE:** Investigators should ensure that all study enrollment criteria have been met at screening. If a participant's clinical status changes (including any available laboratory results or receipt of additional medical records) after screening but before the Week -1 liver biopsy or before the first dose of study intervention is given such that he or she no longer meets all eligibility criteria, then the participant should be excluded from participation in the study. The required source documentation to support meeting the enrollment criteria are noted in Section 10.3, Appendix 3, Regulatory, Ethical, and Study Oversight Considerations.

# 5.3. Lifestyle Considerations

Potential participants must be willing and able to adhere to the following lifestyle restrictions during the course of the study to be eligible for participation:

- 1. Agree to follow all requirements as outlined in Section 6.5 (details regarding prohibited and restricted therapy during the study).
- 2. Agree to follow all requirements that must be met during the study as noted in the Inclusion and Exclusion Criteria (eg, contraceptive requirements).

#### 5.4. Screen Failures

**NOTE:** Retesting of abnormal laboratory values that may lead to exclusion will be allowed once. Retesting will take place during an unscheduled visit in the screening phase.

## Participant Identification, Enrollment, and Screening Logs

The investigator agrees to complete a participant identification and enrollment log to permit easy identification of each participant during and after the study. This document will be reviewed by the sponsor study-site contact for completeness.

The participant identification and enrollment log will be treated as confidential and will be filed by the investigator in the study file. To ensure participant confidentiality, no copy will be made. All reports and communications relating to the study will identify participants by participant identification and age at initial informed consent. In cases where the participant is not randomized into the study, the date seen and age at initial informed consent will be used.

Individuals who do not meet the criteria for participation in this study (screen failure) may not be rescreened without the sponsor's agreement.

### 6. STUDY INTERVENTION

## 6.1. Study Intervention(s) Administered

# **Physical Description of Study Interventions**

The JNJ-3989 supplied for this study will be provided as an aqueous clear, colorless to light yellow solution with 200 mg/mL of JNJ-3989 (containing the two RNAi triggers, JNJ-3976 and JNJ-3924) for SC injection, containing CCI

(CCI

Note that as of Protocol Amendment 5, JNJ-6379 is no longer included as part of the study intervention in this study.

Prior to implementation of Protocol Amendment 5, the JNJ-6379 supplied for this study was formulated as oral tablets containin [CCI] mg (CCI) and [CCI] mg (CCI) JNJ-56136379-AAA. The JNJ-6379 tablets had to be swallowed as a whole.

JNJ-3989 and JNJ-6379 will be/was to be provided under the responsibility of the sponsor. Refer to the IBs and addenda for a list of excipients. 14 16,39

The NAs ETV, tenofovir disoproxil, and TAF formulated as oral film-coated tablets of 0.5-mg, 245-mg, and 25-mg strength, respectively, will be provided by the sponsor.

PegIFN- $\alpha$ 2a formulated as solution for subcutaneous injection in a prefilled syringe with 180  $\mu$ g/0.5 mL of PegIFN- $\alpha$ 2a, will be provided by the sponsor. Refer to the prescribing information for a list of excipients.

#### **Packaging and Labeling**

All study interventions will be packaged with each unit labeled with a unique medication ID number. Packaging and labeling of JNJ-3989, JNJ-6379, PegIFN- $\alpha$ 2a, and the NAs will be/was to be done in an open label way. Commercial supplies of NAs and PegIFN- $\alpha$ 2a will be sourced and a clinical study label will be applied. Study intervention labels will contain information to meet the applicable regulatory requirements.

JNJ-6379 was to be dispensed in child-resistant packaging. Nucleos(t)ide analog and PegIFN- $\alpha$ 2a treatment may also be repackaged into child-resistant packaging if this is not already the case.

No study interventions can be repacked or relabeled without prior approval from the sponsor.

#### **Study Intervention Administration**

Study intervention administration must be captured in the source documents and the CRF.

JNJ-3989 injections will be administered SC (preferably in the abdomen) at the study site.

In between study visits, participants will take their oral study intervention (NA treatment) at home and they will bring their oral study intervention with them to each study visit. At study visits, the

oral study intervention should be taken on site to allow biochemistry and renal biomarker samples to be taken in fasted conditions.

During the study, virologically suppressed participants will continue the same NA treatment they were receiving at time of screening (and during at least 3 months prior to screening). In case participants experienced toxicity to ETV, tenofovir disoproxil, or TAF prior to screening, they should be treated with one of the other two NAs during this study.

Participants who are not receiving any HBV treatment at screening will receive tenofovir disoproxil at start of intervention.

If clinically indicated, switching from one NA treatment (ETV, tenofovir disoproxil, or TAF) to another NA treatment (ETV, tenofovir disoproxil, or TAF) during the study is allowed for all participants after consultation with the sponsor.

For PegIFN- $\alpha$ 2a, administration should be done SC in the thigh or abdomen, preferably in the evening by self-injection. Used PegIFN-a2a syringes should be separated from the needle via the sharps container and then placed into their original box and returned to the site, if allowed per local guidelines and regulations. The used needles in the sharps container will be returned to the study site after completion of treatment with PegIFN-  $\alpha$ 2a or disposed of following local standard procedures. If desired, participants can also choose to have the weekly administration of PegIFN- $\alpha$ 2a performed at the study site irrespective of the time of day.

If JNJ-3989 and PegIFN- $\alpha$ 2a are both injected in the abdomen, they should be injected into different areas of the abdomen and approximate location should be recorded.

For a definition of study intervention overdose, refer to Section 8.5.7.

# **Description of Interventions**

| Intervention name | JNJ-3989 | JNJ-6379**** | PegIFN-α2a | Entecavir (ETV)<br>monohydrate | Tenofovir<br>disoproxil | Tenofovir<br>alafenamide (TAF)* |
|---|---|---|---|---|---|---|
| Туре | Drug | Drug | Drug | Drug | Drug | Drug |
| Dosage formulation | Solution for injection | Tablets | Solution for injection | Film coated tablets | Film coated tablets | Film coated tablets |
| Unit dose strength(s) | 200 mg/vial | 25 and 100 mg | 180 μg/0.5 mL | 0.5 mg | 245 mg | 25 mg |
| Dosage level | 200 mg once every<br>4 weeks (Q4W) | 250 mg once daily (qd) | 180 μg once weekly (QW)** | Nucleoside naïve patients: 0.5 mg qd Lamivudine refractory patients: 1 mg* qd (but should preferably be treated with tenofovir disoproxil or TAF instead) | 245 mg qd | 25 mg qd |
| | | | | Other indications: 1 mg* qd (must be agreed upon by the sponsor) | | |
| Route of administration | Subcutaneous injection preferably in the abdomen | Oral | Subcutaneous injection (in the thigh or abdomen) | Oral | Oral | Oral |
| Use | Investigational intervention | Investigational intervention | Investigational intervention | Background intervention | Background intervention | Background intervention |
| Sourcing | Provided centrally by the sponsor | Provided centrally by the sponsor | Provided centrally by the Sponsor*** | Provided centrally by the sponsor | Provided centrally by the sponsor | Provided centrally by the sponsor |
| Packaging and<br>Labeling | Each unit will be labeled with unique medication ID number | Each unit will be labeled with unique medication ID number | Commercial supplies will be sourced. Each unit will be labeled with unique medication ID number*** | Commercial supplies<br>will be sourced. Each<br>unit will be labeled with<br>unique medication ID<br>number | Commercial supplies will be sourced. Each unit will be labeled with unique medication ID number | Commercial supplies will be sourced. Each unit will be labeled with unique medication ID number |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Intervention name | JNJ-3989 | JNJ-6379*** | PegIFN-α2a | Entecavir (ETV)<br>monohydrate | Tenofovir<br>disoproxil | Tenofovir<br>alafenamide (TAF)* |
|---|---|---|---|---|---|---|
| | | In child resistant packaging | In child resistant packaging*** | In child resistant packaging | In child resistant packaging | In child resistant packaging |
| | | | Labels will contain information to meet the applicable regulatory requirements. | | | y requirements. |
| Food/Fasting instructions | Regardless of food intake | Regardless of food intake | Per the prescribing information | Per prescribing information | Per prescribing information | Per prescribing information |

Q4W: once every 4 weeks; qd: once daily; QW: once weekly

In countries where TAF is available, it will be one of the NA treatment options.

For PegIFN-α2a, dose adjustment may be applicable for participants who develop laboratory abnormalities during PegIFN-α2a treatment (refer to Section 6.6).

<sup>\*\*\*</sup> May vary based on local regulations.

<sup>\*\*\*\*</sup> Participants enrolled before Protocol Amendment 5 was in effect, may have received JNJ-6379 as part of their study intervention. As of Protocol Amendment 5: study intervention includes JNJ-3989, NA and optionally PegIFN α2a

## 6.2. Preparation/Handling/Storage/Accountability

#### Preparation/Handling/Storage

All study interventions must be stored as specified on the product specific labeling.

Study-site personnel will instruct participants on how to store study intervention for at-home use as indicated for this protocol.

Refer to the pharmacy manual/study site investigational product and procedures manual for additional guidance on study intervention preparation, handling, and storage.

## **Accountability**

The investigator is responsible for ensuring that all study intervention received at the site is inventoried and accounted for throughout the study. The dispensing of JNJ-6379 (prior to Protocol Amendment 5), NA, and PegIFN- $\alpha$ 2a (if applicable) to the participant, and the return of JNJ-6379, NA, and PegIFN- $\alpha$ 2a (if applicable) from the participant, must be documented on the intervention accountability form. Participants must be instructed to return all original containers, whether empty or containing oral study intervention. The JNJ-3989 and, if applicable, PegIFN- $\alpha$ 2a injections administered to the participant must be documented on the intervention accountability form. All study intervention will be stored and disposed of according to the sponsor's instructions. Study-site personnel must not combine contents of the study intervention containers.

Participants who stopped JNJ-6379 per Protocol Amendment 5, must return their JNJ-6379 supply at the next scheduled visit. The return of JNJ-6379 from the participant must be documented on the intervention accountability form.

Study intervention must be handled in strict accordance with the protocol and the container label, and must be stored at the study site in a limited-access area or in a locked cabinet under appropriate environmental conditions. Unused study intervention, and oral study intervention returned by the participant, must be available for verification by the sponsor's study site monitor during on-site monitoring visits. The return to the sponsor of unused study intervention, or used returned study intervention for destruction, will be documented on the intervention return form. When the study site is an authorized destruction unit and study intervention supplies are destroyed on-site, this must also be documented on the intervention return form.

Potentially hazardous materials containing hazardous liquids, such as used ampules, needles, syringes and vials, should be disposed of immediately in a safe manner and therefore will not be retained for intervention accountability purposes. Details on handling of used PegIFN- $\alpha$ 2a syringes are described in Section 6.1, Study Intervention(s) Administered.

Study intervention should be dispensed under the supervision of the investigator or a qualified member of the study-site personnel, or by a hospital/clinic pharmacist. Study intervention will be supplied only to participants participating in the study. Returned study intervention must not be dispensed again, even to the same participant. Whenever a participant brings his or her oral study

intervention to the study site for pill count, this is not seen as a return of supplies. Study intervention may not be relabeled or reassigned for use by other participants. The investigator agrees neither to dispense the study intervention from, nor store it at, any site other than the study sites agreed upon with the sponsor. Further guidance and information for the final disposition of unused study interventions are provided in the Study Reference Manual.

## 6.3. Measures to Minimize Bias: Randomization and Blinding

#### **Intervention Allocation**

## Procedures for Randomization and Stratification

Prior to Protocol Amendment 5, central randomization was implemented in this study. Participants were randomly assigned within each panel to 1 of 2 intervention arms in a 1:1 ratio (Arm 1 [JNJ-3989+JNJ-6379+NA]:Arm 2 [JNJ-3989+NA]) based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor. The randomization was balanced by using randomly permuted blocks and was stratified within each panel by Fibroscan score (<7 kPa vs ≥7 kPa). The interactive web response system (IWRS) assigned a unique intervention code, which dictated the intervention assignment and matching study intervention kit for the participant. The requestor had to use his or her own user identification and personal identification number when contacting the IWRS and had to give the relevant participant details to uniquely identify the participant.

As of Protocol Amendment 5, all participants will enroll without randomization within a study panel. The interactive web response system (IWRS) will assign a unique intervention code with matching study intervention kit for the participant. The requestor must use his or her own user identification and personal identification number when contacting the IWRS and will then give the relevant participant details to uniquely identify the participant.

#### **Blinding**

As this is an open label study, blinding procedures are not applicable.

#### 6.4. Study Intervention Compliance

JNJ-3989 will be administered at the study site as a SC injection by qualified study-site personnel to assure compliance with study requirements.

The participants will be requested to bring unused oral study interventions and empty packaging to the study site at each visit.

Every effort should be made to have the participant take the study interventions as indicated in the Schedule of Activities.

• If an injection of JNJ-3989 was missed, the injection should be given as soon as possible but within 3 weeks after the scheduled time. Otherwise, the injection should be skipped and the next injection should be given at the next scheduled time point per the initial injection schedule.

- If a dose of NA is missed, the participant should follow the guidelines in the package insert.
- If an injection of PegIFN- $\alpha$ 2a is missed, the participant should follow the guidelines in the prescribing information.

If a participant's study intervention intake is not according to the protocol, the investigator will take the necessary measures to ensure future adherence to the protocol.

An optional medication diary to document oral study intervention intake can be made available for participants with an observed or known risk for study intervention non-compliance. The completed diaries are reviewed by the site staff and discussed with the participants for compliance monitoring and counseling. Completed diaries will be returned to the site staff to add to the source documents.

## 6.5. Concomitant Therapy

**Note:** With the removal of JNJ-6379 as study intervention in Protocol Amendment 5, JNJ-6379-specific disallowed medications and concomitant medications to be used with caution are no longer applicable and have been removed.

Prestudy therapies administered up to 30 days before the start of screening must be recorded at screening. If applicable, the participant's last anti-HBV treatment prior to screening must also be recorded.

Concomitant therapies must be recorded throughout the study, from signing of the ICF until completion of the participant's last study-related procedure. Concomitant therapies should also be recorded beyond the last study-related procedure only in conjunction with new or worsening S(AE)s.

All therapies (prescription or over-the-counter medications, including vaccines, vitamins, herbal supplements; non-pharmacologic therapies such as electrical stimulation, acupuncture, special diets, exercise regimens, or other specific categories of interest) different from the study intervention must be recorded in the CRF. Recorded information will include a description of the type of therapy, duration of use, dosing regimen, route of administration, and indication. Modification of an effective preexisting therapy should not be made for the explicit purpose of entering a participant into the study.

Local guidelines on the use of live vaccines in participants receiving PegIFN- $\alpha$ 2a should be followed, including for the second dose of Sputnik V (which contains rAd5, with a theoretical risk of replication competence). Sputnik Light, which is the first dose of Sputnik V (with rAd26) is not considered a live vaccine. See below for further guidance on the use of COVID-19 vaccines.

Note that locally approved COVID-19 vaccines (including those that received emergency use authorization or conditional marketing authorization) are allowed throughout the study. For participants receiving PegIFN- $\alpha$ 2a, the following recommendations should be applied to accommodate COVID-19 vaccination during PegIFN- $\alpha$ 2a treatment:

- COVID-19 vaccine and PegIFN-α2a should not be administered on the same day.
- If required, PegIFN- $\alpha$ 2a injection can be delayed with 2 days. The next PegIFN- $\alpha$ 2a injection should be performed at the scheduled time.
- If required, skipping a PegIFN-α2a injection may be considered after consultation with the Sponsor.
- Vaccination with Sputnik V should take above-mentioned consideration about live vaccines into account.

All COVID-19 vaccination-related data (eg, COVID-19 vaccination, AEs, AE management) should be appropriately captured in the CRF and source documents. Refer to the COVID-19 vaccine and/or PegIFN-α2a prescribing information for more details.

An overview of disallowed medication is provided in Table 4.

#### **Table 4: Disallowed Medication**

#### Disallowed at any time prior to screening until end of follow-up:

• Any CAM and oligonucleotide-based treatment (eg, siRNA and antisense oligonucleotides, nucleic acid polymers, etc.), other than the study intervention taken in the context of this study.

#### Disallowed from 6 months prior to screening until end of follow-up:

Any investigational agent, investigational vaccine, invasive investigational medical device, or investigational biological product (other than the study intervention taken in the context of this study). *Note:* For investigational COVID-19 vaccines administered within 6 months prior to screening, an exception will be made as long as the vaccine has been approved (or received emergency use authorization or conditional marketing authorization) at the time of screening.

### Disallowed from 6 months prior to baseline until end of follow-up:

- For participants currently not being treated: Any anti-HBV drug (including vaccines) other than the study intervention taken in the context of this study.
  - *Note*: Prior hepatic treatment with herbal or nutritional products is allowed but should be stopped at screening.
- Any systemically (eg, intravenously, intramuscularly, orally, subcutaneously) administered medication that directly or indirectly interferes with immune responses (eg, cyclosporine, interleukins, IFN, systemic corticosteroids exceeding 5 mg of prednisolone equivalent/day).

#### Disallowed from 1 month prior to screening until end of follow-up:

Anticoagulants and antiplatelet agents.

*Note:* The use of citrate-based anticoagulant is allowed for participants during the leukapheresis procedure. Use of heparin for anticoagulation is not allowed.

*Note:* The use of ibuprofen or paracetamol is allowed. Use of low-dose aspirin is allowed with exception of 7 days prior to biopsies.

#### Disallowed from screening until end of follow-up:

- Any anti-HBV drug (including vaccines) other than the study intervention taken in the context of this study.
  - *Note:* NA standard of care treatment is allowed for virologically suppressed participants.
- Biotin (>1 mg daily dose), either taken alone or as part of a multivitamin formulation. *Note:* The use of other vitamins is allowed.
- Topical steroids (>7 days) under occlusive dressing.

**Note:** The list of disallowed medication is not exhaustive; for products falling in one of the categories and not mentioned by name, the sponsor should be contacted to determine whether the product can be allowed.

The sponsor must be notified in advance (or as soon as possible thereafter) of any instances in which prohibited therapies are administered.

The prescribing information for ETV, tenofovir disoproxil, TAF, and PegIFN- $\alpha$ 2a should be consulted for any additional prohibited medication. In case of flu-like symptoms after administration of PegIFN- $\alpha$ 2a, paracetamol up to a maximum of 2 g per 24 hours and a maximum of 6 g per week is allowed.

Medications requiring SC injection (other than JNJ-3989 and PegIFN- $\alpha$ 2a; eg, insulin) should be administered away from the JNJ-3989 and PegIFN- $\alpha$ 2a injection sites.

#### 6.6. Dose Modification

Dose modifications of JNJ-3989 and NA (increase or decrease of dose level) are not permitted during the study.

For PegIFN- $\alpha$ 2a, dose adjustment guidelines are applicable for participants who develop laboratory abnormalities during PegIFN- $\alpha$ 2a treatment, as recommended in the locally approved prescribing information for PegINF- $\alpha$ 2a and upon investigator's assessment.

Refer to the example from the Pegasys USPI and SmPC (see Table 5).

Table 5: PegIFN-α2a Hematological Dose Modification Guidelines

| Laboratory Values | Recommended Dose |
|---|---|
| ANC <750 cells/mm <sup>3</sup> | Reduce to 135µg |
| ANC <500 cells/mm <sup>3</sup> | Discontinue treatment until ANC values return to more than 1,000 cells/mm <sup>3</sup> . |
| | Reinstitute at 90µg and monitor ANC. |
| Platelet <50,000 cells/mm <sup>3</sup> | Reduce to 90µg |
| Platelet <25,000 cells/mm <sup>3</sup> | Discontinue treatment |

ANC: absolute neutrophil count Source: Pegasys USPI and SmPC

For participants who prematurely discontinue PegIFN- $\alpha$ 2a, treatment with PegIFN- $\alpha$ 2a may be restarted according to the recommendations from the locally approved prescribing information for PegIFN- $\alpha$ 2a.

#### 6.6.1. Study Intervention Completion at Week 48

With the implementation of Protocol Amendment 5, all participants had to stop JNJ-6379 treatment immediately.

Participants will complete treatment with JNJ-3989 after a fixed duration of 48 weeks. If all of the below criteria are met based on clinical laboratory tests performed at Week 44, treatment with NA will also be completed at the next scheduled visit (ie, Week 48):

- The participant has ALT <3x ULN, AND
- The participant has HBV DNA <LLOQ, AND
- The participant is HBeAg negative, AND
- The participant has HBsAg <10 IU/mL.

**Note:** In case of ALT elevation  $\ge 3x$  ULN at Week 44 the investigator must consider different potential causes of increased ALT to ensure appropriate work up and management as needed. If the ALT elevation is unrelated to HBV activity and/or  $\le 3x$  ULN by Week 48, NA completion may be considered at the discretion of the investigator and in consultation with the sponsor.

Participants who do not meet the above criteria at Week 48 should continue NA treatment during the 48-week follow-up phase. Participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who have not met NA treatment completion criteria at Week 48 may have NA treatment completion criteria assessed at the end of treatment with PegIFN- $\alpha$ 2a and stop NA if criteria are met.

If a participant prematurely discontinues investigational intervention before Week 48, follow-up assessments should be obtained as per the Schedule of Activities until 48 weeks after the end of investigational intervention unless the participant withdraws consent. In this case, NA treatment may be continued or, in consultation with the sponsor, discontinued, based on the above-mentioned NA treatment completion criteria.

With the implementation of Protocol Amendment 5, the follow-up period will be extended for participants who are receiving optional treatment with PegIFN- $\alpha$ 2a and who meet NA treatment completion criteria at the end of treatment with NA and PegIFN- $\alpha$ 2a to ensure all participants have at least one year of follow-up after NA treatment cessation.

The investigator should consider to re-start NA treatment per local standard of care at the EOS visit (Follow-up Week 48 up to maximum Follow-up Week 72) for participants who met the NA treatment completion criteria at Week 48 or for participants who met NA treatment completion criteria at the end of treatment with PegIFN-α2a during the follow-up phase, who did not re-start NA treatment during the follow-up phase, and who did not achieve and maintain HBsAg seroclearance. NA will not be provided by the sponsor after the final study visit.

# 6.6.2. NA Re-treatment Criteria and Monitoring after Stopping of NA

Participants who meet the NA treatment completion criteria outlined in Section 6.6.1 will be monitored closely during the follow-up phase.

After stopping NA treatment, participants should be monitored as follows:

• Regular monitoring visits will be every 4 weeks during the follow-up phase in accordance with the Schedule of Activities.

- A post-treatment HBV DNA value of >20,000 IU/mL should trigger re-testing of ALT/AST, HBV DNA, and total and direct bilirubin within a maximum of 7 days from receipt of the data and further repeats as necessary (ie, weekly until HBV DNA returns to <20,000 IU/mL).
- A post-treatment HBV DNA value of >2,000 IU/mL (but <20,000 IU/mL) should trigger a retest within 14 days from receipt of the data and further repeats as necessary (ie, every other week until HBV DNA returns to <2,000 IU/mL).
- A post-treatment ALT value of >5x ULN should trigger re-testing of ALT, AST, ALP, total and direct bilirubin, INR, albumin, and HBV DNA on a weekly basis until ALT and AST levels have returned to <5x ULN.

After stopping NA treatment, participants should re-start NA treatment:

- Immediately with signs of decreasing liver function based on laboratory findings (eg, INR, direct bilirubin) or clinical assessment (eg, ascites, hepatic encephalopathy),
- Immediately with an HBV DNA value of >100,000 IU/mL (irrespective of confirmation and/or ALT increase).
- With confirmed post-treatment HBeAg seroreversion (HBeAg positive after it was negative at NA completion)
- With confirmed\* post-treatment increases in HBV DNA >2,000 IU/mL and ALT >5x ULN
- With confirmed\* post-treatment increases in HBV DNA >20,000 IU/mL.
- \* At least 4 weeks apart frequency of visits as described above

#### Note:

Additional re-testing and/or earlier restarting of NA treatment is at the investigator's discretion, even if the above cut-offs are not yet met.

To avoid delays in decision making, sites are encouraged to run local re-testing in parallel with central re-testing in the situations described above that require more frequent re-testing. Local test results are to be recorded in the CRF and/or source documents, including information on the HBV DNA assay used. In addition, to avoid delays in NA re-treatment, it should be considered to dispense NA to participants who potentially met the NA re-treatment criteria (eg, pending confirmation) and who will not be available to come to the study site immediately at the time the confirmatory test results will become available. This should ensure that the participant can immediately re-start NA treatment if indicated, upon direct confirmation by the investigator.

In case NA treatment is re-started, participants will be followed until the end of the study or until clinical stabilization, whichever comes later.

Refer to Appendix 12 in Section 10.12 for a graphical representation.

## 6.7. Study Intervention After the End of the Study

Participants will be instructed that study intervention will not be made available to them after they have completed/discontinued study intervention and that they should return to their primary physician to determine standard of care.

The investigator should consider to re-start NA treatment per local standard of care at the EOS visit (Follow-up Week 48 up to maximum Follow-up Week 72) for participants who met the NA treatment completion criteria at Week 48 or for participants who met NA treatment completion criteria at the end of treatment with PegIFN-α2a during the follow-up phase, who did not re-start NA treatment during the follow-up phase, and who did not achieve and maintain HBsAg seroclearance. NA will not be provided by the sponsor after the final study visit.

# 7. DISCONTINUATION OF INVESTIGATIONAL INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Intervention

With the implementation of Protocol Amendment 5, all participants had to stop JNJ-6379 treatment immediately.

Treatment with JNJ-3989 and/or PegIFN- $\alpha$ 2a must be discontinued if any of the criteria listed below apply. If JNJ-3989 is discontinued, PegIFN- $\alpha$ 2a should also be discontinued. If PegIFN- $\alpha$ 2a is discontinued, JNJ-3989 should be continued. NA treatment may be continued or, in consultation with the sponsor or discontinued based on investigator judgement.

- The participant withdraws consent to receive study intervention.
- The investigator believes that for safety reasons or tolerability reasons (eg, AE) it is in the best interest of the participant to discontinue JNJ-3989 (and, if applicable, PegIFN-α2a).
- The participant becomes pregnant.
- The participant has a ≥grade 3 rash (see Section 10.5, Appendix 5, Rash Management) or allergic reaction (see Section 8.5.7.2).
- The participant has signs of hepatic decompensation (ie, clinical evidence of ascites, bleeding varices, or hepatic encephalopathy) or an increase in direct bilirubin >1.5x ULN in combination with INR  $\ge 1.5x$  ULN or albumin <3.0 g/dL.
- The participant has a confirmed ≥grade 3 eGFR<sub>cr</sub> abnormality and a drop from baseline of >10 mL/min/1.73 m², considered at least possibly related to JNJ-3989 (or PegIFN-α2a) that persists despite changing tenofovir disoproxil to ETV or TAF (if the patient was receiving tenofovir disoproxil) (see Section 8.5.6.4).
- The participant has a confirmed QTcF prolongation (defined as a QTcF value of >500 ms, or an increase from baseline of >60 ms) at any given time point.
- The participant requires  $\geq$ 7 days of treatment with any of the disallowed medications listed in Section 6.5 and does not intend to discontinue treatment with the disallowed medication.

The participant has confirmed HBV virologic breakthrough (ie, confirmed on-treatment HBV DNA increase by >1 log<sub>10</sub> IU/mL from nadir or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had HBV DNA level <LLOQ of the HBV DNA assay). In case of virologic breakthrough, the same assessments will be done at an unscheduled visit as will be done in case of an ALT flare, but no PBMC sample will be taken (see Section 8.5.6.1 and Schedule of Activities), changing the NA should be considered in consultation with the sponsor.

If virologic breakthrough occurs during JNJ-3989 and PegIFN- $\alpha$ 2a administration, this does not automatically lead to stop of JNJ-3989 and/or PegIFN- $\alpha$ 2a but should be assessed/discussed with the Sponsor.

In case of virologic breakthrough, a viral sequencing sample will be collected at the next visit.

- The participant has ALT/AST elevations, as described in Section 8.5.6.2.
- The participant has confirmed ≥grade 3 hematologic abnormalities as described in Section 8.5.6.5.

**NOTE:** The grades are based on the DAIDS Toxicity Grading Scale (see Section 10.9, Appendix 9, DAIDS Table).

In addition, PegIFN- $\alpha$ 2a (if applicable) must immediately be discontinued for any of the following reasons:

- Participant has platelet count <25,000 cells/mm<sup>3</sup>
- Participant has ANC <500 cells/mm<sup>3</sup>

*Note:* PegIFN- $\alpha$ 2a treatment can be restarted when ANC values return to more than 1,000 cells/mm<sup>3</sup> (see details in Section 6.6, Dose Modification)

- Participant develops evidence of hepatic decompensation during treatment, or ALT increase clinically significant or accompanied by direct bilirubin increase
- Participant develops thyroid disorders or diabetes during treatment and cannot be controlled with medication
- Participant develops new or worsening ophthalmologic disorders
- Participant develops any deterioration of cardiovascular status
- Participant develops serious, acute hypersensitivity reaction (eg, urticaria, angioedema, bronchoconstriction, anaphylaxis)
- Participant develops serious infection (bacterial, viral, fungal) and/or sepsis
- Participant develops persistent or unexplained pulmonary infiltrates or pulmonary function impairment
- Participant with onset or worsening of psoriatic lesion
- Participant develops moderate or severe depression, or other psychiatric symptoms (for mild depression, treatment discontinuation may be considered)

*Note:* Participants who develop a neuropsychiatric AE during optional PegIFN- $\alpha$ 2a treatment, will be monitored closely until the neuropsychiatric AE resolves, with frequent (at least weekly) follow-up phone calls.

- Participant develops colitis symptoms (such as but not limited to abdominal pain, bloody diarrhea, and fever)
- Participant develops symptoms or signs suggestive of pancreatitis

If a participant discontinues investigational intervention for any reason before Week 48, then the early withdrawal assessments should be obtained. The participant will enter the follow-up phase and complete the follow-up schedule unless the participant withdraws consent. Participants who withdraw consent will be offered an optional safety follow-up visit to occur on the day of consent withdrawal. Study intervention assigned to the participant who discontinued study intervention may not be assigned to another participant.

In case a participant withdraws consent for the second biopsy, the study participant may continue the study intervention and visit schedule as outlined in the Schedule of Activities.

# 7.2. Participant Discontinuation/Withdrawal From the Study

A participant will NOT be automatically withdrawn from the study if he or she has to discontinue study intervention before Week 48.

A participant will be withdrawn from the study for any of the following reasons:

- Lost to follow-up,
- Withdrawal of consent,
- Death.

When a participant withdraws before study completion, the reason for withdrawal is to be documented in the CRF and in the source document. If the reason for withdrawal from the study is withdrawal of consent then no additional assessments are allowed. No additional participants will be enrolled in case a participant withdraws from the study.

#### Withdrawal of Consent

A participant declining to return for scheduled visits does not necessarily constitute withdrawal of consent. Alternate follow-up mechanisms that the participant agreed to when signing the consent form apply as local regulations permit.

## 7.2.1. Withdrawal From the Use of Research Samples

### Withdrawal From the Use of Samples in Future Research

The participant may withdraw consent for use of samples for research (refer to Long-Term Retention of Samples for Additional Future Research in Section 10.3, Appendix 3, Regulatory, Ethical, and Study Oversight Considerations). In such a case, samples will be destroyed after they

are no longer needed for the clinical study. Details of the sample retention for research are presented in the main ICF and in the separate ICF for optional research samples.

## 7.3. Lost to Follow-up

To reduce the chances of a participant being deemed lost to follow-up, prior to randomization attempts should be made to obtain contact information from each participant, eg, home, work, and mobile telephone numbers and email addresses for both the participant as well as appropriate family members.

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. A participant cannot be deemed lost to follow-up until all reasonable efforts made by the study-site personnel to contact the participant are deemed futile. The following actions must be taken if a participant fails to return to the study site for a required study visit:

- The study-site personnel must attempt to contact the participant to reschedule the missed visit as soon as possible, to counsel the participant on the importance of maintaining the assigned visit schedule, to ascertain whether the participant wishes to or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every reasonable effort to regain contact with the participant (where possible, 3 telephone calls, emails, fax, and, if necessary, a certified letter to the participant's last known mailing address, or local equivalent methods). These contact attempts should be documented in the participant's medical records.
- Should the participant continue to be unreachable, he or she will be considered to have withdrawn from the study.

Should a study site close, eg, for operational, financial, or other reasons, and the investigator cannot reach the participants to inform them, their contact information will be transferred to another study site.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

#### **Overview**

The Schedule of Activities summarizes the frequency and timing of efficacy, PK, PD, immune, biomarker, pharmacogenomic and safety measurements applicable to this study.

If applicable, ECGs should be completed before any tests, procedures, or other consultations for that visit. Blood collections for PK and PD assessments should be kept as close to the specified time as possible. Samples obtained within 20% of the nominal time from dosing (eg,  $\pm 12$  minutes of a 60-minute time point) will not be captured as a protocol deviation if the exact time of the sample collection is noted on the source document and CRF. Other measurements may be done earlier than specified time points if needed. Actual dates and times of assessments will be recorded in the source documentation and CRF.

Additional serum or urine pregnancy tests may be performed, as determined necessary by the investigator or required by local regulation, to establish the absence of pregnancy at any time during the participation in the study.

The amount of blood drawn from each participant over the entire course of this study will be approximately 1200 mL.

During the leukapheresis procedure, WBCs will be separated from the blood, while the rest of the blood is returned to circulation. This process typically yields approximately 200 ml of cells. For participants undergoing all 3 optional leukapheresis procedures, approximately 600 ml will be collected.

For participants receiving optional PegIFN- $\alpha$ 2a treatment, an additional amount of maximum 50 mL of blood will be drawn. In case participants continue NA treatment during the optional PegIFN- $\alpha$ 2a treatment, an additional amount of maximum 200 mL of blood will be drawn during additional visits every 4 weeks to ensure at least one year of follow-up after NA treatment cessation (extended follow-up phase up to 72 weeks).

Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

## Sample Collection and Handling

The actual dates and times of sample collection, as well as the actual start and stop times of the leukapheresis procedure, must be recorded in the CRF or laboratory requisition form.

Refer to the Schedule of Activities for the timing and frequency of all sample collections.

Instructions for the collection, handling, storage, and shipment of samples are found in the laboratory manual that will be provided. Collection, handling, storage, and shipment of samples must be under the specified, and where applicable, controlled temperature conditions as indicated in the laboratory manual.

#### **Study-specific Materials**

The investigator will be provided with the following supplies:

- IB and any addenda for JNJ-3989,
- Prescribing Information for ETV, tenofovir disoproxil, TAF, and PegIFN-α2a,
- Pharmacy manual/study site investigational product and procedures manual,
- Laboratory manuals,
- IWRS Manual,
- CRF Completion Guidelines,
- Sample ICF,

• Contact information page(s).

## 8.1. Liver Biopsy and Fine Needle Aspiration Biopsy

Percutaneous core liver biopsies and FNABs will be performed at the time points indicated in the Schedule of Activities. If participants agree to undergo an optional liver biopsy, additional FNAB and/or core liver biopsy samples may be taken at the selected location at Follow-up Week 24 or at the time points clinically indicated.

Following local standard practice the biopsy location will be identified with ultrasound (which will also be used to rule out contraindicating conditions for a biopsy) and after application of local anesthesia the FNAB samples and core liver biopsy samples will be collected.

The liver biopsy procedure should be preceded and followed by standard medical monitoring according to local medical practice. This may include an overnight stay at the investigator's discretion. The use of low-dose aspirin is allowed with exception of 7 days prior to biopsies (see Section 6.5).

The liver tissue will be used to assess HBsAg. Changes from baseline in the proportion of HBsAg positive hepatocytes under therapy will be assessed.

In addition, the liver tissue may also be used to assess other HBV markers in the liver such as, but not limited to, total intracellular HBV RNA and DNA, HBeAg, and HBc. Changes in the quantity and potentially changes in the spatial distribution of these markers (including HBsAg) under therapy may be assessed. Viral genome (RNA or DNA) or transcript sequencing/analyses as well as assessment of HBV integrants in the host genome may be performed.

Intrahepatic immune status at baseline and response to treatment will be assessed. Both innate and adaptive immune compartment will be characterized, by measuring the relative number of specific cells and the expression of functional markers in each cell population using various single cell approaches, such as single cell transcriptomics in FNABs and Immunofluorescence staining, and transcriptomics and proteomics profiling in core needle biopsies. Depending on the latest platform developments (spatial transcriptomics, *in situ* sequencing approaches, etc.), methods for immune cells characterization might be adjusted.

Hepatitis B virus-specific T-cells, although very rare in FNABs, may be characterized and counted by multimers binding assays, staining and sorting for positive cells. Downstream profiling of collected HBV-specific T-cells may be performed by T-cell receptor sequencing and RNA sequencing.

Infiltrating immune cells will be used for the evaluation of innate and adaptive immune responses, which can be compared to responses in PBMCs.

Intrahepatic virologic status at baseline and response to treatment will be assessed with a range of methods.

Hepatitis B virus cccDNA levels may be assessed using quantitative polymerase chain reaction (qPCR) methods on a single cell level using laser capture microdissection or bulk analyses. The exact protocol of cccDNA measurement will be determined based on the latest method available considering the performance characteristics and the validation status of the assay. Southern Blot-based methods or novel methods for cccDNA detection (eg, fluorescent in situ hybridization [FiSH]) might be used depending on the availability of sample and established methodology. Quantification of intracellular pre-genomic HBV RNA can be used to determine transcriptional activity of HBV cccDNA by assessing the ratio of pgRNA levels over cccDNA levels.

Immune and virologic markers in the liver and/or changes thereof under therapy will be used to assess association with blood markers and/or treatment response and outcome.

Remaining samples may be used for determination of liver JNJ-3989 (ie, JNJ-3976 and JNJ-3924) and/or JNJ-6379 concentrations and/or research on viral and host biomarkers and immune markers at the viral and/or host RNA/DNA, protein, and cell level.

Samples can only be used for research related to JNJ-3989, JNJ-6379, NA, chronic HBV infection, or chronic HBV infection related disease or may be used to develop tests/assays related to JNJ-3989, JNJ-6379, NA, or chronic HBV infection.

These latter exploratory analyses will be performed at the sponsor's discretion and will always be under the sponsor's supervision.

# 8.2. Blood Efficacy Assessments

Efficacy assessments will be performed at the time points indicated in the Schedule of Activities.

Qualitative and quantitative HBsAg and HBeAg, and quantitative HBcrAg as well as antibodies against HBsAg and HBeAg will be determined using validated serologic assays in a central laboratory. Samples for the determination of HBsAg and HBeAg will be processed in real-time. Samples for the determination of HBcrAg can be analyzed in batch and at the sponsor's discretion.

Hepatitis B virus DNA and HBV RNA will be quantified at central laboratories using validated assays for the quantification of HBV DNA and HBV RNA. Samples for the determination of HBV DNA will be processed in real-time. Samples for the determination of HBV RNA can be analyzed in batch and at the sponsor's discretion.

Hepatitis B virus DNA, HBsAg, HBeAg, anti-HBs, and anti-HBe antibody testing results will be provided to the investigator and the sponsor from screening until the end of follow-up.

It is the responsibility of the investigator:

- To monitor HBV DNA results and ensure that investigational intervention is discontinued in participants with virologic breakthrough (see Section 7.1),
- To assess if NA treatment completion criteria are met (see Section 6.6.1),
- To assess whether re-start of NA treatment during follow-up is needed (see Section 6.6.2).

In participants enrolled at a site with an on-site Fibroscan device, Fibroscan assessments will be performed to determine changes in fibrosis levels.

Samples may be used by the sponsor for additional exploratory assessments analyzing the serologic and virologic characteristics of HBV infection and efficacy or safety of the study intervention.

## 8.2.1. Sequencing

Viral genome sequence analysis will be performed to evaluate mutations associated with the study intervention.

Sequencing of the HBV genome will be performed to monitor HBV variants present at the time points indicated in the Schedule of Activities. The sequencing of samples may be triggered by the sponsor virologist based on changes in HBV DNA levels observed in each individual participant and the limits of the sequencing assay.

Samples may be used by the sponsor for additional assessments analyzing the serologic and virologic characteristics of the HBV infection and efficacy of the study intervention, including viral genotypic and phenotypic assessments.

#### 8.3. Blood Immune Assessments

## 8.3.1. Peripheral Blood Mononuclear Cell Immune Analyses

Samples for PBMC immune analyses will be collected during the study intervention and follow-up phases and will be analyzed centrally for HBV-specific responses by enzyme-linked immunospot (ELISpot) and/or intracellular cytokine staining (ICS) after stimulation with HBV-specific antigens. ELISpot detects T-cells that secrete gamma interferon (IFN- $\gamma$ ) in response to a specific antigenic stimulation, whereas ICS determines the frequency of CD4+ and CD8+ T-cells secreting cytokines such as IFN- $\gamma$ , interleukin (IL)-2 and tumor necrosis factor (TNF)- $\alpha$  in response to a specific antigenic stimulation. Hepatitis B virus-specific T-cells may be characterized in PBMCs by binding assays (multimer staining) combined with downstream TCR and transcriptome profiling.

Additional experiments may be performed to further phenotypically and functionally characterize PBMCs using proliferation or cytotoxic assays or other methods such as cytometry by time of flight to evaluate innate and adaptive immune responses. Leftover samples may be used at the sponsor's discretion for additional exploratory research related to HBV infection or study intervention (safety/efficacy).

Additional PBMC samples may be taken in case of ALT flare, upon discussion with the sponsor, which may require an unscheduled visit.

## 8.3.2. Leukapheresis (Optional With Separate Consent)

Leukapheresis allows to selectively collect higher quantities of PBMCs from participants without withdrawing large volumes of blood.

Leukapheresis will only be performed for participants who consent separately to this component of the study. Participants may withdraw such consent at any time without affecting their participation in other aspects of the study.

Leukapheresis may be done at least 1 week (and up to 3 weeks) after the liver biopsies (see Schedule of Activities). Prior to the procedure, the participant's wellbeing will be checked and leukapheresis will only be offered if there is no clinical reason against it. If a participant has had a recent febrile illness, the leukapheresis should be postponed until body temperature is normal for at least 72 hours.

The leukapheresis procedure should mainly follow local standard procedures. Additional guidelines will be provided via a separate manual in order to standardize this process across sites.

One leukapheresis session is expected to last between 1.5 - 5 hours.

During the procedure, the participant will receive intravenous saline infusions and citrate-based anticoagulant. Use of heparin for anticoagulation is not allowed. A specialized leukapheresis trained research nurse or physician will be in attendance and in charge of the participant's immediate medical care to monitor the leukapheresis.

After completion of the leukapheresis procedure, participants will stay at the site for at least 30 minutes to monitor for any relevant safety events. Additional safety procedures may be performed at the discretion of the site staff. Participants are advised to refrain from exercise and strenuous activities for 3 day after the leukapheresis visit.

### 8.4. Safety Assessments

Safety and tolerability will be assessed throughout the study from the time that the ICF is signed until completion of the last study-related activity, which may include contact for follow-up of safety. The evaluations of safety and tolerability will include monitoring of (S)AEs, physical examinations (including body weight), vital signs measurements, triplicate 12-lead ECGs, and clinical laboratory tests (including hematology, blood biochemistry, blood coagulation, urinalysis, urine chemistry, and renal biomarkers) at predefined time points as specified in the Schedule of Activities. Any clinically relevant changes occurring during the study must be recorded on the Adverse Event section of the CRF.

Adverse events will be reported and followed by the investigator as specified in Section 8.5 and Section 10.4, Appendix 4, Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting.

Specific toxicity management plans in line with the known pharmacological profile of the study intervention (and the drug classes) evaluated in this study are implemented (Sections 8.5.6 and 8.5.7).

Any clinically significant abnormalities persisting at the end of the study/early withdrawal will be followed by the investigator until resolution or until a clinically stable condition is reached.

Details regarding the IFLEP are provided in Section 9.6 and in the Committees Structure in Section 10.3, Appendix 3, Regulatory, Ethical, and Study Oversight Considerations.

## 8.4.1. Physical Examinations

A complete physical examination (including height [at screening only], body weight, skin examination, and other body systems) will be performed at screening, Week 24, and Week 48. A symptom-directed physical examination (including body weight) will be performed at the time points indicated in the Schedule of Activities.

A complete physical examination includes the following: general appearance, eyes, ears, nose, throat, cardiovascular system, respiratory system, gastro-intestinal system, head, neck, thyroid, and skin and mucous membranes. A neurological and musculoskeletal examination will be performed, as well as an examination of the lymph nodes. Body weight and temperature will be measured. Height will be measured at the screening visit only.

## 8.4.2. Vital Signs

Body temperature, pulse rate, and supine SBP and DBP will be assessed at the time points indicated in the Schedule of Activities.

Blood pressure and pulse rate measurements will be assessed with a completely automated device. Manual techniques will be used only if an automated device is not available.

Blood pressure and pulse/heart rate measurements should be preceded by at least 5 minutes of rest in a quiet setting without distractions (eg, television, cell phones).

Clinically relevant abnormalities in vital signs are defined in Section 10.7, Appendix 7, Cardiovascular Safety Abnormalities.

# 8.4.3. Electrocardiograms

Twelve-lead triplicate ECGs will be collected at the time points indicated in the Schedule of Activities and when clinically indicated.

During the collection of ECGs, participants should be in a quiet setting without distractions (eg, television, cell phones). Participants should rest in a supine position for at least 5 minutes before ECG collection and should refrain from talking or moving arms or legs.

At each time point at which triplicate ECGs are required, 3 individual ECG tracings should be obtained as closely as possible in succession, but no more than 2 minutes apart. The full set of triplicates should be completed in less than 10 minutes.

Evaluation of the triplicate 12-lead ECGs will be based on the mean value of the triplicate parameters.

All ECGs will be read centrally. Only on Day 1, pre-dose ECG assessment will also be done locally on-site. Preferably, all ECGs will be read and interpreted under supervision of one and the same qualified person.

Clinically relevant abnormalities in ECG are defined in Section 10.7, Appendix 7, Cardiovascular Safety Abnormalities.

## 8.4.4. Clinical Safety Laboratory Assessments

Blood samples for serum chemistry and hematology and a urine sample for urinalysis will be collected as noted in Section 10.2, Appendix 2, Clinical Laboratory Tests. The investigator must review the laboratory results, document this review, and record any clinically relevant changes occurring during the study in the adverse event section of the CRF. The laboratory reports must be filed with the source documents.

Participants need to have fasted for at least 10 hours before biochemistry samples are taken for measurement of phosphate, calcium, creatinine, and lipids. Participants are to bring their oral study intervention with them to each study visit and have that day's intake at the site.

In case a grade 3 or grade 4 laboratory abnormality occurs, that is considered to be clinically significant by the investigator, a confirmatory test must be performed preferably within 48 hours but no later than 72 hours after the results have become available.

For this study, the laboratory abnormality of cholesterol increase is identified as laboratory abnormality of interest.

Note: cholesterol increase is a laboratory abnormality of interest specific for JNJ-6379, which was part of the study intervention up to Protocol Amendment 4. Because participants who were enrolled before Protocol Amendment 5 was in effect, also received JNJ-6379 as part of their study intervention, monitoring of cholesterol increases will be continued.

## 8.5. Adverse Events and Serious Adverse Events

Special attention will be paid to those participants who discontinue the study for an AE, or who experience an AE of at least grade 3, or an SAE. The grades are based on the DAIDS Toxicity Grading Scale (Section 10.9, Appendix 9, DAIDS Table).

Timely, accurate, and complete reporting and analysis of safety information from clinical studies are crucial for the protection of participants, investigators, and the sponsor, and are mandated by regulatory agencies worldwide. The sponsor has established Standard Operating Procedures in

conformity with regulatory requirements worldwide to ensure appropriate reporting of safety information; all clinical studies conducted by the sponsor or its affiliates will be conducted in accordance with those procedures.

Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally acceptable representative) for the duration of the study.

For further details on AEs and SAEs (Definitions and Classifications; Attribution Definitions; Severity Criteria; Special Reporting Situations; Procedures) as well as product quality complaints, refer to Section 10.4, Appendix 4, Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting.

# 8.5.1. Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information

#### All Adverse Events

All adverse events and special reporting situations, whether serious or non-serious, will be reported from the time a signed and dated ICF is obtained until completion of the participant's last study-related procedure, which may include contact for follow-up of safety. SAEs, including those spontaneously reported to the investigator within 30 days after the last dose of study intervention, must be reported using the SAE Form. The sponsor will evaluate any safety information that is spontaneously reported by an investigator beyond the time frame specified in the protocol.

#### **Serious Adverse Events**

All SAEs occurring during the study must be reported to the appropriate sponsor contact person by study-site personnel immediately and within 24 hours of their knowledge of the event.

Information regarding SAEs will be transmitted to the sponsor using the SAE Form, which must be completed and signed by a physician from the study site, and transmitted to the sponsor within 24 hours. The initial and follow-up reports of a SAE should be made by facsimile (fax).

# 8.5.2. Method of Detecting Adverse Events and Serious Adverse Events

Care will be taken not to introduce bias when detecting AEs or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about adverse event occurrence.

#### **Solicited Adverse Events**

Solicited AEs are predefined local (at the injection site) for which the participant is specifically questioned. Information on ISRs (Section 8.5.6.1) will be solicited.

### **Unsolicited Adverse Events**

Unsolicited adverse events are all adverse events for which the participant is not specifically questioned.

## 8.5.3. Follow-up of Adverse Events and Serious Adverse Events

Adverse events, including pregnancy, will be followed by the investigator as specified in Section 10.4, Appendix 4, Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting.

## 8.5.4. Regulatory Reporting Requirements for Serious Adverse Events

The sponsor assumes responsibility for appropriate reporting of adverse events to the regulatory authorities. The sponsor will also report to the investigator (and the head of the investigational institute where required) all suspected unexpected serious adverse reactions (SUSARs). The investigator (or sponsor where required) must report SUSARs to the appropriate Independent Ethics Committee/Institutional Review Board (IEC/IRB) that approved the protocol unless otherwise required and documented by the IEC/IRB.

## 8.5.5. Pregnancy

All initial reports of pregnancy in female participants or partners of male participants must be reported to the sponsor by the study-site personnel within 24 hours of their knowledge of the event using the appropriate pregnancy notification form. Abnormal pregnancy outcomes (eg, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs and must be reported using the SAE Form. Any participant who becomes pregnant during the study must discontinue further investigational intervention (JNJ-3989).

Follow-up information regarding the outcome of the pregnancy and any postnatal sequelae in the infant will be required.

### 8.5.6. Adverse Events of Special Interest

Events of Special Interest are significant AEs that are judged to be of special interest because of clinical importance, known class effects or based on nonclinical signals. Events of Special Interest that will be carefully monitored during the study include ISRs, ALT/AST elevations, renal complications, hematological abnormalities, and events related to cholesterol increase (Section 8.4.4, Clinical Safety Laboratory Assessments). In addition, the following toxicities will also be carefully monitored: rash and acute systemic allergic reactions.

For participants reporting ALT/AST elevations, rash, ISRs, acute systemic allergic reactions, renal complications, and hematological abnormalities as specified in the DAIDS Toxicity Grading Scale (see Section 10.9, Appendix 9, DAIDS Table), the following should be done.

Note: renal complications and cholesterol increase are AESIs specific for JNJ-6379, which was part of the study intervention up to Protocol Amendment 4 and has been removed with the implementation of Protocol Amendment 5. Because participants who were enrolled before Protocol Amendment 5 was in effect, also received JNJ-6379 as part of their study intervention, the AESIs have not been revised with the removal of JNJ-6379. For all participants having received at least one dose of JNJ-6379, renal safety monitoring will be continued.
## 8.5.6.1. Injection Site Reactions

At the time points specified in the Schedule of Activities or at an unscheduled visit if needed, an evaluation of the injection site will be performed based on participant's description and/or physical examination. Evaluations will be recorded in the source documents and will include at a minimum the time of occurrence, time of resolution and a description of the abnormality including its maximal diameter. For each ISR, information on pain, erythema, induration and pruritus should be obtained as specified in the DAIDS scale (see Section 10.9, Appendix 9, DAIDS Table).

All ISRs (including ISRs below grade 1) should be recorded in the special events section of the CRF.

Digital pictures will be taken when considered appropriate; all efforts should be made to collect images in case of grade 3 and 4 ISRs. Digital pictures will only be taken and collected from participants who consent separately to this component of the study. If digital pictures are required, they should be de-identified and provided to the sponsor.

## 8.5.6.2. Intervention-emergent ALT/AST Elevations

Elevated liver enzyme activity can be triggered by the underlying HBV disease as well as by the study intervention.

Management of intervention-emergent ALT/AST elevations is presented graphically in Section 10.6, Appendix 6, Intervention-emergent ALT/AST Elevations, and is described below.

Any intervention-emergent elevation of ALT and/or AST≥3x ULN and≥3x nadir (ie, lowest value during study participation) should trigger an assessment of confounding factors (alcohol intake, change in concomitant medication, and comorbidities) and should trigger a confirmatory study visit to repeat laboratory testing of ALT, AST, ALP, AFP, bilirubin (total and direct), INR, albumin, and HBV DNA. Additional tests should be considered based on clinical judgement (refer to Section 10.6, Appendix 6, Intervention-emergent ALT/AST Elevations). The confirmatory visit should be scheduled as soon as possible, preferably within 7 days of the receipt of the initial ALT/AST results. In case the repeat laboratory testing shows an isolated ALT/AST elevation (ie, with stable albumin, bilirubin [total and direct], and INR) the participant may continue study intervention. In case of confirmed ALT elevation >1,000 U/L and ≥3x the baseline value, JNJ-3989 (and PegIFN-α2a, if applicable) should be discontinued. In both cases, NA treatment should be continued. The participant will be monitored on a weekly basis (laboratory testing of ALT, AST, ALP, AFP, bilirubin [total and direct], INR, albumin, and HBV DNA) until ALT and AST levels have returned to <5x ULN and HBV DNA is <20,000 IU/mL.

If the ALT and/or AST level is  $\ge 3x$  ULN and  $\ge 3x$  nadir and is associated with any of the following laboratory results or clinical symptoms:

- INR ≥1.5, OR
- direct bilirubin >1.5x ULN, OR
- serum albumin <3.0 g/dL, OR

- ascites, hepatic encephalopathy, or liver-related symptoms (eg, severe fatigue, nausea, vomiting, right upper quadrant pain in the absence of an alternative medical explanation), OR
- other indication of reduced liver function

the participant should discontinue JNJ-3989 (and PegIFN- $\alpha$ 2a, if applicable) and should be monitored on a weekly basis or as per good clinical practice until ALT and AST levels have returned to <5x ULN and HBV DNA is <20,000 IU/mL and, if present, liver-related symptoms have improved. NA treatment should be continued. Additional tests should be considered based on clinical judgement (refer to Section 10.6, Appendix 6, Intervention-emergent ALT/AST Elevations).

In case of prolonged ALT elevation >3x ULN AND >2x nadir, which lasts at least 12 weeks, the decision to continue JNJ-3989 and/or PegIFN- $\alpha$ 2a should be based upon virologic parameters (eg, HBsAg, HBV DNA) and should be made in consultation with the sponsor.

PegIFN- $\alpha$ 2a may need to be discontinued in clinically significant cases of ALT increase or in combined increase of ALT and direct bilirubin. Refer to the prescribing information for PegIFN- $\alpha$ 2a. 41,42

The NA re-treatment criteria during follow-up are presented in Section 6.6.2.

## 8.5.6.3. Complications From Liver Biopsy

Participants should be closely monitored for liver biopsy complications. Infection and internal bleeding and/or puncture of other internal organs (gall bladder, lung, intestine or kidney) can lead to serious complications (uncommon 1 in 1000 to 1 in 100) including the need for emergency surgery, blood transfusion or removal of organs. Deaths directly related to liver biopsy occur rarely (approximately 1 in every 10,000 biopsies). Criteria for participant selection and laboratory assessments are in place to minimize these risks. Additional investigations can be performed at the investigator's discretion. Participants must be treated as clinically appropriate.

## 8.5.6.4. Renal Complications

If renal complications develop, participants should be closely monitored for disturbances in creatinine clearance. Additional investigations can be performed at the investigator's discretion. Participants must be treated as clinically appropriate.

Participants who develop confirmed grade 3 or 4 eGFR<sub>cr</sub> abnormalities with reduction from baseline by at least 10 mL/min/1.73 m<sup>2</sup> will change their NA from tenofovir disoproxil to ETV or TAF (if the patient was receiving tenofovir disoproxil), according to the prescribing information. If the abnormality persists despite change of NA or if the patient is not receiving tenofovir disoproxil, he or she will permanently discontinue the intake of JNJ-3989 (and PegIFN- $\alpha$ 2a, if applicable) if the abnormality is considered at least possibly related to JNJ-3989, and should be followed appropriately until resolution of AE or toxicity. Rechallenge is not allowed.

For all participants having received at least one dose of JNJ-6379, renal safety monitoring will be continued.

## 8.5.6.5. Hematologic Abnormalities

Mild thrombocytopenia was observed in recently conducted non-clinical toxicology studies with the combination of JNJ-3989 and JNJ-6379. In addition, in a 3-month combination study with 80 rats, 1 rat developed pancytopenia related to bone marrow depletion after 23 days of dosing. Previously, in a 9-month dog study in 24 dogs treated with JNJ-6379 alone, pancytopenia which correlated with a marked increase in plasma cell-like cells in the bone marrow was observed in 1 dog after 60 days of dosing.

No thrombocytopenia or pancytopenia has been observed in the ongoing JADE study (56136379HPB2001) investigating JNJ-6379/Placebo with or without NA treatment. All 232 participants have completed at least 24 weeks of study intervention. In a Phase 1 study with JNJ-3989, mild (Grade 1) transient thrombocytopenia was observed in 6 out of 84 participants receiving 3 SC injections of JNJ-3989 alone over a period of up to 12 weeks with background of NA. The transient thrombocytopenia was not considered clinically significant. No thrombocytopenia or pancytopenia was observed in 12 participants when JNJ-3989 and JNJ-6379 were given in combination over a 12-week period.

Based on the non-clinical findings, any relevant abnormalities in hematologic parameters will be carefully monitored as described below:

- Platelet counts: <100, 000 cells/mm³ (at least Grade 2 [DAIDS]) or <100 GI/L or reduction from baseline by at least 50% baseline
- Hemoglobin: Decrease from baseline of at least 2 g/dL from baseline or at least Grade 2 (DAIDS)
- Reticulocyte count: Reduction to <0.5% of the RBC count
- Neutrophil count: Treatment-emergent reduction to at least Grade 2 (DAIDS)

In case any one of the above criteria are met, a confirmatory visit should be scheduled as soon as possible, preferably within 7 days of the receipt of the initial results. Confirmation of the results will trigger weekly or biweekly (every other week) unscheduled visits until improvement or stabilization of the respective parameter(s). Stabilization is defined as no further significant reduction over two consecutive visits.

In case of confirmed Grade 3 or Grade 4 hematologic abnormalities, discontinuation of JNJ-3989 (and PegIFN- $\alpha$ 2a, if applicable]) should be considered. In case of discontinuation, NA treatment should be continued.

## 8.5.7. Other Toxicities

#### 8.5.7.1. Rash

Participants should be informed that they should contact their doctor immediately when they notice any generalized skin reaction. This skin reaction should be evaluated in the clinic the same day (if possible) or the next day.

All rash events should be captured in the special events section of the CRF. A set of separate Rash pages will be completed in case of a rash event.

Monitoring of the evolution of rash events will be performed as described in Table 6 in Section 10.5, Appendix 5, Rash Management.

When safety blood samples are drawn as per the rash management guidelines, these should be processed by the local laboratory. The following parameters will need to be tested: AST, ALT, sedimentation rate, complete blood cell count (including hemoglobin, hematocrit, RBC count, WBC count, differential count [neutrophils, lymphocytes, monocytes, eosinophils, and basophils], and platelet count), and creatinine. The values of the local laboratory assessments need to be transcribed in the CRF by the study site personnel.

The participant may be treated symptomatically until the rash resolves. Oral antihistamines (eg, cetirizine, levocetirizine) and/or topical corticosteroids may provide symptomatic relief but effectiveness of these measures has not been established. If systemic corticosteroids exceeding 5 mg of prednisolone equivalent/day are required for treatment of rash, JNJ-3989 (and PegIFN- $\alpha$ 2a, if applicable) needs to be permanently discontinued. NA treatment can be continued. If the rash is considered to be most likely due to concomitant illness or non-study interventions, standard management, including discontinuation of the likely causative agent, should be undertaken.

## 8.5.7.2. Acute Systemic Allergic Reactions

## Grade 1 (Localized Urticaria [Wheals] With no Medical Intervention Indicated)

Participants may continue the intake of study interventions.

Cetirizine, levocetirizine, topical corticosteroids or antipruritic agents may be prescribed.

Participants should be advised to contact the investigator immediately if there is any worsening of the acute systemic allergic reaction.

# Grade 2 (Localized Urticaria With Intervention Indicated, or Mild Angioedema With no Intervention Indicated)

Participants may continue the intake of study interventions.

Cetirizine, levocetirizine, topical corticosteroids or antipruritic agents may be prescribed.

Participants should be advised to contact the investigator immediately if there is any worsening of the acute systemic allergic reaction, in which case the participant will permanently discontinue the intake of JNJ-3989 (and PegIFN- $\alpha$ 2a, if applicable). Rechallenge is not allowed. The participant's NA treatment may be discontinued based on investigator judgement in consultation with the sponsor.

# Grade 3 (Generalized Urticaria, Angioedema With Intervention Indicated, or Symptoms of Mild Bronchospasm) and Grade 4 (Acute Anaphylaxis, Life-Threatening Bronchospasm, or Laryngeal Edema)

Participants will permanently discontinue the intake of JNJ-3989 (and PegIFN- $\alpha$ 2a, if applicable). Rechallenge is not allowed. The participant's NA treatment may be discontinued based on investigator judgement in consultation with the sponsor.

Participants will be treated as clinically appropriate. Participants should be followed until resolution of the AE and standard management should be undertaken.

## 8.6. Treatment of Overdose

For this study, any dose of JNJ-3989 greater than the protocol-specified dose (refer to Section 6.1) will be considered an overdose; any dose of NA (ETV, tenofovir disoproxil, or TAF) and PegIFN-α2a greater than the prescribed dose will be considered an overdose. The sponsor does not recommend specific therapeutic intervention for an overdose.

In the event of an overdose, the investigator or treating physician should:

- Contact the Medical Monitor immediately.
- Closely monitor the participant for AE/SAE and laboratory abnormalities.
- Obtain a plasma sample for PK analysis as soon as possible from the date of the last dose of study intervention if requested by the Medical Monitor (determined on a case-by-case basis).
- Document the quantity of the excess dose as well as the duration of the overdosing in the CRF.

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the Medical Monitor based on the clinical evaluation of the participant.

#### 8.7. Pharmacokinetics

Plasma samples will be used to evaluate the PK of JNJ-3989 (ie, JNJ-3976 and JNJ-3924), and, optionally, JNJ-6379, NA and/or PegIFN-α2a, as applicable. Serum collected for PK may additionally be used to evaluate safety or efficacy aspects that address concerns arising during or after the study period. Genetic analyses will not be performed on these samples. Participant confidentiality will be maintained.

## 8.7.1. Evaluations

Venous blood samples will be collected for measurement of plasma concentrations of JNJ-3976, JNJ-3924, NA (ETV, TAF, or tenofovir) and PegIFN- $\alpha$ 2a, as applicable, at time points specified in the Schedule of Activities. Bioanalysis of NA and PegIFN- $\alpha$ 2a is optional at the discretion of the sponsor. Bioanalysis of JNJ-6379 may also be done on samples collected from participants who received JNJ-6379 up to Protocol Amendment 4.

All participants will have sparse PK sampling on Day 1 and at Weeks 4, 12, and 24 (and at early withdrawal). All participants who consent to participate in the intensive PK substudy (optional)

will undergo intensive PK sampling at Week 4. If necessary (eg, for operational reasons), this visit may be scheduled at Week 8, 12, or 16.

## 8.7.2. Analytical Procedures

## **Pharmacokinetics**

Plasma samples will be analyzed to determine concentrations of JNJ-3976 and JNJ-3924 using a validated, specific, and sensitive liquid chromatography-fluorescence hybridization method under the supervision of the sponsor.

At the sponsor's discretion, plasma samples may be analyzed to determine concentrations of JNJ-6379 and/or NA and/or PegIFN- $\alpha$ 2a using a validated, specific, and sensitive liquid chromatography-mass spectrometry method under the supervision of the sponsor.

Plasma PK samples may be stored for future exploratory analysis of protein binding or the metabolite profile. Genetic analyses will not be performed on these plasma samples. Participant confidentiality will be maintained.

## 8.7.3. Pharmacokinetic Parameters and Evaluations

#### **Parameters**

Plasma concentration-time data for JNJ-3989 (ie, JNJ-3976 and JNJ-3924) and, optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a will be analyzed via noncompartmental methods for all participants who underwent intensive PK sampling. The main PK parameter will be area under the plasma concentration-time curve over 24 hours (AUC<sub>24h</sub>),  $C_{max}$ ,  $t_{max}$ , plasma trough concentration ( $C_{0h}$ ), plasma concentration at the end of the dosing interval ( $\tau$ ) ( $C_{\tau}$ ), and minimum plasma concentration ( $C_{min}$ ). Additional exposure parameters may be calculated if applicable.

Data from this study may be combined with data from a selection of Phase 1 and 2 studies via population PK modelling. Individual estimates of PK parameters may be generated from the population PK analysis for potential use in exposure-response analysis.

## 8.8. Pharmacokinetics/Pharmacodynamics

Relationships of individual PK parameters for JNJ-3976, JNJ-3924, and, optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a, with selected liver and blood biomarkers, and/or with selected safety endpoints may be evaluated.

## 8.9. Host Genetics

A pharmacogenomic blood sample will be collected (preferably at baseline) to allow for the identification of genetic factors that may influence the efficacy, safety, or PK of the study intervention, to identify genetic factors associated with HBV infection, or to develop assays for the study intervention or HBV infection.

A blood sample will be taken for HLA typing as indicated in the Schedule of Activities. In addition, host DNA blood samples to allow for epigenetic analyses will be collected.

#### 8.10. Host Biomarkers

The study includes collection of blood samples for exploratory analysis of host blood biomarkers at the host RNA, protein, and cell level. Sampling will be performed in all participants at the time points indicated in the Schedule of Activities.

Samples can only be used for research related to study intervention or HBV infection or may be used to develop tests/assays related to study intervention or HBV infection.

Blood samples will be taken at the time points indicated in the Schedule of Activities which can be used to explore immunogenicity of JNJ-3989. The emergence of antibodies to JNJ-3989 (antidrug antibodies) might be analyzed using assays such as an enzyme-linked immunosorbent assay.

## 8.11. Medical Encounters

Eventual medical encounters will be collected in the CRF by the investigator and study site personnel for all participants throughout the study.

## 9. STATISTICAL CONSIDERATIONS

Statistical analysis will be done by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be used to analyze the efficacy and safety data is outlined below. Specific details will be provided in the Statistical Analysis Plan.

The primary analysis will be performed at the time when all participants have completed Week 48 or discontinued earlier. The final analysis will be performed when all participants have completed the last study visit (Follow-up Week 48) or discontinued earlier. For the IAs, please refer to Section 9.5.

## 9.1. Statistical Hypotheses

As this is an exploratory study, no hypothesis will be tested.

## 9.2. Sample Size Determination

This study aims to enroll 18 to 24 participants in total across Panels 1 and 2, ie, 8 to 12 participants per study panel.

Due to the exploratory nature of the study, the sample size was determined based on clinical and feasibility considerations related to the liver biopsy procedures performed multiple times during the study, rather than a formal statistical calculation. Nevertheless, a sample size of 8 to 12 participants each in Panel 1 and 2 is considered sufficient to provide adequate precision of the estimate of the primary endpoint (change from baseline to Week 40 in the proportion of HBsAgpositive hepatocytes) as estimated by the 80% confidence interval (CI).

For the estimation of the absolute change in the proportion of HBsAg-positive hepatocytes from baseline to Week 40 for the overall study population (Panels 1 and 2 combined), the following assumptions were made. Assuming an absolute reduction of 70% in Panel 1 (75% at baseline

versus 5% at Week 40) and 29% in Panel 2 (30% at baseline versus to 1% at Week 40), and assuming an inter-subject variability of the change equal to 0.5 on the logit scale in both panels, a binomial model<sup>40</sup> including visit as covariate with normal random effects provides an expected width of the 80% CI of 16.7% for N 24, a width of 17.9% for N 20, and a width of 20.3% for N 16. The point estimates (two-sided 80% CI) are 50.8% (42.5%; 59.1%) with N 24, 50.7% (41.8%; 59.7%) with N 20, and 50.6% (40.5%; 60.8%) with N 16.

For the between-panel difference in the absolute reduction in the proportion of HBsAg-positive hepatocytes from baseline to Week 40 using the binomial model described above augmented with panel as an additional covariate and the same inter-subject variability, the estimated width of the two-sided 80% CI around the difference (Panel 1 Panel 2) is 17.6% for N 24 (12 per panel), 19.3% for N 20 (10 per panel), and 21.2% for N 16 (8 per panel). The point estimates (80% CI) are 40.4% (31.5%; 49.2%) for N 24, 39.2% (29.6%; 48.9%) for N 20, and 39.4% (28.8%; 50.0%) for N 16.

In addition, N 20 would also be sufficient to provide adequate precision for a between-panel difference in the relative change from baseline of at least 26% in case of large inter-subject variability.

Assuming a drop rate of 20%, the sample size will be therefore set to 12 participants per panel for Panels 1 and 2.

## 9.3. Populations for Analyses

For purposes of analysis, the following populations are defined:

| Population | Description |
|---|---|
| Randomized | All participants who were randomized in the study |
| Enrolled | All participants who were enrolled in the study |
| Intent-to-treat | All participants who were either randomly assigned or enrolled to an intervention arm and |
| (ITT) | received at least 1 dose of study intervention. Participants will be analyzed according to the |
| | study intervention they were randomly assigned or enrolled to. |
| Safety | All participants who received at least 1 dose of study intervention. Participants will be |
| | analyzed according to the study intervention they actually received. |

## 9.4. Statistical Analyses

The Statistical Analysis Plan will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints.

Given the exploratory nature of the study and the limited sample size per panel, no statistical testing will be performed. All data will be summarized descriptively including 80% confidence intervals as appropriate.

## 9.4.1. Analysis of Efficacy and Antiviral Activity

To evaluate the efficacy and antiviral activity in blood and liver, the primary analysis set will be the ITT population. Efficacy and antiviral activity will be assessed for participants in Panels 1

and 2. For all efficacy and antiviral activity endpoints, unless specified otherwise, the following comparisons will be addressed:

1. Overall population, pooling all participants regardless of panels.

Between Panels 1 and 2: HBeAg-positive patients who are not currently being treated versus HBeAg-negative patients being virologically suppressed by NA treatment.

All efficacy summaries will be presented with descriptive statistics, overall and by study panel.

If the endpoint is continuous, the descriptive statistics will include the number of participants, mean, standard deviation (SD), median, range, and interquartile range. If the endpoint is binary or categorical, the frequency distribution with the number and percentage of participants in each category will be calculated.

Graphic displays will also be used to summarize the data and to visualize trends by study panel.

Where applicable, additional specifics for analyses of primary, secondary, and exploratory endpoints are detailed below.

## 9.4.1.1. Analysis of the Primary Endpoint

The primary endpoint is the change between baseline and on-treatment liver biopsy (Week 40) in terms of the proportion of HBsAg positive hepatocytes. The primary endpoint will be summarized descriptively and modelled with an appropriate statistical model accounting for the number of hepatocytes sampled in each liver biopsy. The change from baseline will be summarized for the overall study population and within each panel, together with the between-panel difference in the change..

No imputation rule will be applied for the analysis on the ITT population since only complete cases will be considered. In addition, the treatment policy strategy will be followed to account for the occurrence of intercurrent events, such as treatment discontinuation prior to Week 40, ie, all biopsies collected at Week 40 will be used, regardless of occurrence of treatment discontinuation prior to Week 40. This strategy is supported by the small sample size, the exploratory nature of the study and ethical considerations.

In addition, a sensitivity analysis on the ITT population will be combining a treatment policy strategy with the Baseline Observation Carried Forward (BOCF) approach.

## 9.4.1.2. Analysis of Secondary Endpoints

Secondary endpoints will be analyzed on the ITT population.

## **Changes in Intrahepatic Immune Response**

Variation in proportion of major cell populations, such as but not limited to CD45+ T-cells, CD4+ T-cells, CD8+ T-cells, Natural Killer cells, and dendritic cells, defined by single cell

transcriptomics (in FNABs) and immunofluorescence staining (in core needle biopsies), will be assessed at Week 40 and compared to baseline, overall and by study panel.

The functional characterization of major cell populations will be assessed by transcriptomics and/or proteomics for major cell populations of interest at Week 40 and compared to baseline similarly.

## **Changes in Intrahepatic Viral Nucleic Acids and Proteins**

Changes from baseline in cccDNA level and/or transcriptional activity will be assessed using the general considerations outlined above.

Furthermore, the difference in the level of infected hepatocytes at baseline will be assessed by comparing cccDNA level and/or transcriptional activity.

Analyses of other viral markers will be performed descriptively. Statistical analyses will depend on the assay technology applied and the scope of the analyses.

## 9.4.1.3. Analysis of Exploratory Endpoints

Exploratory endpoints will be analyzed on the ITT population.

The association between intrahepatic markers and blood (immune and viral) markers will be explored both at baseline and on-treatment by study panel using graphical displays and relevant correlation coefficients.

Impact of baseline characteristics on selected efficacy variables and their association with intrahepatic and blood markers will also be evaluated using similar methods.

Identification of markers (either intrahepatic or blood) that could potentially be associated with selected efficacy variables (such as decrease in blood HBsAg levels, intrahepatic cccDNA levels or any other relevant variables) will be conducted. Impact of treatment on different blood and hepatic markers will also be evaluated.

## 9.4.2. Safety Analyses

All safety analyses will be made on the Safety Population (Section 9.3).

Safety will be evaluated by means of descriptive summaries of AEs including AEs of special interest to any of the study interventions, clinical laboratory tests, ECGs, vital signs, and physical examinations. The safety analysis will be done by study phase. Results will be presented in tabular format and/or graphically over time, as appropriate.

#### **Adverse Events**

The verbatim terms used in the CRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Intervention-emergent AEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that has worsened since baseline. All reported intervention-emergent AEs will be included in the

analysis. For each AE, the percentage of participants who experience at least 1 occurrence of the given event will be summarized.

Summaries, listings, datasets, or participant narratives may be provided, as appropriate, for those participants who die, who discontinue intervention due to an AE, or who experience a severe or a serious AE.

Adverse Events Related to the Applied Study Procedures

Summaries, listings, datasets, or participant narratives will be provided, as appropriate, for those enrolled participants who die, or who experience an AE or a severe or a serious AE related to the applied study procedures.

All AE's linked to the study procedure will be evaluated in conjunction with other systemic symptoms and laboratory abnormalities: information on time of onset, duration of events, time to resolution, concomitant therapies, and relationship to study procedures (eg, liver biopsies, blood collection and leukapheresis) will be summarized and described in the report.

## **Clinical Laboratory Tests**

Laboratory data will be summarized by type of laboratory test. Descriptive statistics will be calculated for each laboratory analyte at baseline and for observed values and changes from baseline at each scheduled time point by study phase. A graphical presentation of changes from baseline over time in selected laboratory tests will be also used.

The laboratory abnormalities will be determined according to the criteria specified in the DAIDS Toxicity Grading Scale (see Section 10.9, Appendix 9, DAIDS Table) or in accordance with the normal ranges of the clinical laboratory if no gradings are available. The number and percentage of the participants who experience (worst) laboratory abnormalities will be tabulated by intervention arm and study phase. Shifts in toxicity grades will be tabulated by study phase.

## Electrocardiogram

Electrocardiogram data will be summarized by ECG parameter. Descriptive statistics will be calculated at baseline and for observed values and changes from baseline at each scheduled time point. Frequency tabulations of the abnormalities will be made.

The ECG variables that will be analyzed are heart rate, PR interval, QRS interval, QT interval, and QTcF.<sup>13</sup>

Descriptive statistics of QTc intervals and changes from baseline will be summarized at each scheduled time point. The percentage of participants with QTc interval >450 milliseconds, >480 milliseconds, or >500 milliseconds will be summarized, as will the percentage of participants with QTc interval increases from baseline >30 milliseconds or >60 milliseconds. Shifts in QTc interval categories will be tabulated by study phase.

All clinically relevant abnormalities in ECG waveform that are changes from the baseline readings will be reported (eg, changes in T-wave morphology or the occurrence of U-waves.

## **Vital Signs**

Vital signs including temperature, pulse rate, and supine blood pressure (SBP and DBP) will be summarized over time, using descriptive statistics and/or graphically. The percentage of participants with values beyond clinically important limits will be summarized.

## **Physical Examinations**

Physical examination findings will be summarized at each scheduled time point. Descriptive statistics will be calculated at baseline and for observed values and changes from baseline at each scheduled time point. Frequency tabulations of the abnormalities will be made.

## 9.4.3. Other Analyses

## **Pharmacokinetic Analyses**

Descriptive statistics (number of participants, mean, SD, coefficient of variation, geometric mean, median, minimum, and maximum) will be calculated for the plasma concentrations of JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN-α2a, as applicable, and for the derived plasma PK parameters (noncompartmental analysis).

Special attention will be paid to the plasma concentrations and PK parameters of those participants who discontinued the study for an AE, or who experienced an AE  $\geq$ Grade 3 or an SAE.

For each participant with intensive PK sampling, plasma concentration-time data of JNJ-3976, JNJ-3924, and/or JNJ-6379, and/or NA and/or PegIFN-α2a will be graphically presented. Similarly, graphs of the mean plasma concentration-time profiles and overlay graphs with combined individual plasma concentration time profiles will be produced. Pharmacokinetic parameters will be subjected to an exploratory graphical analysis, including various transformations, to get a general overview.

Population PK analysis of plasma concentration-time data of JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a may be performed using nonlinear mixed-effects modeling. Data may be combined with those from Phase 1 and/or 2 studies to support a relevant structural model. Available baseline characteristics (eg, demographics, laboratory variables, genotypes) may be included in the model as necessary. Details will be given in a population PK analysis plan and results of the population PK analysis, if applied, will be presented in a separate report.

Individual estimates of PK parameters may be generated from the population PK analysis for potential use in exposure-response analysis.

## Pharmacokinetic/Pharmacodynamic Analyses

Relationships of PK parameters for JNJ-3976, JNJ-3924, and optionally, JNJ-6379, NA and/or PegIFN- $\alpha$ 2a with selected efficacy and with selected safety endpoints may be evaluated and graphically displayed.

Modeling of key PD parameters (eg, HBsAg, HBV DNA) may be performed using population PK/PD. If PK/PD modeling of key efficacy endpoints is performed, treatment effect and possible covariates such as disease progression may be investigated. Other biomarkers may be explored at the sponsor's discretion.

## **Resistance Analysis**

The results of HBV viral sequencing will be evaluated by the sponsor virologist. Relevant changes in amino acid and/or nucleic acid variations (eg, substitutions) in the HBV genome will be tabulated and described.

Additional exploratory characterization of the HBV viral sequence and phenotype may be performed and reported separately.

## Pharmacogenomic Analysis

The statistical approach for analyzing the exploratory host DNA research, including epigenetic analyses, may depend on the objective of the analyses (efficacy, safety, and PK) and possibly relevant genes at the time of analysis. Analyses will be conducted at the sponsor's discretion, will always be under the sponsor's supervision, and results will be presented either in the clinical study report or a separate report.

## **Host Exploratory Biomarker Analysis**

Statistical approaches to explore correlations between treatment response/clinical outcome and blood and liver biomarkers vary and depend on the different data types of the applied technology platforms, as well as on the extent of observed differences between participants. Analyses will be conducted at the sponsor's discretion, will always be under the sponsor's supervision, and results will be presented either in the clinical study report or a separate report.

## 9.5. Interim Analysis

Two IAs may be performed: when all participants have completed Week 20 in the intervention phase (or discontinued earlier) and when they have completed Week 72 in the follow-up phase (ie, Follow-up Week 24) (or discontinued earlier). These IAs will be performed by the sponsor to support interactions with health authorities, as well as to support internal decisions about additional studies and/or investigation of other combination regimens.

Both primary and interim analyses will be based on all data available at the predefined cut-off time points and may include data at later time points for those participants who have reached subsequent visits.

## 9.6. Independent Flare Expert Panel

An IFLEP will be appointed for this study. The IFLEP is composed of 3 independent medical experts with experience and expertise in hepatitis B and its treatment. The IFLEP will monitor ALT flares and will make recommendations regarding flare management based on an analysis of aggregate data.

In order to allow for an unbiased assessment, members of the committee will not serve as study investigators.

Further details on the IFLEP process will be included in the IFLEP charter.

## 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

## 10.1. Appendix 1: Abbreviations and Definitions of Terms

AE adverse event
AFP alpha-fetoprotein
ALP alkaline phosphatase
ALT alanine aminotransferase
AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

AUC<sub>0-xh</sub> area under the plasma concentration-time curve from administration to x h

AUC<sub>0-last</sub> area under the plasma concentration-time curve from administration to last quantifiable sampling

point

 $AUC_{\tau}$  area under the plasma concentration-time curve over the dose interval (tau) at steady-state

AUC<sub>∞</sub> area under the plasma concentration-time curve to last sampling point from time zero extrapolated

to infinity

bpm beats per minute

CAM capsid assembly modulator

cccDNA covalently closed circular deoxyribonucleic acid CKD-EPI Chronic Kidney Disease Epidemiology Collaboration

CL/F total apparent oral clearance C<sub>max</sub> maximum plasma concentration

CRF case report form
CT computed tomography
CYP cytochrome P450

DAIDS Division of Acquired Immunodeficiency Syndrome

DBP diastolic blood pressure
DDI drug-drug interaction
DNA deoxyribonucleic acid

EASL European Association for the Study of the Liver

ECG electrocardiogram
eDC electronic data capture
EFD embryofetal development

eGFR estimated glomerular filtration rate

eGFR<sub>cr</sub> estimated glomerular filtration rate based on serum creatinine

ELISpot enzyme-linked immunospot

EOS end of study

EOSI end of study intervention

ETV entecavir

FNAB fine needle aspiration biopsy FSH Follicle-stimulating hormone

FU Wx Follow-up Week x
GCP Good Clinical Practice
GLP Good Laboratory Practice
HBc hepatitis B core protein

HBcrAg hepatitis B core-related antigen HBe hepatitis B e

HBeAg hepatitis B e antigen
HBs hepatitis B surface
HBsAg hepatitis B surface antigen

HBV hepatitis B virus

HCC hepatocellular carcinoma

HCV hepatitis C virus HDV hepatitis D virus HEV hepatitis E virus

HIV-1(-2) human immunodeficiency virus type 1 (type 2)

HLA human leukocyte antigen HRT hormonal replacement therapy IA interim analysis
IB Investigator's Brochure
ICF informed consent form

ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for

Human Use

ICMJE International Committee of Medical Journal Editors

ICS intracellular cytokine staining
IEC Independent Ethics Committee
IFLEP Independent Flare Expert Panel

IFN interferon
IFN-γ gamma interferon
IgM immunoglobulin M

IL interleukin

INR International Normalized Ratio IRB Institutional Review Board ISR injection site reaction

ITT Intent-to-treat

IU/mL International Units Per Milliliter IWRS interactive web response system

LLN lower limit of normal LLOQ lower limit of quantification

MoA mode of action

MRI magnetic resonance imaging

NA nucleos(t)ide analog

NOAEL no observed adverse effect level

(q)PCR (quantitative) polymerase chain reaction

PD pharmacodynamic(s)

PegIFN-α2a pegylated interferon alpha-2a

PK pharmacokinetic(s)

PBMC peripheral blood mononuclear cell pgRNA pre-genomic ribonucleic acid PQC Product Quality Complaint

Q4W once every 4 weeks

qd once daily

QTcF QT interval corrected for heart rate according to Fridericia

RBC red blood cell RNA ribonucleic acid

RNAi ribonucleic acid interference SAE serious adverse event SBP systolic blood pressure

SC subcutaneous SD standard deviation siRNA small interfering RNA

SUSAR suspected unexpected serious adverse reaction

 $t_{1/2 term}$  terminal half-life

T4 thyroxine

 $t_{max}$  time to reach the maximum plasma concentration

TAF tenofovir alafenamide

TEAE treatment-emergent adverse event

TNF tumor necrosis factor

TSH thyroid-stimulating hormone
ULN upper limit of normal
WBC white blood cell

## **Definitions of Terms**

Study intervention Prior to Protocol Amendment 5: JNJ-73763989 (JNJ-3989), JNJ-56136379 (JNJ-6379) and

NA (either ETV, tenofovir disoproxil, or TAF)

As of Protocol Amendment 5: JNJ-73763989 (JNJ-3989) and NA (either ETV, tenofovir

disoproxil, or TAF)

Functional cure HBsAg seroclearance 24 weeks after end of treatment

HBsAg or HBeAg seroclearance

HBsAg or HBeAg negativity, respectively, based on the assay used

HBsAg or HBeAg seroconversion

HBsAg or HBeAg negativity and anti-HBs or anti-HBe antibody positivity, respectively

Virologic breakthrough

Confirmed on-treatment HBV DNA increase by >1 log<sub>10</sub> IU/mL from nadir or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had HBV DNA level

<LLOQ of the HBV DNA assay

ALT/AST nadir Lowest ALT/AST value during study participation

## 10.2. Appendix 2: Clinical Laboratory Tests

The following tests will be performed according to the Schedule of Activities by the central laboratory:

## **Protocol-Required Safety Laboratory Assessments**

| Laboratory | Parameters | | | |
|---|---|---|---|---|
| Assessments | Platelet count | DDC I-di | | White Disease Call (WDC) |
| Hematology | | RBC Indices: | | White Blood Cell (WBC) |
| | RBC count | Mean corpuscular volume | | count with Differential: |
| | Hemoglobin | Mean corpuscular | | Neutrophils |
| | Hematocrit | hemoglobin | | Lymphocytes |
| | Reticulocyte count | Mean corpuso | | Monocytes |
| | Reticulocyte index | hemoglobin c | oncentration | Eosinophils<br>Basophils |
| | Note: A WBC evaluation may include any abnormal cells, which will then be reported | | | |
| | by the laboratory. An RBC | evaluation may | include abno | rmalities in the RBC count, |
| | RBC parameters, or RBC me | orphology, whi | ch will then be | e reported by the laboratory. |
| | In addition, any other abnormal cells in a blood smear will also be reported. | | | |
| Clinical | Sodium | Lactic acid dehydrogenase | | |
| Chemistry | Potassium | | Uric acid | |
| | Chloride | | Calcium | |
| | Bicarbonate | | Phosphate | |
| | Blood urea nitrogen | | Albumin | |
| | Creatinine | | Total protein | |
| | Glucose | | Total cholesterol | |
| | AST/Serum glutamic-oxaloa | | High-density lipoprotein cholesterol | |
| | ALT/Serum glutamic-oxaloa | | Low-density lipoprotein cholesterol | |
| | Gamma-glutamyltransferase | | Triglycerides | |
| | Total, conjugated and uncon | jugated | Magnesium | |
| | bilirubin | | Lipase | |
| | Alkaline phosphatase | Amylase | | |
| | Creatine phosphokinase | | | |
| | Note: Creatinine clearance (eGFR <sub>cr</sub> calculated by the CKD-EPI formula) | | | |
| | assessed. | | | |
| | <i>Note:</i> Reflex testing of pancreatic amylase should be done in case of amylase or lipase | | | |
| | increase from screening onwards. | | | |
| Routine | Dipstick | | Sediment (if | dipstick result is abnormal) |
| Urinalysis | Specific gravity | | RBCs | |
| | pH | | WBCs | |
| | Glucose | | Epithelial ce | lls |
| | Protein | | Crystals | |
| | Blood | | Casts | |
| | Ketones | | Bacteria | |
| | Bilirubin | | | |
| | Urobilinogen | | | |
| | Nitrite | | | |
| | Leukocyte esterase | | | |

| | In case of a positive dipstick result, a urine sample will be set aside for additional | |
|---|---|---|
| | examination of the positive parameter at the central laboratory (eg, quantification as applicable). | |
| Urine | Creatinine | Glucose |
| Chemistry | Sodium | Protein |
| (quantitative | Phosphate | Albumin |
| measurement) | | |
| Renal | Retinol binding protein | |
| Biomarkers | Beta-2-microglobulin | |
| | <i>Note:</i> These renal biomarkers are to assess proximal renal tubular function. | |
| Other Tests | Serum pregnancy testing for women of childbearing potential at screening. | |
| | • Urine pregnancy testing for women of childbearing potential at the time points indicated in the Schedule of Activities. | |
| | Follicle-stimulating hormone (FSH) testing for postmenopausal women at screening. | |
| | • Testing for hepatitis A, B, C, D, and E virus and HIV-1 and -2 at screening. | |
| | • Testing for HBsAg, HBeAg, HBcrAg, and anti-HBs and anti-HBe antibodies at the time points indicated in the Schedule of Activities. | |
| | • Determination of coagulation parameters will be performed at the time points indicated in the Schedule of Activities. International Normalized Ratio (INR) will be calculated by the central laboratory. | |
| | Alpha-fetoprotein at screening. | |
| Other optional | • Testing for HIV-1 and -2, and hepatit | is A, C, D, and E. |
| tests in | Testing for CMV, HSV, EBV infection. | |
| response to ALT flare | | |
| (refer to | Ig-electrophoresis | |
| Section 10.6, | | |
| Appendix 6, | | |
| Intervention- | | |
| emergent | | |
| ALT/AST | | |
| Elevations) | | |
| Thyroid | TSH | |
| function tests | T4 | |

## 10.3. Appendix 3: Regulatory, Ethical, and Study Oversight Considerations

#### REGULATORY AND ETHICAL CONSIDERATIONS

## **Investigator Responsibilities**

The investigator is responsible for ensuring that the study is performed in accordance with the protocol, current International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guidelines on Good Clinical Practice (GCP), and applicable regulatory and country-specific requirements.

Good Clinical Practice is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human participants. Compliance with this standard provides public assurance that the rights, safety, and well-being of study participants are protected, consistent with the principles that originated in the Declaration of Helsinki, and that the study data are credible.

## **Protocol Amendments**

Neither the investigator nor the sponsor will modify this protocol without a formal amendment by the sponsor. All protocol amendments must be issued by the sponsor, and signed and dated by the investigator. Protocol amendments must not be implemented without prior IEC/IRB approval, or when the relevant competent authority has raised any grounds for non-acceptance, except when necessary to eliminate immediate hazards to the participants, in which case the amendment must be promptly submitted to the IEC/IRB and relevant competent authority. Documentation of amendment approval by the investigator and IEC/IRB must be provided to the sponsor. When the change(s) involve only logistic or administrative aspects of the study, the IEC/IRB (where required) only needs to be notified.

During the course of the study, in situations where a departure from the protocol is unavoidable, the investigator or other physician in attendance will contact the appropriate sponsor representative listed in the Contact Information page(s), which will be provided as a separate document. Except in emergency situations, this contact should be made before implementing any departure from the protocol. In all cases, contact with the sponsor must be made as soon as possible to discuss the situation and agree on an appropriate course of action. The data recorded in the CRF and source documents will reflect any departure from the protocol, and the source documents will describe this departure and the circumstances requiring it.

## Regulatory Approval/Notification

This protocol and any amendment(s) must be submitted to the appropriate regulatory authorities in each respective country, if applicable. A study may not be initiated until all local regulatory requirements are met.

## **Required Prestudy Documentation**

The following documents must be provided to the sponsor before shipment of study intervention to the study site:

- Protocol and amendment(s), if any, signed and dated by the principal investigator
- A copy of the dated and signed (or sealed, where appropriate per local regulations), written IEC/IRB approval of the protocol, amendments, ICF, any recruiting materials, and if applicable, participant compensation programs. This approval must clearly identify the specific protocol by title and number and must be signed (or sealed, where appropriate per local regulations) by the chairman or authorized designee.
- Name and address of the IEC/IRB, including a current list of the IEC/IRB members and their function, with a statement that it is organized and operates according to GCP and the applicable laws and regulations. If accompanied by a letter of explanation, or equivalent, from the IEC/IRB, a general statement may be substituted for this list. If an investigator or a member of the study-site personnel is a member of the IEC/IRB, documentation must be obtained to state that this person did not participate in the deliberations or in the vote/opinion of the study.
- Regulatory authority approval or notification, if applicable
- Signed and dated statement of investigator (eg, Form FDA 1572), if applicable
- Documentation of investigator qualifications (eg, curriculum vitae)
- Completed investigator financial disclosure form from the principal investigator, where required
- Signed and dated clinical trial agreement, which includes the financial agreement
- Any other documentation required by local regulations

The following documents must be provided to the sponsor before enrollment of the first participant:

- Completed investigator financial disclosure forms from all subinvestigators
- Documentation of subinvestigator qualifications (eg, curriculum vitae)
- Name and address of any local laboratory conducting tests for the study, and a dated copy of current laboratory normal ranges for these tests, if applicable
- Local laboratory documentation demonstrating competence and test reliability (eg, accreditation/license), if applicable

## **Independent Ethics Committee or Institutional Review Board**

Before the start of the study, the investigator (or sponsor where required) will provide the IEC/IRB with current and complete copies of the following documents (as required by local regulations):

- Final protocol and, if applicable, amendments
- Sponsor-approved ICF (and any other written materials to be provided to the participants)

- IB (or equivalent information) and amendments/addenda
- Sponsor-approved participant recruiting materials
- Information on compensation for study-related injuries or payment to participants for participation in the study, if applicable
- Investigator's curriculum vitae or equivalent information (unless not required, as documented by the IEC/IRB)
- Information regarding funding, name of the sponsor, institutional affiliations, other potential conflicts of interest, and incentives for participants
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after the IEC/IRB has given full approval of the final protocol, amendments (if any, excluding the ones that are purely administrative, with no consequences for participants, data or study conduct, unless required locally), the ICF, applicable recruiting materials, and participant compensation programs, and the sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the IEC/IRB and the documents being approved.

Approval for the collection of optional samples for research and for the corresponding ICF must be obtained from the IEC/IRB. Approval for the protocol can be obtained independent of this optional research component.

During the study the investigator (or sponsor where required) will send the following documents and updates to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments (excluding the ones that are purely administrative, with no consequences for participants, data or study conduct)
- Revision(s) to ICF and any other written materials to be provided to participants
- If applicable, new or revised participant recruiting materials approved by the sponsor
- Revisions to compensation for study-related injuries or payment to participants for participation in the study, if applicable
- New edition(s) of the IB and amendments/addenda
- Summaries of the status of the study at intervals stipulated in guidelines of the IEC/IRB (at least annually)
- Reports of adverse events that are serious, unlisted/unexpected, and associated with the study intervention
- New information that may adversely affect the safety of the participants or the conduct of the study
- Deviations from or changes to the protocol to eliminate immediate hazards to the participants
- Report of deaths of participants under the investigator's care
- Notification if a new investigator is responsible for the study at the site

- Development Safety Update Report and Line Listings, where applicable
- Any other requirements of the IEC/IRB

For all protocol amendments (excluding the ones that are purely administrative, with no consequences for participants, data or study conduct), the amendment and applicable ICF revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will be asked to review and reapprove this study, where required.

At the end of the study, the investigator (or sponsor where required) will notify the IEC/IRB about the study completion.

## **Country Selection**

This study will only be conducted in those countries where the intent is to launch or otherwise help ensure access to the developed product if the need for the product persists, unless explicitly addressed as a specific ethical consideration in Section 4.2.1.

## **Other Ethical Considerations**

For study-specific ethical design considerations, refer to Section 4.2.1.

## FINANCIAL DISCLOSURE

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information in accordance with local regulations to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

Refer to Required Prestudy Documentation (above) for details on financial disclosure.

#### INFORMED CONSENT PROCESS

Each participant must give written consent according to local requirements after the nature of the study has been fully explained. The ICF(s) must be signed before performance of any study-related activity. The ICF(s) that is/are used must be approved by both the sponsor and by the reviewing IEC/IRB and be in a language that the participant can read and understand. The informed consent should be in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and sponsor policy.

Before enrollment in the study, the investigator or an authorized member of the study-site personnel must explain to potential participants the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort participation in the study may entail. Participants will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the participant will receive for the treatment of his or her disease. Participants will

be told that alternative treatments are available if they refuse to take part and that such refusal will not prejudice future treatment. Finally, they will be told that the investigator will maintain a participant identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized sponsor personnel without violating the confidentiality of the participant, to the extent permitted by the applicable law(s) or regulations. By signing the ICF the participant is authorizing such access. It also denotes that the participant agrees to allow his or her study physician to recontact the participant for the purpose of obtaining consent for additional safety evaluations, and subsequent disease-related treatments, if needed.

The participant will be given sufficient time to read the ICF and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the participant's personally dated signature. After having obtained the consent, a copy of the ICF must be given to the participant.

Where local regulations require, a separate ICF may be used for the required DNA component of the study.

If the participant is unable to read or write, an impartial witness should be present for the entire informed consent process (which includes reading and explaining all written information) and should personally date and sign the ICF after the oral consent of the participant is obtained.

## **DATA PROTECTION**

## **Privacy of Personal Data**

The collection and processing of personal data from participants enrolled in this study will be limited to those data that are necessary to fulfill the objectives of the study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of participants confidential.

The informed consent obtained from the participant includes explicit consent for the processing of personal data and for the investigator/institution to allow direct access to his or her original medical records (source data/documents) for study-related monitoring, audit, IEC/IRB review, and regulatory inspection. This consent also addresses the transfer of the data to other entities and to other countries.

The participant has the right to request through the investigator access to his or her personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps will be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Exploratory DNA, PK/PD, and biomarker research is not conducted under standards appropriate for the return of data to participants. In addition, the sponsor cannot make decisions as to the significance of any findings resulting from exploratory research. Therefore, exploratory research data will not be returned to participants or investigators, unless required by law or local regulations. Privacy and confidentiality of data generated in the future on stored samples will be protected by the same standards applicable to all other clinical data.

## LONG-TERM RETENTION OF SAMPLES FOR ADDITIONAL FUTURE RESEARCH

Samples collected in this study may be stored for up to 15 years (or according to local regulations) for additional research. Samples will only be used to understand JNJ-3989 and JNJ-6379,the NAs (ETV, tenofovir disoproxil, and TAF), and PegIFN-α2a, to understand chronic HBV infection, to understand differential intervention responders, and to develop tests/assays related to JNJ-3989 and JNJ-6379 the NAs (ETV, tenofovir disoproxil, and TAF), and chronic HBV infection. The research may begin at any time during the study or the post-study storage period.

Stored samples will be coded throughout the sample storage and analysis process and will not be labeled with personal identifiers. Participants may withdraw their consent for their samples to be stored for research (refer to Section 7.2.1).

#### **COMMITTEES STRUCTURE**

## **Independent Flare Expert Panel**

An IFLEP will be appointed for this study. The IFLEP is composed of 3 independent medical experts with experience and expertise in hepatitis B and its treatment. The IFLEP will monitor ALT flares and will make recommendations regarding flare management based on an analysis of aggregate data.

In order to allow for an unbiased assessment, members of the committee will not serve as study investigators

Further details on the IFLEP process will be included in the IFLEP charter.

#### PUBLICATION POLICY/DISSEMINATION OF CLINICAL STUDY DATA

All information, including but not limited to information regarding JNJ-3989 and JNJ-6379 or the sponsor's operations (eg, patent application, formulas, manufacturing processes, basic scientific data, prior clinical data, formulation information) supplied by the sponsor to the investigator and not previously published, and any data, including pharmacogenomic or exploratory biomarker research data, generated as a result of this study, are considered confidential and remain the sole property of the sponsor. The investigator agrees to maintain this information in confidence and use this information only to accomplish this study and will not use it for other purposes without the sponsor's prior written consent.

The investigator understands that the information developed in the study will be used by the sponsor in connection with the continued development of JNJ-3989 and JNJ-6379, and thus may

be disclosed as required to other clinical investigators or regulatory agencies. To permit the information derived from the clinical studies to be used, the investigator is obligated to provide the sponsor with all data obtained in the study.

The results of the study will be reported in a Clinical Study Report generated by the sponsor and will contain data from all study sites that participated in the study as per protocol. Recruitment performance or specific expertise related to the nature and the key assessment parameters of the study will be used to determine a coordinating investigator for the study. Results of pharmacogenomic or exploratory biomarker analyses performed after the Clinical Study Report has been issued will be reported in a separate report and will not require a revision of the Clinical Study Report.

Study participant identifiers will not be used in publication of results. Any work created in connection with performance of the study and contained in the data that can benefit from copyright protection (except any publication by the investigator as provided for below) shall be the property of the sponsor as author and owner of copyright in such work.

Consistent with Good Publication Practices and International Committee of Medical Journal Editors (ICMJE) guidelines, the sponsor shall have the right to publish such primary (multicenter) data and information without approval from the investigator. The investigator has the right to publish study site-specific data after the primary data are published. If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application. In the event that issues arise regarding scientific integrity or regulatory compliance, the sponsor will review these issues with the investigator. The sponsor will not mandate modifications to scientific content and does not have the right to suppress information. For multicenter study designs and sub-study approaches, secondary results generally should not be published before the primary endpoints of a study have been published. Similarly, investigators will recognize the integrity of a multicenter study by not submitting for publication data derived from the individual study site until the combined results from the completed study have been submitted for publication, within 18 months after the study end date, or the sponsor confirms there will be no multicenter study publication. Authorship of publications resulting from this study will be based on the guidelines on authorship, such as those described in the ICMJE Recommendations for the Conduct, Reporting, Editing and Publication of Scholarly Work in Medical Journals, which state that the named authors must have made a significant contribution to the conception or design of the work; or the acquisition, analysis, or interpretation of the data for the work; and drafted the work or revised it critically for important intellectual content; and given final approval of the version to be published; and agreed to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

## Registration of Clinical Studies and Disclosure of Results

The sponsor will register and disclose the existence of and the results of clinical studies as required by law. The disclosure of the final study results will be performed after the end of study in order to ensure the statistical analyses are relevant.

## **DATA QUALITY ASSURANCE**

## **Data Quality Assurance/Quality Control**

Steps to be taken to ensure the accuracy and reliability of data include the selection of qualified investigators and appropriate study sites, review of protocol procedures with the investigator and study-site personnel before the study, periodic monitoring visits by the sponsor, and direct transmission of clinical laboratory data from a central laboratory to the sponsor's data base. Written instructions will be provided for collection, handling, storage, and shipment of samples.

Guidelines for CRF completion will be provided and reviewed with study-site personnel before the start of the study.

The sponsor will review CRF for accuracy and completeness during on-site monitoring visits and after transmission to the sponsor; any discrepancies will be resolved with the investigator or designee, as appropriate. After upload of the data into the study database they will be verified for accuracy and consistency with the data sources.

## CASE REPORT FORM COMPLETION

Case report forms are prepared and provided by the sponsor for each participant in electronic format. All data relating to the study must be recorded in CRF. All CRF entries, corrections, and alterations must be made by the investigator or authorized study-site personnel. The investigator must verify that all data entries in the CRF are accurate and correct.

The study data will be transcribed by study-site personnel from the source documents onto an electronic CRF, if applicable. Study-specific data will be transmitted in a secure manner to the sponsor.

Worksheets may be used for the capture of some data to facilitate completion of the CRF. Any such worksheets will become part of the participant's source documents. Data must be entered into CRF in English. The CRF must be completed as soon as possible after a participant visit and the forms should be available for review at the next scheduled monitoring visit.

All participative measurements (eg, pain scale information or other questionnaires) will be completed by the same individual who made the initial baseline determinations whenever possible.

If necessary, queries will be generated in the electronic data capture (eDC) tool. If corrections to a CRF are needed after the initial entry into the CRF, this can be done in either of the following ways:

- Investigator and study-site personnel can make corrections in the eDC tool at their own initiative or as a response to an auto query (generated by the eDC tool).
- Sponsor or sponsor delegate can generate a query for resolution by the investigator and study-site personnel.

#### SOURCE DOCUMENTS

At a minimum, source documents consistent in the type and level of detail with that commonly recorded at the study site as a basis for standard medical care must be available for the following: participant identification, eligibility, and study identification; study discussion and date of signed informed consent; dates of visits; dates of blood collection, date and time of start and end of leukapheresis, results of safety and efficacy parameters as required by the protocol; record of all adverse events and follow-up of adverse events; concomitant medication; intervention receipt/dispensing/return records; study intervention administration information; and date of study completion and reason for early discontinuation of investigational intervention or withdrawal from the study, if applicable.

The author of an entry in the source documents should be identifiable.

Specific details required as source data for the study and source data collection methods will be reviewed with the investigator before the study and will be described in the monitoring guidelines (or other equivalent document).

The following data will be recorded directly into the CRF and will be considered source data:

- Race
- Blood pressure and pulse/heart rate
- Height and weight
- Details of physical examination

The minimum source documentation requirements for Section 5.1 and Section 5.2 that specify a need for documented medical history are as follows:

- Referral letter from treating physician or
- Complete history of medical notes at the site
- Discharge summaries

Inclusion and exclusion criteria not requiring documented medical history must be verified at a minimum by participant interview or other protocol required assessment (eg, physical examination, laboratory assessment) and documented in the source documents.

An eSource system may be utilized, which contains data traditionally maintained in a hospital or clinic record to document medical care (eg, electronic source documents) as well as the clinical study-specific data fields as determined by the protocol. This data is electronically extracted for

use by the sponsor. If eSource is utilized, references made to the CRF in the protocol include the eSource system but information collected through eSource may not be limited to that found in the CRF.

#### **MONITORING**

The sponsor will use a combination of monitoring techniques (central, remote, or on-site monitoring) to monitor this study.

The sponsor will perform on-site monitoring visits as frequently as necessary. The monitor will record dates of the visits in a study site visit log that will be kept at the study site. The first post-initiation visit will be made as soon as possible after enrollment has begun. At these visits, the monitor will compare the data entered into the CRF with the source documents (eg, hospital/clinic/physician's office medical records); a sample may be reviewed. The nature and location of all source documents will be identified to ensure that all sources of original data required to complete the CRF are known to the sponsor and study-site personnel and are accessible for verification by the sponsor study-site contact. If electronic records are maintained at the study site, the method of verification must be discussed with the study-site personnel.

Direct access to source documents (medical records) must be allowed for the purpose of verifying that the recorded data are consistent with the original source data. Findings from this review will be discussed with the study-site personnel. The sponsor expects that, during monitoring visits, the relevant study-site personnel will be available, the source documents will be accessible, and a suitable environment will be provided for review of study-related documents. The monitor will meet with the investigator on a regular basis during the study to provide feedback on the study conduct.

In addition to on-site monitoring visits, remote contacts can occur. It is expected that during these remote contacts, study-site personnel will be available to provide an update on the progress of the study at the site.

Central monitoring will take place for data identified by the sponsor as requiring central review.

## **ON-SITE AUDITS**

Representatives of the sponsor's clinical quality assurance department may visit the study site at any time during or after completion of the study to conduct an audit of the study in compliance with regulatory guidelines and company policy. These audits will require access to all study records, including source documents, for inspection. Participant privacy must, however, be respected. The investigator and study-site personnel are responsible for being present and available for consultation during routinely scheduled study-site audit visits conducted by the sponsor or its designees.

Similar auditing procedures may also be conducted by agents of any regulatory body, either as part of a national GCP compliance program or to review the results of this study in support of a

regulatory submission. The investigator should immediately notify the sponsor if he or she has been contacted by a regulatory agency concerning an upcoming inspection.

#### RECORD RETENTION

In compliance with the ICH/GCP guidelines, the investigator/institution will maintain all CRF and all source documents that support the data collected from each participant, as well as all study documents as specified in ICH/GCP Section 8, Essential Documents for the Conduct of a Clinical Trial, and all study documents as specified by the applicable regulatory requirement(s). The investigator/institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained.

If the responsible investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the investigator relocate or dispose of any study documents before having obtained written approval from the sponsor.

If it becomes necessary for the sponsor or the appropriate regulatory authority to review any documentation relating to this study, the investigator/institution must permit access to such reports.

#### STUDY AND SITE START AND CLOSURE

#### First Act of Recruitment

The first site open is considered the first act of recruitment and it becomes the study start date.

## **Study Termination**

The sponsor reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IEC/IRB or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further study intervention development

## 10.4. Appendix 4: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

## ADVERSE EVENT DEFINITIONS AND CLASSIFICATIONS

#### **Adverse Event**

An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. (Definition per ICH)

This includes any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.

Note: The sponsor collects adverse events starting with the signing of the ICF (refer to All Adverse Events under Section 8.5.1 for time of last AE recording).

## **Serious Adverse Event**

A SAE based on ICH and EU Guidelines on Pharmacovigilance for Medicinal Products for Human Use is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (The participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect
- Is a suspected transmission of any infectious agent via a medicinal product
- Is Medically Important\*

\*Medical and scientific judgment should be exercised in deciding whether expedited reporting is also appropriate in other situations, such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. These should usually be considered serious.

If a serious and unexpected adverse event occurs for which there is evidence suggesting a causal relationship between the study intervention and the event (eg, death from anaphylaxis), the event must be reported as a serious and unexpected suspected adverse reaction even if it is a component of the study endpoint (eg, all-cause mortality).

## Unlisted (Unexpected) Adverse Event/Reference Safety Information

An adverse event is considered unlisted if the nature or severity is not consistent with the applicable product reference safety information. For JNJ-3989 and JNJ-6379, the expectedness of an adverse event will be determined by whether or not it is listed in the IB. For ETV, tenofovir disoproxil, and TAF with a marketing authorization, the expectedness of an adverse event will be determined by whether or not it is listed in the package insert.

#### ATTRIBUTION DEFINITIONS

## **Assessment of Causality**

The causal relationship to study intervention is determined by the Investigator. The following selection should be used to assess all AEs.

#### Related

There is a reasonable causal relationship between study intervention administration and the AE.

#### **Not Related**

There is not a reasonable causal relationship between study intervention administration and the AE.

The term "reasonable causal relationship" means there is evidence to support a causal relationship.

## **SEVERITY CRITERIA**

An assessment of severity grade will be made by the investigator using the general categorical descriptors outlined in the DAIDS Toxicity Grading Scale (see Section 10.9, Appendix 9, DAIDS Table).

## SPECIAL REPORTING SITUATIONS

Safety events of interest on a sponsor study intervention in an interventional study that may require expedited reporting or safety evaluation include, but are not limited to:

- Overdose of a sponsor study intervention
- Suspected abuse/misuse of a sponsor study intervention
- Accidental or occupational exposure to a sponsor study intervention
- Medication error, intercepted medication error, or potential medication error involving a sponsor medicinal product (with or without patient exposure to the sponsor medicinal product, eg, product name confusion, product label confusion, intercepted prescribing or dispensing errors)
- Exposure to a sponsor study intervention from breastfeeding

Special reporting situations should be recorded in the CRF. Any special reporting situation that meets the criteria of a SAE should be recorded on the SAE page of the CRF.

## **PROCEDURES**

#### **All Adverse Events**

All adverse events, regardless of seriousness, severity, or presumed relationship to study intervention, must be recorded using medical terminology in the source document and the CRF. Whenever possible, diagnoses should be given when signs and symptoms are due to a common etiology (eg, cough, runny nose, sneezing, sore throat, and head congestion should be reported as "upper respiratory infection"). Investigators must record in the CRF their opinion concerning the relationship of the adverse event to study therapy. All measures required for adverse event management must be recorded in the source document and reported according to sponsor instructions.

In the context of this study, AEs and SAEs associated with/triggered by the liver biopsies, leukapheresis, or blood collection procedures are to be reported to the sponsor.

For all studies with an outpatient phase, including open-label studies, the participant must be provided with a "wallet (study) card" and instructed to carry this card with them for the duration of the study indicating the following:

- Study number
- Statement, in the local language(s), that the participant is participating in a clinical study
- Investigator's name and 24-hour contact telephone number
- Local sponsor's name and 24-hour contact telephone number (for medical personnel only)
- Site number
- Participant number
- Any other information that is required to do an emergency breaking of the blind

## **Serious Adverse Events**

All SAEs that have not resolved by the end of the study, or that have not resolved upon discontinuation of the participant's participation in the study, must be followed until any of the following occurs:

- The event resolves
- The event stabilizes
- The event returns to baseline, if a baseline value/status is available
- The event can be attributed to agents other than the study intervention or to factors unrelated to study conduct
- It becomes unlikely that any additional information can be obtained (participant or health care practitioner refusal to provide additional information, lost to follow-up after demonstration of due diligence with follow-up efforts)

Suspected transmission of an infectious agent by a medicinal product will be reported as a SAE. Any event requiring hospitalization (or prolongation of hospitalization) that occurs during the course of a participant's participation in a study must be reported as a SAE, except hospitalizations for the following:

- Hospitalizations not intended to treat an acute illness or adverse event (eg, social reasons such as pending placement in long-term care facility)
- Surgery or procedure planned before entry into the study (must be documented in the CRF). Note: Hospitalizations that were planned before the signing of the ICF, and where the underlying condition for which the hospitalization was planned has not worsened, will not be considered SAEs. Any adverse event that results in a prolongation of the originally planned hospitalization is to be reported as a new SAE.

The cause of death of a participant in a study, whether or not the event is expected or associated with the study intervention, is considered an SAE.

#### CONTACTING SPONSOR REGARDING SAFETY

The names (and corresponding telephone numbers) of the individuals who should be contacted regarding safety issues or questions regarding the study are listed in the Contact Information page(s), which will be provided as a separate document.

#### PRODUCT QUALITY COMPLAINT HANDLING

A product quality complaint (PQC) is defined as any suspicion of a product defect related to manufacturing, labeling, or packaging, ie, any dissatisfaction relative to the identity, quality, durability, or reliability of a product, including its labeling or package integrity. A PQC may have an impact on the safety and efficacy of the product. Timely, accurate, and complete reporting and analysis of PQC information from studies are crucial for the protection of participants, investigators, and the sponsor, and are mandated by regulatory agencies worldwide. The sponsor has established procedures in conformity with regulatory requirements worldwide to ensure appropriate reporting of PQC information; all studies conducted by the sponsor or its affiliates will be conducted in accordance with those procedures.

#### **Procedures**

All initial PQCs must be reported to the sponsor by the study-site personnel within 24 hours after being made aware of the event.

If the defect is combined with a SAE, the study-site personnel must report the PQC to the sponsor according to the SAE reporting timelines (refer to Section 8.5.1). A sample of the suspected product should be maintained for further investigation if requested by the sponsor.

## **Contacting Sponsor Regarding Product Quality**

The names (and corresponding telephone numbers) of the individuals who should be contacted regarding product quality issues are listed in the Contact Information page(s), which will be provided as a separate document.

## 10.5. Appendix 5: Rash Management

Status: Approved, Date: 25 November 2021

Table 6: Management of Rash Events by Severity Grade

| | Definition | Study<br>Intervention<br>Action | Activities by Day <sup>a</sup> | Referral to<br>Dermatologist and<br>Dermatology Activities |
|---|---|---|---|---|
| Grade 1 rash<br>(with or<br>without<br>pruritus) <sup>b</sup> | Erythema | Study intervention intake may be continued at the investigator's discretion | <u>Day 0</u> : optional on site visit for initial rash evaluation may be performed at the investigator's discretion. | Not required |
| | | | Safety laboratory assessments may be performed at the investigator's discretion (recommended if visit occurs). | |
| | | | Digital pictures* of skin lesions may be taken at the investigator's discretion. | |
| | | | Determine if participant was adhering to the recommended sun-<br>protective measures. If appropriate, provide sun protection<br>counseling. | |
| | | | <u>Day 1 and thereafter</u> : appropriate follow-up visits at the investigator's discretion until resolution of rash. | |
| | | | Safety laboratory assessments and photography (digital pictures* of skin lesions) may be performed at the investigator's discretion. | |
| | | | * Digital pictures to be taken at the clinical site upon consent of the participant. | |
| Grade 2 rash<br>(with or without<br>pruritus) <sup>b</sup> | Diffuse,<br>maculopapular rash,<br>or dry desquamation | Study intervention intake may be continued at the investigator's discretion | <u>Day 0</u> : required on-site visit (if a visit is not possible, telephone contact with the participant should take place to collect information and give advice on the necessary measures to be taken). | Referral to dermatologist<br>at the discretion of the<br>investigator <sup>c</sup> |
| | | | Safety laboratory assessments may be performed at the investigator's discretion (recommended). | Biopsy not required, but<br>may be performed at the<br>dermatologist's<br>discretion |
| | | | Digital pictures* of skin lesions may be taken at the investigator's discretion. Digital pictures* of skin lesions are recommended in case consultation of a dermatologist is required. Determine if participant was adhering to the recommended sun-protective measures. If appropriate, provide sun protection counseling. | |
| | | | <u>Day 1 and thereafter</u> : appropriate follow-up visits at the investigator's discretion until resolution of rash or until clinical stability is reached. | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.
**Table 6:** Management of Rash Events by Severity Grade

| | Definition | Study<br>Intervention<br>Action | Activities by Day <sup>a</sup> | Referral to<br>Dermatologist and<br>Dermatology Activities |
|---|---|---|---|---|
| | | | Safety laboratory assessments are required on Day 1 and are required thereafter only if the previous values were abnormal (but may be performed at the investigator's discretion). If the rash progresses to a higher grade, safety laboratory assessments of the higher grade should be followed. | |
| | | | Digital pictures* of skin lesions may be taken at the investigator's discretion. | |
| | | | * Digital pictures to be taken at the clinical site upon consent of the participant. | |
| Grade 3 rash <sup>b</sup> | Vesiculation, moist | Must permanently | Day 0: required on-site visit. | Required <sup>c</sup> |
| | desquamation, or ulceration OR Any cutaneous event with 1 of the following: - Elevations in AST/ALT | discontinue JNJ-3989; no rechallenge allowed NA treatment may be discontinued based on | Safety laboratory assessments required to be performed. | Biopsy not required, but<br>may be performed at the<br>dermatologist's<br>discretion. |
| | | | Digital pictures* of skin lesions may be taken at the investigator's discretion (recommended). | |
| | | | Determine if participant was adhering to the recommended sun-<br>protective measures. If appropriate, provide sun protection<br>counseling. | |
| | >2×baseline | investigator judgement in | <u>Day 1</u> : required on-site visit. | |
| | value<br>- Fever >38°C or | consultation with | Safety laboratory assessments required to be performed. | |
| | 100°F - Eosinophils >1.00×10³/μL - Serum sickness- like reaction | the sponsor | Digital pictures* of skin lesions may be taken at the investigator's discretion (recommended). | |
| | | | <u>Further visit(s)</u> : appropriate follow-up required until resolution of rash or until clinical stability is reached. | |
| | | | Safety laboratory assessments and photography (digital pictures* of skin lesions) are recommended to be performed until the rash severity resolves to grade 2 or grade 1. | |
| | | | * Digital pictures to be taken at the clinical site upon consent of the participant. | |

| Table 6: | Management of Rash Even | ts by Severity Grade |
|----------|-------------------------|----------------------|
|----------|-------------------------|----------------------|

| | Definition | Study<br>Intervention<br>Action | Activities by Day <sup>a</sup> | Referral to<br>Dermatologist and<br>Dermatology Activities |
|---|---|---|---|---|
| Grade 4 rash | Exfoliative | Must permanently | <u>Day 0</u> : required on-site visit. | Required <sup>c</sup> |
| | dermatitis OR | discontinue<br>JNJ-3989; no | Safety laboratory assessments required to be performed. | Biopsy required and to |
| | Mucous membrane involvement in at least 2 distinct sites | rechallenge<br>allowed | Digital pictures* of skin lesions may be taken at the investigator's discretion (recommended). | be performed as soon as possible after the onset of the rash. |
| | OR | NA treatment may | Determine if participant was adhering to the recommended sun- | |
| | Erythema multiforme major OR | be discontinued<br>based on<br>investigator<br>judgement in<br>consultation with<br>the sponsor | protective measures. If appropriate, provide sun protection counseling. | |
| | Stevens-Johnson | | <u>Day 1</u> : required on-site visit. | |
| | syndrome OR | | Safety laboratory assessments required to be performed. | |
| | Toxic epidermal necrolysis OR | | Digital pictures* of skin lesions may be taken at the investigator's discretion (recommended). | |
| | Necrosis requiring surgery | | <u>Further visit(s)</u> : appropriate follow-up required until resolution of rash or until clinical stability is reached. | |
| | | Safety laboratory assessments and photography (digital pictures* of skin lesions) are recommended to be performed until the rash severity resolves to grade 2 or grade 1. | | |
| | | | * Digital pictures to be taken at the clinical site upon consent of the participant. | |

AE: adverse event; ALT: alanine aminotransferase; AST: aspartate aminotransferase; NA: nucleos(t)ide analog.

- Day 0 of the rash is the first day of investigator assessment and not the first day of rash as reported by the participant. The initial visit should be conducted as soon as possible after the participant contacts the investigator to report the AE (ie, preferably on Day 0). The initial visit and subsequent visits to manage the rash may require unscheduled visit(s).
- b The participant should be advised to contact the investigator immediately if there is any worsening of the rash, if any systemic signs or symptoms appear, or if mucosal involvement develops. In case the rash evolves to a higher grade than that first observed, management of the rash should follow the guidelines indicated for the higher grade.
- <sup>c</sup> If applicable, dermatologist visit should occur preferably within 24 hours after onset of rash.

#### Notes:

- Local laboratory assessments are to be used for rash management. The values of the local laboratory assessments need to be transcribed in the eCRF by the study site personnel.
- Digital pictures that are collected, dermatological consultation reports or biopsy reports that become available, should be de-identified and provided to the sponsor.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

# 10.6. Appendix 6: Intervention-emergent ALT/AST Elevations



- <sup>a</sup> Additional tests may be considered based on clinical judgement in case of confirmed ALT flares:
  - Hepatitis A, D, C, E: IgM anti-HAV; delta IgM, IgG & PCR, HCV RNA, IgM & IgG anti-HEV, HEV RNA
  - CMV, HSV, EBV infection: IgM & IgG anti-CMV, IgM & IgG anti-HSV; IgM & IgG anti-EBV, PCR
  - HIV
  - Ig-electrophoresis

# 10.7. Appendix 7: Cardiovascular Safety Abnormalities

## **ECG**

All important abnormalities from the ECG readings will be listed.

| | | ECG parameter | | |
|---|---|---|---|---|
| <b>Abnormality Code</b> | <b>Heart Rate</b> | PR | QRS | QTcorrected |
| Abnormalities on actual values | | | | |
| Abnormally low | <45 bpm | NAP | - | - |
| Abnormally high | ≥120 bpm | >220 ms | ≥120 ms | - |
| Borderline prolonged QT | - | - | - | 450 ms < QTc ≤480 ms |
| Prolonged QT | - | - | - | $480 \text{ ms} < \text{QTc} \leq 500 \text{ ms}$ |
| Pathologically prolonged QT | - | - | = | QTc >500 ms |
| Abnormalities on changes from bas | eline (ΔQTc) | | | |
| Normal QTc change | - | - | - | ΔQTc <30 ms |
| Borderline QTc change | - | - | - | $30 \text{ ms} \leq \Delta \text{QTc} \leq 60 \text{ ms}$ |
| Abnormally high QTc change | - | - | - | $\Delta QTc > 60 \text{ ms}$ |

ECG: electrocardiogram; NAP = not applicable

For absolute QTc parameters the categories are defined based on the ICH E14 GuidanceF<sup>a</sup>

# Vital Signs<sup>b</sup>

The following abnormalities will be defined for vital signs:

| | Vital Signs parameter | | |
|---|---|---|---|
| <b>Abnormality Code</b> | Pulse | DBP | SBP |
| Abnormalities on actual values | | | |
| Abnormally low | ≤45 bpm | ≤50 mmHg | ≤90 mmHg |
| Grade 1 or mild | - | >90 mmHg - <100 mmHg | >140 mmHg - <160 mmHg |
| Grade 2 or moderate | - | ≥100 mmHg - <110 mmHg | ≥160 mmHg - <180 mmHg |
| Grade 3 or severe | - | ≥110 mmHg | ≥180 mmHg |
| Abnormally high | ≥120 bpm | = | = |

DBP: diastolic blood pressure; SBP: systolic blood pressure

<sup>&</sup>lt;sup>a</sup> The clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs CHMP/ICH/2/04, May 2005.

<sup>&</sup>lt;sup>b</sup> The classification of AEs related to hypotension and hypertension will be done according to the DAIDS grading scale.

# 10.8. Appendix 8: Contraceptive and Barrier Guidance and Collection of Pregnancy Information

Participants must follow contraceptive measures as outlined in Section 5.1. Pregnancy information will be collected and reported as noted in Section 8.5.5 and Section 10.4, Appendix 4 Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting.

#### **Definitions**

# Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

# Woman Not of Childbearing Potential

## premenarchal

A premenarchal state is one in which menarche has not yet occurred.

## postmenopausal

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level (>40 IU/L or mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT), however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. If there is a question about menopausal status in women on HRT, the woman will be required to use one of the non-estrogen-containing hormonal highly effective contraceptive methods if she wishes to continue HRT during the study.

# • permanently sterile

Permanent sterilization methods include hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.

**Note:** If the childbearing potential changes after start of the study (eg, a premenarchal woman experiences menarche) or the risk of pregnancy changes (eg, a woman who is not heterosexually active becomes active), a woman must begin a highly effective method of contraception, as described throughout the inclusion criteria.

If reproductive status is questionable, additional evaluation should be considered.

Contraceptive (birth control) use by men or women should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.

Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants in clinical studies.

## **Examples of Contraceptives**

## EXAMPLES OF CONTRACEPTIVES<sup>a</sup> ALLOWED DURING THE STUDY INCLUDE:

#### **USER INDEPENDENT**

**Highly Effective Methods That Are User Independent** *Failure rate of* <1% *per year when used consistently and correctly.* 

- Implantable progestogen-only hormone contraception associated with inhibition of ovulation<sup>b</sup>
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)
- Tubal closure (eg, bilateral tubal occlusion, bilateral tubal ligation)
- Azoospermic partner (vasectomized or due to medical cause)

(Vasectomized partner is a highly effective contraceptive method provided that the partner is the sole sexual partner of the woman of childbearing potential and the absence of sperm has been confirmed. If not, additional highly effective method of contraception should be used. Spermatogenesis cycle is approximately 74 days.)

#### USER DEPENDENT

**Highly Effective Methods That Are User Dependent** *Failure rate of* <1% *per year when used consistently and correctly.* 

• Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>b</sup>

ora1

intravaginal

transdermal

injectable

Progestogen-only hormone contraception associated with inhibition of ovulation<sup>b</sup>

oral

injectable

Sexual abstinence

(Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.)

a) Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants in clinical studies.

## 10.9. Appendix 9: DAIDS Table

# DIVISION OF AIDS (DAIDS) TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS, VERSION 2.1, PUBLISH DATE: JULY, 2017

The DAIDS grading table is a descriptive terminology to be utilized for AE reporting in this study. A grading (severity) scale is provided for each AE term.

# **General Instructions**

# Grading Adult and Pediatric Adverse Events

When a single parameter is not appropriate for grading an AE in both adult and pediatric populations, separate parameters with specified age ranges are provided. If there is no distinction between adult and pediatric populations, the listed parameter should be used for grading an AE in both populations.

## Determining Severity Grade for Parameters Between Grades

If the severity of an AE could fall under either 1 of 2 grades (eg, the severity of an AE could be either grade 2 or grade 3), sites should select the higher of the 2 grades.

Laboratory normal ranges should be taken into consideration to assign gradings to a laboratory value.

#### **Definitions**

| Basic self-care functions | Adults: activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding |
|---|---|
| | Young children: activities that are age and culturally appropriate (eg, feeding self with culturally appropriate eating implements) |
| Usual social & functional activities | Activities which adults and children perform on a routine basis and those which are part of regular activities of daily living, for example: |
| | Adults: adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, or pursuing a hobby |
| | Young Children: activities that are age and culturally appropriate (eg, social interactions, play activities, learning tasks) |
| Intervention | Medical, surgical, or other procedures recommended or provided by a healthcare professional for the treatment of an AE. |

## Estimating Severity Grade for Parameters not Identified in the Grading Table

The functional table below should be used to grade the severity of an AE that is not specifically identified in the grading table. In addition, all deaths related to an AE are to be classified as grade 5.

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Clinical AE NOT identified elsewhere in the grading table | Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated | Moderate symptoms<br>causing greater than<br>minimal interference<br>with usual social &<br>functional activities<br>with intervention<br>indicated | Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated | Potentially<br>life threatening<br>symptoms causing<br>inability to perform<br>basic self care<br>functions with<br>intervention indicated<br>to prevent permanent<br>impairment, persistent<br>disability, or death |

**NOTE:** Laboratory abnormalities may have their grading defined in the DAIDS table below, however, all laboratory abnormalities do not necessarily represent an AE. If a laboratory abnormality is considered an AE, the AE need not have the same grade as the laboratory abnormality itself. The AE grade for a laboratory abnormality should be defined by the table above.

| | MAJ | OR CLINICAL CONDIT | TIONS | * |
|---|---|---|---|---|
| | | CARDIOVASCULAR | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Arrhythmia (by ECG or physical examination) Specify type, if applicable | No symptoms AND<br>No intervention<br>indicated | No symptoms AND<br>Non urgent<br>intervention indicated | Non life threatening<br>symptoms AND Non<br>urgent intervention<br>indicated | Life threatening<br>arrhythmia OR Urgent<br>intervention indicated |
| Blood Pressure Abnormalities <sup>a</sup> Hypertension (with the lowest reading taken after repeat testing during a visit) aged ≥18 years | 140 to <160 mmHg<br>systolic OR 90 to<br><100 mmHg diastolic | ≥160 to <180 mmHg<br>systolic OR ≥100 to<br><110 mmHg diastolic | ≥180 mmHg systolic<br>OR ≥110 mmHg<br>diastolic | Life threatening consequences in a participant not previously diagnosed with hypertension (eg, malignant hypertension) OR Hospitalization indicated |
| aged <18 years | >120/80 mmHg | ≥95 <sup>th</sup> to <99 <sup>th</sup> percentile + 5 mmHg adjusted for age, height, and gender (systolic and/or diastolic) | ≥99 <sup>th</sup> percentile<br>+ 5 mmHg adjusted for<br>age, height, and gender<br>(systolic and/or<br>diastolic) | Life threatening consequences in a participant not previously diagnosed with hypertension (eg, malignant hypertension) OR Hospitalization indicated |
| Hypotension | No symptoms | Symptoms corrected<br>with oral fluid<br>replacement | Symptoms AND IV fluids indicated | Shock requiring use of<br>vasopressors or<br>mechanical assistance<br>to maintain blood<br>pressure |
| Cardiac Ischemia or<br>Infarction<br>Report only I | NAP | NAP | New symptoms with<br>ischemia (stable<br>angina) OR New<br>testing consistent with<br>ischemia | Unstable angina OR<br>Acute myocardial<br>infarction |

ECG: electrocardiogram; IV: intravenous; NAP: not applicable

Blood pressure norms for children aged <18 years can be found in: Expert Panel on Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents. Pediatrics 2011;128;S213; originally published online November 14, 2011; DOI: 10.1542/peds.2009 2107C.

| | MAJ | OR CLINICAL CONDIT | TIONS | |
|---|---|---|---|---|
| | | CARDIOVASCULAR | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Heart Failure | No symptoms AND<br>Laboratory or cardiac<br>imaging abnormalities | Symptoms with mild<br>to moderate activity or<br>exertion | Symptoms at rest or<br>with minimal activity<br>or exertion<br>(eg, hypoxemia) OR<br>Intervention indicated<br>(eg, oxygen) | Life threatening consequences OR Urgent intervention indicated (eg, vasoactive medications, ventricular assist device, heart transplant) |
| Hemorrhage<br>(with significant acute<br>blood loss) | NAP | Symptoms AND No transfusion indicated | Symptoms AND<br>Transfusion of ≤2 units<br>packed RBCs indicated | Life threatening<br>hypotension OR<br>Transfusion of >2 units<br>packed RBCs (for<br>children, packed RBCs<br>>10 cc/kg) indicated |
| Prolonged PR Interval or AV Block Report only 1 aged >16 years | PR interval 0.21 to <0.25 seconds | PR interval ≥0.25 seconds OR Type I 2 <sup>nd</sup> degree AV block | Type II 2 <sup>nd</sup> degree AV<br>block OR Ventricular<br>pause ≥3.0 seconds | Complete AV block |
| aged ≤16 years | 1st degree AV block<br>(PR interval > normal<br>for age and rate) | Type I 2 <sup>nd</sup> degree AV<br>block | Type II 2 <sup>nd</sup> degree AV<br>block OR Ventricular<br>pause ≥3.0 seconds | Complete AV block |
| Prolonged QTc<br>Interval as per<br>Fridericia's formula <sup>b</sup> | 0.45 to 0.47 seconds | >0.47 to 0.50 seconds | >0.50 seconds OR<br>≥0.06 seconds above<br>baseline | Life threatening<br>consequences<br>(eg, TdP, other<br>associated serious<br>ventricular<br>dysrhythmia) |
| Thrombosis or<br>Embolism<br>Report only I | NAP | Symptoms AND No intervention indicated | Symptoms AND<br>Intervention indicated | Life threatening<br>embolic event<br>(eg, pulmonary<br>embolism, thrombus) |

AV: atrioventricular; NAP: not applicable; RBC: red blood cell; TdP: Torsades de Pointes b Modified by the sponsor.

| | | DERMATOLOGIC | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Alopecia (scalp only) | Detectable by participant, representative, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | NAP | NAP |
| Bruising | Localized to 1 area | Localized to more than 1 area | Generalized | NAP |
| Cellulitis | NAP | Nonparenteral<br>treatment indicated<br>(eg, oral antibiotics,<br>antifungals, antivirals) | IV treatment indicated<br>(eg, IV antibiotics,<br>antifungals, antivirals) | Life threatening<br>consequences<br>(eg, sepsis, tissue<br>necrosis) |
| Hyperpigmentation | Slight or localized<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities | Marked or generalized causing greater than minimal interference with usual social & functional activities | NAP | NAP |
| Hypopigmentation | Slight or localized<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities | Marked or generalized causing greater than minimal interference with usual social & functional activities | NAP | NAP |
| Petechiae | Localized to 1 area | Localized to more than 1 area | Generalized | NAP |
| Pruritus <sup>c</sup> (without skin lesions) | Itching causing no or<br>minimal interference<br>with usual social &<br>functional activities | Itching causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Itching causing inability to perform usual social & functional activities | NAP |
| Rash<br>Specify type, if<br>applicable | Localized rash | Diffuse rash OR Target<br>lesions | Diffuse rash AND<br>Vesicles or limited<br>number of bullae OR<br>superficial ulcerations<br>of mucous membrane<br>limited to 1 site | Extensive or<br>generalized bullous<br>lesions OR Ulceration<br>of mucous membrane<br>involving 2 or more<br>distinct mucosal sites<br>OR Stevens Johnson<br>syndrome OR Toxic<br>epidermal necrolysis |

IV: intravenous; NAP: not applicable

For pruritus associated with injections or infusions, refer to the SITE REACTIONS TO INJECTIONS AND INFUSIONS section.

| | END | OCRINE AND METABO | OLIC | *- |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Diabetes Mellitus | Controlled without medication | Controlled with<br>medication OR<br>Modification of current<br>medication regimen | Uncontrolled despite<br>treatment modification<br>OR Hospitalization for<br>immediate glucose<br>control indicated | Life threatening<br>consequences<br>(eg, ketoacidosis,<br>hyperosmolar<br>nonketotic coma, end<br>organ failure) |
| Gynecomastia | Detectable by participant, representative, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing pain with greater than minimal interference with usual social & functional activities | Disfiguring changes<br>AND Symptoms<br>requiring intervention<br>or causing inability to<br>perform usual social &<br>functional activities | NAP |
| Hyperthyroidism | No symptoms AND<br>Abnormal laboratory<br>value | Symptoms causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life threatening consequences (eg, thyroid storm) |
| Hypothyroidism | No symptoms AND<br>Abnormal laboratory<br>value | Symptoms causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life threatening<br>consequences<br>(eg, myxedema coma) |
| Lipoatrophy <sup>d</sup> | Detectable by participant, representative, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | Disfiguring changes | NAP |
| Lipohypertrophy | Detectable by participant, representative, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | Disfiguring changes | NAP |

A disorder characterized by fat loss in the face, extremities, and buttocks.

A disorder characterized by abnormal fat accumulation on the back of the neck, breasts, and abdomen.

| | | GASTROINTESTINAL | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite<br>associated with<br>decreased oral intake<br>without significant<br>weight loss | Loss of appetite<br>associated with<br>significant weight loss | Life threatening<br>consequences OR<br>Aggressive<br>intervention indicated<br>(eg, tube feeding, total<br>parenteral nutrition) |
| Ascites | No symptoms | Symptoms AND<br>Intervention indicated<br>(eg, diuretics,<br>therapeutic<br>paracentesis) | Symptoms recur or persist despite intervention | Life threatening consequences |
| Bloating or<br>Distension<br>Report only 1 | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NAP |
| Cholecystitis | NAP | Symptoms AND<br>Medical intervention<br>indicated | Radiologic,<br>endoscopic, or<br>operative intervention<br>indicated | Life threatening<br>consequences<br>(eg, sepsis,<br>perforation) |
| Constipation | NAP | Persistent constipation<br>requiring regular use<br>of dietary<br>modifications,<br>laxatives, or enemas | Obstipation with manual evacuation indicated | Life threatening consequences (eg, obstruction) |
| Diarrhea<br>aged ≥1 year | Transient or intermittent episodes of unformed stools OR Increase of ≤3 stools over baseline per 24 hour period | Persistent episodes of<br>unformed to watery<br>stools OR Increase of<br>4 to 6 stools over<br>baseline per 24 hour<br>period | Increase of ≥7 stools<br>per 24 hour period OR<br>IV fluid replacement<br>indicated | Life threatening consequences (eg, hypotensive shock) |
| aged <1 year | Liquid stools (more<br>unformed than usual)<br>but usual number of<br>stools | Liquid stools with<br>increased number of<br>stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Life threatening<br>consequences<br>(eg, liquid stools<br>resulting in severe<br>dehydration,<br>hypotensive shock) |
| Dysphagia or<br>Odynophagia<br>Report only 1 and<br>specify location | Symptoms but able to eat usual diet | Symptoms causing<br>altered dietary intake<br>with no intervention<br>indicated | Symptoms causing<br>severely altered dietary<br>intake with<br>intervention indicated | Life threatening reduction in oral intake |
| Gastrointestinal<br>Bleeding | Not requiring intervention other than iron supplement | Endoscopic intervention indicated | Transfusion indicated | Life threatening<br>consequences<br>(eg, hypotensive<br>shock) |

IV: intravenous; NAP: not applicable

| | | GASTROINTESTINAL | | <i>**</i> |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Mucositis or<br>Stomatitis<br>Report only 1 and<br>specify location | Mucosal erythema | Patchy<br>pseudomembranes or<br>ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Life threatening<br>consequences<br>(eg, aspiration,<br>choking) OR Tissue<br>necrosis OR Diffuse<br>spontaneous mucosal<br>bleeding |
| Nausea | Transient (<24 hours) or intermittent AND No or minimal interference with oral intake | Persistent nausea<br>resulting in decreased<br>oral intake for 24 to<br>48 hours | Persistent nausea<br>resulting in minimal<br>oral intake for<br>>48 hours OR<br>Rehydration indicated<br>(eg, IV fluids) | Life threatening<br>consequences<br>(eg, hypotensive<br>shock) |
| Pancreatitis | NAP | Symptoms with hospitalization not indicated | Symptoms with<br>hospitalization<br>indicated | Life threatening<br>consequences<br>(eg, circulatory<br>failure, hemorrhage,<br>sepsis) |
| Perforation<br>(colon or rectum) | NAP | NAP | Intervention indicated | Life threatening consequences |
| Proctitis | Rectal discomfort with<br>no intervention<br>indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social & functional activities OR Operative intervention indicated | Life threatening<br>consequences<br>(eg, perforation) |
| Rectal Discharge | Visible discharge | Discharge requiring the use of pads | NAP | NAP |
| Vomiting | Transient or intermittent AND No or minimal interference with oral intake | Frequent episodes with<br>no or mild dehydration | Persistent vomiting<br>resulting in orthostatic<br>hypotension OR<br>Aggressive rehydration<br>indicated (eg, IV<br>fluids) | Life threatening<br>consequences<br>(eg, hypotensive<br>shock) |

IV: intravenous; NAP: not applicable

| | | MUSCULOSKELETAL | | ** |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Arthralgia | Joint pain causing no or<br>minimal interference<br>with usual social &<br>functional activities | Joint pain causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain<br>causing inability to<br>perform basic self care<br>functions |
| Arthritis | Stiffness or joint<br>swelling causing no or<br>minimal interference<br>with usual social &<br>functional activities | Stiffness or joint<br>swelling causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Stiffness or joint<br>swelling causing<br>inability to perform<br>usual social &<br>functional activities | Disabling joint<br>stiffness or swelling<br>causing inability to<br>perform basic self care<br>functions |
| Myalgia (generalized) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain<br>causing inability to<br>perform basic self care<br>functions |
| Osteonecrosis | NAP | No symptoms but with<br>radiographic findings<br>AND No operative<br>intervention indicated | Bone pain with<br>radiographic findings<br>OR Operative<br>intervention indicated | Disabling bone pain<br>with radiographic<br>findings causing<br>inability to perform<br>basic self care<br>functions |
| Osteopenia <sup>f</sup> | D1 (D) | N/A D | WAR | N/A D |
| aged ≥30 years<br>aged <30 years | BMD t score 2.5 to 1<br>BMD z score 2 to 1 | NAP<br>NAP | NAP<br>NAP | NAP<br>NAP |
| Osteoporosis <sup>f</sup> aged ≥30 years | NAP | BMD t score < 2.5 | Pathologic fracture<br>(eg, compression<br>fracture causing loss of<br>vertebral height) | Pathologic fracture causing life threatening consequences |
| aged <30 years | NAP | BMD z score < 2 | Pathologic fracture<br>(eg, compression<br>fracture causing loss of<br>vertebral height) | Pathologic fracture<br>causing<br>life threatening<br>consequences |

BMD: bone mineral density; NAP: not applicable

Bone mineral density t and z scores can be found in: Kanis JA on behalf of the World Health Organization Scientific Group (2007). Assessment of osteoporosis at the primary health care level. Technical Report. World Health Organization Collaborating Centre for Metabolic Bone Diseases, University of Sheffield, UK. 2007: Printed by the University of Sheffield.

| | NEUROLOGIC | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acute CNS Ischemia | NAP | NAP | Transient ischemic attack | Cerebral vascular<br>accident (eg, stroke<br>with neurological<br>deficit) |
| Altered Mental Status (for Dementia, refer to Cognitive, Behavioral, or Attentional Disturbance below) | Changes causing no or<br>minimal interference<br>with usual social &<br>functional activities | Mild lethargy or<br>somnolence causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR<br>Obtundation OR Coma |
| Ataxia | Symptoms causing no or minimal interference with usual social & functional activities OR No symptoms with ataxia detected on examination | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Disabling symptoms<br>causing inability to<br>perform basic self care<br>functions |
| Cognitive, Behavioral, or Attentional Disturbance (includes dementia and attention deficit disorder) Specify type, if applicable | Disability causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities OR<br>Specialized resources<br>not indicated | Disability causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities OR<br>Specialized resources<br>on part time basis<br>indicated | Disability causing inability to perform usual social & functional activities OR Specialized resources on a full time basis indicated | Disability causing inability to perform basic self care functions OR Institutionalization indicated |
| Developmental Delay<br>Specify type, if<br>applicable<br>aged <18 years | Mild developmental<br>delay, either motor or<br>cognitive, as<br>determined by<br>comparison with a<br>developmental<br>screening tool<br>appropriate for the<br>setting | Moderate<br>developmental delay,<br>either motor or<br>cognitive, as<br>determined by<br>comparison with a<br>developmental<br>screening tool<br>appropriate for the<br>setting | Severe developmental<br>delay, either motor or<br>cognitive, as<br>determined by<br>comparison with a<br>developmental<br>screening tool<br>appropriate for the<br>setting | Developmental regression, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting |
| Headache CNS: control por course suct | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self care functions OR Hospitalization indicated OR Headache with significant impairment of alertness or other neurologic function |

CNS: central nervous system; NAP: not applicable

| | | NEUROLOGIC | | * |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Neuromuscular<br>Weakness<br>(includes myopathy<br>and neuropathy)<br>Specify type, if<br>applicable | Minimal muscle weakness causing no or minimal interference with usual social & functional activities OR No symptoms with decreased strength on examination | Muscle weakness<br>causing greater than<br>minimal interference<br>with usual social &<br>functional activities | Muscle weakness<br>causing inability to<br>perform usual social &<br>functional activities | Disabling muscle<br>weakness causing<br>inability to perform<br>basic self care<br>functions OR<br>Respiratory muscle<br>weakness impairing<br>ventilation |
| Neurosensory Alteration (includes paresthesia and painful neuropathy) Specify type, if applicable | Minimal paresthesia<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities OR No<br>symptoms with<br>sensory alteration on<br>examination | Sensory alteration or<br>paresthesia causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Sensory alteration or<br>paresthesia causing<br>inability to perform<br>usual social &<br>functional activities | Disabling sensory<br>alteration or<br>paresthesia causing<br>inability to perform<br>basic self care<br>functions |
| Seizures New Onset Seizure aged ≥18 years | NAP | NAP | 1 to 3 seizures | Prolonged and<br>repetitive seizures<br>(eg, status epilepticus)<br>OR Difficult to control<br>(eg, refractory<br>epilepsy) |
| aged <18 years<br>(includes new or<br>pre existing<br>febrile seizures) | Seizure lasting <5 minutes with <24 hours postictal state | Seizure lasting 5 to<br><20 minutes with<br><24 hours postictal<br>state | Seizure lasting ≥20 minutes OR >24 hours postictal state | Prolonged and<br>repetitive seizures<br>(eg, status epilepticus)<br>OR Difficult to control<br>(eg, refractory<br>epilepsy) |
| Pre existing Seizure | NAP | Increased frequency<br>from previous level of<br>control without change<br>in seizure character | Change in seizure<br>character either in<br>duration or quality (eg,<br>severity or focality) | Prolonged and<br>repetitive seizures<br>(eg, status epilepticus)<br>OR Difficult to control<br>(eg, refractory<br>epilepsy) |
| Syncope | Near syncope without<br>loss of consciousness<br>(eg, pre syncope) | Loss of consciousness with no intervention indicated | Loss of consciousness<br>AND Hospitalization<br>or intervention<br>required | NAP |

NAP: not applicable

| | PREGNANCY, PUERPERIUM, AND PERINATAL | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Stillbirth<br>(report using mother's<br>participant ID)<br>Report only 1 | NAP | NAP | Fetal death occurring at ≥20 weeks gestation | NAP |
| Preterm Birth<br>(report using mother's<br>participant ID) | Live birth at 34 to <37 weeks gestational age | Live birth at 28 to<br><34 weeks gestational<br>age | Live birth at 24 to <28 weeks gestational age | Live birth at <24 weeks gestational age |
| Abortion or Miscarriage <sup>g</sup> (report using mother's participant ID) Report only 1 | Chemical pregnancy | Uncomplicated spontaneous abortion or miscarriage | Complicated spontaneous abortion or miscarriage | NAP |

ID: identity, NAP: not applicable

g A pregnancy loss occurring at <20 weeks gestational age.

| | PSYCHIATRIC | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Insomnia | Mild difficulty falling<br>asleep, staying asleep,<br>or waking up early<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities | Moderate difficulty<br>falling asleep, staying<br>asleep, or waking up<br>early causing more<br>than minimal<br>interference with usual<br>social & functional<br>activities | Severe difficulty falling asleep, staying asleep, or waking up early causing inability to perform usual social & functional activities requiring intervention or hospitalization | NAP |
| Psychiatric Disorders<br>(includes anxiety,<br>depression, mania, and<br>psychosis)<br>Specify disorder | Symptoms with intervention not indicated OR Behavior causing no or minimal interference with usual social & functional activities | Symptoms with intervention indicated OR Behavior causing greater than minimal interference with usual social & functional activities | Symptoms with<br>hospitalization<br>indicated OR Behavior<br>causing inability to<br>perform usual social &<br>functional activities | Threatens harm to self<br>or others OR Acute<br>psychosis OR<br>Behavior causing<br>inability to perform<br>basic self care<br>functions |
| Suicidal Ideation or<br>Attempt<br>Report only 1 | Preoccupied with<br>thoughts of death AND<br>No wish to kill oneself | Preoccupied with<br>thoughts of death AND<br>Wish to kill oneself<br>with no specific plan<br>or intent | Thoughts of killing<br>oneself with partial or<br>complete plans but no<br>attempt to do so OR<br>Hospitalization<br>indicated | Suicide attempted |

NAP: not applicable

| | | RESPIRATORY | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acute Bronchospasm | Forced expiratory<br>volume in 1 second or<br>peak flow reduced to<br>≥70% to <80% OR<br>Mild symptoms with<br>intervention not<br>indicated | Forced expiratory volume in 1 second or peak flow 50% to <70% OR Symptoms with intervention indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Forced expiratory<br>volume in 1 second or<br>peak flow 25% to<br><50% OR Symptoms<br>causing inability to<br>perform usual social<br>& functional activities | Forced expiratory volume in 1 second or peak flow <25% OR Life threatening respiratory or hemodynamic compromise OR Intubation |
| Dyspnea or<br>Respiratory Distress<br>Report only 1 | Dyspnea on exertion with no or minimal interference with usual social & functional activities OR Wheezing OR Minimal increase in respiratory rate for age | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities OR Nasal flaring OR Intercostal retractions OR Pulse oximetry 90% to <95% | Dyspnea at rest<br>causing inability to<br>perform usual social<br>& functional activities<br>OR Pulse oximetry<br><90% | Respiratory failure with<br>ventilator support<br>indicated (eg, CPAP,<br>BPAP, intubation) |

BPAP: biphasic positive airway pressure; CPAP: continuous positive airway pressure; NAP: not applicable

| | | SENSORY | | * |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Hearing Loss aged ≥12 years | NAP | Hearing aid or intervention not indicated | Hearing aid or intervention indicated | Profound bilateral<br>hearing loss (>80 dB at<br>2 kHz and above) OR<br>Nonserviceable<br>hearing (ie, >50 dB<br>audiogram and <50%<br>speech discrimination) |
| aged <12 years<br>(based on a 1, 2,<br>3, 4, 6, and 8 kHz<br>audiogram) | >20 dB hearing loss at ≤4 kHz | >20 dB hearing loss at<br>>4 kHz | >20 dB hearing loss at<br>≥3 kHz in 1 ear with<br>additional speech<br>language related<br>services indicated<br>(where available) OR<br>Hearing loss sufficient<br>to indicate therapeutic<br>intervention, including<br>hearing aids | Audiologic indication<br>for cochlear implant<br>and additional speech<br>language related<br>services indicated<br>(where available) |
| Tinnitus | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities with<br>intervention not<br>indicated | Symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated | Symptoms causing inability to perform usual social & functional activities | NAP |
| Uveitis | No symptoms AND<br>Detectable on<br>examination | Anterior uveitis with<br>symptoms OR Medical<br>intervention indicated | Posterior or<br>pan uveitis OR<br>Operative intervention<br>indicated | Disabling visual loss in affected eye(s) |
| Vertigo | Vertigo causing no or<br>minimal interference<br>with usual social &<br>functional activities | Vertigo causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo<br>causing inability to<br>perform basic self care<br>functions |
| Visual Changes<br>(assessed from<br>baseline) | Visual changes<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities | Visual changes causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Visual changes<br>causing inability to<br>perform usual social &<br>functional activities | Disabling visual loss in affected eye(s) |

dB: decibel; kHz: kilohertz; NAP: not applicable

| | SYSTEMIC | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acute Allergic<br>Reaction | Localized urticaria<br>(wheals) with no<br>medical intervention<br>indicated | Localized urticaria<br>with intervention<br>indicated OR Mild<br>angioedema with no<br>intervention indicated | Generalized urticaria<br>OR Angioedema with<br>intervention indicated<br>OR Symptoms of mild<br>bronchospasm | Acute anaphylaxis OR<br>Life threatening<br>bronchospasm OR<br>Laryngeal edema |
| Chills | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities | Symptoms causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Symptoms causing inability to perform usual social & functional activities | NAP |
| Cytokine Release<br>Syndrome <sup>h</sup> | Mild signs and<br>symptoms AND<br>Therapy (ie, antibody<br>infusion) interruption<br>not indicated | Therapy (ie, antibody infusion) interruption indicated AND Responds promptly to symptomatic treatment OR Prophylactic medications indicated for ≤24 hours | Prolonged severe signs<br>and symptoms OR<br>Recurrence of<br>symptoms following<br>initial improvement | Life threatening<br>consequences<br>(eg, requiring pressor<br>or ventilator support) |
| Fatigue or Malaise<br>Report only 1 | Symptoms causing no<br>or minimal<br>interference with usual<br>social & functional<br>activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating<br>symptoms of fatigue or<br>malaise causing<br>inability to perform<br>basic self care<br>functions |
| Fever<br>(non axillary<br>temperatures only) | 38.0°C to <38.6°C or<br>100.4°F to <101.5°F | ≥38.6°C to <39.3°C or<br>≥101.5°F to <102.7°F | ≥39.3°C to <40.0°C or<br>≥102.7°F to <104.0°F | ≥40.0°C or ≥104.0°F |
| Pain <sup>1</sup> (not associated with study intervention injections and not specified elsewhere) Specify location | Pain causing no or<br>minimal interference<br>with usual social &<br>functional activities | Pain causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Pain causing inability<br>to perform usual social<br>& functional activities | Disabling pain causing inability to perform basic self care functions OR Hospitalization indicated |
| Serum Sickness <sup>J</sup> | Mild signs and symptoms | Moderate signs and<br>symptoms AND<br>Intervention indicated<br>(eg, antihistamines) | Severe signs and<br>symptoms AND<br>Higher level<br>intervention indicated<br>(eg, steroids or IV<br>fluids) | Life threatening<br>consequences<br>(eg, requiring pressor<br>or ventilator support) |

IV: intravenous; NAP: not applicable

<sup>&</sup>lt;sup>h</sup> A disorder characterized by nausea, headache, tachycardia, hypotension, rash, and/or shortness of breath.

For pain associated with injections or infusions, refer to the SITE REACTIONS TO INJECTIONS AND INFUSIONS section.

A disorder characterized by fever, arthralgia, myalgia, skin eruptions, lymphadenopathy, marked discomfort, and/or dyspnea.

| | | SYSTEMIC | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Underweight <sup>k</sup> aged >5 to 19 years | WHO BMI z score<br>< 1 to 2 | WHO BMI z score < 2 to 3 | WHO BMI z score < 3 | WHO BMI z score < 3<br>with life threatening<br>consequences |
| aged 2 to 5 years | WHO Weight for<br>height z score<br>< 1 to 2 | WHO Weight for<br>height z score<br>< 2 to 3 | WHO Weight for<br>height z score < 3 | WHO Weight for<br>height z score < 3 with<br>life threatening<br>consequences |
| aged <2 years | WHO Weight for<br>length z score<br>< 1 to 2 | WHO Weight for<br>length z score<br>< 2 to 3 | WHO Weight for<br>length z score < 3 | WHO Weight for<br>length z score < 3 with<br>life threatening<br>consequences |
| Unintentional Weight<br>Loss<br>(excludes postpartum<br>weight loss) | NAP | 5% to <9% loss in<br>body weight from<br>baseline | ≥9% to <20% loss in<br>body weight from<br>baseline | ≥20% loss in body<br>weight from baseline<br>OR Aggressive<br>intervention indicated<br>(eg, tube feeding, total<br>parenteral nutrition) |

BMI: body mass index; NAP: not applicable; WHO: World Health Organization

k WHO reference tables may be accessed by clicking the desired age range or h WHO reference tables may be accessed by clicking the desired age range or by accessing the following URLs: http://www.who.int/growthref/who2007 bmi for age/en/ for participants aged >5 to 19 years and http://www.who.int/childgrowth/standards/chart catalogue/en/ for those aged ≤5 years.

| URINARY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Urinary Tract<br>Obstruction | NAP | Signs or symptoms of<br>urinary tract<br>obstruction without<br>hydronephrosis or renal<br>dysfunction | Signs or symptoms of<br>urinary tract<br>obstruction with<br>hydronephrosis or<br>renal dysfunction | Obstruction causing life threatening consequences |

NAP: not applicable

| | SITE REACTIO | ONS TO INJECTIONS A | ND INFUSIONS | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Injection Site Pain or<br>Tenderness<br>Report only 1 | Pain or tenderness<br>causing no or minimal<br>limitation of use of<br>limb | Pain or tenderness<br>causing greater than<br>minimal limitation of<br>use of limb | Pain or tenderness<br>causing inability to<br>perform usual social &<br>functional activities | Pain or tenderness<br>causing inability to<br>perform basic self care<br>function OR<br>Hospitalization<br>indicated |
| Injection Site<br>Erythema or Redness <sup>1</sup><br>Report only 1<br>aged >15 years | 2.5 to <5 cm in<br>diameter OR 6.25 to<br><25 cm² surface area<br>AND Symptoms<br>causing no or minimal<br>interference with<br>usual social &<br>functional activities | ≥5 to <10 cm in<br>diameter OR ≥25 to<br><100 cm² surface area<br>OR Symptoms causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | ≥10 cm in diameter OR ≥100 cm² surface area OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage OR Symptoms causing inability to perform usual social & functional activities | Potentially life threatening consequences (eg, abscess, exfoliative dermatitis, necrosis involving dermis or deeper tissue) |
| aged ≤15 years | ≤2.5 cm in diameter | >2.5 cm in diameter<br>with <50% surface area<br>of the extremity<br>segment involved<br>(eg, upper arm or thigh) | ≥50% surface area of<br>the extremity segment<br>involved (eg, upper<br>arm or thigh) OR<br>Ulceration OR<br>Secondary infection<br>OR Phlebitis OR<br>Sterile abscess OR<br>Drainage | Potentially<br>life threatening<br>consequences<br>(eg, abscess,<br>exfoliative dermatitis,<br>necrosis involving<br>dermis or deeper<br>tissue) |
| Injection Site Induration or Swelling Report only 1 aged >15 years | Same as for Injection<br>Site Erythema or<br>Redness, aged<br>>15 years | Same as for Injection<br>Site Erythema or<br>Redness, aged<br>>15 years | Same as for Injection<br>Site Erythema or<br>Redness, aged<br>>15 years | Same as for Injection<br>Site Erythema or<br>Redness, aged<br>>15 years |
| aged ≤15 years | Same as for Injection<br>Site Erythema or<br>Redness, aged<br>≤15 years | Same as for Injection Site Erythema or Redness, aged ≤15 years | Same as for Injection Site Erythema or Redness, aged ≤15 years | Same as for Injection Site Erythema or Redness, aged ≤15 years |
| Injection Site Pruritus | Itching localized to<br>the injection site that<br>is relieved<br>spontaneously or in<br><48 hours of<br>treatment | Itching beyond the injection site that is not generalized OR Itching localized to the injection site requiring ≥48 hours treatment | Generalized itching causing inability to perform usual social & functional activities | NAP |

NAP: not applicable
Injection Site Error

Injection Site Erythema or Redness should be evaluated and graded using the greatest single diameter or measured surface area.

| | LABORATORY VALUES <sup>m</sup> CHEMISTRIES | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acidosis | NAP | pH ≥7.3 to <lln< td=""><td>pH &lt;7.3 without<br/>life threatening<br/>consequences</td><td>pH &lt;7.3 with<br/>life threatening<br/>consequences</td></lln<> | pH <7.3 without<br>life threatening<br>consequences | pH <7.3 with<br>life threatening<br>consequences |
| Albumin, Low (g/dL; g/L) | 3.0 to <lln<br>30 to <lln< td=""><td>≥2.0 to &lt;3.0<br/>≥20 to &lt;30</td><td>&lt;2.0<br/>&lt;20</td><td>NAP</td></lln<></lln<br> | ≥2.0 to <3.0<br>≥20 to <30 | <2.0<br><20 | NAP |
| ALP, High | 1.25 to <2.5×ULN | 2.5 to <5.0×ULN | 5.0 to <10.0×ULN | ≥10.0×ULN |
| Alkalosis | NAP | pH >ULN to ≤7.5 | pH >7.5 without life threatening consequences | pH >7.5 with<br>life threatening<br>consequences |
| ALT or SGPT, High<br>Report only 1 | 1.25 to <2.5×ULN | 2.5 to <5.0×ULN | 5.0 to <10.0×ULN | ≥10.0×ULN |
| Amylase (Pancreatic)<br>or Amylase (Total),<br>High<br>Report only 1 | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| AST or SGOT, High<br>Report only 1 | 1.25 to <2.5×ULN | 2.5 to <5.0×ULN | 5.0 to <10.0×ULN | ≥10.0×ULN |
| Bicarbonate, Low<br>(mEq/L; mmol/L) | 16.0 to <lln<br>16.0 to <lln< td=""><td>11.0 to &lt;16.0<br/>11.0 to &lt;16.0</td><td>8.0 to &lt;11.0<br/>8.0 to &lt;11.0</td><td>&lt;8.0<br/>&lt;8.0</td></lln<></lln<br> | 11.0 to <16.0<br>11.0 to <16.0 | 8.0 to <11.0<br>8.0 to <11.0 | <8.0<br><8.0 |
| Bilirubin<br>Direct Bilirubin,"<br>High<br>aged > 28 days | NAP | NAP | >ULN with other signs<br>and symptoms of<br>hepatotoxicity | >ULN with<br>life threatening<br>consequences<br>(eg, signs and<br>symptoms of liver<br>failure) |
| aged ≤28 days | ULN to ≤1 mg/dL | >1 to ≤1.5 mg/dL | >1.5 to ≤2 mg/dL | >2 mg/dL |
| Total Bilirubin, High<br>aged >28 days | 1,1 to <1.6×ULN | 1.6 to <2.6×ULN | 2.6 to <5.0×ULN | ≥5.0×ULN |
| aged ≤28 days | Refer to Appendix A <sup>o</sup> | Refer to Appendix A <sup>o</sup> | Refer to Appendix A <sup>o</sup> | Refer to Appendix A <sup>o</sup> |

ALP: alkaline phosphatase; ALT: alanine aminotransferase; AST: aspartate aminotransferase; LLN: lower limit of normal; mEq: milliequivalent; NAP: not applicable; SGOT: serum glutamic oxaloacetic transaminase; SGPT: serum glutamate pyruvate transaminase; ULN: upper limit of normal

Reminder: An asymptomatic abnormal laboratory finding without an accompanying AE should not be reported to DAIDS in an expedited time frame unless it meets protocol specific reporting requirements.

Direct bilirubin >1.5 mg/dL in a participant aged <28 days should be graded as grade 2, if <10% of the total bilirubin. Appendix A "Total Bilirubin Table for Term and Preterm Neonates" is provided together with the DAIDS table corrected version 2.1 at the following URL: https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf. Appendix A is not applicable for this study.

| LABORATORY VALUES | | | | |
|---|---|---|---|---|
| | CHEMISTRIES | | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Calcium, High (mg/dL; mmol/L) aged ≥7 days aged <7 days | 10.6 to <11.5<br>2.65 to <2.88<br>11.5 to <12.4<br>2.88 to <3.10 | 11.5 to <12.5<br>2.88 to <3.13<br>12.4 to <12.9<br>3.10 to <3.23 | 12.5 to <13.5<br>3.13 to <3.38<br>12.9 to <13.5<br>3.23 to <3.38 | ≥13.5<br>≥3.38<br>≥13.5<br>≥3.38 |
| Calcium (Ionized),<br>High<br>(mg/dL; mmol/L) | >ULN to <6.0<br>>ULN to <1.5 | 6.0 to <6.4<br>1.5 to <1.6 | 6.4 to <7.2<br>1.6 to <1.8 | ≥7.2<br>≥1.8 |
| Calcium, Low<br>(mg/dL; mmol/L)<br>aged ≥7 days | 7.8 to <8.4<br>1.95 to <2.10 | 7.0 to <7.8<br>1.75 to <1.95 | 6.1 to <7.0<br>1.53 to <1.75 | <6.1<br><1.53 |
| aged <7 days | 6.5 to <7.5<br>1.63 to <1.88 | 6.0 to <6.5<br>1.50 to <1.63 | 5.50 to <6.0<br>1.38 to <1.50 | <5.50<br><1.38 |
| Calcium (Ionized),<br>Low<br>(mg/dL; mmol/L) | <lln 4.0<br="" to=""><lln 1.0<="" td="" to=""><td>3.6 to &lt;4.0<br/>0.9 to &lt;1.0</td><td>3.2 to &lt;3.6<br/>0.8 to &lt;0.9</td><td>&lt;3.2<br/>&lt;0.8</td></lln></lln> | 3.6 to <4.0<br>0.9 to <1.0 | 3.2 to <3.6<br>0.8 to <0.9 | <3.2<br><0.8 |
| Cardiac Troponin I,<br>High | NAP | NAP | NAP | Levels consistent with<br>myocardial infarction<br>or unstable angina as<br>defined by the local<br>laboratory |
| Creatine Kinase,<br>High | 3 to <6×ULN | 6 to <10×ULN | 10 to <20×ULN | ≥20×ULN |
| Creatinine, High<br>Report only 1 <sup>p</sup> | 1.1 to 1.3×ULN | >1.3 to 1.8×ULN OR<br>Increase to 1.3 to<br><1.5×participant's<br>baseline | >1.8 to <3.5×ULN OR<br>Increase to 1.5 to<br><2.0×participant's<br>baseline | ≥3.5×ULN OR<br>Increase of<br>≥2.0×participant's<br>baseline |
| Creatinine<br>Clearance <sup>q</sup> or eGFR,<br>Low<br>Report only 1 <sup>p</sup> | NAP | <90 to 60 ml/min or<br>ml/min/1.73 m <sup>2</sup> OR<br>10% to <30% decrease<br>from participant's<br>baseline | <60 to 30 ml/min or<br>ml/min/1.73 m <sup>2</sup> OR<br>30% to <50% decrease<br>from participant's<br>baseline | <30 ml/min or<br>ml/min/1.73 m² OR<br>≥50% decrease from<br>participant's baseline<br>or dialysis needed |
| Glucose<br>(mg/dL; mmol/L)<br>Fasting, High | 110 to 125<br>6.11 to <6.95 | >125 to 250<br>6.95 to <13.89 | >250 to 500<br>13.89 to <27.75 | >500<br>≥27.75 |
| Nonfasting, High | 116 to 160<br>6.44 to <8.89 | >160 to 250<br>8.89 to <13.89 | >250 to 500<br>13.89 to <27.75 | >500<br>≥27.75 |
| Glucose, Low<br>(mg/dL; mmol/L)<br>aged ≥1 month | 55 to 64<br>3.05 to <3.55 | 40 to <55<br>2.22 to <3.05 | 30 to <40<br>1.67 to <2.22 | <30<br><1.67 |
| aged <1 month | 50 to 54<br>2.78 to <3.00 | 40 to <50<br>2.22 to <2.78 | 30 to <40<br>1.67 to <2.22 | <30<br><1.67 |
| Lactate, High | ULN to <2.0×ULN without acidosis | ≥2.0×ULN without acidosis | Increased lactate with pH <7.3 without life threatening consequences | Increased lactate with pH <7.3 with life threatening consequences |

eGFR: estimated glomerular filtration rate; LLN: lower limit of normal; NAP: not applicable; ULN: upper limit of normal P Reminder: Choose the method that selects for the higher grade.

<sup>&</sup>lt;sup>q</sup> Use the applicable formula (ie, Cockcroft Gault in mL/min or Schwartz, modification of diet in renal disease study [MDRD], or Chronic Kidney Disease Epidemiology Collaboration [CKD EPI] in mL/min/1.73m<sup>2</sup>). Sites should choose the method defined in their study and when not specified, use the method most relevant to the study population.

| | LABORATORY VALUES CHEMISTRIES | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Lipase, High | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| Lipid Disorders<br>(mg/dL; mmol/L)<br>Cholesterol, Fasting,<br>High<br>aged ≥18 years | 200 to <240<br>5.18 to <6.19 | 240 to <300<br>6.19 to <7.77 | ≥300<br>≥7.77 | NAP |
| aged < 18 years | 170 to <200<br>4.40 to <5.15 | 200 to <300<br>5.15 to <7.77 | ≥300<br>≥7.77 | NAP |
| LDL, Fasting, High | 130 to <160 | 160 to <190 | ≥190 | NAP |
| aged ≥18 years | 3.37 to <4.12 | 4.12 to <4.90 | ≥4.90 | |
| aged > 2 to | 110 to <130 | 130 to <190 | ≥190 | NAP |
| <18 years | 2.85 to <3.34 | 3.34 to <4.90 | ≥4.90 | |
| Triglycerides, | 150 to 300 | >300 to 500 | >500 to 1,000 | >1,000 |
| Fasting, High | 1.71 to 3.42 | >3.42 to 5.7 | >5.7 to 11.4 | >11.4 |
| Magnesium <sup>r</sup> , Low (mEq/L; mmol/L) | 1.2 to <1.4 | 0.9 to <1.2 | 0.6 to <0.9 | <0.6 |
| | 0.60 to <0.70 | 0.45 to <0.60 | 0.30 to <0.45 | <0.30 |
| Phosphate, Low<br>(mg/dL; mmol/L)<br>aged > 14 years | 2.0 to <lln<br>0.65 to <lln< td=""><td>1.4 to &lt;2.0<br/>0.45 to &lt;0.65</td><td>1.0 to &lt;1.4<br/>0.32 to &lt;0.45</td><td>&lt;1.0<br/>&lt;0.32</td></lln<></lln<br> | 1.4 to <2.0<br>0.45 to <0.65 | 1.0 to <1.4<br>0.32 to <0.45 | <1.0<br><0.32 |
| aged 1 to | 3.0 to <3.5 | 2.5 to <3.0 | 1.5 to <2.5 | <1.5 |
| 14 years | 0.97 to <1.13 | 0.81 to <0.97 | 0.48 to <0.81 | <0.48 |
| aged < 1 year | 3.5 to <4.5 | 2.5 to <3.5 | 1.5 to <2.5 | <1.5 |
| | 1.13 to <1.45 | 0.81 to <1.13 | 0.48 to <0.81 | <0.48 |
| Potassium, High | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| (mEq/L; mmol/L) | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| Potassium, Low (mEq/L; mmol/L) | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| Sodium, High | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| (mEq/L; mmol/L) | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| Sodium, Low | 130 to <135 | 125 to <130 | 120 to <125 | <120 |
| (mEq/L; mmol/L) | 130 to <135 | 125 to <130 | 120 to <125 | < <i>I20</i> |
| Uric Acid, High | 7.5 to <10.0 | 10.0 to <12.0 | 12.0 to <15.0 | ≥15.0 |
| (mg/dL; mmol/L) | 0.45 to <0.59 | 0.59 to <0.71 | 0.71 to <0.89 | ≥0.89 |

LDL: low density lipoprotein; LLN: lower limit of normal; mEq: milliequivalent; NAP: not applicable; ULN: upper limit of normal

 $<sup>^{\</sup>rm r}$  To convert a magnesium value from mg/dL to mmol/L, laboratories should multiply by 0.4114.

| LABORATORY VALUES | | | | |
|---|---|---|---|---|
| | | HEMATOLOGY | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Absolute CD4 <sup>+</sup> Count, Low (cells/mm³; cells/L) aged >5 years (not HIV infected) | 300 to <400<br>0.300×10 <sup>9</sup> to<br><0.400×10 <sup>9s</sup> | 200 to <300<br>0.200×10 <sup>9</sup> to<br><0.300×10 <sup>9</sup> 8 | 100 to <200<br>0.100×10 <sup>9</sup> to<br><0.200×10 <sup>9</sup> s | <100<br><0.100×10 <sup>9s</sup> |
| Absolute Lymphocyte<br>Count, Low<br>(cells/mm³; cells/L)<br>aged >5 years<br>(not HIV infected) | 600 to <650<br>0.600×10 <sup>9</sup> to<br><0.650×10 <sup>9</sup> | 500 to <600<br>0.500×10 <sup>9</sup> to<br><0.600×10 <sup>9</sup> | 350 to <500<br>0.350×10 <sup>9</sup> to<br><0.500×10 <sup>9</sup> | <350<br><0.350×10 <sup>9</sup> |
| Absolute Neutrophil<br>Count, Low<br>(cells/mm³; cells/L)<br>aged >7 days | 800 to 1,000<br>0.800×10 <sup>9</sup> to<br>1.000×10 <sup>9</sup> | 600 to 799<br>0.600×10 <sup>9</sup> to<br>0.799×10 <sup>9</sup> | 400 to 599<br>0.400×10 <sup>9</sup> to<br>0.599×10 <sup>9</sup> | <400<br><0.400×10 <sup>9</sup> |
| aged 2 to 7 days | 1,250 to 1,500<br>1.250×10 <sup>9</sup> to<br>1.500×10 <sup>9</sup> | 1,000 to 1,249<br>1.000×10 <sup>9</sup> to<br>1.249×10 <sup>9</sup> | 750 to 999<br>0.750×10 <sup>9</sup> to<br>0.999×10 <sup>9</sup> | <750<br><0.750×10 <sup>9</sup> |
| aged ≤1 day | 4,000 to 5,000<br>4.000×10 <sup>9</sup> to<br>5.000×10 <sup>9</sup> | 3,000 to 3,999<br>3.000×10 <sup>9</sup> to<br>3.999×10 <sup>9</sup> | 1,500 to 2,999<br>1.500×10 <sup>9</sup> to<br>2.999×10 <sup>9</sup> | <1,500<br><1.500×10° |
| Fibrinogen,<br>Decreased<br>(mg/dL; g/L) | 100 to <200<br>1.00 to <2.00<br>OR<br>0.75 to <1.00×LLN | 75 to <100<br>0.75 to <1.00<br>OR<br>≥0.50 to <0.75×LLN | 50 to <75<br>0.50 to <0.75<br>OR<br>0.25 to <0.50×LLN | <50<br><0.50<br>OR<br><0.25×LLN<br>OR Associated with<br>gross bleeding |
| Hemoglobin <sup>t</sup> , Low<br>(g/dL; mmol/L) <sup>u</sup><br>aged ≥13 years<br>(male only) | 10.0 to 10.9<br>6.19 to 6.76 | 9.0 to <10.0<br>5.57 to <6.19 | 7.0 to <9.0<br>4.34 to <5.57 | <7.0<br><4.34 |
| aged ≥13 years<br>(female only) | 9.5 to 10.4<br>5.88 to 6.48 | 8.5 to <9.5<br>5.25 to <5.88 | 6.5 to <8.5<br>4.03 to <5.25 | <6.5<br><4.03 |
| aged 57 days to<br><13 years (male<br>and female) | 9.5 to 10.4<br>5.88 to 6.48 | 8.5 to <9.5<br>5.25 to <5.88 | 6.5 to <8.5<br>4.03 to <5.25 | <6.5<br><4.03 |
| aged 36 to 56 days<br>(male and female) | 8.5 to 9.6<br>5.26 to 5.99 | 7.0 to <8.5<br>4.32 to <5.26 | 6.0 to <7.0<br>3.72 to <4.32 | <6.0<br><3.72 |
| aged 22 to 35 days (male and female) | 9.5 to 11.0<br>5.88 to 6.86 | 8.0 to <9.5<br>4.94 to <5.88 | 6.7 to <8.0<br>4.15 to <4.94 | <6.7<br><4.15 |
| aged 8 to $\leq$ 21 days (male and female) | 11.0 to 13.0<br>6.81 to 8.10 | 9.0 to <11.0<br>5.57 to <6.81 | 8.0 to <9.0<br>4.96 to <5.57 | <8.0<br><4.96 |
| aged ≤7 days (male<br>and female)<br>HIV: human immunodefic | 13.0 to 14.0<br>8.05 to 8.72 | 10.0 to <13.0<br>6.19 to <8.05 | 9.0 to <10.0<br>5.59 to <6.19 | <9.0<br><5.59 |

HIV: human immunodeficiency virus; LLN: lower limit of normal

<sup>8</sup> Revised by the sponsor.

Male and female sex are defined as sex at birth. For transgender participants aged ≥13 years who have been on hormone therapy for more than 6 consecutive months, grade hemoglobin based on the gender with which they identify (ie, a transgender female should be graded using the female sex at birth hemoglobin laboratory values).

The most commonly used conversion factor to convert g/dL to mmol/L is 0.6206. For grading hemoglobin results obtained by an analytic method with a conversion factor other than 0.6206, the result must be converted to g/dL using the appropriate conversion factor for the particular laboratory.

| | | LABORATORY VALU | ES | |
|---|---|---|---|---|
| | | HEMATOLOGY | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| INR, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.5×ULN | 1.5 to <2.0×ULN | 2.0 to <3.0×ULN | ≥3.0×ULN |
| Methemoglobin<br>(% hemoglobin) | 5.0% to <10.0% | 10.0% to <15.0% | 15.0% to <20.0% | ≥20.0% |
| PTT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.66×ULN | 1.66 to <2.33×ULN | 2.33 to <3.00×ULN | ≥3.00×ULN |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to <125,000<br>100.000×10 <sup>9</sup> to<br><125.000×10 <sup>9</sup> | 50,000 to <100,000<br>50.000×10 <sup>9</sup> to<br><100.000×10 <sup>9</sup> | 25,000 to <50,000<br>25.000×10 <sup>9</sup> to<br><50.000×10 <sup>9</sup> | <25,000<br><25.000×10 <sup>9</sup> |
| PT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.25×ULN | 1.25 to <1.50×ULN | 1.50 to <3.00×ULN | ≥3.00×ULN |
| WBC, Decreased<br>(cells/mm³; cells/L)<br>aged >7 days | 2,000 to 2,499<br>2.000×10° to<br>2.499×10° | 1,500 to 1,999<br>1.500×10 <sup>9</sup> to<br>1.999×10 <sup>9</sup> | 1,000 to 1,499<br>1.000×10 <sup>9</sup> to<br>1.499×10 <sup>9</sup> | <1,000<br><1.000×10 <sup>9</sup> |
| aged ≤7 days | 5,500 to 6,999<br>5.500×10 <sup>9</sup> to<br>6.999×10 <sup>9</sup> | 4,000 to 5,499<br>4.000×10 <sup>9</sup> to<br>5.499×10 <sup>9</sup> | 2,500 to 3,999<br>2.500×10 <sup>9</sup> to<br>3.999×10 <sup>9</sup> | <2,500<br><2.500×10 <sup>9</sup> |

INR: International Normalized Ratio; NAP: not applicable; PT: prothrombin time; PTT: partial thromboplastin time; ULN: upper limit of normal; WBC: white blood cell

| | | LABORATORY VALUE | S | |
|---|---|---|---|---|
| | | URINALYSIS | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Glycosuria<br>(random collection<br>tested by dipstick) | Trace to 1+ or ≤250 mg | 2+ or >250 to ≤500 mg | >2+ or >500 mg | NAP |
| Hematuria (not to be reported based on dipstick findings or on blood believed to be of menstrual origin) | 6 to <10 RBCs per<br>high power field | ≥10 RBCs per high<br>power field | Gross, with or without<br>clots OR With RBC<br>casts OR Intervention<br>indicated | Life threatening consequences |
| Proteinuria<br>(random collection<br>tested by dipstick) | 1+ | 2+ | 3+ or higher | NAP |

NAP: not applicable; RBC: red blood cell

# 10.10. Appendix 10: Protocol Amendment History

The Protocol Amendment Summary of Changes Table for the current amendment is located directly before the Table of Contents (TOC).

## Amendment 5 (01 October 2021)

**Overall Rationale for the Amendment:** The primary reasons for this amendment are to remove JNJ-6379 as study intervention, to add a new nucleos(t)ide analog (NA) re-treatment criterion for participants who discontinued NA treatment during follow-up, and to include more frequent monitoring for participants who discontinued NA treatment during follow-up.

Based on emerging data from recent interim analyses of the REEF-1 (73763989HPB2001) and REEF-2 (73763989PAHPB2002) studies, the benefit-risk profile of JNJ-6379 in combination with JNJ-3989+NA is unfavorable compared to JNJ-3989+NA.

In the primary REEF-1 analysis (Week 48, end of treatment) the mean reduction of hepatitis B surface antigen (HBsAg) in the triple arm (JNJ-6379+JNJ-3989 100mg+NA) appeared to be less than in the dual arm (JNJ-3989 100mg+NA). More recent interim results of the REEF-2 study (Week 48, end of treatment) confirmed this observation when the effect of JNJ-6379+JNJ-3989 200mg+NA on mean HBsAg level reduction in REEF-2 study is compared to JNJ-3989 200mg+NA in the REEF-1 study. To match with the REEF-2 population, this cross-study comparison focused on the REEF-1 subpopulation of hepatitis B e antigen (HBeAg) negative, virologically suppressed participants with chronic hepatitis B. Pharmacokinetic-pharmacodynamic modelling analyses accounting for variability in baseline characteristics further support this observation. Therefore, a negative impact of JNJ-6379 on the HBsAg lowering effect of JNJ-3989+NA is suspected.

From a safety perspective, transient reductions of eGFR based on creatinine (eGFRcr) in JNJ-6379 containing treatment arms with fast recovery after end of treatment had been described in the Jade study (56136379HPB2001) and was confirmed in the REEF-1 study. In absence of a pattern of increased biomarkers of proximal tubulo-toxicity (the beta-2microglobulin/creatinine and the retinol binding protein/creatinine ratios), the eGFRcr reduction during treatment was interpreted as transporter inhibition at the level of creatinine excretion from the proximal tubule rather than renal toxicity.

Recent data from REEF-2 confirm the transient pattern of eGFRcr declines but, in addition, show an increase of the beta-2microglobulin/creatinine and the retinol binding protein/creatinine ratios in some participants when tenofovir disoproxil fumarate (TDF) treatment was continued and combined with JNJ-6379+JNJ-3989. These new data are suggesting that JNJ-6379 in combination with TDF may contribute to renal tubulo-toxicity. There was no apparent increase in the beta-2-microglobulin/creatinine or retinol binding protein/creatinine ratios in participants receiving ETV (active or control arm), nor in participants receiving TDF+placebo.

The negative impact of JNJ-6379, when combined with JNJ-3989 + NA, on HBsAg reduction taken together with the adverse renal profile leads to conclusion of an unfavorable benefit-risk balance of JNJ-6379 in combination with JNJ-3989+NA, compared to JNJ-3989+NA alone. Therefore, the Sponsor has decided to discontinue treatment with JNJ-6379 in all ongoing clinical studies effective immediately. Participants currently on treatment with JNJ-6379 will be contacted and requested to stop taking JNJ-6379, while continuing treatment with NA, JNJ-3989 and optional PegIFN- $\alpha$ 2a. For newly enrolled participants, JNJ-6379 will be no longer included in the treatment regimen.

In addition, a new NA re-treatment criterion and more frequent monitoring for participants who discontinued NA treatment during follow-up were added. The reason for these changes is a severe clinical alanine aminotransferase (ALT) flare that was reported following discontinuation of NA treatment in a virologically suppressed HBeAg negative participant on long-term TDF treatment who was randomized to the control arm (placebo + placebo + NA) in the REEF-2 study. The participant presented with hepatitis B

virus (HBV) DNA levels that increased rapidly, before any relevant changes in liver markers were noted. Discontinuation of NA treatment followed the protocol-defined criteria and was in line with recent European Association for the Study of the Liver (EASL) treatment guidelines.<sup>5</sup> Flares following NA discontinuation are not unexpected, but the rapid evolution and clinical deterioration seen in this participant who was anti-HBe antibody positive at screening and had no history or evidence of liver cirrhosis was unforeseeable. Therefore, to protect safety of participants, the protocol was amended as detailed below.

In addition, based on Health Authority request, it has been clarified that the follow-up phase of 48 weeks will be extended to ensure that all study participants have at least one year of follow-up after NA treatment cessation.

Furthermore, the eligibility criteria, the PegIFN- $\alpha$ 2a discontinuation criteria, and the monitoring of neuropsychiatric adverse events during PegIFN- $\alpha$ 2a treatment were amended to be consistent with the PegIFN- $\alpha$ 2a prescribing information.

Other changes, clarifications and corrections were also made as detailed below.

| <b>Description of Change</b> | Brief Rationale | Section Number and Name |
|---|---|---|
| Throughout the protocol, JNJ-6379 has been removed as study intervention. Participants enrolled before Protocol Amendment 5 and who are being treated with JNJ-3989+JNJ-6379+NA (Arm 1 in Panel 1 and Panel 2) had to stop JNJ-6379 treatment immediately. They will continue with JNJ-3989+NA treatment up to the end of the 48-week open-label study intervention phase and will then enter the follow-up phase during which they stop treatment with JNJ-3989 and NA if completion criteria are met. Throughout the protocol, elements specific for JNJ-6379 have been modified. | Based on emerging data from recent interim analyses of the REEF-1 and REEF-2 studies, showing that the benefit-risk profile of JNJ-6379 in combination with JNJ-3989+NA is unfavorable compared to JNJ-3989+NA. | 1.1 Synopsis 1.2 Schema 1.3.1 Schedule of Activities Screening and Study Intervention Phase 2 INTRODUCTION 2.1 Study Rationale 2.2 Background 2.3 Benefit-Risk Assessment 2.3.2.2.2 Potential Risks for JNJ-6379 2.3.3 Benefit-risk Assessment for Study Participation 3 OBJECTIVES AND ENDPOINTS 4.1 Overall Design 4.2 Scientific Rationale for Study Design 4.3 Justification for Dose 4.3.2 JNJ-6379 5.1 Inclusion Criteria 5.2 Exclusion Criteria 6.1 Study Intervention(s) Administered 6.2 Preparation/Handling/Storage/Accountability 6.3 Measures to Minimize Bias: Randomization and Blinding 6.4 Study Intervention Compliance 6.5 Concomitant Therapy 6.6 Dose Modification 6.6.1 Study Intervention Completion at Week 48 7.1 Discontinuation of Study Intervention 8 STUDY ASSESSMENTS AND PROCEDURES 8.4.4 Clinical Safety Laboratory Assessments8.5.5 Pregnancy8.5.6 Adverse Events of Special Interest 8.5.7 Other Toxicities 8.6 Treatment of Overdose 8.7 Pharmacokinetics 8.7.1 Evaluations |

| A new NA re-treatment criterion was added for participants who discontinued NA treatment during follow-up. | To ensure that participants with significant HBV DNA increases during treatment-free follow-up are monitored at least weekly and/or immediately re-start NA treatment irrespective of ALT levels. | 8.7.3 Pharmacokinetic Parameters and Evaluations 8.8 Pharmacokinetics/Pharmacodynamics 9.2 Sample Size Determination 9.3 Populations for Analyses 9.4 Statistical Analyses 9.4.1 Analysis of Efficacy and Antiviral Activity 9.4.2 Safety Analyses 9.4.3 Other Analyses 10.1 Appendix 1: Abbreviations and Definitions of Terms 10.5 Appendix 5: Rash Management 10.6 Appendix 6: Intervention-emergent ALT/AST Elevations 1.1 Synopsis 1.3.2 Schedule of Activities Follow-up Phase 4.2 Scientific Rationale for Study Design 6.6.2 NA Re-treatment Criteria During Follow-up 7.1 Discontinuation of Study Intervention 8.5.6.2 Intervention-emergent ALT/AST Elevations 10.12 Appendix 12: NA Re-treatment During |
|---|---|---|
| Participants who discontinue NA treatment during follow-up, will be monitored more frequently, with a study visit at least once every 4 weeks. The visit frequency for participants who continue NA treatment or have restarted NA treatment during the follow-up period and for whom the HBV DNA and ALT values are stable remains at least once every 12 weeks. For participants with increased follow-up, the total blood volume to be collected during | To further protect the safety of participants. | Follow-up 1.3.2 Schedule of Activities Follow-up Phase 2.3.2.2 Potential Risks 6.7 Study Intervention After the End of the Study 7.1 Discontinuation of Study Intervention 8 STUDY ASSESSMENTS AND PROCEDURES |
| the study will increase. A note has been added to clarify that the follow-up phase of 48 weeks will be extended with a maximum of 24 weeks (ie, up to Follow-up Week 72) to ensure that all study participants have at least one year of follow-up after NA treatment cessation. The end of study definition and study completion definitions were updated to include this possible extension. For participants with extended follow-up, the total blood | Upon Health authority request. | 1.1 Synopsis 1.2 Schema 1.3.2 Schedule of Activities Follow-up Phase 4.1 Overall Design 4.2 Scientific Rationale for Study Design 4.4 End of Study Definition 6.6.1 Study Intervention Completion at Week 48 8 STUDY ASSESSMENTS AND PROCEDURES |

| | | AMENDMENT |
|---|---|---|
| volume to be collected during | | |
| the study was updated. | | |
| The PegIFN-α2a | Upon Health Authority | 1.3.1 Schedule of Activities Screening and |
| discontinuation criteria were | request and to be consistent | Study Intervention Phase |
| updated to clarify that | with the PegIFN-α2a | 1.3.3 Schedule of Activities – Optional |
| participants with moderate or | prescribing information | PegIFN-α2a Treatment |
| severe depression or other | | 5.2 Exclusion Criteria |
| psychiatric symptoms should | | 7.1 Discontinuation of Study Intervention |
| immediately discontinue | | |
| PegIFN-α2a treatment. | | |
| In addition, participants will be | | |
| closely monitored for | | |
| neuropsychiatric adverse events | | |
| during the optional PegIFN-α2a | | |
| treatment period. | | |
| Participants who develop a | | |
| neuropsychiatric adverse event | | |
| during optional PegIFN-α2a | | |
| treatment will be monitored | | |
| closely until the | | |
| neuropsychiatric adverse event | | |
| resolves, with frequent (at least | | |
| weekly) follow-up phone calls. | | |
| Furthermore, exclusion | | |
| criterion 31 was amended to | | |
| exclude participants with a | | |
| history of a severe psychiatric | | |
| disorder. | | |
| The Contraceptive and Barrier | Upon Health Authority | 5.1 Inclusion Criteria |
| Guidance and Collection of | request and to align with the | 10.8 Appendix 8: Contraceptive and Barrier |
| Pregnancy Information section | latest version of the | Guidance and Collection of Pregnancy |
| was updated: the list of | sponsor's protocol template. | Information |
| examples which are not | sponsor's protocor template. | |
| allowed as sole method of | | |
| contraception during the study | | |
| and the footnote concerning | | |
| possible interaction between | | |
| hormonal contraception and the | | |
| study intervention have been | | |
| removed. Additional | | |
| clarifications were also made. | | |
| Recommendations regarding | Clarification considering the | 6.5 Concomitant Therapy |
| the use of live vaccines during | second dose concerns a life- | 10.11 Appendix 11: Covid Appendix |
| the study were added. | attenuated virus. | |
| It was clarified that venous | Clarification. | 1.1 Synopsis |
| blood samples will be collected | | 1.3.1 Schedule of Activities Screening and |
| for measurement of JNJ-3989, | | Study Intervention Phase |
| NA, and PegIFN-α2a. | | 3 OBJECTIVES AND ENDPOINTS |
| However, bioanalysis of NA | | 8.7 Pharmacokinetics |
| and PegIFN-α2a is optional at | | 8.7.1 Evaluations |
| the discretion of the sponsor. | | |
| Bioanalysis of JNJ-6379 may | | |
| also be done on samples | | |
| and de done on bumples | L | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| collected from participants who received JNJ-6379 up to Protocol Amendment 4. | | |
|---|---|---|
| Exclusion criterion 1 was adapted to clarify that participants with a positive HIV-1 or HIV-2 antibody/antigen test at screening should have a confirmatory HIV RNA test, to rule out false positive results. They can be enrolled if they have a negative HIV RNA test at screening. It was also clarified that participants with evidence of HIV-1 or HIV-2 infection who are on antiretroviral treatment are excluded. | Clarification upon Health<br>Authority request | 5.2 Exclusion Criteria |
| It was clarified that the use of low-dose aspirin is allowed with exception of 7 days prior to biopsies. | Clarification upon investigator's request. | 1.1 Synopsis 6.5 Concomitant Therapy 8.1 Liver Biopsy and Fine Needle Aspiration Biopsy |
| Minor errors were corrected and minor clarifications were made. | Correction and clarification. | Throughout the protocol |

## **Amendment 4 (30 July 2021)**

Overall Rationale for the Amendment: The primary reason for this amendment is to offer participants optional treatment with PegIFN-α2a for either 12 or 24 weeks starting after the Week 40 biopsy (or after the optional leukapheresis if applicable), to investigate whether addition of PegIFN-α2a towards the end of the treatment regimen may enhance response to treatment. This change is based on the availability of preliminary 48-week treatment data from the Phase 2b study REEF-1 (73763989HPB2001) and new data presented during the European Association for the Study of the Liver (EASL) conference of 2021 showing that HBsAg declines with siRNA treatment can be increased when combined with PegIFN. <sup>43</sup>

The REEF-1 study is evaluating the efficacy of 3 doses of JNJ-3989 (40, 100, or 200 mg Q4W) + NA, of JNJ-3989 100 mg Q4W + JNJ-6379 + NA, of JNJ-6379 + NA, and of NA alone. Data showed that all regimens were safe and well-tolerated through end of treatment at Week 48. The JNJ-3989 200 mg dose achieved the highest response rate (19.1%) for the primary endpoint of meeting the NA treatment completion criteria at Week 48 (ie, ALT <3x ULN, HBV DNA <LLOQ, HBeAg-negative [<LLOQ], and HBsAg <10 IU/mL). No participant in the JNJ-6379 + NA arm and 1 participant in the NA alone arm achieved the primary endpoint. The largest mean (SD) decline at Week 48 of 3.56 (1.328) log<sub>10</sub> IU/mL was observed in the JNJ-3989 200 mg + NA arm in the HBeAg positive currently not treated participants. The mean HBsAg decline followed a biphasic pattern, with a steeper decline during the first 24 weeks followed by a more shallow decline between Week 24 and Week 48. At Week 48, a limited number of participants reached HBsAg seroclearance.

This amendment will allow to investigate whether addition of PegIFN- $\alpha$ 2a for 12 or 24 weeks at or after the Week 40 biopsy increases the participant's chances to achieve HBsAg loss.

| <b>Description of Change</b> | Brief Rationale | Section Number and Name |
|---|---|---|
| In addition to the study | To investigate whether | 1.1 Synopsis |
| intervention participants are | addition of PegIFN-α2a | 1.2 Schema |
| randomized to, they may also | towards the end of the | 1.3.3 Schedule of Activities – Optional |
| receive optional treatment with | treatment regimen increases | PegIFN-α2a Treatment |
| PegIFN-α2a after the Week 40 | the participant's chances to | 2 INTRODUCTION |
| biopsy (or after the optional | achieve HBsAg loss. | 2.1 Study Rationale |
| leukapheresis if applicable) but | delife ve 11251 ig 1655. | 2.2.1.3 Combination of JNJ-3989 with |
| before the Week 48 visit. The | | PegIFN-α2a |
| duration (either 12 or 24 | | 2.2.1.4 Combination of JNJ-6379 with |
| weeks) will be at the | | PegIFN-α2a |
| , | | 2.2.2.3 Combination of JNJ-3989 and JNJ- |
| investigator's discretion. | | 6379 with PegIFN-α2a<br>2.3 Benefit-Risk Assessment |
| | | 3 OBJECTIVES AND ENDPOINTS |
| | | 4.1 Overall Design |
| | | 5.2 Exclusion Criteria |
| | | 6.1 Study Intervention(s) Administered |
| | | 6.2 |
| | | Preparation/Handling/Storage/Accountability |
| | | 6.4 Study Intervention Compliance |
| | | 6.5 Concomitant Therapy |
| | | 6.6 Dose Modification |
| | | 7.1 Discontinuation of Study Intervention |
| | | 8 STUDY ASSESSMENTS AND |
| | | PROCEDURES |
| | | 8.5.6 Adverse Events of Special Interest |
| | | 8.6 Treatment of Overdose |
| | | 8.7 Pharmacokinetics |
| | | 8.8 Pharmacokinetics/Pharmacodynamics |
| | | 9.4.3 Other Analyses |
| | | 10.1 Appendix 1: Abbreviations and |
| | | Definitions of Terms |
| | | 10.2 Appendix 2: Clinical Laboratory Tests<br>10.3 Appendix 3: Regulatory, Ethical, and |
| | | Study Oversight Considerations |
| | | 10.11 Appendix 11: Covid Appendix |
| | | 11 REFERENCES |
| | | TI KLI EKLIVELS |
| ALT elevations were added as | To ensure the safety of | 2.3.2.2.1 Potential Risks for JNJ-3989 |
| a potential risk and the section | participants during treatment | 8.5.6.1 Injection Site Reactions |
| on management of ALT | with JNJ-3989, based on | 10.6 Appendix 6: Intervention-emergent |
| elevations was updated. | emerging data from studies | ALT/AST Elevations |
| cicvations was updated. | REEF-1 and REEF-D. | |
| Updates were made to the | For increased precision of | 1.1 Symonesis |
| assumed statistical distribution | <u> </u> | 1.1 Synopsis 9.2 Sample Size Determination |
| | the estimation of the | 9.4.1.1 Analysis of the Primary Endpoint |
| and model-based approach that | primary efficacy endpoint | 11 REFERENCES |
| will be used in the analysis of | and its variability. | 11 REI EREINOES |
| the primary efficacy endpoint | | |
| and also used to justify the | | |
| planned sample size. | | |
| Removal of the mITT | The same approach for | 1.1 Synopsis |
| population. | complete case analysis can | 9.3 Populations for Analyses |
| | be implemented using the | 9.4.1 Analysis of Efficacy and Antiviral |
| | ITT population (including | Activity |
| | 111 population (including | <u> </u> |

| | | AMENDMENT |
|---|---|---|
| | all panels) and therefore | |
| | mITT can be removed. | |
| Description of efficacy and | For clarification and | 9.4.1 Analysis of Efficacy and Antiviral |
| antiviral activity analyses were | completeness. | Activity |
| added to clarify the | | |
| explorations of interest which | | |
| include the statistical analyses | | |
| overall for the entire study | | |
| population, the comparisons | | |
| between panels regardless of | | |
| intervention arm, between | | |
| intervention arms within panel, | | |
| and between intervention arms | | |
| across panels. | | |
| Updates were made to the | For completeness. | 2.2.2.1 JNJ-3989 and JNJ-6379 |
| clinical background section as | i or compressions. | 2.2.2.2 Combination of JNJ-3989 and JNJ- |
| more data have become | | 6379 with Entecavir, Tenofovir Disoproxil, or |
| available. | | Tenofovir Alafenamide |
| avanasie. | | 2.3.3 Benefit-risk Assessment for Study |
| | | Participation |
| | | 11 REFERENCES |
| Update of follow-up procedures | For clarification. | 4.2 Scientific Rationale for Study Design |
| and criteria for re-initiation of | | 6.6.2 NA Re-treatment Criteria During Follow- |
| NA treatment. | | up |
| | | 10.12 Appendix 12: NA Re-treatment During Follow-up |
| A study intervention | For completeness. | 7.1 Discontinuation of Study Intervention |
| discontinuation criterion was | For completeness. | 7.1 Discontinuation of Study Intervention |
| added for participants who | | |
| withdraw consent. | | |
| Study intervention | For clarification. | 7.1 Discontinuation of Study Intervention |
| discontinuation criteria on | For Clarification. | 8.5.6.4 Renal Complications |
| hepatic decompensation and | | 0.5.0.4 Renar Complications |
| eGFR <sub>cr</sub> abnormality were | | |
| updated. | | |
| 1 | For completeness | 7.1 Discontinuation of Study Intervention |
| The study intervention discontinuation criterion on | For completeness. | 7.1 Discontinuation of Study Intervention |
| virologic breakthrough was | | |
| updated. | | |
| * | Correction. | 1.2.1 Sahadula of Activities Saragning and |
| Local platelet aggregation | Correction. | 1.3.1 Schedule of Activities Screening and Study Intervention Phase |
| testing was added to the schedule of activities instead of | | 1.3.2 Schedule of Activities Follow-up Phase |
| | | 1.5.2 Senedate of rectivities 1 onlow up 1 hase |
| only mentioned in a footnote. | Comment's an | 121 61 11 16 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 |
| The footnotes related to HBeAg | Correction. | 1.3.1 Schedule of Activities Screening and |
| testing were corrected. | T | Study Intervention Phase |
| Language on urine pregnancy | To provide additional | 1.3.2 Schedule of Activities Follow-up Phase |
| testing for at-home use was | guidance on urine pregnancy | 10.11 Appendix 11: Covid Appendix |
| updated. | testing at home. | 52F 1 .: C.:. |
| Exclusion criterion 1 | For clarification. | 5.2 Exclusion Criteria |
| (concerning evidence of HIV-1 | | |
| or HIV-2 infection at | | |
| screening) and criterion 2 were | | |
| updated. | | |
| It was clarified that JNJ-3989 should preferably be administered via subcutaneous injection in the abdomen. | For clarification. | 1.1 Synopsis 6.1 Study Intervention(s) Administered |
|---|---|---|
| Head, neck, and thyroid were added to complete physical examination. | For completeness. | 8.4.1 Physical Examinations |
| Language was added on medical encounters. | For completeness. | 8.11 Medical Encounters |
| Management of rash and acute systemic allergic reactions were moved under a separate subheader. | For correction and clarification as rash and acute systemic allergic reactions are not considered AESIs for JNJ-3989 or JNJ-6379. | 8.5.6 Adverse Events of Special Interest |
| Minor errors were corrected and minor clarifications were made. | Correction and clarification. | Throughout the protocol |

# Amendment 3 (14 August 2020)

Overall Rationale for the Amendment: The sample size justification section was updated.

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 9.2 Sample Size Determination | More details were added on the | For clarification |
| 11 REFERENCES | justification for sample size | |
| | determination | |
| 1.3.2 Schedule of | Optional biopsy was delinked from | The leukapheresis procedure was |
| Activities - Follow-up Phase | the leukapheresis procedure | incorrectly linked with the optional |
| | | biopsy |
| 10.11 Appendix 11: Covid | Guidance on study conduct during | Options for study-related |
| Appendix | the COVID-19 pandemic was | participant management are being |
| | added | provided in the event of disruption |
| | | to the study conduct due to the |
| | | COVID-19 pandemic |

# **Amendment 2 (07 May 2020)**

**Overall Rationale for the Amendment:** Following Health Authority (HA) feedback the protocol was amended as specified below

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| 1.1 Synopsis, 9.3 Populations for | An additional population (mITT) | Per HA request, the modified ITT |
| Analyses | was added. | (mITT) analysis set, restricted to |
| | | participants with biopsy data at |
| | | both Baseline and Week 40, was |
| | | defined as the primary analysis |
| | | population for consistency with the |
| | | planned observed cases analysis of |
| | | the primary efficacy endpoint |
| | | described in section 9.4.1.1. |

| 9.4.1 Analysis of Efficacy and<br>Antiviral Activity, 9.4.1.1 Analysis<br>of the Primary Endpoint, 9.4.1.2<br>Analysis of Secondary Endpoints,<br>9.4.1.3 Analysis of Exploratory<br>Endpoints | The mITT analysis set was added to the ITT set for the purpose of the efficacy analyses. | Per HA request, in order to evaluate<br>the potential bias in using complete<br>case analysis, both mITT as<br>primary analysis set and ITT as<br>secondary analysis set will be used. |
|---|---|---|
| Title page and footer | Updated confidentiality statement | In line with the latest protocol template |

# Amendment 1 (10 April 2020)

**Overall Rationale for the Amendment:** Following Health Authority (HA) feedback the protocol was amended as specified below

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| 9.4.1.1 Analysis of the Primary | Methods for handling missing data | Per HA request the approach to |
| Endpoint | were added to the protocol. | handle missing data in the primary |
| | | analysis of the primary endpoint |
| | | was added. |
| 2.3.2.3.1 Potential Risks and | The risk language regarding | Per HA request the complications |
| Inconvenience Associated with the | possible serious complications of | from a liver biopsy are now |
| Liver Biopsy Procedures | liver biopsies has been updated. | described in the protocol. |
| 8.5.6.3 Complications From Liver | | |
| Biopsy | | |
| 1.3.1 Schedule of | Additional timepoints were added | Correction |
| Activities - Screening and Study | for whole blood single cell | |
| Intervention Phase | profiling. | |
| Schedule of Activities - Follow-up | | |
| Phase | | |

## 10.11. Appendix 11: Covid Appendix

#### GUIDANCE ON STUDY CONDUCT DURING THE COVID-19 PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including hospitals; study-site personnel being reassigned to critical tasks.

In alignment with recent health authority guidance, the sponsor is providing options for study-related participant management in the event of disruption to the conduct of the study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health and well-being of participants and site staff and maintain oversight of delegated trial activities. If, at any time, a participant's safety is considered at risk, study intervention will be discontinued, and study follow-up will be conducted.

Scheduled visits that cannot be conducted in person at the study site will be performed to the extent possible remotely/virtually or delayed until such time that on-site visits can be resumed. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible. Participants will also be questioned regarding general health status to fulfill any physical examination requirement.

Every effort should be made to adhere to protocol-specified assessments for participants on study intervention, including follow-up. Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, or the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the CR).

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance. If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical officer to discuss plans for study intervention and follow-up. Modifications made to the study conduct as a result of the COVID-19 pandemic should be summarized in the clinical study report.

#### GUIDANCE SPECIFIC TO THIS PROTOCOL

The following emergency provisions are meant to ensure participant safety on study while site capabilities are compromised by COVID-19 related restrictions. Remote medical consultation and alternatives to study intervention dispensing, administration, and clinical laboratory assessments may allow continued study participation for participants in this trial. Before implementing any of these emergency provisions, the sponsor should be consulted to perform a benefit-risk analysis and to ensure the measures are executed and documented correctly.

As restrictions are lifted and the acute phase of the COVID-19 pandemic resolves, sites should revert to original protocol conduct as soon as feasible and in accordance with any country-specific regulatory requirements.

## Dispensing/administration of study intervention:

- For participants able to visit the study site, but who request to reduce visit frequency, or for whom limited access to the site is expected, an additional supply of oral study intervention can be provided.
- For participants unable to visit the study site, direct-to-patient (DTP) shipment or handover to a caregiver or delegate of oral study intervention may be implemented, where allowed per local regulations and if requested by the treating study physician. Where DTP shipments or handover to delegates are deemed necessary, the process must be coordinated between the site and sponsor staff following standard DTP procedures for arranging shipment and adhering to associated approvals and documentation requirements.
- JNJ-3989 should always be administered by a nurse at the study site or, if site visits are not possible, at the participant's home. Per the protocol, if a scheduled injection of JNJ-3989 was missed, the injection should be given as soon as possible but within 3 weeks after the scheduled time. Otherwise, the injection should be skipped and the next injection should be given at the next scheduled time point per the initial injection schedule.

## **Continuation of study intervention:**

- Any issue with continuation and/or provision of study intervention should be discussed with the sponsor and should be well documented.
- Study intervention should be continued if, in the assessment of the investigator, it does not result in risk to the participant. If at any time the participant's safety is considered at risk due to study intervention, study intervention will be temporarily or permanently discontinued, while every effort should be made to maintain follow-up on study. The benefit of continuing study intervention should be assessed by the investigator for each individual participant, considering the potential impact of reduced direct clinical supervision on participant safety.
- If a participant develops a SARS-CoV-2 infection, the investigator should contact the sponsor to discuss plans for study intervention and follow-up. A decision to continue study intervention should be made by the investigator depending on symptoms and concomitant medication(s) used for the treatment of COVID-19. Study intervention must be discontinued if prohibited medication is used.

• When a participant, for whom study intervention has been interrupted, recovers from suspected or confirmed SARS-CoV-2 infection or related disease and all AEs related to SARS-CoV-2 infection improve to Grade ≤1, the investigator should discuss with the sponsor about resuming study intervention.

## **COVID-19** vaccination during the study:

Local guidelines on the use of live vaccines in participants receiving PegIFN-α2a should be followed, including for the second dose of Sputnik V (which contains rAd5, with a theoretical risk of replication competence). Sputnik Light, which is the first dose of Sputnik V (with rAd26) is not considered a live vaccine. See below for further guidance on the use of COVID-19 vaccines.

Locally approved COVID-19 vaccines (including those that received emergency use authorization or conditional marketing authorization) are allowed throughout the study. For participants receiving PegIFN- $\alpha$ 2a, the following recommendations should be applied to accommodate COVID-19 vaccination during PegIFN- $\alpha$ 2a treatment:

- COVID-19 vaccine and PegIFN- $\alpha$ 2a should not be administered on the same day.
- If required, PegIFN- $\alpha$ 2a injection can be delayed with 2 days. The next PegIFN- $\alpha$ 2a injection should be performed at the scheduled time.
- If required, skipping a PegIFN-α2a injection may be considered after consultation with the Sponsor.
- Vaccination with Sputnik V should take above-mentioned consideration about live vaccines into account.

All COVID-19 vaccination-related data (eg, COVID-19 vaccination, AEs, AE management) should be appropriately captured in the CRF and source documents. Refer to the COVID-19 vaccine and/or PegIFN-α2a prescribing information for more details.

#### Study visits and assessments:

- If possible, central laboratory testing as outlined in the Schedule of Activities is to be continued. If central laboratory tests cannot be performed, the use of a local laboratory is allowed for study evaluations. A copy of the local laboratory report should be reviewed by the investigator and filed with the source documents, along with reference ranges.
- To safely maintain participants on study intervention while site capabilities are compromised by COVID-19-related restrictions, study visits may be performed by a nurse (who received study-specific training) at the patient's home (home health nurse) until such time that on-site visits can be resumed. The following activities may be completed as required per the Schedule of Activities and as feasible:
  - Sampling, processing and shipping of laboratory samples (as described above)
  - Checking study compliance: medication diary (if available), intake of oral study intervention, storage of oral study intervention
  - Performing ECGs

- If JNJ-3989 is administered at the patient's home, it will need to be done by a nurse (who received study-specific training)
- Delivering oral study interventions and urine pregnancy tests for at-home use
- Any data related to adverse events (AEs), concomitant medication, vital signs, and ECGs will be reviewed and assessed by the investigator.
- In addition, participants may have tele-health visits conducted by qualified site personnel via phone or video conversation as per local regulation. Assessments may include review of AEs (including ISRs), concomitant medications, and study intervention accountability. Participants will also be questioned regarding general health status to fulfill any physical examination requirement.
- Procedures and timings should follow the Schedule of Activities as closely as possible. Standard AE/SAE reporting requirements apply.
- Ultrasound (and Fibroscan where applicable) should be done as close as possible to the time points specified in the Schedule of Activities. However, if this is not possible due to COVID-19 related restrictions, the imaging test should be performed as soon as possible.

#### **Informed consent:**

 Consenting and re-consenting of participants (including also remote consenting by phone or video consultation) will be performed as applicable for the measures taken and according to local guidance for informed consent applicable during the COVID-19 pandemic. The process is to be documented in the source documents.

## Source data verification/monitoring:

• In case on-site monitoring visits are not possible, the site monitor may contact the investigator to arrange monitoring activities remotely (in accordance with site and local requirements). Additional on-site monitoring visits may be needed in the future to catch up on source data verification.

#### Site audits:

 During the COVID-19 pandemic and at the impacted sites, study site GCP audits with direct impact/engagement from the investigator and study-site personnel would not be conducted in order to comply with national, local, and/or organizational social distancing restrictions. Additional quality assurance activities such as remote audits or focused review of study-related documents may take place with limited impact/engagement if possible.

# 10.12. Appendix 12: NA Re-treatment and Monitoring After Stopping of NA

Participants who meet the NA treatment completion critera will be monitored for NA re-treatment during the follow-up phase

#### Frequency of monitoring:

- Regular monitoring visits will be every 4 weeks during the follow up phase in accordance with the schedule of activities (SoA)
- A post-treatment HBV DNA value of >20,000 IU/mL should trigger re-testing of ALT/AST, HBV DNA, and total and direct bilirubin
  within a maximum of 7 days from receipt of the data and further repeats as necessary (ie, weekly until HBV DNA returns to
  <20,000 IU/mL)</li>
- A post-treatment HBV DNA value of >2,000 IU/mL (but <20,000 IU/mL) should trigger a re-test within 14 days from receipt of the
  data and further repeats as necessary (ie, every other week until HBV DNA returns to <2,000 IU/mL)</li>
- A post-treatment ALT value of >5x ULN should trigger re-testing of ALT, AST, ALP, total and direct bilirubin, INR, albumin, and HBV DNA on a weekly basis until ALT and AST levels have returned to <5x ULN</li>

#### Re-start of NA treatment:

Status: Approved, Date: 25 November 2021

- immediately with signs of decreasing liver function based on laboratory findings (eg, INR, direct bilirubin) or clinical assessment (eg, ascites, hepatic encephalopathy)
- immediately with an HBV DNA value of >100,000 IU/mL (irrespective of confirmation and/or ALT increase)
- with confirmed post-treatment HBeAg seroreversion (HBeAg positive after it was negative at NA completion)
- with confirmed\* post-treatment increases in HBV DNA >2,000 IU/mL and ALT >5x ULN
- With confirmed\* post-treatment increases in HBV DNA >20,000 IU/mL

Note: Additional re-testing and/or earlier restarting of NA-treatment is at the investigator's discretion also if the above cut-offs are not yet met.

<sup>\*</sup> At least 4 weeks apart - frequency of visits as described above

#### 11. REFERENCES

- 1. American Red Cross Blood donor eligibility requirements. Available from: http://www.redcrossblood.org/donating-blood/eligibility-requirements. Accessed 28 March 2019.
- 2. Burak KW, Sherman M. Hepatocellular carcinoma: Consensus, controversies and future directions. A report from the Canadian Association for the Study of the Liver Hepatocellular Carcinoma Meeting. Can J Gastroenterol Hepatol. 2015;29(4):178 84.
- 3. Cohen SM, Johansson SL, Arnold LL, Lawson TA. Urinary tract calculi and thresholds in carcinogenesis. Food and Chem Toxicol. 2002;40;793-799.
- 4. Dusheiko G, Wang B, Carey I. HBsAg loss in chronic hepatitis B: pointers to the benefits of curative therapy. Hepatol Int. 2016;10:727 729.
- 5. European Association for the Study of the Liver (EASL) clinical practice guidelines on the management of chronic hepatitis B virus infection. J Hepatol. 2017;67:370-398.
- 6. European Medicines Agency (EMA). Assessment report Vemlidy (Tenofovir alafenamide). https://www.ema.europa.eu/documents/assessment-report/vemlidy-epar-public-assessment-report en.pdf. 10 November 2016. Accessed 29 January 2019.
- 7. Fang Z, Li J, Yu X, et al. Polarization of monocytic myeloid-derived suppressor cells by hepatitis B surface antigen is mediated via ERK/IL-6/STAT3 signaling feedback and restrains the activation of T cells in chronic hepatitis B virus infection. J Immunol. 2015;195(10):4873-4483.
- 8. Gane E, et al. Dose Response with the RNA Interference Therapy JNJ-3989 Combined with Nucleos(t)ide Analogue Treatment in Expanded Cohorts of Patients with Chronic Hepatitis B. The Liver Meeting, Boston 2019, Poster 0696.
- 9. Gehring AJ, Protzer U. Targeting Innate and Adaptive Immune Responses to Cure Chronic HBV Infection. Gastroenterology. 2019 Jan;156(2):325-337.
- 10. Gill US, Pallett LJ, Kennedy PTF, et al. Liver sampling: a vital window into HBV pathogenesis on the path to functional cure. Gut 2018;67:767-775.
- 11. Gill US, Pallett LJ, Thomas N, et al. Fine needle aspirates comprehensively sample intrahepatic immunity. Gut 2019;68:1493-1503.
- 12. Henry SP, Johnson M, Zanardi TA, Fey R, Auyeung D, Lappin PB, Levin AA. Renal uptake and tolerability of a 2'-O-methoxyethyl modified antisense oligonucleotide (ISIS 113715) in monkey. Toxicology. 2012;301(1 3):13-20.
- 13. International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartite Guideline E14: Clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs. ICH 12 May 2005.
- 14. Investigator's Brochure: JNJ-56136379 Edition 6. Janssen Research & Development (February 2021).
- 15. Investigator's Brochure: JNJ-73763989 Edition 5. Janssen Research & Development (April 2021).
- 16. Investigator's Brochure: JNJ-73763989 Edition 5, Addendum 1. Janssen Research & Development (July 2021).
- 17. Janas MM, Harbison CE, Perry VK, et al. The nonclinical safety profile of GalNac-conjugated RNAi therapeutics in subacute studies. Toxicol. Pathol. 2018;46(7):735-745.
- 18. Janssen HLA, Arif A. Averting hepatocellular carcinoma in chronic hepatitis B with antiviral therapy: tipping the balance or not yet? Gastroentology. 2014;147:24 26.
- 19. Jeng W-J, Chen Y-C, Chien R-N, Sheen I-S, Liaw Y-F. Incidence and predictors of hepatitis B surface antigen seroclearance after cessation of nucleos(t)ide analogue therapy in hepatitis B e antigen-negative chronic hepatitis B. Hepatology. 2018;68:425-434.
- 20. Li H, Zhai N, Wang Z, et al. Regulatory NK cells mediated between immunosuppressive monocytes and dysfunctional T cells in chronic HBV infection. Gut. 2018;67(11):2035-2044.

- 21. Lok AS, Zoulim F, Dusheiko G, Ghany MG. Hepatitis B cure: from discovery to regulatory approval. J Hepatol. 2017;67(4):847-861.
- 22. Magalhães-Costa P, Lebre L, Peixe P, Santos S, Chagas C. Hepatocellular carcinoma in chronic hepatitis B patients on third generation nucleos(t)ides analogs: Risk factors and performance of a risk score. GE Port J Gastroenterol. 2016;23:233-242.
- 23. Memorandum to Advisory Committee Members and Guests from Entecavir Review Team. Briefing document for NDA 21-797, entecavir 0.5 and 1 mg tablets and NDA 21-798, entecavir oral solution 0.05 mg/mL, 10 February 2005.
- 24. Memorandum to Advisory Committee Members and Guests from Tenofovir Review Team. Background Package for NDA 21-356: VIREAD (tenofovir disoproxil fumarate), 6 September 2001.
- 25. Papatheodoridis GV, Chan HLY, Hansen BE, et al. Risk of hepatocellular carcinoma in chronic hepatitis B: Assessment and modification with current antiviral therapy. J Hepatol. 2015;62:956 967.
- 26. Papatheodoridis GV, Rigopoulou EI, Papatheodoridi M, et al. DARING-B: discontinuation of effective entecavir or tenofovir disoproxil fumarate long-term therapy before HBsAg loss in non-cirrhotic HBeAg negative chronic hepatitis B. Antivir Ther. 2018;23(8):677-685.
- PEGASYS Summary of Product Characteristics.
   http://www.ema.europa.eu/docs/en GB/document library/EPAR Product Information/human/000395/WC500039195.pdf. Accessed 22 November 2019
- 28. Polaris Observatory Conservatory. Global prevalence, treatment, and prevention of hepatitis B virus infection in 2016: a modelling study. Lancet Gastroenterol Hepatol 2018;3:383–403.
- 29. Rehermann B, Thimme R. Insights From Antiviral Therapy Into Immune Responses to Hepatitis B and C Virus Infection. Gastroenterology. 2019;156(2):369–383.
- 30. Sarin KS, Kumar M, Lau GK, et al. Asian-Pacific clinical practice guidelines on the management of hepatitis B: A 2015 update. Hepatol Int. 2016;10:1-98.
- 31. Stanaway JD, Flaxman AD, Naghavi M, et al. The global burden of viral hepatitis from 1990 to 2013: findings from the global burden of disease Study 2013. Lancet. 2016;388(10049):1081-1088.
- 32. Tannehill-Gregg SH, Dominick MA, Reisinger AJ, et al. Strain-related Differences in Urine Composition of Male Rats of Potential Relevance to Urolithiasis. Toxicol Pathol. 2009;37:293-305.
- 33. Terrault NA, Bzowej NH, Chang K, et al. AASLD guidelines for treatment of chronic hepatitis B. Hepatology. 2016;63(1):261 283.
- 34. Wang S, Chen Z, Hu C, et al. Hepatitis B virus surface antigen selectively inhibits TLR2 ligand-induced IL-12 production in monocytes/macrophages by interfering with JNK activation. J Immunol. 2013;190(10):5142 5151.
- 35. Wooddell CI, Yuen MF, Chan HL, et al. RNAi-based treatment of chronically infected patients and chimpanzees reveals that integrated hepatitis B virus DNA is a source of HBsAg. Sci. Transl. Med. 2017; 9: 409.
- 36. Yuen MF, Chen DS, Dusheiko GM, et al. Hepatitis B virus infection. Nat Rev Dis Prim. 2018; 4: Article number 18035.
- 37. Yuen MF, et al. First Clinical Experience with RNA Interference-based Triple Combination Therapy in Chronic Hepatitis B: JNJ-3989, JNJ-6379 and a Nucleos(t)ide Analogue. The Liver Meeting, Boston 2019, LB Poster 4.
- 38. Newcombe RG. Interval estimation for the difference between independent proportions: comparison of eleven methods. Stat Med. 1998; 17, 873-890.
- 39. Investigator's Brochure: JNJ-56136379 Edition 6, Addendum 1. Janssen Research & Development (July 2021).
- 40. Kassahun W, Neysens T, Molenbergh G, Faes C, Verbeke G. Modeling overdispersed longitudinal binary data using a combined beta and normal random-effects model. Arch Public Health. 2012;70(1):7

- 41. PEGASYS Summary of Product Characteristics. Roche Registration GmbH. Revised July 2020. Available at https://www.ema.europa.eu/en/documents/product-information/pegasys-epar-product-information en.pdf. Accessed 4 September 2020.
- 42. PEGASYS United States Prescribing Information. Hoffmann-La Roche, Inc. Revised October 2017. Available at https://www.accessdata.fda.gov/drugsatfda\_docs/label/2017/103964s5270lbl.pdf. Accessed 4 September 2020.
- 43. Yuen MF, et al. Preliminary on-treatment data from a phase 2 study evaluating VIR-2218 in combination with pegylated interferon alfa-2a in participants with chronic hepatitis B infection. EASL 2021. PO-824

## **INVESTIGATOR AGREEMENT**

I have read this protocol and agree that it contains all necessary details for carrying out this study. I will conduct the study as outlined herein and will complete the study within the time designated.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure that they are fully informed regarding the study intervention, the conduct of the study, and the obligations of confidentiality.

| Coordinating Investigato | r (wnere requirea): | | |
|---|---|---|---|
| Name (typed or printed): | | | |
| Institution and Address: | | | |
| Signature: | | Date: | |
| | | | (Day Month Year) |
| Principal (Site) Investigation | tor: | | |
| Name (typed or printed): | _ | | |
| Institution and Address: | | | |
| Telephone Number: | _ | | |
| rerephone runnoer. | | | |
| Signature: | | Date: | |
| | | | (Day Month Year) |
| Consula Damenalla M | alfaal Office | | |
| Sponsor's Responsible M | | | |
| Name (typed or printed): | PPD | | |
| Institution: | Janssen Research & Development | | |
| Signature: _electronic sig | nature appended at the end of the protocol | Date: | |
| | | | (Day Month Year) |

**Note:** If the address or telephone number of the investigator changes during the study, written notification will be provided by the investigator to the sponsor, and a protocol amendment will not be required.

# **Signature**

| User | Date | Reason |
|------|----------------------------------|-------------------|
| PPD | 25-Nov-2021<br>10:27:57<br>(GMT) | Document Approval |